CLINICAL TRIAL: NCT03504397
Title: A Phase 3, Global, Multi-Center, Double-Blind, Randomized, Efficacy Study of Zolbetuximab (IMAB362) Plus mFOLFOX6 Compared With Placebo Plus mFOLFOX6 as First-line Treatment of Subjects With Claudin (CLDN)18.2-Positive, HER2-Negative, Locally Advanced Unresectable or Metastatic Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma
Brief Title: A Study to Compare Zolbetuximab (IMAB362) and Chemotherapy With Placebo and Chemotherapy in Adults With Gastric Cancer.
Acronym: Spotlight
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8951-CL-0301; 2017-002567-17 (EudraCT Number); CTR20190258 (Registry Identifier: ChinaDrugTrials.org.cn); jRCT2080224032 (Other: jRCT); 2024-511365-11-00 (Other: EU(CTIS))
Expanded Access: NCT06048081 (Available)
Record Dates: First submitted 2018-04-12; First posted 2018-04-20 (Actual); Results first posted 2025-02-26 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Locally Advanced Unresectable Gastroesophageal Junction (GEJ) Adenocarcinoma or Cancer; Locally Advanced Unresectable Gastric Adenocarcinoma or Cancer; Metastatic Gastric Adenocarcinoma or Cancer; Metastatic Gastroesophageal Junction (GEJ) Adenocarcinoma
Keywords: HER2; IMAB362; leucovorin; fluorouracil; Gastric cancer; claudiximab; zolbetuximab; oxaliplatin; adenocarcinoma; Gastro-Esophageal Junction cancer; HER2 Negative mFOLFOX6
MeSH Terms: conditions — Adenocarcinoma; Neoplasms; Stomach Neoplasms | interventions — zolbetuximab; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- mFOLFOX6 + Zolbetuximab (Experimental): Participants received intravenous (IV) infusion (minimum 2-hour) of zolbetuximab at a loading dose of 800 milligrams per square meter (mg/m^2) on cycle1 day1(C1D1) followed by 600 mg/m^2 every 3 weeks starting from C1D22 until study treatment discontinuation criteria were met. Participants also received upto 12 treatments of mFOLFOX6 (or components if some were discontinued due to toxicity) over 4/more cycles. mFOLFOX6 was administered on Days 1, 15 & 29 of each cycle (5-FU:400mg/m^2 IV bolus over 5-15 minutes followed by 2400mg/m^2 over 46-48 hours continuous IV infusion every 2 weeks for 4 cycles. Folinic acid: 400mg/m^2 IV infusion over 2 hours; oxaliplatin: 85mg/m^2 IV infusion over 2 hours) A maximum of 12 doses of oxaliplatin was permitted. After mFOLFOX6 treatments, participants continued to receive 5-FU & Folinic acid on Days 1, 15 & 29 of each cycle at the investigator discretion or until study treatment discontinuation criteria were met. Each cycle was approximately 42 days.
  Interventions: Drug: zolbetuximab; Drug: oxaliplatin; Drug: folinic acid; Drug: fluorouracil
- Placebo plus mFOLFOX6 (Placebo Comparator): Participants received an IV infusion (minimum 2-hour infusion) of placebo matched to zolbetuximab on C1D1, followed by subsequent doses every 3 weeks starting from C1D22 until study treatment discontinuation criteria were met. Participants also received up to 12 treatments of mFOLFOX6 (or components if some were discontinued due to toxicity) over 4 or more cycles. mFOLFOX6 was administered on Days 1, 15, and 29 of each cycle (5-fluorouracil: 400 mg/m^2 IV bolus over 5-15 minutes followed by 2400mg/m^2 over 46-48 hours continuous IV infusion every 2 weeks for 4 cycles. Folinic acid: 400 mg/m^2 IV infusion over 2 hours; oxaliplatin: 85 mg/m^2 IV infusion over 2 hours). A maximum of 12 doses of oxaliplatin was permitted. After mFOLFOX6 treatments, participants could continue to receive 5-FU and folinic acid on Days 1, 15, and 29 of each cycle at the investigator's discretion or until study treatment discontinuation criteria were met. Each cycle was approximately 42 days.
  Interventions: Drug: placebo; Drug: oxaliplatin; Drug: folinic acid; Drug: fluorouracil

INTERVENTIONS:
Drug: zolbetuximab — Participants received an IV infusion (as a minimum of 2-hour infusion) of zolbetuximab at a loading dose of 800 mg/m^2 on C1D1 followed by subsequent doses of 600 mg/m^2 every 3 weeks starting from C1D22 until participant meets study treatment discontinuation criteria. Each cycle was approximately 42 days.
  Other Names: IMAB362
  Arms: mFOLFOX6 + Zolbetuximab
Drug: placebo — Participants received an IV infusion (as a minimum of 2-hour infusion) of placebo matched to zolbetuximab on C1D1 followed by subsequent doses every 3 weeks starting from C1D22 until participant met study treatment discontinuation criteria. Each cycle was approximately 42 days.
  Arms: Placebo plus mFOLFOX6
Drug: oxaliplatin — Participants received up to 12 treatments of oxaliplatin administered 85 mg/m^2 IV infusion over 2 hours) on Days 1, 15 and 29 of each cycle.. A maximum of 12 doses of oxaliplatin was permitted. Each cycle was approximately 42 days.
Drug: folinic acid — Participants received up to 12 treatments of folinic acid administered 400 mg/m^2 IV infusion over 2 hours 4 or more cycles on Days 1, 15 and 29 of each cycle. participants could continue to receive folinic acid on Days 1, 15 and 29 of each cycle at the investigator's discretion or until the participant met the study treatment discontinuation criteria. Each cycle was approximately 42 days.
Drug: fluorouracil — Participants received up to 12 treatments of 5-fluorouracil over 4 or more cycles administered by IV bolus 400 mg/m^2 over 5 to 15 minutes followed by 2400mg/m^2 over 46-48 hours continuous IV infusion every 2 weeks for 4 cycles. Participants could continue to receive 5-fluorouracil on Days 1, 15 and 29 of each cycle at the investigator's discretion or until the participant met the study treatment discontinuation criteria. Each cycle was approximately 42 days.

SUMMARY:
Zolbetuximab is being studied in people with cancer in and around the stomach or where the food pipe (esophagus) joins the stomach, called gastroesophageal junction (GEJ) cancer. Most people with this type of cancer have a protein called Claudin 18.2 in their tumor. Zolbetuximab is thought to work by attaching to the Claudin 18.2 protein in their tumor, which switches on the body's immune system to attack the tumor. There is an unmet medical need to treat people with advanced stomach cancer or GEJ cancer. This study will give more information about how well zolbetuximab works when given with chemotherapy in adults with advanced stomach cancer or GEJ cancer. In this study, adults with advanced stomach cancer or GEJ cancer will either be given zolbetuximab with chemotherapy or a placebo with chemotherapy. A placebo looks like zolbetuximab but doesn't have any medicine in it. Zolbetuximab with chemotherapy has already been approved to treat gastric cancer and GEJ cancer in some countries. This study is being done in countries where zolbetuximab has not yet been approved for use. If zolbetuximab becomes approved for use in those countries taking part in this study, the study doctor will switch study treatment in those countries to the licensed zolbetuximab. If this happens, people taking part in those countries will leave this study and receive licensed zolbetuximab.

The main aim of the study is to check if zolbetuximab and chemotherapy can prevent or delay the worsening of people's gastric cancer and GEJ cancer compared to placebo and chemotherapy.

Adults with advanced stomach cancer or GEJ cancer can take part. Locally advanced means the cancer has spread to nearby tissue. Unresectable means the cancer cannot be removed by surgery. Metastatic means the cancer has spread to other parts of the body. A tumor sample of their cancer will also have the Claudin 18.2 protein. They may have been previously treated with certain standard therapies, but have not been treated with chemotherapy for their cancer. People cannot take part if they need to take medicines to suppress their immune system, have blockages or bleeding in their gut, have specific uncontrollable cancers such as symptomatic or untreated cancers in the nervous system, or have a specific heart condition, or infections.

The study treatments are either zolbetuximab with chemotherapy, or placebo with chemotherapy. People who take part will receive just 1 of the study treatments by chance. Study treatment will be double-blinded. That means that the people in the study and the study doctors will not know who takes which of the study treatments. Study treatment will be given in cycles. The study treatment is given to people slowly through a tube into a vein. This is called an infusion. People will have 4 infusions in 6-week (42-day) cycles as follows:

* Zolbetuximab or placebo - 2 infusions in a cycle.
* Chemotherapy (called modified FOLFOX6 or mFOLFOX6) - 3 infusions in a cycle. The first infusion is combined with zolbetuximab or placebo on day 1 of each cycle. People may receive zolbetuximab or placebo until their cancer worsens, they cannot tolerate the study treatment, or they need to start another cancer treatment. People will receive mFOLFOX6 for up to 6 months (4 study treatment cycles). After the 6 months people may receive chemotherapy containing folinic acid and fluorouracil instead of mFOLFOX6. People may receive folinic acid and fluorouracil chemotherapy for more than 6 months, or until their cancer worsens, they cannot tolerate the study treatment, or they need to start another cancer treatment. People will visit the clinic on certain days during their study treatment. The study doctors will check if people had any medical problems from taking zolbetuximab or the other study treatments. Also, people in the study will have health checks. On some visits they will have scans to check for any changes in their cancer. People will have the option of giving a tumor sample after their study treatment has finished. People will visit the clinic after they stop their study treatment. People who start treatment with licensed zolbetuximab or mFOLFOX6 outside of this study will not need to visit the clinic. People will be asked about any medical problems and will have a health check. People will visit the clinic at 1 month after they stop their study treatment. People will continue to have scans every 9 or 12 weeks to check for any changes in their cancer. People will have telephone health checks every 3 months. The number of visits and checks done at each visit will depend on the health of each person and whether they completed their study treatment or not.

DETAILED DESCRIPTION:
After the marketing approval in Japan on 26 Mar 2024, this study continued as "post marketing clinical study" in Japan. In the rest of the countries which participated in this study, this study continued as clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Female subject eligible to participate if she is not pregnant (negative serum pregnancy test at screening; female subjects with elevated serum beta human chorionic gonadotropin and a demonstrated non-pregnant status through additional testing are eligible) and at least one of the following conditions applies:

  * Not a woman of child-bearing potential (WOCBP) OR
  * WOCBP who agrees to follow the contraceptive guidance throughout the treatment period and for at least 9 months after the final administration of oxaliplatin and 6 months after the final administration of all other study drugs
* Female subject must agree not to breastfeed starting at screening and throughout the study period, and for 6 months after the final study drug administration.
* Female subject must not donate ova starting at screening and throughout the study period, and for 9 months after the final administration of oxaliplatin and 6 months after the final administration of all other study drugs.
* A sexually active male subject with a female partner(s) who is of child-bearing potential must agree to use contraception during the treatment period and for at least 6 months after the final study drug administration.
* Male subject must agree not to donate sperm starting at screening and throughout the study period, and for 6 months after the final study drug administration.
* Male subject with a pregnant or breastfeeding partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy or time partner is breastfeeding throughout the study period and for 6 months after the final study drug administration.
* Subject has histologically confirmed diagnosis of Gastric or GEJ adenocarcinoma.
* Subject has radiologically confirmed locally advanced unresectable or metastatic disease within 28 days prior to randomization.
* Subject has radiologically evaluable disease (measurable and/or non-measurable disease according to RECIST 1.1), per local assessment, ≤ 28 days prior to randomization. For subjects with only 1 evaluable lesion and prior radiotherapy ≤ 3 months before randomization, the lesion must either be outside the field of prior radiotherapy or have documented progression following radiation therapy.
* Subject's tumor expresses CLDN18.2 in ≥ 75% of tumor cells demonstrating moderate to strong membranous staining as determined by central immunohistochemistry (IHC) testing.
* Subject has a HER2-Negative tumor as determined by local or central testing on a gastric or GEJ tumor specimen. (Unique to China: Subject has a known HER2-negative gastric or GEJ tumor.)
* Subject has ECOG performance status 0 to 1.
* Subject has predicted life expectancy ≥ 12 weeks.
* Subject must meet all of the following criteria based on the centrally or locally analyzed laboratory tests collected within 14 days prior to randomization. In the case of multiple sample collections within this period, the most recent sample collection with available results should be used to determine eligibility.

  * Hemoglobin (Hgb) ≥ 9 g/dL. Subjects requiring transfusions are eligible if they have a post-transfusion Hgb ≥ 9 g/dL.
  * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
  * Platelets ≥ 100 x 10^9/L
  * Albumin ≥ 2.5 g/dL
  * Total bilirubin ≤ 1.5 x upper limit of normal (ULN) without liver metastases (or < 3.0 x ULN if liver metastases are present)
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN without liver metastases (or ≤ 5 x ULN if liver metastases are present)
  * Estimated creatinine clearance ≥ 30 mL/min
  * Prothrombin time (PT)/international normalized ratio (INR) and partial thromboplastin time (PTT) ≤ 1.5 x ULN (except for subjects receiving anticoagulation therapy)

Exclusion Criteria:

* Subject has received prior systemic chemotherapy for locally advanced unresectable or metastatic gastric or GEJ adenocarcinoma. However, subject may have received either neo-adjuvant or adjuvant chemotherapy, immunotherapy or other systemic anticancer therapies, as long as it was completed at least 6 months prior to randomization. Subject may have received treatment with herbal medications that have known antitumor activity > 28 days prior to randomization.
* Subject has received radiotherapy for locally advanced unresectable or metastatic gastric or GEJ adenocarcinoma ≤ 14 days prior to randomization and has not recovered from any related toxicity.
* Subject has received systemic immunosuppressive therapy, including systemic corticosteroids within 14 days prior to randomization. Subjects using a physiologic replacement dose of hydrocortisone or its equivalent (defined as up to 30 mg per day of hydrocortisone or up to 10 mg per day of prednisone), receiving a single dose of systemic corticosteroids or receiving systemic corticosteroids as premedication for radiologic imaging contrast use are allowed.
* Subject has received other investigational agents or devices within 28 days prior to randomization.
* Subject has prior severe allergic reaction or intolerance to known ingredients of zolbetuximab or other monoclonal antibodies, including humanized or chimeric antibodies.
* Subject has known immediate or delayed hypersensitivity, intolerance or contraindication to any component of study treatment.
* Subject has prior severe allergic reaction or intolerance to any component of mFOLFOX6.
* Subject has known dihydropyrimidine dehydrogenase deficiency.
* Subject has a complete gastric outlet syndrome or a partial gastric outlet syndrome with persistent/recurrent vomiting.
* Subject has significant gastric bleeding and/or untreated gastric ulcers that would exclude the subject from participation.
* Subject has a known history of a positive test for human immunodeficiency virus (HIV) infection or known active hepatitis B (positive hepatitis B surface antigen (HBs Ag)) or C infection. NOTE: Screening for these infections should be conducted per local requirements.

  * For subjects who are negative for HBs Ag, but hepatitis B core antibody (HBc Ab) positive, an HB deoxyribonucleic acid (DNA) test will be performed and if positive, the subject will be excluded.
  * Subjects with positive hepatitis C virus (HCV) serology, but negative HCV ribonucleic acid (RNA) test are eligible.
  * Subjects treated for HCV with undetectable viral load results are eligible.
* Subject has an active autoimmune disease that has required systemic treatment within the past 3 months prior to randomization.
* Subject has active infection requiring systemic therapy that has not completely resolved within 7 days prior to randomization.
* Subject has significant cardiovascular disease, including any of the following:

  * Congestive heart failure (defined as New York Heart Association Class III or IV), myocardial infarction, unstable angina, coronary angioplasty, stenting, coronary artery bypass graft, cerebrovascular accident (CVA) or hypertensive crisis within 6 months prior to randomization.
  * History of clinically significant ventricular arrhythmias (i.e., sustained ventricular tachycardia, ventricular fibrillation or Torsades de Pointes)
  * QTc interval > 450 msec for male subjects; QTc interval > 470 msec for female subjects
  * History or family history of congenital long QT syndrome
  * Cardiac arrhythmias requiring anti-arrhythmic medications (Subject with rate controlled atrial fibrillation for > 1 month prior to randomization are eligible).
* Subject has a history of central nervous system metastases and/or carcinomatous meningitis from gastric/GEJ cancer.
* Subject has known peripheral sensory neuropathy > Grade 1 unless the absence of deep tendon reflexes is the sole neurological abnormality.
* Subject has had a major surgical procedure ≤ 28 days prior to randomization.

  * Subject is without complete recovery from a major surgical procedure ≤ 14 days prior to randomization.
* Subject has psychiatric illness or social situations that would preclude study compliance.
* Subject has another malignancy for which treatment is required.
* Subject has any concurrent disease, infection or comorbid condition that interferes with the ability of the subject to participate in the study, which places the subject at undue risk or complicates the interpretation of data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 565 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2026-03-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Global Medical Lead, Study Director — Astellas Pharma Global Development, Inc.
Locations (220):
- United States (51):
  - University of Arizona, Phoenix, Arizona
  - The University of Arizona Medical Center, Tucson, Arizona
  - CBCC Global Research, Inc. at Comprehensive Blood and Cancer, Bakersfield, California
  - City of Hope Nat'l Medical Center, Duarte, California
  - St. Jude Hospital Yorba Linda, Fullerton, California
  - Pacific Shores Medical Group, Huntington Beach, California
  - Loma Linda University, Loma Linda, California
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - University of California Davis, Sacramento, California
  - University of California - San Francisco, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Memorial Sloan Kettering Cancer Center, Middletown, Connecticut
  - Memorial Cancer Institute - West, Hollywood, Florida
  - University of Miami, Miami, Florida
  - Orlando Health Inc, Orlando, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Cancer Treatment Centers of America, Atlanta, Newnan, Georgia
  - Northwestern University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
  - University of Maryland Medical Center(UMMC)Transplant Center, Baltimore, Maryland
  - Maryland Oncology Hematology, Brandywine, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Health Partners Institute, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Memorial Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center, Montvale, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, Commack, New York
  - Memorial Sloan Kettering Cancer Center, Harrison, New York
  - Mount Sinai School of Medicine, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Memorial Sloan Kettering Cancer Center, Uniondale, New York
  - The Ohio State University Medical Center, Columbus, Ohio
  - Precision Cancer Research -Dayton Physicians Network, Middletown, Ohio
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - Earle A. Chiles Research Institute, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Cancer Treatment Centers of America, Philadelphia, Philadelphia, Pennsylvania
  - Rhode Island Hospital-Lifespan Cancer Institute, Providence, Rhode Island
  - Sanford Cancer Center, Sioux Falls, South Dakota
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Inova Dwight and Martha Schar Cancer Institute, Fairfax, Virginia
  - MultiCare Regional Cancer Center - Gig Harbor, Auburn, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (5):
  - Site AU61002, Douglas, Queensland
  - Site AU61011, Tugun, Queensland
  - Site AU61008, Adelaide, South Australia
  - Site AU61006, East Bentleigh, Victoria
  - Site AU61007, Kogarah
- Belgium (10):
  - Site BE32007, Edegem, Antwerpen
  - Site BE32001, Brussels, Bruxelles-Capitale, Région de
  - Site BE32008, Mons, Hainaut
  - Site BE32002, Brussels, Liege
  - Site BE32012, Ghent, Oost-Vlaanderen
  - Site BE32006, Leuven, Vlaams Brabant
  - Site BE32005, Bruges
  - Site BE32004, Brussels
  - Site BE32011, Charleroi
  - Site BE32010, Haine-Saint-Paul
- Brazil (12):
  - Site BR55010, Brasília, Federal District
  - Site BR55006, Lajeado, Rio Grande do Sul
  - Site BR55002, Itajaí, Santa Catarina
  - Site BR55007, Barretos, São Paulo
  - Site BR55003, Santo André, São Paulo
  - Site BR55005, São José do Rio Preto, São Paulo
  - Site BR55017, Belo Horizonte
  - Site BR55016, Passo Fundo
  - Site BR55015, Rio de Janeiro
  - Site BR55018, Santa Catarina
  - Site BR55009, São Paulo
  - Site BR55004, São Paulo
- Canada (5):
  - Site CA15005, Edmonton, Alberta
  - Site CA15009, Saint John, New Brunswick
  - Site CA15011, Toronto, Ontario
  - Site CA15002, Montreal, Quebec
  - Site CA15008, Montreal, Quebec
- Chile (4):
  - Site CL56003, Providencia, Santiago Metropolitan
  - Site CL56008, Providencia
  - Site CL56005, Santiago
  - Site CL56007, Valdivia
- China (8):
  - Site CN86003, Haerbin, Heilongjiang
  - Site CN86006, Nanjing, Jiangsu
  - Site CN86004, Hangzhou, Zhejiang
  - Site CN86009, Beijing
  - Site CN86002, Beijing
  - Site CN86005, Hefei
  - Site CN86001, Xiamen
  - Site CN86008, Zhengzhou
- Colombia (6):
  - Site CO57006, Medellín, Antioquia
  - Site CO57009, Bogotá, DC
  - Site CO57007, Montería, Departamento de Córdoba
  - Site CO57005, Cali, Valle del Cauca Department
  - Site CO57001, Cali
  - Site CO57002, Medellín
- France (13):
  - Site FR33009, Dijon, Bourgogne-Franche-Comté
  - Site FR33010, Brest, Brittany Region
  - Site FR33001, Rennes, Brittany Region
  - Site FR33008, Besançon, Franche-Comte
  - Site FR33011, Montpellier, Languedoc-Roussillon
  - Site FR33002, Paris, Paris
  - Site FR33101, Saint-Herblain, Pays de la Loire Region
  - Site FR33005, Nice, Provence-Alpes-Côte d'Azur Region
  - Site FR33003, Lyon, Rhone
  - Site FR33006, Poitiers, Vienne
  - Site FR33103, Créteil
  - Site FR33007, Nice
  - Site FR33104, Saint-Priest-en-Jarez
- Germany (11):
  - Site DE49008, Munich, Bavaria
  - Site DE49007, München, Bavaria
  - Site DE49002, Mainz, Rhineland-Palatinate
  - Site DE49010, Dresden, Saxony
  - Site DE49004, Leipzig, Saxony
  - Site DE49021, Halle, Saxony-Anhalt
  - Site DE49015, Magdeburg, Saxony-Anhalt
  - Site DE49012, Berlin
  - Site DE49011, Berlin
  - Site DE49018, Dresden
  - Site DE49019, Heilbronn
- Israel (6):
  - Site IL97206, Kfar Saba, Central District
  - Site IL97210, HaDarom
  - Site IL97201, Haifa
  - Site IL97209, Holon
  - Site IL97202, Jerusalem
  - Site IL97203, Tel Aviv
- Italy (18):
  - Site IT39011, Meldola, Forli
  - Site IT39020, Monza, Lombardy
  - Site IT39023, Vicenza, VI
  - Site IT39013, Ancona
  - Site IT39004, Bergamo
  - Site IT39009, Cremona
  - Site IT39006, Milan
  - Site IT39008, Milan
  - Site IT39021, Modena
  - Site IT39016, Padua
  - Site IT39012, Parma
  - Site IT39018, Perugia
  - Site IT39003, Piacenza
  - Site IT39019, Pisa
  - Site IT39022, Reggio Emilia
  - Site IT39015, Roma
  - Site IT39026, Terni
  - Site IT39024, Turin to
- Japan (15):
  - Site JP81009, Nagoya, Aichi-ken
  - Site JP81003, Kashiwa, Chiba
  - Site JP81002, Matsuyama, Ehime
  - Site JP81007, Sapporo, Hokkaido
  - Site JP81014, Kobe, Hyōgo
  - Site JP81001, Suita, Osaka
  - Site JP81015, Hidaka, Saitama
  - Site JP81010, Kitaadachi-gun, Saitama
  - Site JP81012, Sunto-gun, Shizuoka
  - Site JP81013, Bunkyo-ku, Tokyo
  - Site JP81006, Chuo-ku, Tokyo
  - Site JP81008, Koto-ku, Tokyo
  - Site JP81005, Fukuoka
  - Site JP81004, Osaka
  - Site JP81011, Osaka
- Mexico (8):
  - Site MX52002, Mexico City, Mexico City
  - Site MX52007, Mexico City, Mexico City
  - Site MX52010, Veracruz, Ver, Veracruz
  - Site MX52001, Aguascalientes
  - Site MX52003, Distrito Federal
  - Site MX52009, Jalisco
  - Site MX52004, Oaxaca City
  - Site MX52008, San Luis de Potosi
- Peru (5):
  - Site PE51004, San Isidro, Lima region
  - Site PE51003, Arequipa
  - Site PE51005, Lima
  - Site PE51006, Lima
  - Site PE51001, Lima
- Poland (5):
  - Site PL48004, Lublin, Lubusz Voivodeship
  - Site PL48007, Ostrołęka, Masovian Voivodeship
  - Site PL48005, Wieliszew, Masovian Voivodeship
  - Site PL48002, Brzozów, Podkarpackie Voivodeship
  - Site PL48009, Warsaw
- South Korea (8):
  - Site KR82002, Seongnam-si, Gyeonggi-do
  - Site KR82009, Suwon, Gyeonggido [Kyonggi-do]
  - Site KR82004, Seoul, Seoul Teugbyeolsi
  - Site KR82008, Incheon
  - Site KR82003, Seoul
  - Site KR82005, Seoul
  - Site KR82007, Seoul
  - Site KR82006, Seoul
- Spain (13):
  - Site ES34013, Badalona, Barcelona
  - Site ES34010, Ávila, Castille and León
  - Site ES34011, Alcorcón, Madrid
  - Site ES34005, Barcelona
  - Site ES34016, Barcelona
  - Site ES34015, Barcelona
  - Site ES34019, Burgos
  - Site ES34008, Madrid
  - Site ES34017, Madrid
  - Site ES34004, Madrid
  - Site ES34003, Murcia
  - Site ES34018, Seville
  - Site ES34006, Zaragoza
- Taiwan (7):
  - Site TW88605, Kwei-Shan, Taoyuan
  - Site TW88608, Kaohsiung City
  - Site TW88604, Kaohsiung City
  - Site TW88603, Taichung
  - Site TW88607, Tainan
  - Site TW88606, Taipei
  - Site TW88601, Taipei
- United Kingdom (10):
  - Site GB44003, Aberdeen, Aberdeenshire
  - Site GB44101, London, London, City of
  - Site GB44102, Sutton, Surrey
  - Site GB44103, Cambridge
  - Site GB44009, Coventry
  - Site GB44104, Dundee
  - Site GB44008, Leeds
  - Site GB44002, London
  - Site GB44004, London
  - Site GB44001, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Shitara K, Shah MA, Lordick F, Bang YJ, Ilson D, Van Cutsem E, Enzinger P, Kim SS, Klempner SJ, Moran D, Park JW, Bhattacharya P, Ajani JA, Xu RH. Zolbetuximab plus chemotherapy for locally advanced unresectable or metastatic stomach or gastroesophageal junction cancers: a plain language summary. Future Oncol. 2024;20(26):1861-1877. doi: 10.1080/14796694.2024.2342107. Epub 2024 May 24. PMID 38861294
- [Derived] Shitara K, Lordick F, Bang YJ, Enzinger P, Ilson D, Shah MA, Van Cutsem E, Xu RH, Aprile G, Xu J, Chao J, Pazo-Cid R, Kang YK, Yang J, Moran D, Bhattacharya P, Arozullah A, Park JW, Oh M, Ajani JA. Zolbetuximab plus mFOLFOX6 in patients with CLDN18.2-positive, HER2-negative, untreated, locally advanced unresectable or metastatic gastric or gastro-oesophageal junction adenocarcinoma (SPOTLIGHT): a multicentre, randomised, double-blind, phase 3 trial. Lancet. 2023 May 20;401(10389):1655-1668. doi: 10.1016/S0140-6736(23)00620-7. Epub 2023 Apr 15. PMID 37068504

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with claudin (CLDN)18.2-positive, human epidermal growth factor receptor 2 (HER2) -negative locally advanced unresectable or metastatic gastric and gastroesophageal junction (GEJ) adenocarcinoma.
Pre-assignment Details: Participants who met all inclusion criteria and none of the exclusion criteria were enrolled in the study. Randomization was stratified by region (Asia vs Non-Asia), number of organs with metastatic sites (0 to 2 vs ≥ 3) and prior gastrectomy (Yes or No).
Groups:
- mFOLFOX6+ Placebo: Participants received an IV infusion (minimum 2-hour infusion) of placebo matched to zolbetuximab on C1D1, followed by subsequent doses every 3 weeks starting from C1D22 until study treatment discontinuation criteria were met. Participants also received up to 12 treatments of mFOLFOX6 (or components if some were discontinued due to toxicity) over 4 or more cycles. mFOLFOX6 was administered on Days 1, 15, and 29 of each cycle (5-fluorouracil: 400 mg/m^2 IV bolus over 5-15 minutes followed by 2400mg/m^2 over 46-48 hours continuous IV infusion every 2 weeks for 4 cycles. Folinic acid: 400 mg/m^2 IV infusion over 2 hours; oxaliplatin: 85 mg/m^2 IV infusion over 2 hours). A maximum of 12 doses of oxaliplatin was permitted. After mFOLFOX6 treatments, participants could continue to receive 5-FU and folinic acid on Days 1, 15, and 29 of each cycle at the investigator's discretion or until study treatment discontinuation criteria were met. Each cycle was approximately 42 days.
Period: Overall Study
Arm/Group | mFOLFOX6 + Zolbetuximab | mFOLFOX6+ Placebo
Started | 283 | 282
Participants Who Received at Least One Dose of Study Drug | 279 | 278
Completed | 26 | 17
Not Completed | 257 | 265
Not completed — Progressive Disease | 151 | 199
Not completed — Withdrawal by Subject | 29 | 17
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 14 | 16
Not completed — Adverse Event | 40 | 14
Not completed — miscellaneous | 17 | 15
Not completed — Protocol deviation | 1 | 0
Not completed — Participants who did not take the study drug | 4 | 4

BASELINE CHARACTERISTICS:
Population: Full analysis set(FAS) included all participants who were randomized to 1 of the treatment arms.
Groups:
- mFOLFOX6 + Zolbetuximab: Participants received an IV infusion (as a minimum of 2-hour infusion) of zolbetuximab at a loading dose of 800 mg/m^2 on C1D1 followed by subsequent doses of 600 mg/m^2 every 3 weeks starting from C1D22 until participant meets study treatment discontinuation criteria. Participants also received up to 12 treatments of 5-fluorouracil, folinic acid and oxaliplatin (mFOLFOX6) (or components of mFOLFOX6 if some components were discontinued due to toxicity) over 4 or more cycles in which mFOLFOX6 was administered on Days 1, 15 and 29 of each cycle (5-fluorouracil administered by IV bolus 400 mg/m^2 over 5 to 15 minutes followed by 2400mg/m^2 over 46-48 hours continuous IV infusion every 2 weeks for 4 cycles. Folinic acid administered 400 mg/m^2 IV infusion over 2 hours; oxaliplatin administered 85 mg/m^2 IV infusion over 2 hours). A maximum of 12 doses of oxaliplatin was permitted. After mFOLFOX6 treatments, participants could continue to receive 5-FU and folinic acid on Days 1, 15 and 29 of each cycle at the investigator's discretion or until the participant met the study treatment discontinuation criteria. Each cycle was approximately 42 days.
- mFOLFOX6+Placebo: Participants received an IV infusion (minimum 2-hour infusion) of placebo matched to zolbetuximab on C1D1, followed by subsequent doses every 3 weeks starting from C1D22 until study treatment discontinuation criteria were met. Participants also received up to 12 treatments of mFOLFOX6 (or components if some were discontinued due to toxicity) over 4 or more cycles. mFOLFOX6 was administered on Days 1, 15, and 29 of each cycle (5-fluorouracil: 400 mg/m^2 IV bolus over 5-15 minutes followed by 2400mg/m^2 over 46-48 hours continuous IV infusion every 2 weeks for 4 cycles. Folinic acid: 400 mg/m^2 IV infusion over 2 hours; oxaliplatin: 85 mg/m^2 IV infusion over 2 hours). A maximum of 12 doses of oxaliplatin was permitted. After mFOLFOX6 treatments, participants could continue to receive 5-FU and folinic acid on Days 1, 15, and 29 of each cycle at the investigator's discretion or until study treatment discontinuation criteria were met. Each cycle was approximately 42 days.
- Total: Total of all reporting groups
Arm/Group | mFOLFOX6 + Zolbetuximab | mFOLFOX6+Placebo | Total
Number analyzed (Participants) | 283 | 282 | 565
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.7 (11.7) | 58.8 (13.0) | 59.3 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 107 | 214
  Male | 176 | 175 | 351
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 37 | 73
  Not Hispanic or Latino | 225 | 213 | 438
  Unknown or Not Reported | 22 | 32 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 8 | 17
  Asian | 96 | 97 | 193
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 140 | 134 | 274
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 33 | 41 | 74
Region (Asia vs Non-Asia) [Number; unit: Participants]
  Asia | 88 | 89 | 177
  Non- Asia | 195 | 193 | 388
Number of organs with metastatic sites [Number; unit: Participants]
  0-2 metastatic sites | 219 | 219 | 438
  >=3 metastatic sites | 64 | 63 | 127
Prior Gastrectomy [Number; unit: Participants]
  YES | 84 | 82 | 166
  NO | 199 | 200 | 399

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of randomization until the date of radiological progressive disease (PD) (per Response Evaluation Criteria in Solid Tumors [RECIST] 1.1 by independent review committee [IRC]) or death from any cause, whichever was earliest. PD was defined as development of new, or progression of existing metastases to the primary cancer under the study. Kaplan -Meier (KM) estimates was used.
Time Frame: From date of randomization until the date of first documented radiological progression or date of death from any cause, whichever occurred first (up to 62 months and 18 days)
Population: FAS
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | mFOLFOX6 + Zolbetuximab | mFOLFOX6+ Placebo
Number analyzed (Participants) | 283 | 282
Months | 11.04 [9.69 to 12.52] | 8.94 [8.21 to 10.41]
Statistical Analysis 1: Comparison: mFOLFOX6 + Zolbetuximab vs mFOLFOX6+ Placebo; Test type: Superiority; p = 0.0024, Log Rank — Log-rank test stratified by: * Region (Asia vs Non-Asia) * Number of organs with metastatic sites (0 to 2 vs ≥ 3) * Prior gastrectomy (Yes or No); Hazard Ratio (HR) = 0.734, 95% CI 2-sided [0.591 to 0.910]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization until the date of death from any cause. Kaplan-Meier estimates was used.
Time Frame: From the date of randomization until 62 months and 18 days
Population: FAS
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | mFOLFOX6 + Zolbetuximab | mFOLFOX6+ Placebo
Number analyzed (Participants) | 283 | 282
Months | 18.23 [16.13 to 20.63] | 15.57 [13.67 to 16.92]
Statistical Analysis 1: Comparison: mFOLFOX6 + Zolbetuximab vs mFOLFOX6+ Placebo; Test type: Superiority; p = 0.0075, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.784, 95% CI 2-sided [0.644 to 0.954]

3. Secondary Outcome: Time to Confirmed Deterioration (TTCD) Using Physical Functioning (PF) as Measured by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core Questionnaire (EORTC QLQ-C30)
Description: TTCD: time from randomization to first clinically meaning full deterioration (CMD) that was confirmed at next scheduled visit. EORTC-QLQ-C30 was a 30-item cancer-specific instrument consisting of 5 functional scales (physical,role,emotional,social & cognitive), 9 symptom scales (fatigue, nausea/vomiting,general pain,dyspnea,insomnia,appetite loss,constipation,diarrhea,financial difficulties) & global health status scale. Most items were scored 1(not at all) to 4(very much) except for items contributing to global health status/QoL, which were scored 1(very poor) to 7(excellent). All raw domain scores were linearly transformed to 0-100scale with higher scores on symptoms indicate worse health state. CMD was defined if a participant's change from baseline exceeded a pre-specified threshold of -13. This was derived from an Exit Survey conducted using Patient Global Impression of Severity/Change(PGIS/PGIC) questionnaires as an anchor for estimating meaningful change. KM estimates was used.
Time Frame: From the date of randomization until 62 months and 18 days
Population: FAS
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | mFOLFOX6 + Zolbetuximab | mFOLFOX6+ Placebo
Number analyzed (Participants) | 283 | 282
Months | 9.89 [6.01 to NA] — Data was not estimable because less than 50% of participants had event (data was estimated using KM and it requires at least 50% of event to be able to calculate time using KM. | 12.32 [9.26 to NA] — Data was not estimable because less than 50% of participants had event (data was estimated using KM and it requires at least 50% of event to be able to calculate time using KM.
Statistical Analysis 1: Comparison: mFOLFOX6 + Zolbetuximab vs mFOLFOX6+ Placebo; Test type: Superiority; p = 0.0280, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.295, 95% CI 2-sided [0.994 to 1.687]

4. Secondary Outcome: Time to Confirmed Deterioration (TTCD) Using Oesophago-gastric Questionnaire (OG25) on Abdominal Pain and Discomfort as Measured by EORTC QLQ-OG25
Description: TTCD: time from randomization to first CMD that was confirmed at next scheduled visit. EORTC QLQ-OG25 evaluated gastric and GEJ cancer specific symptoms. A 25 item instrument with 6 scales: dysphagia (3 items), eating restrictions (4 ), reflux (2), odynophagia (2), pain and discomfort (2), anxiety (2), as well as 10 single items: eating in front of others, dry mouth, trouble with taste, body image, trouble swallowing saliva, choked when swallowing, trouble with coughing, trouble talking, weight and hair loss. Items were scored:1: not at all; 2: a little, 3: quite a bit, 4: very much, and were transformed linearly into scores (0 to 100) with higher scores indicating worse symptoms. CMD was defined if a participant's change from baseline exceeded a pre-specified threshold of 16.67. This was derived from an Exit Survey conducted to use PGIS/PGIC questionnaires as an anchor for estimating the meaningful change. KM estimates was used.
Time Frame: From the date of randomization until 62 months and 18 days
Population: FAS
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | mFOLFOX6 + Zolbetuximab | mFOLFOX6+ Placebo
Number analyzed (Participants) | 283 | 282
Months | NA [NA to NA] — Data was not estimable because less than 50% of participants had event (data was estimated using KM and it requires at least 50% of event to be able to calculate time using KM ) | NA [15.67 to NA] — Data was not estimable because less than 50% of participants had event (data was estimated using KM and it requires at least 50% of event to be able to calculate time using KM )
Statistical Analysis 1: Comparison: mFOLFOX6 + Zolbetuximab vs mFOLFOX6+ Placebo; Test type: Superiority; p = 0.0508, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.713, 95% CI 2-sided [0.475 to 1.071]

5. Secondary Outcome: Time to Confirmed Deterioration (TTCD) Using Global Health Status as Measured by EORTC QLQ-C30
Description: TTCD: time from randomization to first CMD that was confirmed at the next scheduled visit. The EORTC-QLQ-C30 was a 30-item cancer-specific instrument consisting of 5 functional scales (physical, role, emotional, social and cognitive), 9 symptom scales/items (fatigue, nausea/vomiting, general pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties) and a global health status scale. Most items were scored 1 ("not at all") to 4 ("very much") except for the items contributing to the global health status/QoL, which were scored 1 ("very poor") to 7 ("excellent"). All raw domain scores were linearly transformed to a 0-100 scale with higher scores on symptoms indicate a worse health state. CMD was defined if a participant's change from baseline exceeded a pre-specified threshold of -10. This was derived from an Exit Survey conducted to use PGIS/PGIC questionnaires as an anchor for estimating the meaningful change. KM estimates was used.
Time Frame: From the date of randomization until 62 months and 18 days
Population: FAS
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | mFOLFOX6 + Zolbetuximab | mFOLFOX6+ Placebo
Number analyzed (Participants) | 283 | 282
Months | 15.44 [7.06 to 23.89] | 11.83 [9.23 to 15.08]
Statistical Analysis 1: Comparison: mFOLFOX6 + Zolbetuximab vs mFOLFOX6+ Placebo; Test type: Superiority; p = 0.1685, Log Rank; Hazard Ratio (HR) = 1.142, 95% CI 2-sided [0.874 to 1.492] — Log-rank test stratified by: * Region (Asia vs Non-Asia) * Number of organs with metastatic sites (0 to 2 vs ≥ 3) * Prior gastrectomy (Yes or No)

6. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants who had best overall response (BOR) of complete response (CR) or partial response (PR) as was assessed by IRC per RECIST 1.1. CR was defined as complete resolution of all attributable clinical symptoms and physical findings. PR was defined as partial resolution of at Least some of the clinical symptoms and physical findings.
Time Frame: From the date of randomization until 62 months and 18 days
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | mFOLFOX6 + Zolbetuximab | mFOLFOX6+ Placebo
Number analyzed (Participants) | 283 | 282
Percentage of participants | 48.1 [42.11 to 54.05] | 47.5 [41.56 to 53.52]
Statistical Analysis 1: Comparison: mFOLFOX6 + Zolbetuximab vs mFOLFOX6+ Placebo; Test type: Superiority; p = 0.4536, Cochran-Mantel-Haenszel; Based on 1-sided Cochran-Mantel-Haenszel (CMH) test. Stratification factors were Region, Number of Metastatic Sites and Prior Gastrectomy

7. Secondary Outcome: Duration Of Response (DOR)
Description: DOR was defined as the time from the date of the first response (CR/PR) until the date of PD as assessed by IRC per RECIST 1.1 or date of death from any cause, whichever is earliest.CR was defined as complete resolution of all attributable clinical symptoms and physical findings. PR was defined as partial resolution of at Least some of the clinical symptoms and physical findings.PD was defined as development of new, or progression of existing metastases to the primary cancer under the sudy.
Time Frame: From date of first response (CR/PR) until 62 months and 18 day
Population: FAS - All Objective Responders
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | mFOLFOX6 + Zolbetuximab | mFOLFOX6+ Placebo
Number analyzed (Participants) | 136 | 134
Months | 9.00 [7.49 to 10.38] | 8.11 [6.47 to 11.37]
Statistical Analysis 1: Comparison: mFOLFOX6 + Zolbetuximab vs mFOLFOX6+ Placebo; Test type: Superiority; p = 0.0721, Log Rank; Hazard Ratio (HR) = 0.789, 95% CI 2-sided [0.573 to 1.087] — [estimate comment as in outcome 5, analysis 1]

8. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An Adverse event (AE) is any untoward medical occurrence in a participant administered a study drug, and which does not have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease (new or exacerbated) temporally associated with the use of a medicinal product, whether or notconsidered related to the medicinal product. TEAE defined as an AE observed after starting administration of the study drug through 30 days after the last dose.
Time Frame: From first dose until 62 months and 18 days
Population: Safety analysis set (SAF) included all participants who received at least 1 dose of any study drug (zolbetuximab/placebo and mFOLFOX6).
Measure: Number; unit: Participants
Arm/Group | mFOLFOX6 + Zolbetuximab | mFOLFOX6+ Placebo
Number analyzed (Participants) | 279 | 278
Participants | 278 | 277

9. Secondary Outcome: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: ECOG grades 0-5, where 0 = Fully active, able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2 = Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours; 3 = Capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4 = Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair and 5 = Dead.
Time Frame: Baseline, cycle (C) 1 day (D) 22, D1 and D22 of C2 through C39
Population: FAS with available data was analyzed.
Measure: Number; unit: Participants
Arm/Group | mFOLFOX6 + Zolbetuximab | mFOLFOX6+ Placebo
Number analyzed (Participants) | 279 | 278
Participants
  Baseline Score 0 | 125 | 115
  Baseline Score 1 | 153 | 163
  Baseline Score 2 | 1 | 0
  Baseline Score 3 | 0 | 0
  Baseline Score 4 | 0 | 0
  Baseline Score 5 | 0 | 0
  C1D22 Score 0: number analyzed (Participants) | 209 | 238
  C1D22 Score 0 | 83 | 102
  C1D22 Score 1: number analyzed (Participants) | 209 | 238
  C1D22 Score 1 | 116 | 133
  C1D22 Score 2: number analyzed (Participants) | 209 | 238
  C1D22 Score 2 | 8 | 3
  C1D22 Score 3: number analyzed (Participants) | 209 | 238
  C1D22 Score 3 | 2 | 0
  C1D22 Score 4: number analyzed (Participants) | 209 | 238
  C1D22 Score 4 | 0 | 0
  C1D22 Score 5: number analyzed (Participants) | 209 | 238
  C1D22 Score 5 | 0 | 0
  C2D1 Score 0: number analyzed (Participants) | 239 | 262
  C2D1 Score 0 | 103 | 112
  C2D1 Score 1: number analyzed (Participants) | 239 | 262
  C2D1 Score 1 | 127 | 144
  C2D1 Score 2: number analyzed (Participants) | 239 | 262
  C2D1 Score 2 | 8 | 6
  C2D1 Score 3: number analyzed (Participants) | 239 | 262
  C2D1 Score 3 | 1 | 0
  C2D1 Score 4: number analyzed (Participants) | 239 | 262
  C2D1 Score 4 | 0 | 0
  C2D1 Score 5: number analyzed (Participants) | 239 | 262
  C2D1 Score 5 | 0 | 0
  C2D22 Score 0: number analyzed (Participants) | 179 | 201
  C2D22 Score 0 | 64 | 78
  C2D22 Score 1: number analyzed (Participants) | 179 | 201
  C2D22 Score 1 | 113 | 123
  C2D22 Score 2: number analyzed (Participants) | 179 | 201
  C2D22 Score 2 | 2 | 0
  C2D22 Score 3: number analyzed (Participants) | 179 | 201
  C2D22 Score 3 | 0 | 0
  C2D22 Score 4: number analyzed (Participants) | 179 | 201
  C2D22 Score 4 | 0 | 0
  C2D22 Score 5: number analyzed (Participants) | 179 | 201
  C2D22 Score 5 | 0 | 0
  C3D1 Score 0: number analyzed (Participants) | 222 | 226
  C3D1 Score 0 | 94 | 91
  C3D1 Score 1: number analyzed (Participants) | 222 | 226
  C3D1 Score 1 | 118 | 132
  C3D1 Score 2: number analyzed (Participants) | 222 | 226
  C3D1 Score 2 | 10 | 3
  C3D1 Score 3: number analyzed (Participants) | 222 | 226
  C3D1 Score 3 | 0 | 0
  C3D1 Score 4: number analyzed (Participants) | 222 | 226
  C3D1 Score 4 | 0 | 0
  C3D1 Score 5: number analyzed (Participants) | 222 | 226
  C3D1 Score 5 | 0 | 0
  C3D22 Score 0: number analyzed (Participants) | 179 | 172
  C3D22 Score 0 | 78 | 65
  C3D22 Score 1: number analyzed (Participants) | 179 | 172
  C3D22 Score 1 | 97 | 104
  C3D22 Score 2: number analyzed (Participants) | 179 | 172
  C3D22 Score 2 | 4 | 3
  C3D22 Score 3: number analyzed (Participants) | 179 | 172
  C3D22 Score 3 | 0 | 0
  C3D22 Score 4: number analyzed (Participants) | 179 | 172
  C3D22 Score 4 | 0 | 0
  C3D22 Score 5: number analyzed (Participants) | 179 | 172
  C3D22 Score 5 | 0 | 0
  C4D1 Score 0: number analyzed (Participants) | 201 | 199
  C4D1 Score 0 | 78 | 79
  C4D1 Score 1: number analyzed (Participants) | 201 | 199
  C4D1 Score 1 | 118 | 115
  C4D1 Score 2: number analyzed (Participants) | 201 | 199
  C4D1 Score 2 | 5 | 5
  C4D1 Score 3: number analyzed (Participants) | 201 | 199
  C4D1 Score 3 | 0 | 0
  C4D1 Score 4: number analyzed (Participants) | 201 | 199
  C4D1 Score 4 | 0 | 0
  C4D1 Score 5: number analyzed (Participants) | 201 | 199
  C4D1 Score 5 | 0 | 0
  C4D22 Score 0: number analyzed (Participants) | 139 | 147
  C4D22 Score 0 | 49 | 54
  C4D22 Score 1: number analyzed (Participants) | 139 | 147
  C4D22 Score 1 | 84 | 89
  C4D22 Score 2: number analyzed (Participants) | 139 | 147
  C4D22 Score 2 | 6 | 3
  C4D22 Score 3: number analyzed (Participants) | 139 | 147
  C4D22 Score 3 | 0 | 1
  C4D22 Score 4: number analyzed (Participants) | 139 | 147
  C4D22 Score 4 | 0 | 0
  C4D22 Score 5: number analyzed (Participants) | 139 | 147
  C4D22 Score 5 | 0 | 0
  C5D1 Score 0: number analyzed (Participants) | 179 | 173
  C5D1 Score 0 | 70 | 70
  C5D1 Score 1: number analyzed (Participants) | 179 | 173
  C5D1 Score 1 | 101 | 101
  C5D1 Score 2: number analyzed (Participants) | 179 | 173
  C5D1 Score 2 | 8 | 1
  C5D1 Score 3: number analyzed (Participants) | 179 | 173
  C5D1 Score 3 | 0 | 1
  C5D1 Score 4: number analyzed (Participants) | 179 | 173
  C5D1 Score 4 | 0 | 0
  C5D1 Score 5: number analyzed (Participants) | 179 | 173
  C5D1 Score 5 | 0 | 0
  C5D22 Score 0: number analyzed (Participants) | 129 | 136
  C5D22 Score 0 | 57 | 53
  C5D22 Score 1: number analyzed (Participants) | 129 | 136
  C5D22 Score 1 | 67 | 82
  C5D22 Score 2: number analyzed (Participants) | 129 | 136
  C5D22 Score 2 | 5 | 1
  C5D22 Score 3: number analyzed (Participants) | 129 | 136
  C5D22 Score 3 | 0 | 0
  C5D22 Score 4: number analyzed (Participants) | 129 | 136
  C5D22 Score 4 | 0 | 0
  C5D22 Score 5: number analyzed (Participants) | 129 | 136
  C5D22 Score 5 | 0 | 0
  C6D1 Score 0: number analyzed (Participants) | 152 | 144
  C6D1 Score 0 | 66 | 57
  C6D1 Score 1: number analyzed (Participants) | 152 | 144
  C6D1 Score 1 | 82 | 84
  C6D1 Score 2: number analyzed (Participants) | 152 | 144
  C6D1 Score 2 | 3 | 3
  C6D1 Score 3: number analyzed (Participants) | 152 | 144
  C6D1 Score 3 | 1 | 0
  C6D1 Score 4: number analyzed (Participants) | 152 | 144
  C6D1 Score 4 | 0 | 0
  C6D1 Score 5: number analyzed (Participants) | 152 | 144
  C6D1 Score 5 | 0 | 0
  C6D22 Score 0: number analyzed (Participants) | 121 | 110
  C6D22 Score 0 | 51 | 50
  C6D22 Score 1: number analyzed (Participants) | 121 | 110
  C6D22 Score 1 | 67 | 59
  C6D22 Score 2: number analyzed (Participants) | 121 | 110
  C6D22 Score 2 | 3 | 1
  C6D22 Score 3: number analyzed (Participants) | 121 | 110
  C6D22 Score 3 | 0 | 0
  C6D22 Score 4: number analyzed (Participants) | 121 | 110
  C6D22 Score 4 | 0 | 0
  C6D22 Score 5: number analyzed (Participants) | 121 | 110
  C6D22 Score 5 | 0 | 0
  C7D1 Score 0: number analyzed (Participants) | 139 | 113
  C7D1 Score 0 | 65 | 55
  C7D1 Score 1: number analyzed (Participants) | 139 | 113
  C7D1 Score 1 | 70 | 58
  C7D1 Score 2: number analyzed (Participants) | 139 | 113
  C7D1 Score 2 | 3 | 0
  C7D1 Score 3: number analyzed (Participants) | 139 | 113
  C7D1 Score 3 | 1 | 0
  C7D1 Score 4: number analyzed (Participants) | 139 | 113
  C7D1 Score 4 | 0 | 0
  C7D1 Score 5: number analyzed (Participants) | 139 | 113
  C7D1 Score 5 | 0 | 0
  C7D22 Score 0: number analyzed (Participants) | 105 | 90
  C7D22 Score 0 | 46 | 45
  C7D22 Score 1: number analyzed (Participants) | 105 | 90
  C7D22 Score 1 | 56 | 45
  C7D22 Score 2: number analyzed (Participants) | 105 | 90
  C7D22 Score 2 | 3 | 0
  C7D22 Score 3: number analyzed (Participants) | 105 | 90
  C7D22 Score 3 | 0 | 0
  C7D22 Score 4: number analyzed (Participants) | 105 | 90
  C7D22 Score 4 | 0 | 0
  C7D22 Score 5: number analyzed (Participants) | 105 | 90
  C7D22 Score 5 | 0 | 0
  C8D1 Score 0: number analyzed (Participants) | 117 | 98
  C8D1 Score 0 | 53 | 52
  C8D1 Score 1: number analyzed (Participants) | 117 | 98
  C8D1 Score 1 | 62 | 46
  C8D1 Score 2: number analyzed (Participants) | 117 | 98
  C8D1 Score 2 | 2 | 0
  C8D1 Score 3: number analyzed (Participants) | 117 | 98
  C8D1 Score 3 | 0 | 0
  C8D1 Score 4: number analyzed (Participants) | 117 | 98
  C8D1 Score 4 | 0 | 0
  C8D1 Score 5: number analyzed (Participants) | 117 | 98
  C8D1 Score 5 | 0 | 0
  C8D22 Score 0: number analyzed (Participants) | 87 | 78
  C8D22 Score 0 | 37 | 43
  C8D22 Score 1: number analyzed (Participants) | 87 | 78
  C8D22 Score 1 | 47 | 35
  C8D22 Score 2: number analyzed (Participants) | 87 | 78
  C8D22 Score 2 | 3 | 0
  C8D22 Score 3: number analyzed (Participants) | 87 | 78
  C8D22 Score 3 | 0 | 0
  C8D22 Score 4: number analyzed (Participants) | 87 | 78
  C8D22 Score 4 | 0 | 0
  C8D22 Score 5: number analyzed (Participants) | 87 | 78
  C8D22 Score 5 | 0 | 0
  C9D1 Score 0: number analyzed (Participants) | 97 | 74
  C9D1 Score 0 | 45 | 40
  C9D1 Score 1: number analyzed (Participants) | 97 | 74
  C9D1 Score 1 | 48 | 34
  C9D1 Score 2: number analyzed (Participants) | 97 | 74
  C9D1 Score 2 | 4 | 0
  C9D1 Score 3: number analyzed (Participants) | 97 | 74
  C9D1 Score 3 | 0 | 0
  C9D1 Score 4: number analyzed (Participants) | 97 | 74
  C9D1 Score 4 | 0 | 0
  C9D1 Score 5: number analyzed (Participants) | 97 | 74
  C9D1 Score 5 | 0 | 0
  C9D22 Score 0: number analyzed (Participants) | 76 | 65
  C9D22 Score 0 | 33 | 37
  C9D22 Score 1: number analyzed (Participants) | 76 | 65
  C9D22 Score 1 | 42 | 28
  C9D22 Score 2: number analyzed (Participants) | 76 | 65
  C9D22 Score 2 | 1 | 0
  C9D22 Score 3: number analyzed (Participants) | 76 | 65
  C9D22 Score 3 | 0 | 0
  C9D22 Score 4: number analyzed (Participants) | 76 | 65
  C9D22 Score 4 | 0 | 0
  C9D22 Score 5: number analyzed (Participants) | 76 | 65
  C9D22 Score 5 | 0 | 0
  C10D1 Score 0: number analyzed (Participants) | 82 | 63
  C10D1 Score 0 | 40 | 34
  C10D1 Score 1: number analyzed (Participants) | 82 | 63
  C10D1 Score 1 | 41 | 29
  C10D1 Score 2: number analyzed (Participants) | 82 | 63
  C10D1 Score 2 | 1 | 0
  C10D1 Score 3: number analyzed (Participants) | 82 | 63
  C10D1 Score 3 | 0 | 0
  C10D1 Score 4: number analyzed (Participants) | 82 | 63
  C10D1 Score 4 | 0 | 0
  C10D1 Score 5: number analyzed (Participants) | 82 | 63
  C10D1 Score 5 | 0 | 0
  C10D22 Score 0: number analyzed (Participants) | 67 | 48
  C10D22 Score 0 | 29 | 25
  C10D22 Score 1: number analyzed (Participants) | 67 | 48
  C10D22 Score 1 | 38 | 23
  C10D22 Score 2: number analyzed (Participants) | 67 | 48
  C10D22 Score 2 | 0 | 0
  C10D22 Score 3: number analyzed (Participants) | 67 | 48
  C10D22 Score 3 | 0 | 0
  C10D22 Score 4: number analyzed (Participants) | 67 | 48
  C10D22 Score 4 | 0 | 0
  C10D22 Score 5: number analyzed (Participants) | 67 | 48
  C10D22 Score 5 | 0 | 0
  C11D1 Score 0: number analyzed (Participants) | 77 | 52
  C11D1 Score 0 | 36 | 23
  C11D1 Score 1: number analyzed (Participants) | 77 | 52
  C11D1 Score 1 | 39 | 29
  C11D1 Score 2: number analyzed (Participants) | 77 | 52
  C11D1 Score 2 | 2 | 0
  C11D1 Score 3: number analyzed (Participants) | 77 | 52
  C11D1 Score 3 | 0 | 0
  C11D1 Score 4: number analyzed (Participants) | 77 | 52
  C11D1 Score 4 | 0 | 0
  C11D1 Score 5: number analyzed (Participants) | 77 | 52
  C11D1 Score 5 | 0 | 0
  C11D22 Score 0: number analyzed (Participants) | 61 | 39
  C11D22 Score 0 | 26 | 22
  C11D22 Score 1: number analyzed (Participants) | 61 | 39
  C11D22 Score 1 | 35 | 17
  C11D22 Score 2: number analyzed (Participants) | 61 | 39
  C11D22 Score 2 | 0 | 0
  C11D22 Score 3: number analyzed (Participants) | 61 | 39
  C11D22 Score 3 | 0 | 0
  C11D22 Score 4: number analyzed (Participants) | 61 | 39
  C11D22 Score 4 | 0 | 0
  C11D22 Score 5: number analyzed (Participants) | 61 | 39
  C11D22 Score 5 | 0 | 0
  C12D1 Score 0: number analyzed (Participants) | 67 | 47
  C12D1 Score 0 | 28 | 27
  C12D1 Score 1: number analyzed (Participants) | 67 | 47
  C12D1 Score 1 | 37 | 19
  C12D1 Score 2: number analyzed (Participants) | 67 | 47
  C12D1 Score 2 | 2 | 1
  C12D1 Score 3: number analyzed (Participants) | 67 | 47
  C12D1 Score 3 | 0 | 0
  C12D1 Score 4: number analyzed (Participants) | 67 | 47
  C12D1 Score 4 | 0 | 0
  C12D1 Score 5: number analyzed (Participants) | 67 | 47
  C12D1 Score 5 | 0 | 0
  C12D22 Score 0: number analyzed (Participants) | 50 | 33
  C12D22 Score 0 | 24 | 17
  C12D22 Score 1: number analyzed (Participants) | 50 | 33
  C12D22 Score 1 | 25 | 16
  C12D22 Score 2: number analyzed (Participants) | 50 | 33
  C12D22 Score 2 | 1 | 0
  C12D22 Score 3: number analyzed (Participants) | 50 | 33
  C12D22 Score 3 | 0 | 0
  C12D22 Score 4: number analyzed (Participants) | 50 | 33
  C12D22 Score 4 | 0 | 0
  C12D22 Score 5: number analyzed (Participants) | 50 | 33
  C12D22 Score 5 | 0 | 0
  C13D1 Score 0: number analyzed (Participants) | 61 | 39
  C13D1 Score 0 | 26 | 22
  C13D1 Score 1: number analyzed (Participants) | 61 | 39
  C13D1 Score 1 | 34 | 17
  C13D1 Score 2: number analyzed (Participants) | 61 | 39
  C13D1 Score 2 | 1 | 0
  C13D1 Score 3: number analyzed (Participants) | 61 | 39
  C13D1 Score 3 | 0 | 0
  C13D1 Score 4: number analyzed (Participants) | 61 | 39
  C13D1 Score 4 | 0 | 0
  C13D1 Score 5: number analyzed (Participants) | 61 | 39
  C13D1 Score 5 | 0 | 0
  C13D22 Score 0: number analyzed (Participants) | 53 | 26
  C13D22 Score 0 | 23 | 14
  C13D22 Score 1: number analyzed (Participants) | 53 | 26
  C13D22 Score 1 | 29 | 12
  C13D22 Score 2: number analyzed (Participants) | 53 | 26
  C13D22 Score 2 | 1 | 0
  C13D22 Score 3: number analyzed (Participants) | 53 | 26
  C13D22 Score 3 | 0 | 0
  C13D22 Score 4: number analyzed (Participants) | 53 | 26
  C13D22 Score 4 | 0 | 0
  C13D22 Score 5: number analyzed (Participants) | 53 | 26
  C13D22 Score 5 | 0 | 0
  C14D1 Score 0: number analyzed (Participants) | 47 | 36
  C14D1 Score 0 | 23 | 18
  C14D1 Score 1: number analyzed (Participants) | 47 | 36
  C14D1 Score 1 | 24 | 17
  C14D1 Score 2: number analyzed (Participants) | 47 | 36
  C14D1 Score 2 | 0 | 1
  C14D1 Score 3: number analyzed (Participants) | 47 | 36
  C14D1 Score 3 | 0 | 0
  C14D1 Score 4: number analyzed (Participants) | 47 | 36
  C14D1 Score 4 | 0 | 0
  C14D1 Score 5: number analyzed (Participants) | 47 | 36
  C14D1 Score 5 | 0 | 0
  C14D22 Score 0: number analyzed (Participants) | 38 | 22
  C14D22 Score 0 | 18 | 12
  C14D22 Score 1: number analyzed (Participants) | 38 | 22
  C14D22 Score 1 | 19 | 10
  C14D22 Score 2: number analyzed (Participants) | 38 | 22
  C14D22 Score 2 | 1 | 0
  C14D22 Score 3: number analyzed (Participants) | 38 | 22
  C14D22 Score 3 | 0 | 0
  C14D22 Score 4: number analyzed (Participants) | 38 | 22
  C14D22 Score 4 | 0 | 0
  C14D22 Score 5: number analyzed (Participants) | 38 | 22
  C14D22 Score 5 | 0 | 0
  C15D1 Score 0: number analyzed (Participants) | 43 | 30
  C15D1 Score 0 | 19 | 15
  C15D1 Score 1: number analyzed (Participants) | 43 | 30
  C15D1 Score 1 | 24 | 15
  C15D1 Score 2: number analyzed (Participants) | 43 | 30
  C15D1 Score 2 | 0 | 0
  C15D1 Score 3: number analyzed (Participants) | 43 | 30
  C15D1 Score 3 | 0 | 0
  C15D1 Score 4: number analyzed (Participants) | 43 | 30
  C15D1 Score 4 | 0 | 0
  C15D1 Score 5: number analyzed (Participants) | 43 | 30
  C15D1 Score 5 | 0 | 0
  C15D22 Score 0: number analyzed (Participants) | 36 | 20
  C15D22 Score 0 | 15 | 12
  C15D22 Score 1: number analyzed (Participants) | 36 | 20
  C15D22 Score 1 | 21 | 8
  C15D22 Score 2: number analyzed (Participants) | 36 | 20
  C15D22 Score 2 | 0 | 0
  C15D22 Score 3: number analyzed (Participants) | 36 | 20
  C15D22 Score 3 | 0 | 0
  C15D22 Score 4: number analyzed (Participants) | 36 | 20
  C15D22 Score 4 | 0 | 0
  C15D22 Score 5: number analyzed (Participants) | 36 | 20
  C15D22 Score 5 | 0 | 0
  C16D1 Score 0: number analyzed (Participants) | 41 | 25
  C16D1 Score 0 | 20 | 13
  C16D1 Score 1: number analyzed (Participants) | 41 | 25
  C16D1 Score 1 | 21 | 12
  C16D1 Score 2: number analyzed (Participants) | 41 | 25
  C16D1 Score 2 | 0 | 0
  C16D1 Score 3: number analyzed (Participants) | 41 | 25
  C16D1 Score 3 | 0 | 0
  C16D1 Score 4: number analyzed (Participants) | 41 | 25
  C16D1 Score 4 | 0 | 0
  C16D1 Score 5: number analyzed (Participants) | 41 | 25
  C16D1 Score 5 | 0 | 0
  C16D22 Score 0: number analyzed (Participants) | 32 | 16
  C16D22 Score 0 | 14 | 9
  C16D22 Score 1: number analyzed (Participants) | 32 | 16
  C16D22 Score 1 | 18 | 7
  C16D22 Score 2: number analyzed (Participants) | 32 | 16
  C16D22 Score 2 | 0 | 0
  C16D22 Score 3: number analyzed (Participants) | 32 | 16
  C16D22 Score 3 | 0 | 0
  C16D22 Score 4: number analyzed (Participants) | 32 | 16
  C16D22 Score 4 | 0 | 0
  C16D22 Score 5: number analyzed (Participants) | 32 | 16
  C16D22 Score 5 | 0 | 0
  C17D1 Score 0: number analyzed (Participants) | 34 | 19
  C17D1 Score 0 | 15 | 10
  C17D1 Score 1: number analyzed (Participants) | 34 | 19
  C17D1 Score 1 | 18 | 9
  C17D1 Score 2: number analyzed (Participants) | 34 | 19
  C17D1 Score 2 | 1 | 0
  C17D1 Score 3: number analyzed (Participants) | 34 | 19
  C17D1 Score 3 | 0 | 0
  C17D1 Score 4: number analyzed (Participants) | 34 | 19
  C17D1 Score 4 | 0 | 0
  C17D1 Score 5: number analyzed (Participants) | 34 | 19
  C17D1 Score 5 | 0 | 0
  C17D22 Score 0: number analyzed (Participants) | 23 | 9
  C17D22 Score 0 | 9 | 5
  C17D22 Score 1: number analyzed (Participants) | 23 | 9
  C17D22 Score 1 | 13 | 4
  C17D22 Score 2: number analyzed (Participants) | 23 | 9
  C17D22 Score 2 | 1 | 0
  C17D22 Score 3: number analyzed (Participants) | 23 | 9
  C17D22 Score 3 | 0 | 0
  C17D22 Score 4: number analyzed (Participants) | 23 | 9
  C17D22 Score 4 | 0 | 0
  C17D22 Score 5: number analyzed (Participants) | 23 | 9
  C17D22 Score 5 | 0 | 0
  C18D1 Score 0: number analyzed (Participants) | 30 | 17
  C18D1 Score 0 | 13 | 8
  C18D1 Score 1: number analyzed (Participants) | 30 | 17
  C18D1 Score 1 | 17 | 9
  C18D1 Score 2: number analyzed (Participants) | 30 | 17
  C18D1 Score 2 | 0 | 0
  C18D1 Score 3: number analyzed (Participants) | 30 | 17
  C18D1 Score 3 | 0 | 0
  C18D1 Score 4: number analyzed (Participants) | 30 | 17
  C18D1 Score 4 | 0 | 0
  C18D1 Score 5: number analyzed (Participants) | 30 | 17
  C18D1 Score 5 | 0 | 0
  C18D22 Score 0: number analyzed (Participants) | 22 | 11
  C18D22 Score 0 | 11 | 6
  C18D22 Score 1: number analyzed (Participants) | 22 | 11
  C18D22 Score 1 | 10 | 5
  C18D22 Score 2: number analyzed (Participants) | 22 | 11
  C18D22 Score 2 | 1 | 0
  C18D22 Score 3: number analyzed (Participants) | 22 | 11
  C18D22 Score 3 | 0 | 0
  C18D22 Score 4: number analyzed (Participants) | 22 | 11
  C18D22 Score 4 | 0 | 0
  C18D22 Score 5: number analyzed (Participants) | 22 | 11
  C18D22 Score 5 | 0 | 0
  C19D1 Score 0: number analyzed (Participants) | 26 | 16
  C19D1 Score 0 | 9 | 8
  C19D1 Score 1: number analyzed (Participants) | 26 | 16
  C19D1 Score 1 | 17 | 7
  C19D1 Score 2: number analyzed (Participants) | 26 | 16
  C19D1 Score 2 | 0 | 1
  C19D1 Score 3: number analyzed (Participants) | 26 | 16
  C19D1 Score 3 | 0 | 0
  C19D1 Score 4: number analyzed (Participants) | 26 | 16
  C19D1 Score 4 | 0 | 0
  C19D1 Score 5: number analyzed (Participants) | 26 | 16
  C19D1 Score 5 | 0 | 0
  C19D22 Score 0: number analyzed (Participants) | 21 | 12
  C19D22 Score 0 | 9 | 6
  C19D22 Score 1: number analyzed (Participants) | 21 | 12
  C19D22 Score 1 | 12 | 6
  C19D22 Score 2: number analyzed (Participants) | 21 | 12
  C19D22 Score 2 | 0 | 0
  C19D22 Score 3: number analyzed (Participants) | 21 | 12
  C19D22 Score 3 | 0 | 0
  C19D22 Score 4: number analyzed (Participants) | 21 | 12
  C19D22 Score 4 | 0 | 0
  C19D22 Score 5: number analyzed (Participants) | 21 | 12
  C19D22 Score 5 | 0 | 0
  C20D1 Score 0: number analyzed (Participants) | 26 | 16
  C20D1 Score 0 | 9 | 8
  C20D1 Score 1: number analyzed (Participants) | 26 | 16
  C20D1 Score 1 | 16 | 8
  C20D1 Score 2: number analyzed (Participants) | 26 | 16
  C20D1 Score 2 | 1 | 0
  C20D1 Score 3: number analyzed (Participants) | 26 | 16
  C20D1 Score 3 | 0 | 0
  C20D1 Score 4: number analyzed (Participants) | 26 | 16
  C20D1 Score 4 | 0 | 0
  C20D1 Score 5: number analyzed (Participants) | 26 | 16
  C20D1 Score 5 | 0 | 0
  C20D22 Score 0: number analyzed (Participants) | 19 | 11
  C20D22 Score 0 | 7 | 7
  C20D22 Score 1: number analyzed (Participants) | 19 | 11
  C20D22 Score 1 | 11 | 4
  C20D22 Score 2: number analyzed (Participants) | 19 | 11
  C20D22 Score 2 | 1 | 0
  C20D22 Score 3: number analyzed (Participants) | 19 | 11
  C20D22 Score 3 | 0 | 0
  C20D22 Score 4: number analyzed (Participants) | 19 | 11
  C20D22 Score 4 | 0 | 0
  C20D22 Score 5: number analyzed (Participants) | 19 | 11
  C20D22 Score 5 | 0 | 0
  C21D1 Score 0: number analyzed (Participants) | 23 | 16
  C21D1 Score 0 | 8 | 9
  C21D1 Score 1: number analyzed (Participants) | 23 | 16
  C21D1 Score 1 | 14 | 7
  C21D1 Score 2: number analyzed (Participants) | 23 | 16
  C21D1 Score 2 | 1 | 0
  C21D1 Score 3: number analyzed (Participants) | 23 | 16
  C21D1 Score 3 | 0 | 0
  C21D1 Score 4: number analyzed (Participants) | 23 | 16
  C21D1 Score 4 | 0 | 0
  C21D1 Score 5: number analyzed (Participants) | 23 | 16
  C21D1 Score 5 | 0 | 0
  C21D22 Score 0: number analyzed (Participants) | 15 | 9
  C21D22 Score 0 | 4 | 5
  C21D22 Score 1: number analyzed (Participants) | 15 | 9
  C21D22 Score 1 | 10 | 4
  C21D22 Score 2: number analyzed (Participants) | 15 | 9
  C21D22 Score 2 | 1 | 0
  C21D22 Score 3: number analyzed (Participants) | 15 | 9
  C21D22 Score 3 | 0 | 0
  C21D22 Score 4: number analyzed (Participants) | 15 | 9
  C21D22 Score 4 | 0 | 0
  C21D22 Score 5: number analyzed (Participants) | 15 | 9
  C21D22 Score 5 | 0 | 0
  C22D1 Score 0: number analyzed (Participants) | 17 | 13
  C22D1 Score 0 | 6 | 4
  C22D1 Score 1: number analyzed (Participants) | 17 | 13
  C22D1 Score 1 | 10 | 9
  C22D1 Score 2: number analyzed (Participants) | 17 | 13
  C22D1 Score 2 | 1 | 0
  C22D1 Score 3: number analyzed (Participants) | 17 | 13
  C22D1 Score 3 | 0 | 0
  C22D1 Score 4: number analyzed (Participants) | 17 | 13
  C22D1 Score 4 | 0 | 0
  C22D1 Score 5: number analyzed (Participants) | 17 | 13
  C22D1 Score 5 | 0 | 0
  C22D22 Score 0: number analyzed (Participants) | 11 | 9
  C22D22 Score 0 | 3 | 5
  C22D22 Score 1: number analyzed (Participants) | 11 | 9
  C22D22 Score 1 | 7 | 4
  C22D22 Score 2: number analyzed (Participants) | 11 | 9
  C22D22 Score 2 | 1 | 0
  C22D22 Score 3: number analyzed (Participants) | 11 | 9
  C22D22 Score 3 | 0 | 0
  C22D22 Score 4: number analyzed (Participants) | 11 | 9
  C22D22 Score 4 | 0 | 0
  C22D22 Score 5: number analyzed (Participants) | 11 | 9
  C22D22 Score 5 | 0 | 0
  C23D1 Score 0: number analyzed (Participants) | 16 | 13
  C23D1 Score 0 | 5 | 5
  C23D1 Score 1: number analyzed (Participants) | 16 | 13
  C23D1 Score 1 | 10 | 8
  C23D1 Score 2: number analyzed (Participants) | 16 | 13
  C23D1 Score 2 | 1 | 0
  C23D1 Score 3: number analyzed (Participants) | 16 | 13
  C23D1 Score 3 | 0 | 0
  C23D1 Score 4: number analyzed (Participants) | 16 | 13
  C23D1 Score 4 | 0 | 0
  C23D1 Score 5: number analyzed (Participants) | 16 | 13
  C23D1 Score 5 | 0 | 0
  C23D22 Score 0: number analyzed (Participants) | 14 | 7
  C23D22 Score 0 | 4 | 3
  C23D22 Score 1: number analyzed (Participants) | 14 | 7
  C23D22 Score 1 | 9 | 4
  C23D22 Score 2: number analyzed (Participants) | 14 | 7
  C23D22 Score 2 | 1 | 0
  C23D22 Score 3: number analyzed (Participants) | 14 | 7
  C23D22 Score 3 | 0 | 0
  C23D22 Score 4: number analyzed (Participants) | 14 | 7
  C23D22 Score 4 | 0 | 0
  C23D22 Score 5: number analyzed (Participants) | 14 | 7
  C23D22 Score 5 | 0 | 0
  C24D1 Score 0: number analyzed (Participants) | 16 | 10
  C24D1 Score 0 | 6 | 4
  C24D1 Score 1: number analyzed (Participants) | 16 | 10
  C24D1 Score 1 | 10 | 6
  C24D1 Score 2: number analyzed (Participants) | 16 | 10
  C24D1 Score 2 | 0 | 0
  C24D1 Score 3: number analyzed (Participants) | 16 | 10
  C24D1 Score 3 | 0 | 0
  C24D1 Score 4: number analyzed (Participants) | 16 | 10
  C24D1 Score 4 | 0 | 0
  C24D1 Score 5: number analyzed (Participants) | 16 | 10
  C24D1 Score 5 | 0 | 0
  C24D22 Score 0: number analyzed (Participants) | 9 | 6
  C24D22 Score 0 | 2 | 3
  C24D22 Score 1: number analyzed (Participants) | 9 | 6
  C24D22 Score 1 | 7 | 3
  C24D22 Score 2: number analyzed (Participants) | 9 | 6
  C24D22 Score 2 | 0 | 0
  C24D22 Score 3: number analyzed (Participants) | 9 | 6
  C24D22 Score 3 | 0 | 0
  C24D22 Score 4: number analyzed (Participants) | 9 | 6
  C24D22 Score 4 | 0 | 0
  C24D22 Score 5: number analyzed (Participants) | 9 | 6
  C24D22 Score 5 | 0 | 0
  C25D1 Score 0: number analyzed (Participants) | 14 | 8
  C25D1 Score 0 | 4 | 3
  C25D1 Score 1: number analyzed (Participants) | 14 | 8
  C25D1 Score 1 | 10 | 5
  C25D1 Score 2: number analyzed (Participants) | 14 | 8
  C25D1 Score 2 | 0 | 0
  C25D1 Score 3: number analyzed (Participants) | 14 | 8
  C25D1 Score 3 | 0 | 0
  C25D1 Score 4: number analyzed (Participants) | 14 | 8
  C25D1 Score 4 | 0 | 0
  C25D1 Score 5: number analyzed (Participants) | 14 | 8
  C25D1 Score 5 | 0 | 0
  C25D22 Score 0: number analyzed (Participants) | 11 | 6
  C25D22 Score 0 | 2 | 2
  C25D22 Score 1: number analyzed (Participants) | 11 | 6
  C25D22 Score 1 | 9 | 4
  C25D22 Score 2: number analyzed (Participants) | 11 | 6
  C25D22 Score 2 | 0 | 0
  C25D22 Score 3: number analyzed (Participants) | 11 | 6
  C25D22 Score 3 | 0 | 0
  C25D22 Score 4: number analyzed (Participants) | 11 | 6
  C25D22 Score 4 | 0 | 0
  C25D22 Score 5: number analyzed (Participants) | 11 | 6
  C25D22 Score 5 | 0 | 0
  C26D1 Score 0: number analyzed (Participants) | 13 | 6
  C26D1 Score 0 | 3 | 2
  C26D1 Score 1: number analyzed (Participants) | 13 | 6
  C26D1 Score 1 | 10 | 4
  C26D1 Score 2: number analyzed (Participants) | 13 | 6
  C26D1 Score 2 | 0 | 0
  C26D1 Score 3: number analyzed (Participants) | 13 | 6
  C26D1 Score 3 | 0 | 0
  C26D1 Score 4: number analyzed (Participants) | 13 | 6
  C26D1 Score 4 | 0 | 0
  C26D1 Score 5: number analyzed (Participants) | 13 | 6
  C26D1 Score 5 | 0 | 0
  C26D22 Score 0: number analyzed (Participants) | 8 | 3
  C26D22 Score 0 | 2 | 0
  C26D22 Score 1: number analyzed (Participants) | 8 | 3
  C26D22 Score 1 | 6 | 3
  C26D22 Score 2: number analyzed (Participants) | 8 | 3
  C26D22 Score 2 | 0 | 0
  C26D22 Score 3: number analyzed (Participants) | 8 | 3
  C26D22 Score 3 | 0 | 0
  C26D22 Score 4: number analyzed (Participants) | 8 | 3
  C26D22 Score 4 | 0 | 0
  C26D22 Score 5: number analyzed (Participants) | 8 | 3
  C26D22 Score 5 | 0 | 0
  C27D1 Score 0: number analyzed (Participants) | 13 | 6
  C27D1 Score 0 | 3 | 2
  C27D1 Score 1: number analyzed (Participants) | 13 | 6
  C27D1 Score 1 | 10 | 4
  C27D1 Score 2: number analyzed (Participants) | 13 | 6
  C27D1 Score 2 | 0 | 0
  C27D1 Score 3: number analyzed (Participants) | 13 | 6
  C27D1 Score 3 | 0 | 0
  C27D1 Score 4: number analyzed (Participants) | 13 | 6
  C27D1 Score 4 | 0 | 0
  C27D1 Score 5: number analyzed (Participants) | 13 | 6
  C27D1 Score 5 | 0 | 0
  C27D22 Score 0: number analyzed (Participants) | 9 | 4
  C27D22 Score 0 | 2 | 1
  C27D22 Score 1: number analyzed (Participants) | 9 | 4
  C27D22 Score 1 | 7 | 3
  C27D22 Score 2: number analyzed (Participants) | 9 | 4
  C27D22 Score 2 | 0 | 0
  C27D22 Score 3: number analyzed (Participants) | 9 | 4
  C27D22 Score 3 | 0 | 0
  C27D22 Score 4: number analyzed (Participants) | 9 | 4
  C27D22 Score 4 | 0 | 0
  C27D22 Score 5: number analyzed (Participants) | 9 | 4
  C27D22 Score 5 | 0 | 0
  C28D1 Score 0: number analyzed (Participants) | 13 | 6
  C28D1 Score 0 | 4 | 2
  C28D1 Score 1: number analyzed (Participants) | 13 | 6
  C28D1 Score 1 | 9 | 4
  C28D1 Score 2: number analyzed (Participants) | 13 | 6
  C28D1 Score 2 | 0 | 0
  C28D1 Score 3: number analyzed (Participants) | 13 | 6
  C28D1 Score 3 | 0 | 0
  C28D1 Score 4: number analyzed (Participants) | 13 | 6
  C28D1 Score 4 | 0 | 0
  C28D1 Score 5: number analyzed (Participants) | 13 | 6
  C28D1 Score 5 | 0 | 0
  C28D22 Score 0: number analyzed (Participants) | 9 | 1
  C28D22 Score 0 | 2 | 0
  C28D22 Score 1: number analyzed (Participants) | 9 | 1
  C28D22 Score 1 | 7 | 1
  C28D22 Score 2: number analyzed (Participants) | 9 | 1
  C28D22 Score 2 | 0 | 0
  C28D22 Score 3: number analyzed (Participants) | 9 | 1
  C28D22 Score 3 | 0 | 0
  C28D22 Score 4: number analyzed (Participants) | 9 | 1
  C28D22 Score 4 | 0 | 0
  C28D22 Score 5: number analyzed (Participants) | 9 | 1
  C28D22 Score 5 | 0 | 0
  C29D1 Score 0: number analyzed (Participants) | 10 | 5
  C29D1 Score 0 | 4 | 2
  C29D1 Score 1: number analyzed (Participants) | 10 | 5
  C29D1 Score 1 | 6 | 3
  C29D1 Score 2: number analyzed (Participants) | 10 | 5
  C29D1 Score 2 | 0 | 0
  C29D1 Score 3: number analyzed (Participants) | 10 | 5
  C29D1 Score 3 | 0 | 0
  C29D1 Score 4: number analyzed (Participants) | 10 | 5
  C29D1 Score 4 | 0 | 0
  C29D1 Score 5: number analyzed (Participants) | 10 | 5
  C29D1 Score 5 | 0 | 0
  C29D22 Score 0: number analyzed (Participants) | 7 | 3
  C29D22 Score 0 | 2 | 1
  C29D22 Score 1: number analyzed (Participants) | 7 | 3
  C29D22 Score 1 | 5 | 2
  C29D22 Score 2: number analyzed (Participants) | 7 | 3
  C29D22 Score 2 | 0 | 0
  C29D22 Score 3: number analyzed (Participants) | 7 | 3
  C29D22 Score 3 | 0 | 0
  C29D22 Score 4: number analyzed (Participants) | 7 | 3
  C29D22 Score 4 | 0 | 0
  C29D22 Score 5: number analyzed (Participants) | 7 | 3
  C29D22 Score 5 | 0 | 0
  C30D1 Score 0: number analyzed (Participants) | 10 | 5
  C30D1 Score 0 | 3 | 2
  C30D1 Score 1: number analyzed (Participants) | 10 | 5
  C30D1 Score 1 | 7 | 3
  C30D1 Score 2: number analyzed (Participants) | 10 | 5
  C30D1 Score 2 | 0 | 0
  C30D1 Score 3: number analyzed (Participants) | 10 | 5
  C30D1 Score 3 | 0 | 0
  C30D1 Score 4: number analyzed (Participants) | 10 | 5
  C30D1 Score 4 | 0 | 0
  C30D1 Score 5: number analyzed (Participants) | 10 | 5
  C30D1 Score 5 | 0 | 0
  C30D22 Score 0: number analyzed (Participants) | 7 | 0
  C30D22 Score 0 | 1 |
  C30D22 Score 1: number analyzed (Participants) | 7 | 0
  C30D22 Score 1 | 6 |
  C30D22 Score 2: number analyzed (Participants) | 7 | 0
  C30D22 Score 2 | 0 |
  C30D22 Score 3: number analyzed (Participants) | 7 | 0
  C30D22 Score 3 | 0 |
  C30D22 Score 4: number analyzed (Participants) | 7 | 0
  C30D22 Score 4 | 0 |
  C30D22 Score 5: number analyzed (Participants) | 7 | 0
  C30D22 Score 5 | 0 |
  C31D1 Score 0: number analyzed (Participants) | 8 | 4
  C31D1 Score 0 | 3 | 2
  C31D1 Score 1: number analyzed (Participants) | 8 | 4
  C31D1 Score 1 | 5 | 2
  C31D1 Score 2: number analyzed (Participants) | 8 | 4
  C31D1 Score 2 | 0 | 0
  C31D1 Score 3: number analyzed (Participants) | 8 | 4
  C31D1 Score 3 | 0 | 0
  C31D1 Score 4: number analyzed (Participants) | 8 | 4
  C31D1 Score 4 | 0 | 0
  C31D1 Score 5: number analyzed (Participants) | 8 | 4
  C31D1 Score 5 | 0 | 0
  C31D22 Score 0: number analyzed (Participants) | 5 | 1
  C31D22 Score 0 | 1 | 1
  C31D22 Score 1: number analyzed (Participants) | 5 | 1
  C31D22 Score 1 | 4 | 0
  C31D22 Score 2: number analyzed (Participants) | 5 | 1
  C31D22 Score 2 | 0 | 0
  C31D22 Score 3: number analyzed (Participants) | 5 | 1
  C31D22 Score 3 | 0 | 0
  C31D22 Score 4: number analyzed (Participants) | 5 | 1
  C31D22 Score 4 | 0 | 0
  C31D22 Score 5: number analyzed (Participants) | 5 | 1
  C31D22 Score 5 | 0 | 0
  C32D1 Score 0: number analyzed (Participants) | 6 | 2
  C32D1 Score 0 | 1 | 0
  C32D1 Score 1: number analyzed (Participants) | 6 | 2
  C32D1 Score 1 | 5 | 2
  C32D1 Score 2: number analyzed (Participants) | 6 | 2
  C32D1 Score 2 | 0 | 0
  C32D1 Score 3: number analyzed (Participants) | 6 | 2
  C32D1 Score 3 | 0 | 0
  C32D1 Score 4: number analyzed (Participants) | 6 | 2
  C32D1 Score 4 | 0 | 0
  C32D1 Score 5: number analyzed (Participants) | 6 | 2
  C32D1 Score 5 | 0 | 0
  C32D22 Score 0: number analyzed (Participants) | 5 | 0
  C32D22 Score 0 | 1 |
  C32D22 Score 1: number analyzed (Participants) | 5 | 0
  C32D22 Score 1 | 4 |
  C32D22 Score 2: number analyzed (Participants) | 5 | 0
  C32D22 Score 2 | 0 |
  C32D22 Score 3: number analyzed (Participants) | 5 | 0
  C32D22 Score 3 | 0 |
  C32D22 Score 4: number analyzed (Participants) | 5 | 0
  C32D22 Score 4 | 0 |
  C32D22 Score 5: number analyzed (Participants) | 5 | 0
  C32D22 Score 5 | 0 |
  C33D1 Score 0: number analyzed (Participants) | 4 | 2
  C33D1 Score 0 | 1 | 1
  C33D1 Score 1: number analyzed (Participants) | 4 | 2
  C33D1 Score 1 | 3 | 1
  C33D1 Score 2: number analyzed (Participants) | 4 | 2
  C33D1 Score 2 | 0 | 0
  C33D1 Score 3: number analyzed (Participants) | 4 | 2
  C33D1 Score 3 | 0 | 0
  C33D1 Score 4: number analyzed (Participants) | 4 | 2
  C33D1 Score 4 | 0 | 0
  C33D1 Score 5: number analyzed (Participants) | 4 | 2
  C33D1 Score 5 | 0 | 0
  C33D22 Score 0: number analyzed (Participants) | 3 | 0
  C33D22 Score 0 | 1 |
  C33D22 Score 1: number analyzed (Participants) | 3 | 0
  C33D22 Score 1 | 2 |
  C33D22 Score 2: number analyzed (Participants) | 3 | 0
  C33D22 Score 2 | 0 |
  C33D22 Score 3: number analyzed (Participants) | 3 | 0
  C33D22 Score 3 | 0 |
  C33D22 Score 4: number analyzed (Participants) | 3 | 0
  C33D22 Score 4 | 0 |
  C33D22 Score 5: number analyzed (Participants) | 3 | 0
  C33D22 Score 5 | 0 |
  C34D1 Score 0: number analyzed (Participants) | 3 | 2
  C34D1 Score 0 | 1 | 1
  C34D1 Score 1: number analyzed (Participants) | 3 | 2
  C34D1 Score 1 | 2 | 1
  C34D1 Score 2: number analyzed (Participants) | 3 | 2
  C34D1 Score 2 | 0 | 0
  C34D1 Score 3: number analyzed (Participants) | 3 | 2
  C34D1 Score 3 | 0 | 0
  C34D1 Score 4: number analyzed (Participants) | 3 | 2
  C34D1 Score 4 | 0 | 0
  C34D1 Score 5: number analyzed (Participants) | 3 | 2
  C34D1 Score 5 | 0 | 0
  C34D22 Score 0: number analyzed (Participants) | 2 | 0
  C34D22 Score 0 | 1 |
  C34D22 Score 1: number analyzed (Participants) | 2 | 0
  C34D22 Score 1 | 1 |
  C34D22 Score 2: number analyzed (Participants) | 2 | 0
  C34D22 Score 2 | 0 |
  C34D22 Score 3: number analyzed (Participants) | 2 | 0
  C34D22 Score 3 | 0 |
  C34D22 Score 4: number analyzed (Participants) | 2 | 0
  C34D22 Score 4 | 0 |
  C34D22 Score 5: number analyzed (Participants) | 2 | 0
  C34D22 Score 5 | 0 |
  C35D1 Score 0: number analyzed (Participants) | 2 | 1
  C35D1 Score 0 | 0 | 0
  C35D1 Score 1: number analyzed (Participants) | 2 | 1
  C35D1 Score 1 | 2 | 1
  C35D1 Score 2: number analyzed (Participants) | 2 | 1
  C35D1 Score 2 | 0 | 0
  C35D1 Score 3: number analyzed (Participants) | 2 | 1
  C35D1 Score 3 | 0 | 0
  C35D1 Score 4: number analyzed (Participants) | 2 | 1
  C35D1 Score 4 | 0 | 0
  C35D1 Score 5: number analyzed (Participants) | 2 | 1
  C35D1 Score 5 | 0 | 0
  C35D22 Score 0: number analyzed (Participants) | 1 | 1
  C35D22 Score 0 | 0 | 0
  C35D22 Score 1: number analyzed (Participants) | 1 | 1
  C35D22 Score 1 | 1 | 1
  C35D22 Score 2: number analyzed (Participants) | 1 | 1
  C35D22 Score 2 | 0 | 0
  C35D22 Score 3: number analyzed (Participants) | 1 | 1
  C35D22 Score 3 | 0 | 0
  C35D22 Score 4: number analyzed (Participants) | 1 | 1
  C35D22 Score 4 | 0 | 0
  C35D22 Score 5: number analyzed (Participants) | 1 | 1
  C35D22 Score 5 | 0 | 0
  C36D1 Score 0: number analyzed (Participants) | 2 | 1
  C36D1 Score 0 | 0 | 0
  C36D1 Score 1: number analyzed (Participants) | 2 | 1
  C36D1 Score 1 | 2 | 1
  C36D1 Score 2: number analyzed (Participants) | 2 | 1
  C36D1 Score 2 | 0 | 0
  C36D1 Score 3: number analyzed (Participants) | 2 | 1
  C36D1 Score 3 | 0 | 0
  C36D1 Score 4: number analyzed (Participants) | 2 | 1
  C36D1 Score 4 | 0 | 0
  C36D1 Score 5: number analyzed (Participants) | 2 | 1
  C36D1 Score 5 | 0 | 0
  C36D22 Score 0: number analyzed (Participants) | 1 | 1
  C36D22 Score 0 | 0 | 0
  C36D22 Score 1: number analyzed (Participants) | 1 | 1
  C36D22 Score 1 | 1 | 1
  C36D22 Score 2: number analyzed (Participants) | 1 | 1
  C36D22 Score 2 | 0 | 0
  C36D22 Score 3: number analyzed (Participants) | 1 | 1
  C36D22 Score 3 | 0 | 0
  C36D22 Score 4: number analyzed (Participants) | 1 | 1
  C36D22 Score 4 | 0 | 0
  C36D22 Score 5: number analyzed (Participants) | 1 | 1
  C36D22 Score 5 | 0 | 0
  C37D1 Score 0: number analyzed (Participants) | 2 | 0
  C37D1 Score 0 | 0 |
  C37D1 Score 1: number analyzed (Participants) | 2 | 0
  C37D1 Score 1 | 2 |
  C37D1 Score 2: number analyzed (Participants) | 2 | 0
  C37D1 Score 2 | 0 |
  C37D1 Score 3: number analyzed (Participants) | 2 | 0
  C37D1 Score 3 | 0 |
  C37D1 Score 4: number analyzed (Participants) | 2 | 0
  C37D1 Score 4 | 0 |
  C37D1 Score 5: number analyzed (Participants) | 2 | 0
  C37D1 Score 5 | 0 |
  C37D22 Score 0: number analyzed (Participants) | 1 | 0
  C37D22 Score 0 | 0 |
  C37D22 Score 1: number analyzed (Participants) | 1 | 0
  C37D22 Score 1 | 1 |
  C37D22 Score 2: number analyzed (Participants) | 1 | 0
  C37D22 Score 2 | 0 |
  C37D22 Score 3: number analyzed (Participants) | 1 | 0
  C37D22 Score 3 | 0 |
  C37D22 Score 4: number analyzed (Participants) | 1 | 0
  C37D22 Score 4 | 0 |
  C37D22 Score 5: number analyzed (Participants) | 1 | 0
  C37D22 Score 5 | 0 |
  C38D1 Score 0: number analyzed (Participants) | 1 | 0
  C38D1 Score 0 | 0 |
  C38D1 Score 1: number analyzed (Participants) | 1 | 0
  C38D1 Score 1 | 1 |
  C38D1 Score 2: number analyzed (Participants) | 1 | 0
  C38D1 Score 2 | 0 |
  C38D1 Score 3: number analyzed (Participants) | 1 | 0
  C38D1 Score 3 | 0 |
  C38D1 Score 4: number analyzed (Participants) | 1 | 0
  C38D1 Score 4 | 0 |
  C38D1 Score 5: number analyzed (Participants) | 1 | 0
  C38D1 Score 5 | 0 |
  C38D22 Score 0: number analyzed (Participants) | 1 | 0
  C38D22 Score 0 | 0 |
  C38D22 Score 1: number analyzed (Participants) | 1 | 0
  C38D22 Score 1 | 1 |
  C38D22 Score 2: number analyzed (Participants) | 1 | 0
  C38D22 Score 2 | 0 |
  C38D22 Score 3: number analyzed (Participants) | 1 | 0
  C38D22 Score 3 | 0 |
  C38D22 Score 4: number analyzed (Participants) | 1 | 0
  C38D22 Score 4 | 0 |
  C38D22 Score 5: number analyzed (Participants) | 1 | 0
  C38D22 Score 5 | 0 |
  C39D1 Score 0: number analyzed (Participants) | 1 | 0
  C39D1 Score 0 | 0 |
  C39D1 Score 1: number analyzed (Participants) | 1 | 0
  C39D1 Score 1 | 1 |
  C39D1 Score 2: number analyzed (Participants) | 1 | 0
  C39D1 Score 2 | 0 |
  C39D1 Score 3: number analyzed (Participants) | 1 | 0
  C39D1 Score 3 | 0 |
  C39D1 Score 4: number analyzed (Participants) | 1 | 0
  C39D1 Score 4 | 0 |
  C39D1 Score 5: number analyzed (Participants) | 1 | 0
  C39D1 Score 5 | 0 |
  C39D22 Score 0: number analyzed (Participants) | 1 | 0
  C39D22 Score 0 | 0 |
  C39D22 Score 1: number analyzed (Participants) | 1 | 0
  C39D22 Score 1 | 1 |
  C39D22 Score 2: number analyzed (Participants) | 1 | 0
  C39D22 Score 2 | 0 |
  C39D22 Score 3: number analyzed (Participants) | 1 | 0
  C39D22 Score 3 | 0 |
  C39D22 Score 4: number analyzed (Participants) | 1 | 0
  C39D22 Score 4 | 0 |
  C39D22 Score 5: number analyzed (Participants) | 1 | 0
  C39D22 Score 5 | 0 |

10. Secondary Outcome: Change From Baseline in Health Related Quality of Life (HRQoL) Measured by the EORTC-QLQ-C30 Questionnaire
Description: The EORTC-QLQ-C30 is a 30-item cancer-specific instrument consisting of 5 functional scales (physical, role, emotional, social and cognitive), 9 symptom scales/items (fatigue, nausea/vomiting, general pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties) and a global health status scale. Most items are scored 1 ("not at all") to 4 ("very much") except for the items contributing to the global health status/QoL, which are scored 1 ("very poor") to 7 ("excellent"). All raw domain scores are linearly transformed to a 0-100 scale with higher scores on symptoms indicate a worse health state.
Time Frame: Baseline, C1D22, D1 and D22 of C2 through C25, C26D1, C27D1,C28D1 30 day follow up, 90 day follow up
Population: FAS with available data was analyzed.
Measure: Mean (Standard Deviation); unit: units on Scale
Arm/Group | mFOLFOX6 + Zolbetuximab | mFOLFOX6+ Placebo
Number analyzed (Participants) | 257 | 258
units on Scale
  Global Health Status Baseline | 64.20 (20.86) | 63.47 (20.63)
  Global Health Status C1D22: number analyzed (Participants) | 177 | 210
  Global Health Status C1D22 | -5.18 (20.75) | 0.48 (17.98)
  Global Health Status C2D1: number analyzed (Participants) | 207 | 225
  Global Health Status C2D1 | 1.61 (20.40) | 5.56 (18.68)
  Global Health Status C2D22: number analyzed (Participants) | 150 | 181
  Global Health Status C2D22 | 0.17 (18.51) | 1.98 (20.79)
  Global Health Status C3D1: number analyzed (Participants) | 190 | 198
  Global Health Status C3D1 | 2.85 (17.89) | 5.77 (19.92)
  Global Health Status C3D22: number analyzed (Participants) | 152 | 149
  Global Health Status C3D22 | -3.13 (19.10) | 3.13 (18.03)
  Global Health Status C4D1: number analyzed (Participants) | 170 | 163
  Global Health Status C4D1 | 0.64 (20.49) | 6.65 (21.04)
  Global Health Status C4D22: number analyzed (Participants) | 123 | 128
  Global Health Status C4D22 | -2.78 (18.16) | 1.50 (22.37)
  Global Health Status C5D1: number analyzed (Participants) | 149 | 145
  Global Health Status C5D1 | -0.62 (20.69) | 4.83 (20.71)
  Global Health Status C5D22: number analyzed (Participants) | 111 | 116
  Global Health Status C5D22 | 0.53 (21.24) | 0.07 (21.52)
  Global Health Status C6D1: number analyzed (Participants) | 123 | 122
  Global Health Status C6D1 | 1.90 (20.66) | 0.07 (21.57)
  Global Health Status C6D22: number analyzed (Participants) | 103 | 94
  Global Health Status C6D22 | 3.48 (18.21) | 2.39 (18.15)
  Global Health Status C7D1: number analyzed (Participants) | 114 | 98
  Global Health Status C7D1 | 0.00 (20.50) | 4.34 (17.64)
  Global Health Status C7D22: number analyzed (Participants) | 81 | 74
  Global Health Status C7D22 | 1.54 (18.50) | 3.38 (20.32)
  Global Health Status C8D1: number analyzed (Participants) | 80 | 83
  Global Health Status C8D1 | 3.12 (19.82) | 4.82 (17.90)
  Global Health Status C8D22: number analyzed (Participants) | 72 | 65
  Global Health Status C8D22 | 1.62 (19.91) | 6.92 (18.67)
  Global Health Status C9D1: number analyzed (Participants) | 75 | 62
  Global Health Status C9D1 | 6.11 (18.09) | 4.57 (15.14)
  Global Health Status C9D22: number analyzed (Participants) | 60 | 55
  Global Health Status C9D22 | 3.33 (19.54) | 3.18 (17.82)
  Global Health Status C10D1: number analyzed (Participants) | 66 | 56
  Global Health Status C10D1 | 3.03 (18.87) | 3.87 (19.20)
  Global Health Status C10D22: number analyzed (Participants) | 57 | 43
  Global Health Status C10D22 | 0.58 (19.47) | 5.43 (17.34)
  Global Health Status C11D1: number analyzed (Participants) | 63 | 46
  Global Health Status C11D1 | 4.37 (16.92) | 3.99 (15.09)
  Global Health Status C11D22: number analyzed (Participants) | 44 | 31
  Global Health Status C11D22 | 2.65 (18.31) | 1.34 (16.12)
  Global Health Status C12D1: number analyzed (Participants) | 53 | 41
  Global Health Status C12D1 | 1.89 (18.82) | 2.64 (14.00)
  Global Health Status C12D22: number analyzed (Participants) | 38 | 25
  Global Health Status C12D22 | -0.88 (17.41) | -3.33 (12.50)
  Global Health Status C13D1: number analyzed (Participants) | 48 | 35
  Global Health Status C13D1 | 3.47 (18.18) | 0.95 (13.52)
  Global Health Status C13D22: number analyzed (Participants) | 41 | 21
  Global Health Status C13D22 | -2.85 (19.24) | -0.79 (13.15)
  Global Health Status C14D1: number analyzed (Participants) | 39 | 30
  Global Health Status C14D1 | -0.85 (23.48) | 0.83 (20.22)
  Global Health Status C14D22: number analyzed (Participants) | 32 | 19
  Global Health Status C14D22 | -1.30 (19.64) | -1.32 (16.26)
  Global Health Status C15D1: number analyzed (Participants) | 35 | 27
  Global Health Status C15D1 | -0.71 (26.69) | 0.93 (16.88)
  Global Health Status C15D22: number analyzed (Participants) | 30 | 17
  Global Health Status C15D22 | -3.89 (22.92) | -3.43 (18.18)
  Global Health Status C16D1: number analyzed (Participants) | 35 | 22
  Global Health Status C16D1 | 1.90 (20.32) | 1.89 (18.17)
  Global Health Status C16D22: number analyzed (Participants) | 29 | 14
  Global Health Status C16D22 | -2.59 (20.18) | -2.38 (14.41)
  Global Health Status C17D1: number analyzed (Participants) | 30 | 18
  Global Health Status C17D1 | -3.89 (28.68) | 0.93 (13.06)
  Global Health Status C17D22: number analyzed (Participants) | 23 | 0
  Global Health Status C17D22 | -6.88 (25.33) |
  Global Health Status C18D1: number analyzed (Participants) | 27 | 16
  Global Health Status C18D1 | 0.00 (24.57) | -1.56 (13.68)
  Global Health Status C18D22: number analyzed (Participants) | 21 | 10
  Global Health Status C18D22 | -7.14 (21.94) | -1.67 (12.30)
  Global Health Status C19D1: number analyzed (Participants) | 23 | 15
  Global Health Status C19D1 | -3.62 (24.60) | -6.11 (14.25)
  Global Health Status C19D22: number analyzed (Participants) | 20 | 11
  Global Health Status C19D22 | -4.58 (20.32) | -7.58 (12.05)
  Global Health Status C20D1: number analyzed (Participants) | 23 | 15
  Global Health Status C20D1 | -2.54 (24.67) | 1.11 (12.94)
  Global Health Status C20D22: number analyzed (Participants) | 18 | 10
  Global Health Status C20D22 | -3.70 (22.18) | -0.83 (15.93)
  Global Health Status C21D1: number analyzed (Participants) | 20 | 14
  Global Health Status C21D1 | 2.08 (20.75) | -1.79 (15.39)
  Global Health Status C21D22: number analyzed (Participants) | 14 | 0
  Global Health Status C21D22 | -4.17 (17.83) |
  Global Health Status C22D1: number analyzed (Participants) | 15 | 12
  Global Health Status C22D1 | -0.56 (24.29) | -6.25 (14.70)
  Global Health Status C22D22: number analyzed (Participants) | 11 | 0
  Global Health Status C22D22 | -10.61 (29.13) |
  Global Health Status C23D1: number analyzed (Participants) | 16 | 13
  Global Health Status C23D1 | -4.17 (29.03) | -0.64 (15.39)
  Global Health Status C23D22: number analyzed (Participants) | 11 | 0
  Global Health Status C23D22 | -3.79 (22.16) |
  Global Health Status C24D1: number analyzed (Participants) | 14 | 0
  Global Health Status C24D1 | -0.60 (26.04) |
  Global Health Status C24D22: number analyzed (Participants) | 0 | 0
  Global Health Status C25D1: number analyzed (Participants) | 12 | 0
  Global Health Status C25D1 | -6.94 (15.82) |
  Global Health Status C25D22: number analyzed (Participants) | 11 | 0
  Global Health Status C25D22 | -3.03 (17.59) |
  Global Health Status C26D1: number analyzed (Participants) | 13 | 0
  Global Health Status C26D1 | 6.41 (23.11) |
  Global Health Status C27D1: number analyzed (Participants) | 11 | 0
  Global Health Status C27D1 | 2.27 (22.39) |
  Global Health Status C28D1: number analyzed (Participants) | 12 | 0
  Global Health Status C28D1 | 0.69 (26.93) |
  Global Health Status 30 Day follow up: number analyzed (Participants) | 72 | 91
  Global Health Status 30 Day follow up | -4.98 (21.20) | -4.03 (20.99)
  Global Health Status 90 Day follow up: number analyzed (Participants) | 86 | 83
  Global Health Status 90 Day follow up | -5.72 (21.55) | -4.62 (22.32)
  Physical Functioning Baseline | 79.71 (20.37) | 78.79 (21.13)
  Physical Functioning C1D22: number analyzed (Participants) | 177 | 210
  Physical Functioning C1D22 | -4.22 (17.23) | -1.49 (15.70)
  Physical Functioning C2D1: number analyzed (Participants) | 207 | 225
  Physical Functioning C2D1 | -1.90 (18.80) | 1.69 (17.92)
  Physical Functioning C2D22: number analyzed (Participants) | 150 | 181
  Physical Functioning C2D22 | -0.98 (17.69) | 1.73 (18.69)
  Physical Functioning C3D1: number analyzed (Participants) | 190 | 198
  Physical Functioning C3D1 | -0.84 (19.51) | 2.66 (18.70)
  Physical Functioning C3D22: number analyzed (Participants) | 152 | 149
  Physical Functioning C3D22 | -1.36 (17.26) | 1.52 (15.88)
  Physical Functioning C4D1: number analyzed (Participants) | 170 | 163
  Physical Functioning C4D1 | 0.12 (19.69) | 1.47 (19.25)
  Physical Functioning C4D22: number analyzed (Participants) | 123 | 128
  Physical Functioning C4D22 | -2.60 (19.87) | -1.51 (19.61)
  Physical Functioning C5D1: number analyzed (Participants) | 149 | 145
  Physical Functioning C5D1 | -3.00 (22.55) | 0.55 (18.86)
  Physical Functioning C5D22: number analyzed (Participants) | 111 | 116
  Physical Functioning C5D22 | -2.52 (22.47) | 0.11 (19.72)
  Physical Functioning C6D1: number analyzed (Participants) | 123 | 122
  Physical Functioning C6D1 | -1.08 (20.91) | -1.26 (18.92)
  Physical Functioning C6D22: number analyzed (Participants) | 103 | 94
  Physical Functioning C6D22 | -2.01 (22.59) | -0.92 (15.96)
  Physical Functioning C7D1: number analyzed (Participants) | 114 | 98
  Physical Functioning C7D1 | -1.35 (21.67) | -0.95 (15.58)
  Physical Functioning C7D22: number analyzed (Participants) | 81 | 74
  Physical Functioning C7D22 | -2.14 (18.67) | 1.89 (19.03)
  Physical Functioning C8D1: number analyzed (Participants) | 80 | 83
  Physical Functioning C8D1 | 0.33 (21.87) | 0.88 (15.85)
  Physical Functioning C8D22: number analyzed (Participants) | 72 | 65
  Physical Functioning C8D22 | 1.02 (18.84) | -0.31 (17.66)
  Physical Functioning C9D1: number analyzed (Participants) | 75 | 62
  Physical Functioning C9D1 | 2.13 (20.33) | 0.43 (17.24)
  Physical Functioning C9D22: number analyzed (Participants) | 60 | 55
  Physical Functioning C9D22 | 2.78 (23.46) | 1.94 (16.61)
  Physical Functioning C10D1: number analyzed (Participants) | 66 | 56
  Physical Functioning C10D1 | 2.53 (21.65) | 0.71 (16.26)
  Physical Functioning C10D22: number analyzed (Participants) | 57 | 43
  Physical Functioning C10D22 | 3.27 (18.61) | -2.48 (19.36)
  Physical Functioning C11D1: number analyzed (Participants) | 63 | 46
  Physical Functioning C11D1 | 3.60 (20.17) | -3.33 (16.91)
  Physical Functioning C11D22: number analyzed (Participants) | 44 | 31
  Physical Functioning C11D22 | 3.33 (18.72) | -6.02 (16.18)
  Physical Functioning C12D1: number analyzed (Participants) | 53 | 41
  Physical Functioning C12D1 | 2.26 (20.08) | -3.58 (14.61)
  Physical Functioning C12D22: number analyzed (Participants) | 38 | 25
  Physical Functioning C12D22 | 2.63 (20.65) | -5.60 (14.74)
  Physical Functioning C13D1: number analyzed (Participants) | 48 | 35
  Physical Functioning C13D1 | 3.06 (20.35) | -6.67 (17.26)
  Physical Functioning C13D22: number analyzed (Participants) | 41 | 21
  Physical Functioning C13D22 | 1.46 (21.63) | -6.98 (19.60)
  Physical Functioning C14D1: number analyzed (Participants) | 39 | 30
  Physical Functioning C14D1 | 4.27 (17.27) | -3.56 (13.30)
  Physical Functioning C14D22: number analyzed (Participants) | 32 | 19
  Physical Functioning C14D22 | 0.42 (19.67) | -1.75 (13.49)
  Physical Functioning C15D1: number analyzed (Participants) | 35 | 27
  Physical Functioning C15D1 | 3.24 (18.39) | -6.42 (18.35)
  Physical Functioning C15D22: number analyzed (Participants) | 30 | 17
  Physical Functioning C15D22 | 3.56 (18.26) | 0.39 (14.43)
  Physical Functioning C16D1: number analyzed (Participants) | 35 | 22
  Physical Functioning C16D1 | 3.43 (20.98) | -4.55 (18.79)
  Physical Functioning C16D22: number analyzed (Participants) | 29 | 14
  Physical Functioning C16D22 | 5.29 (19.39) | -7.14 (14.67)
  Physical Functioning C17D1: number analyzed (Participants) | 30 | 18
  Physical Functioning C17D1 | 3.78 (25.05) | -3.70 (11.93)
  Physical Functioning C17D22: number analyzed (Participants) | 23 | 0
  Physical Functioning C17D22 | -3.19 (26.20) |
  Physical Functioning C18D1: number analyzed (Participants) | 27 | 16
  Physical Functioning C18D1 | 3.46 (21.03) | -2.92 (6.87)
  Physical Functioning C18D22: number analyzed (Participants) | 21 | 10
  Physical Functioning C18D22 | 3.17 (20.83) | 0.00 (7.03)
  Physical Functioning C19D1: number analyzed (Participants) | 23 | 15
  Physical Functioning C19D1 | 3.48 (17.39) | -1.33 (8.05)
  Physical Functioning C19D22: number analyzed (Participants) | 20 | 11
  Physical Functioning C19D22 | -1.00 (18.39) | -4.24 (8.58)
  Physical Functioning C20D1: number analyzed (Participants) | 23 | 15
  Physical Functioning C20D1 | 0.29 (22.43) | -1.78 (8.90)
  Physical Functioning C20D22: number analyzed (Participants) | 18 | 10
  Physical Functioning C20D22 | -1.48 (24.37) | -4.67 (7.73)
  Physical Functioning C21D1: number analyzed (Participants) | 20 | 14
  Physical Functioning C21D1 | 2.33 (15.18) | -1.43 (9.13)
  Physical Functioning C21D22: number analyzed (Participants) | 14 | 0
  Physical Functioning C21D22 | -3.33 (18.07) |
  Physical Functioning C22D1: number analyzed (Participants) | 15 | 12
  Physical Functioning C22D1 | 3.11 (18.83) | -2.22 (6.56)
  Physical Functioning C22D22: number analyzed (Participants) | 11 | 0
  Physical Functioning C22D22 | -5.45 (24.00) |
  Physical Functioning C23D1: number analyzed (Participants) | 16 | 13
  Physical Functioning C23D1 | -3.33 (19.78) | 1.54 (9.49)
  Physical Functioning C23D22: number analyzed (Participants) | 11 | 0
  Physical Functioning C23D22 | 1.82 (15.23) |
  Physical Functioning C24D1: number analyzed (Participants) | 14 | 0
  Physical Functioning C24D1 | -3.81 (21.36) |
  Physical Functioning C24D22: number analyzed (Participants) | 0 | 0
  Physical Functioning C25D1: number analyzed (Participants) | 12 | 0
  Physical Functioning C25D1 | 5.00 (11.42) |
  Physical Functioning C25D22: number analyzed (Participants) | 11 | 0
  Physical Functioning C25D22 | 2.42 (15.28) |
  Physical Functioning C26D1: number analyzed (Participants) | 13 | 0
  Physical Functioning C26D1 | 3.08 (14.56) |
  Physical Functioning C27D1: number analyzed (Participants) | 11 | 0
  Physical Functioning C27D1 | 3.64 (15.88) |
  Physical Functioning C28D1: number analyzed (Participants) | 12 | 0
  Physical Functioning C28D1 | 1.67 (15.86) |
  Physical Functioning 30 Day follow up: number analyzed (Participants) | 72 | 91
  Physical Functioning 30 Day follow up | -9.26 (24.63) | -6.96 (21.73)
  Physical Functioning 90 Day follow up: number analyzed (Participants) | 86 | 83
  Physical Functioning 90 Day follow up | -13.57 (23.77) | -11.49 (25.95)
  Role Functioning Baseline | 74.77 (27.56) | 75.52 (28.02)
  Role Functioning C1D22: number analyzed (Participants) | 177 | 210
  Role Functioning C1D22 | -6.78 (25.09) | -4.13 (24.10)
  Role Functioning C2D1: number analyzed (Participants) | 207 | 225
  Role Functioning C2D1 | -0.64 (26.78) | 0.30 (25.92)
  Role Functioning C2D22: number analyzed (Participants) | 150 | 181
  Role Functioning C2D22 | -1.67 (25.82) | -1.20 (28.44)
  Role Functioning C3D1: number analyzed (Participants) | 190 | 198
  Role Functioning C3D1 | 0.96 (28.02) | 2.19 (26.57)
  Role Functioning C3D22: number analyzed (Participants) | 152 | 149
  Role Functioning C3D22 | -3.73 (25.96) | -0.89 (25.98)
  Role Functioning C4D1: number analyzed (Participants) | 170 | 163
  Role Functioning C4D1 | -1.18 (28.41) | 1.94 (26.92)
  Role Functioning C4D22: number analyzed (Participants) | 123 | 128
  Role Functioning C4D22 | -2.98 (28.39) | -2.73 (24.82)
  Role Functioning C5D1: number analyzed (Participants) | 149 | 145
  Role Functioning C5D1 | -4.25 (29.71) | -2.87 (27.24)
  Role Functioning C5D22: number analyzed (Participants) | 111 | 116
  Role Functioning C5D22 | -2.70 (30.03) | -2.73 (27.88)
  Role Functioning C6D1: number analyzed (Participants) | 123 | 122
  Role Functioning C6D1 | -1.76 (29.94) | -5.46 (26.19)
  Role Functioning C6D22: number analyzed (Participants) | 103 | 94
  Role Functioning C6D22 | -4.21 (29.59) | -2.84 (25.47)
  Role Functioning C7D1: number analyzed (Participants) | 114 | 98
  Role Functioning C7D1 | -5.56 (28.37) | -2.55 (22.75)
  Role Functioning C7D22: number analyzed (Participants) | 81 | 74
  Role Functioning C7D22 | -5.35 (29.68) | -1.58 (24.08)
  Role Functioning C8D1: number analyzed (Participants) | 80 | 83
  Role Functioning C8D1 | -2.92 (29.62) | -0.60 (23.20)
  Role Functioning C8D22: number analyzed (Participants) | 72 | 65
  Role Functioning C8D22 | -1.39 (28.22) | -1.03 (21.83)
  Role Functioning C9D1: number analyzed (Participants) | 75 | 62
  Role Functioning C9D1 | 4.89 (26.53) | -2.96 (22.49)
  Role Functioning C9D22: number analyzed (Participants) | 60 | 55
  Role Functioning C9D22 | -0.83 (30.13) | -0.61 (22.21)
  Role Functioning C10D1: number analyzed (Participants) | 66 | 56
  Role Functioning C10D1 | 0.00 (29.38) | -3.27 (26.1)
  Role Functioning C10D22: number analyzed (Participants) | 57 | 43
  Role Functioning C10D22 | -0.58 (30.37) | -2.71 (26.96)
  Role Functioning C11D1: number analyzed (Participants) | 63 | 46
  Role Functioning C11D1 | 1.32 (32.56) | -0.36 (21.28)
  Role Functioning C11D22: number analyzed (Participants) | 44 | 31
  Role Functioning C11D22 | -3.79 (28.27) | -9.14 (20.11)
  Role Functioning C12D1: number analyzed (Participants) | 53 | 41
  Role Functioning C12D1 | -0.63 (26.55) | -2.85 (21.38)
  Role Functioning C12D22: number analyzed (Participants) | 38 | 25
  Role Functioning C12D22 | -5.26 (28.24) | -4.0 (24.19)
  Role Functioning C13D1: number analyzed (Participants) | 48 | 35
  Role Functioning C13D1 | -1.04 (29.86) | -2.38 (24.30)
  Role Functioning C13D22: number analyzed (Participants) | 41 | 21
  Role Functioning C13D22 | -4.88 (29.40) | 0.00 (19.0)
  Role Functioning C14D1: number analyzed (Participants) | 39 | 30
  Role Functioning C14D1 | -2.99 (26.18) | -5.56 (20.22)
  Role Functioning C14D22: number analyzed (Participants) | 32 | 19
  Role Functioning C14D22 | -3.65 (27.67) | -2.63 (20.23)
  Role Functioning C15D1: number analyzed (Participants) | 35 | 27
  Role Functioning C15D1 | -1.90 (27.94) | -5.56 (24.46)
  Role Functioning C15D22: number analyzed (Participants) | 30 | 17
  Role Functioning C15D22 | -5.00 (31.00) | 5.88 (22.00)
  Role Functioning C16D1: number analyzed (Participants) | 35 | 22
  Role Functioning C16D1 | 0.48 (30.38) | 0.00 (23.00)
  Role Functioning C16D22: number analyzed (Participants) | 29 | 14
  Role Functioning C16D22 | -6.32 (31.94) | -1.19 (20.11)
  Role Functioning C17D1: number analyzed (Participants) | 30 | 18
  Role Functioning C17D1 | -0.56 (33.76) | 0.00 (16.17)
  Role Functioning C17D22: number analyzed (Participants) | 23 | 0
  Role Functioning C17D22 | -11.59 (36.73) |
  Role Functioning C18D1: number analyzed (Participants) | 27 | 16
  Role Functioning C18D1 | -4.32 (28.72) | -1.04 (14.23)
  Role Functioning C18D22: number analyzed (Participants) | 21 | 10
  Role Functioning C18D22 | -3.17 (24.51) | -1.67 (14.59)
  Role Functioning C19D1: number analyzed (Participants) | 23 | 15
  Role Functioning C19D1 | -3.62 (24.60) | -5.56 (19.59)
  Role Functioning C19D22: number analyzed (Participants) | 20 | 11
  Role Functioning C19D22 | -8.33 (18.34) | -3.03 (19.46)
  Role Functioning C20D1: number analyzed (Participants) | 23 | 15
  Role Functioning C20D1 | -5.80 (23.36) | -4.44 (20.38)
  Role Functioning C20D22: number analyzed (Participants) | 18 | 10
  Role Functioning C20D22 | -6.48 (33.40) | -6.67 (11.65)
  Role Functioning C21D1: number analyzed (Participants) | 20 | 14
  Role Functioning C21D1 | 2.50 (21.81) | -1.19 (17.86)
  Role Functioning C21D22: number analyzed (Participants) | 14 | 0
  Role Functioning C21D22 | -5.95 (21.29) |
  Role Functioning C22D1: number analyzed (Participants) | 15 | 12
  Role Functioning C22D1 | -2.22 (15.26) | -2.78 (18.58)
  Role Functioning C22D22: number analyzed (Participants) | 11 | 0
  Role Functioning C22D22 | -13.64 (36.38) |
  Role Functioning C23D1: number analyzed (Participants) | 16 | 13
  Role Functioning C23D1 | -6.25 (28.46) | 1.28 (12.66)
  Role Functioning C23D22: number analyzed (Participants) | 11 | 0
  Role Functioning C23D22 | -4.55 (22.47) |
  Role Functioning C24D1: number analyzed (Participants) | 14 | 0
  Role Functioning C24D1 | -7.14 (26.73) |
  Role Functioning C24D22: number analyzed (Participants) | 0 | 0
  Role Functioning C25D1: number analyzed (Participants) | 12 | 0
  Role Functioning C25D1 | -4.17 (20.26) |
  Role Functioning C25D22: number analyzed (Participants) | 11 | 0
  Role Functioning C25D22 | -12.12 (18.40) |
  Role Functioning C26D1: number analyzed (Participants) | 13 | 0
  Role Functioning C26D1 | -11.54 (19.70) |
  Role Functioning C27D1: number analyzed (Participants) | 11 | 0
  Role Functioning C27D1 | -6.06 (22.70) |
  Role Functioning C28D1: number analyzed (Participants) | 12 | 0
  Role Functioning C28D1 | -6.94 (24.06) |
  Role Functioning 30 Day follow up: number analyzed (Participants) | 72 | 91
  Role Functioning 30 Day follow up | -13.19 (29.46) | -10.99 (30.65)
  Role Functioning 90 Day follow up: number analyzed (Participants) | 86 | 83
  Role Functioning 90 Day follow up | -14.53 (33.90) | -14.26 (29.58)
  Emotional Functioning Baseline | 74.64 (20.71) | 73.45 (21.16)
  Emotional Functioning C1D22: number analyzed (Participants) | 177 | 210
  Emotional Functioning C1D22 | 0.85 (19.08) | 3.33 (15.96)
  Emotional Functioning C2D1: number analyzed (Participants) | 207 | 225
  Emotional Functioning C2D1 | 4.55 (20.49) | 6.15 (17.93)
  Emotional Functioning C2D22: number analyzed (Participants) | 150 | 181
  Emotional Functioning C2D22 | 5.78 (19.36) | 5.85 (18.69)
  Emotional Functioning C3D1: number analyzed (Participants) | 190 | 198
  Emotional Functioning C3D1 | 6.27 (20.28) | 9.43 (18.44)
  Emotional Functioning C3D22: number analyzed (Participants) | 152 | 149
  Emotional Functioning C3D22 | 3.62 (21.14) | 9.06 (19.35)
  Emotional Functioning C4D1: number analyzed (Participants) | 170 | 163
  Emotional Functioning C4D1 | 7.40 (20.20) | 8.13 (18.86)
  Emotional Functioning C4D22: number analyzed (Participants) | 123 | 128
  Emotional Functioning C4D22 | 2.71 (19.46) | 6.84 (20.98)
  Emotional Functioning C5D1: number analyzed (Participants) | 149 | 145
  Emotional Functioning C5D1 | 4.19 (24.21) | 5.80 (20.23)
  Emotional Functioning C5D22: number analyzed (Participants) | 111 | 116
  Emotional Functioning C5D22 | 4.35 (24.04) | 2.95 (18.17)
  Emotional Functioning C6D1: number analyzed (Participants) | 123 | 122
  Emotional Functioning C6D1 | 6.44 (24.56) | 4.92 (17.86)
  Emotional Functioning C6D22: number analyzed (Participants) | 103 | 94
  Emotional Functioning C6D22 | 5.50 (21.44) | 7.54 (17.96)
  Emotional Functioning C7D1: number analyzed (Participants) | 114 | 98
  Emotional Functioning C7D1 | 5.70 (22.24) | 7.99 (19.59)
  Emotional Functioning C7D22: number analyzed (Participants) | 81 | 74
  Emotional Functioning C7D22 | 3.70 (20.20) | 7.66 (18.90)
  Emotional Functioning C8D1: number analyzed (Participants) | 80 | 83
  Emotional Functioning C8D1 | 5.21 (19.64) | 9.14 (19.42)
  Emotional Functioning C8D22: number analyzed (Participants) | 72 | 65
  Emotional Functioning C8D22 | 7.29 (24.58) | 6.41 (20.35)
  Emotional Functioning C9D1: number analyzed (Participants) | 75 | 62
  Emotional Functioning C9D1 | 8.67 (23.86) | 6.99 (16.05)
  Emotional Functioning C9D22: number analyzed (Participants) | 60 | 55
  Emotional Functioning C9D22 | 6.11 (25.25) | 5.76 (18.69)
  Emotional Functioning C10D1: number analyzed (Participants) | 66 | 56
  Emotional Functioning C10D1 | 7.20 (23.97) | 6.85 (18.26)
  Emotional Functioning C10D22: number analyzed (Participants) | 57 | 43
  Emotional Functioning C10D22 | 8.04 (22.27) | 6.20 (20.50)
  Emotional Functioning C11D1: number analyzed (Participants) | 63 | 46
  Emotional Functioning C11D1 | 9.13 (20.83) | 3.99 (21.14)
  Emotional Functioning C11D22: number analyzed (Participants) | 44 | 31
  Emotional Functioning C11D22 | 8.33 (17.88) | 1.88 (22.64)
  Emotional Functioning C12D1: number analyzed (Participants) | 53 | 41
  Emotional Functioning C12D1 | 9.59 (19.57) | 2.44 (18.66)
  Emotional Functioning C12D22: number analyzed (Participants) | 38 | 25
  Emotional Functioning C12D22 | 3.95 (19.25) | 4.33 (18.65)
  Emotional Functioning C13D1: number analyzed (Participants) | 48 | 35
  Emotional Functioning C13D1 | 7.99 (23.44) | 1.43 (24.38)
  Emotional Functioning C13D22: number analyzed (Participants) | 41 | 21
  Emotional Functioning C13D22 | 3.86 (20.34) | -3.17 (19.63)
  Emotional Functioning C14D1: number analyzed (Participants) | 39 | 30
  Emotional Functioning C14D1 | 6.20 (21.61) | 2.22 (18.94)
  Emotional Functioning C14D22: number analyzed (Participants) | 32 | 19
  Emotional Functioning C14D22 | 3.65 (21.27) | -1.75 (18.96)
  Emotional Functioning C15D1: number analyzed (Participants) | 35 | 27
  Emotional Functioning C15D1 | 6.43 (21.49) | 2.47 (18.46)
  Emotional Functioning C15D22: number analyzed (Participants) | 30 | 17
  Emotional Functioning C15D22 | 4.17 (16.63) | -2.45 (20.99)
  Emotional Functioning C16D1: number analyzed (Participants) | 35 | 22
  Emotional Functioning C16D1 | 9.76 (21.81) | -3.41 (21.62)
  Emotional Functioning C16D22: number analyzed (Participants) | 29 | 14
  Emotional Functioning C16D22 | 6.03 (19.02) | -4.76 (20.60)
  Emotional Functioning C17D1: number analyzed (Participants) | 30 | 18
  Emotional Functioning C17D1 | 7.50 (28.90) | 3.70 (19.43)
  Emotional Functioning C17D22: number analyzed (Participants) | 23 | 0
  Emotional Functioning C17D22 | 7.25 (23.21) |
  Emotional Functioning C18D1: number analyzed (Participants) | 27 | 16
  Emotional Functioning C18D1 | 8.33 (20.28) | 2.60 (20.12)
  Emotional Functioning C18D22: number analyzed (Participants) | 21 | 10
  Emotional Functioning C18D22 | 5.95 (18.47) | -5.00 (21.59)
  Emotional Functioning C19D1: number analyzed (Participants) | 23 | 15
  Emotional Functioning C19D1 | 8.70 (23.09) | -2.22 (19.02)
  Emotional Functioning C19D22: number analyzed (Participants) | 20 | 11
  Emotional Functioning C19D22 | 4.17 (24.26) | -3.79 (20.87)
  Emotional Functioning C20D1: number analyzed (Participants) | 23 | 15
  Emotional Functioning C20D1 | 10.51 (17.27) | 2.78 (20.33)
  Emotional Functioning C20D22: number analyzed (Participants) | 18 | 10
  Emotional Functioning C20D22 | 8.80 (17.26) | -6.67 (19.95)
  Emotional Functioning C21D1: number analyzed (Participants) | 20 | 14
  Emotional Functioning C21D1 | 11.25 (18.39) | -2.98 (24.59)
  Emotional Functioning C21D22: number analyzed (Participants) | 14 | 0
  Emotional Functioning C21D22 | 6.55 (16.40) |
  Emotional Functioning C22D1: number analyzed (Participants) | 15 | 12
  Emotional Functioning C22D1 | 11.67 (16.61) | 2.78 (21.42)
  Emotional Functioning C22D22: number analyzed (Participants) | 11 | 0
  Emotional Functioning C22D22 | -2.27 (27.41) |
  Emotional Functioning C23D1: number analyzed (Participants) | 16 | 13
  Emotional Functioning C23D1 | 7.81 (19.36) | 5.13 (21.93)
  Emotional Functioning C23D22: number analyzed (Participants) | 11 | 0
  Emotional Functioning C23D22 | 4.55 (17.62) |
  Emotional Functioning C24D1: number analyzed (Participants) | 14 | 0
  Emotional Functioning C24D1 | 14.88 (20.72) |
  Emotional Functioning C24D22: number analyzed (Participants) | 0 | 0
  Emotional Functioning C25D1: number analyzed (Participants) | 12 | 0
  Emotional Functioning C25D1 | 9.03 (21.75) |
  Emotional Functioning C25D22: number analyzed (Participants) | 11 | 0
  Emotional Functioning C25D22 | 1.52 (22.92) |
  Emotional Functioning C26D1: number analyzed (Participants) | 13 | 0
  Emotional Functioning C26D1 | 10.90 (24.86) |
  Emotional Functioning C27D1: number analyzed (Participants) | 11 | 0
  Emotional Functioning C27D1 | 13.64 (18.36) |
  Emotional Functioning C28D1: number analyzed (Participants) | 12 | 0
  Emotional Functioning C28D1 | 14.58 (21.36) |
  Emotional Functioning 30 Day follow up: number analyzed (Participants) | 72 | 91
  Emotional Functioning 30 Day follow up | -2.55 (22.19) | -2.47 (19.90)
  Emotional Functioning 90 Day follow up: number analyzed (Participants) | 86 | 83
  Emotional Functioning 90 Day follow up | -1.74 (22.69) | -4.02 (23.65)
  Cognitive Functioning Baseline | 87.48 (17.62) | 86.69 (18.35)
  Cognitive Functioning C1D22: number analyzed (Participants) | 177 | 210
  Cognitive Functioning C1D22 | -3.01 (18.04) | -0.32 (14.49)
  Cognitive Functioning C2D1: number analyzed (Participants) | 207 | 225
  Cognitive Functioning C2D1 | -0.16 (19.57) | 0.30 (15.98)
  Cognitive Functioning C2D22: number analyzed (Participants) | 150 | 181
  Cognitive Functioning C2D22 | -1.00 (16.75) | -1.10 (15.38)
  Cognitive Functioning C3D1: number analyzed (Participants) | 190 | 198
  Cognitive Functioning C3D1 | -0.61 (20.67) | -0.17 (16.19)
  Cognitive Functioning C3D22: number analyzed (Participants) | 152 | 149
  Cognitive Functioning C3D22 | -3.07 (18.83) | -0.11 (13.49)
  Cognitive Functioning C4D1: number analyzed (Participants) | 170 | 163
  Cognitive Functioning C4D1 | 0.10 (19.82) | -1.64 (15.85)
  Cognitive Functioning C4D22: number analyzed (Participants) | 123 | 128
  Cognitive Functioning C4D22 | -5.28 (21.59) | -1.82 (16.10)
  Cognitive Functioning C5D1: number analyzed (Participants) | 149 | 145
  Cognitive Functioning C5D1 | -4.03 (21.19) | -3.56 (17.26)
  Cognitive Functioning C5D22: number analyzed (Participants) | 111 | 116
  Cognitive Functioning C5D22 | -4.35 (23.54) | -3.16 (16.14)
  Cognitive Functioning C6D1: number analyzed (Participants) | 123 | 122
  Cognitive Functioning C6D1 | -5.42 (24.00) | -3.13 (17.22)
  Cognitive Functioning C6D22: number analyzed (Participants) | 103 | 94
  Cognitive Functioning C6D22 | -2.27 (23.46) | -0.71 (14.85)
  Cognitive Functioning C7D1: number analyzed (Participants) | 114 | 98
  Cognitive Functioning C7D1 | -2.49 (19.36) | -3.57 (17.46)
  Cognitive Functioning C7D22: number analyzed (Participants) | 81 | 74
  Cognitive Functioning C7D22 | -2.06 (18.33) | -0.45 (16.08)
  Cognitive Functioning C8D1: number analyzed (Participants) | 80 | 83
  Cognitive Functioning C8D1 | -3.75 (21.38) | -2.61 (16.97)
  Cognitive Functioning C8D22: number analyzed (Participants) | 72 | 65
  Cognitive Functioning C8D22 | 1.16 (22.08) | -5.90 (20.92)
  Cognitive Functioning C9D1: number analyzed (Participants) | 75 | 62
  Cognitive Functioning C9D1 | -0.67 (22.67) | -2.15 (17.72)
  Cognitive Functioning C9D22: number analyzed (Participants) | 60 | 55
  Cognitive Functioning C9D22 | -1.67 (24.10) | 0.91 (18.26)
  Cognitive Functioning C10D1: number analyzed (Participants) | 66 | 56
  Cognitive Functioning C10D1 | -0.25 (23.11) | -2.68 (17.05)
  Cognitive Functioning C10D22: number analyzed (Participants) | 57 | 43
  Cognitive Functioning C10D22 | -1.17 (19.63) | -3.10 (21.60)
  Cognitive Functioning C11D1: number analyzed (Participants) | 63 | 46
  Cognitive Functioning C11D1 | 2.12 (19.74) | -2.90 (20.28)
  Cognitive Functioning C11D22: number analyzed (Participants) | 44 | 31
  Cognitive Functioning C11D22 | -2.27 (15.91) | -4.30 (19.71)
  Cognitive Functioning C12D1: number analyzed (Participants) | 53 | 41
  Cognitive Functioning C12D1 | 0.00 (18.20) | -1.63 (18.56)
  Cognitive Functioning C12D22: number analyzed (Participants) | 38 | 25
  Cognitive Functioning C12D22 | -1.75 (19.68) | -6.00 (15.87)
  Cognitive Functioning C13D1: number analyzed (Participants) | 48 | 35
  Cognitive Functioning C13D1 | 1.04 (18.96) | -5.24 (28.23)
  Cognitive Functioning C13D22: number analyzed (Participants) | 41 | 21
  Cognitive Functioning C13D22 | -1.22 (20.20) | -1.59 (25.77)
  Cognitive Functioning C14D1: number analyzed (Participants) | 39 | 30
  Cognitive Functioning C14D1 | 0.43 (18.92) | -3.89 (20.85)
  Cognitive Functioning C14D22: number analyzed (Participants) | 32 | 19
  Cognitive Functioning C14D22 | -4.17 (21.17) | -3.51 (24.58)
  Cognitive Functioning C15D1: number analyzed (Participants) | 35 | 27
  Cognitive Functioning C15D1 | -1.43 (24.04) | 1.23 (15.28)
  Cognitive Functioning C15D22: number analyzed (Participants) | 30 | 17
  Cognitive Functioning C15D22 | -0.56 (17.22) | 3.92 (24.67)
  Cognitive Functioning C16D1: number analyzed (Participants) | 35 | 22
  Cognitive Functioning C16D1 | 1.43 (18.24) | -2.27 (26.38)
  Cognitive Functioning C16D22: number analyzed (Participants) | 29 | 14
  Cognitive Functioning C16D22 | -1.15 (18.86) | -1.19 (17.86)
  Cognitive Functioning C17D1: number analyzed (Participants) | 30 | 18
  Cognitive Functioning C17D1 | -0.56 (25.70) | -2.78 (16.42)
  Cognitive Functioning C17D22: number analyzed (Participants) | 23 | 0
  Cognitive Functioning C17D22 | -2.17 (23.73) |
  Cognitive Functioning C18D1: number analyzed (Participants) | 27 | 16
  Cognitive Functioning C18D1 | -0.62 (19.87) | 0.00 (10.54)
  Cognitive Functioning C18D22: number analyzed (Participants) | 21 | 10
  Cognitive Functioning C18D22 | 0.00 (20.41) | -3.33 (10.54)
  Cognitive Functioning C19D1: number analyzed (Participants) | 23 | 15
  Cognitive Functioning C19D1 | -1.45 (18.74) | -2.22 (10.67)
  Cognitive Functioning C19D22: number analyzed (Participants) | 20 | 11
  Cognitive Functioning C19D22 | -5.00 (20.30) | 1.52 (11.68)
  Cognitive Functioning C20D1: number analyzed (Participants) | 23 | 15
  Cognitive Functioning C20D1 | -2.90 (19.24) | 1.11 (11.73)
  Cognitive Functioning C20D22: number analyzed (Participants) | 18 | 10
  Cognitive Functioning C20D22 | 0.93 (17.59) | 0.00 (7.86)
  Cognitive Functioning C21D1: number analyzed (Participants) | 20 | 14
  Cognitive Functioning C21D1 | 0.00 (15.29) | -2.38 (12.84)
  Cognitive Functioning C21D22: number analyzed (Participants) | 14 | 0
  Cognitive Functioning C21D22 | -2.38 (14.41) |
  Cognitive Functioning C22D1: number analyzed (Participants) | 15 | 12
  Cognitive Functioning C22D1 | 0.00 (16.67) | -1.39 (13.22)
  Cognitive Functioning C22D22: number analyzed (Participants) | 11 | 0
  Cognitive Functioning C22D22 | 4.55 (19.85) |
  Cognitive Functioning C23D1: number analyzed (Participants) | 16 | 13
  Cognitive Functioning C23D1 | -1.04 (17.71) | 2.56 (9.25)
  Cognitive Functioning C23D22: number analyzed (Participants) | 11 | 0
  Cognitive Functioning C23D22 | 1.52 (15.73) |
  Cognitive Functioning C24D1: number analyzed (Participants) | 14 | 0
  Cognitive Functioning C24D1 | 2.38 (18.32) |
  Cognitive Functioning C24D22: number analyzed (Participants) | 0 | 0
  Cognitive Functioning C25D1: number analyzed (Participants) | 12 | 0
  Cognitive Functioning C25D1 | 4.17 (14.43) |
  Cognitive Functioning C25D22: number analyzed (Participants) | 11 | 0
  Cognitive Functioning C25D22 | 0.00 (16.67) |
  Cognitive Functioning C26D1: number analyzed (Participants) | 13 | 0
  Cognitive Functioning C26D1 | 2.56 (19.06) |
  Cognitive Functioning C27D1: number analyzed (Participants) | 11 | 0
  Cognitive Functioning C27D1 | 6.06 (18.67) |
  Cognitive Functioning C28D1: number analyzed (Participants) | 12 | 0
  Cognitive Functioning C28D1 | 4.17 (18.97) |
  Cognitive Functioning 30 Day follow up: number analyzed (Participants) | 72 | 91
  Cognitive Functioning 30 Day follow up | -8.56 (24.54) | -6.41 (17.70)
  Cognitive Functioning 90 Day follow up: number analyzed (Participants) | 86 | 83
  Cognitive Functioning 90 Day follow up | -11.63 (21.25) | -7.83 (20.22)
  Social Functioning Baseline | 75.36 (25.77) | 73.26 (27.18)
  Social Functioning C1D22: number analyzed (Participants) | 177 | 210
  Social Functioning C1D22 | -3.11 (24.13) | 0.48 (23.05)
  Social Functioning C2D1: number analyzed (Participants) | 207 | 225
  Social Functioning C2D1 | -0.32 (24.24) | 3.11 (25.69)
  Social Functioning C2D22: number analyzed (Participants) | 150 | 181
  Social Functioning C2D22 | -2.44 (23.04) | 2.76 (27.47)
  Social Functioning C3D1: number analyzed (Participants) | 190 | 198
  Social Functioning C3D1 | 0.53 (25.31) | 2.44 (26.78)
  Social Functioning C3D22: number analyzed (Participants) | 152 | 149
  Social Functioning C3D22 | -5.70 (25.09) | 3.80 (25.86)
  Social Functioning C4D1: number analyzed (Participants) | 170 | 163
  Social Functioning C4D1 | 0.20 (24.86) | 5.62 (23.88)
  Social Functioning C4D22: number analyzed (Participants) | 123 | 128
  Social Functioning C4D22 | -0.95 (25.28) | 2.73 (22.21)
  Social Functioning C5D1: number analyzed (Participants) | 149 | 145
  Social Functioning C5D1 | -1.57 (29.21) | 1.38 (29.43)
  Social Functioning C5D22: number analyzed (Participants) | 111 | 116
  Social Functioning C5D22 | -0.75 (28.37) | 0.86 (27.26)
  Social Functioning C6D1: number analyzed (Participants) | 123 | 122
  Social Functioning C6D1 | 0.54 (24.51) | 0.27 (26.42)
  Social Functioning C6D22: number analyzed (Participants) | 103 | 94
  Social Functioning C6D22 | 1.29 (24.44) | 3.01 (29.33)
  Social Functioning C7D1: number analyzed (Participants) | 114 | 98
  Social Functioning C7D1 | -1.61 (24.49) | 0.00 (24.87)
  Social Functioning C7D22: number analyzed (Participants) | 81 | 74
  Social Functioning C7D22 | -1.03 (26.66) | 4.50 (26.21)
  Social Functioning C8D1: number analyzed (Participants) | 80 | 83
  Social Functioning C8D1 | -0.83 (21.53) | 3.01 (22.56)
  Social Functioning C8D22: number analyzed (Participants) | 72 | 65
  Social Functioning C8D22 | 1.85 (21.04) | 1.03 (24.09)
  Social Functioning C9D1: number analyzed (Participants) | 75 | 62
  Social Functioning C9D1 | 2.67 (21.05) | 3.23 (25.22)
  Social Functioning C9D22: number analyzed (Participants) | 60 | 55
  Social Functioning C9D22 | 2.78 (21.52) | 3.33 (26.91)
  Social Functioning C10D1: number analyzed (Participants) | 66 | 56
  Social Functioning C10D1 | 3.03 (23.19) | -0.60 (28.60)
  Social Functioning C10D22: number analyzed (Participants) | 57 | 43
  Social Functioning C10D22 | 2.34 (21.69) | -1.55 (30.82)
  Social Functioning C11D1: number analyzed (Participants) | 63 | 46
  Social Functioning C11D1 | 3.70 (21.88) | 1.81 (25.87)
  Social Functioning C11D22: number analyzed (Participants) | 44 | 31
  Social Functioning C11D22 | -0.76 (21.55) | -3.76 (22.65)
  Social Functioning C12D1: number analyzed (Participants) | 53 | 41
  Social Functioning C12D1 | 4.09 (17.87) | 0.00 (26.09)
  Social Functioning C12D22: number analyzed (Participants) | 38 | 25
  Social Functioning C12D22 | -1.32 (21.71) | 4.00 (22.71)
  Social Functioning C13D1: number analyzed (Participants) | 48 | 35
  Social Functioning C13D1 | 2.43 (21.19) | 1.43 (26.62)
  Social Functioning C13D22: number analyzed (Participants) | 41 | 21
  Social Functioning C13D22 | 1.22 (23.39) | 8.73 (22.74)
  Social Functioning C14D1: number analyzed (Participants) | 39 | 30
  Social Functioning C14D1 | 2.99 (22.25) | 0.56 (25.33)
  Social Functioning C14D22: number analyzed (Participants) | 32 | 19
  Social Functioning C14D22 | 0.52 (20.52) | 6.14 (23.71)
  Social Functioning C15D1: number analyzed (Participants) | 35 | 27
  Social Functioning C15D1 | 2.38 (28.34) | -6.17 (24.96)
  Social Functioning C15D22: number analyzed (Participants) | 30 | 17
  Social Functioning C15D22 | 3.89 (20.38) | 0.00 (22.05)
  Social Functioning C16D1: number analyzed (Participants) | 35 | 22
  Social Functioning C16D1 | 3.33 (22.43) | 3.79 (24.09)
  Social Functioning C16D22: number analyzed (Participants) | 29 | 14
  Social Functioning C16D22 | 1.15 (22.24) | 3.57 (26.29)
  Social Functioning C17D1: number analyzed (Participants) | 30 | 18
  Social Functioning C17D1 | 1.67 (26.75) | 4.63 (26.69)
  Social Functioning C17D22: number analyzed (Participants) | 23 | 0
  Social Functioning C17D22 | -3.62 (22.45) |
  Social Functioning C18D1: number analyzed (Participants) | 27 | 16
  Social Functioning C18D1 | 1.85 (21.85) | -1.04 (20.61)
  Social Functioning C18D22: number analyzed (Participants) | 21 | 10
  Social Functioning C18D22 | 2.38 (16.06) | -6.67 (11.65)
  Social Functioning C19D1: number analyzed (Participants) | 23 | 15
  Social Functioning C19D1 | 3.62 (16.63) | -5.56 (16.27)
  Social Functioning C19D22: number analyzed (Participants) | 20 | 11
  Social Functioning C19D22 | 0.83 (11.44) | -4.55 (16.82)
  Social Functioning C20D1: number analyzed (Participants) | 23 | 15
  Social Functioning C20D1 | 2.17 (19.66) | -3.33 (19.11)
  Social Functioning C20D22: number analyzed (Participants) | 18 | 10
  Social Functioning C20D22 | 1.85 (15.00) | 5.00 (13.72)
  Social Functioning C21D1: number analyzed (Participants) | 20 | 14
  Social Functioning C21D1 | 6.67 (16.58) | -11.90 (15.23)
  Social Functioning C21D22: number analyzed (Participants) | 14 | 0
  Social Functioning C21D22 | 7.14 (15.63) |
  Social Functioning C22D1: number analyzed (Participants) | 15 | 12
  Social Functioning C22D1 | 1.11 (20.38) | -4.17 (16.09)
  Social Functioning C22D22: number analyzed (Participants) | 11 | 0
  Social Functioning C22D22 | -4.55 (21.20) |
  Social Functioning C23D1: number analyzed (Participants) | 16 | 13
  Social Functioning C23D1 | 1.04 (17.71) | -2.56 (16.45)
  Social Functioning C23D22: number analyzed (Participants) | 11 | 0
  Social Functioning C23D22 | 4.55 (19.85) |
  Social Functioning C24D1: number analyzed (Participants) | 14 | 0
  Social Functioning C24D1 | 2.38 (23.44) |
  Social Functioning C24D22: number analyzed (Participants) | 0 | 0
  Social Functioning C25D1: number analyzed (Participants) | 12 | 0
  Social Functioning C25D1 | 2.78 (29.16) |
  Social Functioning C25D22: number analyzed (Participants) | 11 | 0
  Social Functioning C25D22 | 3.03 (19.46) |
  Social Functioning C26D1: number analyzed (Participants) | 13 | 0
  Social Functioning C26D1 | 2.56 (21.35) |
  Social Functioning C27D1: number analyzed (Participants) | 11 | 0
  Social Functioning C27D1 | 6.06 (23.89) |
  Social Functioning C28D1: number analyzed (Participants) | 12 | 0
  Social Functioning C28D1 | 5.56 (20.52) |
  Social Functioning 30 Day follow up: number analyzed (Participants) | 72 | 91
  Social Functioning 30 Day follow up | -12.73 (30.45) | -2.56 (26.98)
  Social Functioning 90 Day follow up: number analyzed (Participants) | 86 | 83
  Social Functioning 90 Day follow up | -9.88 (29.64) | -6.02 (27.74)
  Fatigue Baseline | 31.13 (23.94) | 32.69 (23.71)
  Fatigue C1D22: number analyzed (Participants) | 177 | 210
  Fatigue C1D22 | 8.47 (23.12) | 4.50 (20.34)
  Fatigue C2D1: number analyzed (Participants) | 207 | 225
  Fatigue C2D1 | 3.81 (22.20) | -1.48 (22.30)
  Fatigue C2D22: number analyzed (Participants) | 150 | 181
  Fatigue C2D22 | 4.00 (22.75) | -0.06 (21.90)
  Fatigue C3D1: number analyzed (Participants) | 190 | 198
  Fatigue C3D1 | 2.11 (23.61) | -2.13 (21.92)
  Fatigue C3D22: number analyzed (Participants) | 152 | 149
  Fatigue C3D22 | 8.48 (23.15) | -0.37 (21.47)
  Fatigue C4D1: number analyzed (Participants) | 170 | 163
  Fatigue C4D1 | 1.70 (25.04) | -1.30 (23.34)
  Fatigue C4D22: number analyzed (Participants) | 123 | 128
  Fatigue C4D22 | 5.96 (24.03) | -1.48 (22.80)
  Fatigue C5D1: number analyzed (Participants) | 149 | 145
  Fatigue C5D1 | 4.85 (26.79) | 0.38 (24.82)
  Fatigue C5D22: number analyzed (Participants) | 111 | 116
  Fatigue C5D22 | 5.61 (27.94) | 1.82 (25.12)
  Fatigue C6D1: number analyzed (Participants) | 123 | 122
  Fatigue C6D1 | 1.08 (25.66) | 2.00 (22.86)
  Fatigue C6D22: number analyzed (Participants) | 103 | 94
  Fatigue C6D22 | 2.05 (24.74) | -0.35 (21.83)
  Fatigue C7D1: number analyzed (Participants) | 114 | 98
  Fatigue C7D1 | 0.78 (22.74) | -1.81 (21.15)
  Fatigue C7D22: number analyzed (Participants) | 81 | 74
  Fatigue C7D22 | 4.53 (22.21) | -1.35 (21.21)
  Fatigue C8D1: number analyzed (Participants) | 80 | 83
  Fatigue C8D1 | -0.14 (23.95) | -1.34 (23.11)
  Fatigue C8D22: number analyzed (Participants) | 72 | 65
  Fatigue C8D22 | -0.77 (22.71) | -1.03 (23.38)
  Fatigue C9D1: number analyzed (Participants) | 75 | 62
  Fatigue C9D1 | -4.30 (22.81) | -3.58 (21.55)
  Fatigue C9D22: number analyzed (Participants) | 60 | 55
  Fatigue C9D22 | -0.74 (24.28) | -3.23 (23.00)
  Fatigue C10D1: number analyzed (Participants) | 66 | 56
  Fatigue C10D1 | -1.18 (23.88) | -3.97 (23.82)
  Fatigue C10D22: number analyzed (Participants) | 57 | 43
  Fatigue C10D22 | -0.39 (21.92) | 0.26 (22.55)
  Fatigue C11D1: number analyzed (Participants) | 63 | 46
  Fatigue C11D1 | -4.23 (20.30) | -1.21 (20.45)
  Fatigue C11D22: number analyzed (Participants) | 44 | 31
  Fatigue C11D22 | -3.79 (19.31) | -0.36 (21.94)
  Fatigue C12D1: number analyzed (Participants) | 53 | 41
  Fatigue C12D1 | -3.98 (19.13) | 0.54 (20.63)
  Fatigue C12D22: number analyzed (Participants) | 38 | 25
  Fatigue C12D22 | 1.17 (18.04) | 2.67 (22.52)
  Fatigue C13D1: number analyzed (Participants) | 48 | 35
  Fatigue C13D1 | -1.16 (21.77) | 3.17 (23.43)
  Fatigue C13D22: number analyzed (Participants) | 41 | 21
  Fatigue C13D22 | 1.36 (23.07) | 2.65 (16.06)
  Fatigue C14D1: number analyzed (Participants) | 39 | 30
  Fatigue C14D1 | 0.00 (20.71) | 1.48 (20.37)
  Fatigue C14D22: number analyzed (Participants) | 32 | 19
  Fatigue C14D22 | 0.00 (21.49) | -0.58 (20.11)
  Fatigue C15D1: number analyzed (Participants) | 35 | 27
  Fatigue C15D1 | 3.49 (25.25) | 4.94 (23.54)
  Fatigue C15D22: number analyzed (Participants) | 30 | 17
  Fatigue C15D22 | 2.96 (9.12) | -7.19 (21.50)
  Fatigue C16D1: number analyzed (Participants) | 35 | 22
  Fatigue C16D1 | -2.22 (22.51) | 0.51 (21.54)
  Fatigue C16D22: number analyzed (Participants) | 29 | 14
  Fatigue C16D22 | 1.53 (27.33) | 2.38 (23.13)
  Fatigue C17D1: number analyzed (Participants) | 30 | 18
  Fatigue C17D1 | 1.85 (22.24) | -0.62 (23.33)
  Fatigue C17D22: number analyzed (Participants) | 23 | 0
  Fatigue C17D22 | 8.70 (26.58) |
  Fatigue C18D1: number analyzed (Participants) | 27 | 16
  Fatigue C18D1 | -2.88 (18.64) | -2.78 (21.66)
  Fatigue C18D22: number analyzed (Participants) | 21 | 10
  Fatigue C18D22 | -4.23 (17.73) | 1.11 (20.59)
  Fatigue C19D1: number analyzed (Participants) | 23 | 15
  Fatigue C19D1 | -0.48 (23.08) | 2.96 (25.36)
  Fatigue C19D22: number analyzed (Participants) | 20 | 11
  Fatigue C19D22 | -1.11 (19.71) | 3.03 (26.80)
  Fatigue C20D1: number analyzed (Participants) | 23 | 15
  Fatigue C20D1 | 1.45 (26.65) | -1.48 (15.64)
  Fatigue C20D22: number analyzed (Participants) | 18 | 10
  Fatigue C20D22 | 4.32 (29.80) | 2.22 (18.74)
  Fatigue C21D1: number analyzed (Participants) | 20 | 14
  Fatigue C21D1 | -4.44 (15.88) | -0.79 (19.72)
  Fatigue C21D22: number analyzed (Participants) | 14 | 0
  Fatigue C21D22 | 8.73 (21.43) |
  Fatigue C22D1: number analyzed (Participants) | 15 | 12
  Fatigue C22D1 | 5.19 (20.52) | 2.78 (17.81)
  Fatigue C22D22: number analyzed (Participants) | 11 | 0
  Fatigue C22D22 | 9.09 (29.32) |
  Fatigue C23D1: number analyzed (Participants) | 16 | 13
  Fatigue C23D1 | 11.11 (22.22) | -1.71 (19.16)
  Fatigue C23D22: number analyzed (Participants) | 11 | 0
  Fatigue C23D22 | 7.07 (18.10) |
  Fatigue C24D1: number analyzed (Participants) | 14 | 0
  Fatigue C24D1 | 6.35 (22.10) |
  Fatigue C24D22: number analyzed (Participants) | 0 | 0
  Fatigue C25D1: number analyzed (Participants) | 12 | 0
  Fatigue C25D1 | 6.48 (15.32) |
  Fatigue C25D22: number analyzed (Participants) | 11 | 0
  Fatigue C25D22 | 8.08 (20.54) |
  Fatigue C26D1: number analyzed (Participants) | 13 | 0
  Fatigue C26D1 | 3.42 (17.79) |
  Fatigue C27D1: number analyzed (Participants) | 11 | 0
  Fatigue C27D1 | 1.01 (14.45) |
  Fatigue C28D1: number analyzed (Participants) | 12 | 0
  Fatigue C28D1 | 3.70 (15.95) |
  Fatigue 30 Day follow up: number analyzed (Participants) | 72 | 91
  Fatigue 30 Day follow up | 8.02 (26.32) | 6.96 (25.80)
  Fatigue 90 Day follow up: number analyzed (Participants) | 86 | 83
  Fatigue 90 Day follow up | 11.63 (29.12) | 13.25 (25.35)
  Nausea and Vomiting Baseline | 15.37 (23.90) | 17.18 (24.33)
  Nausea and Vomiting C1D22: number analyzed (Participants) | 177 | 210
  Nausea and Vomiting C1D22 | 9.13 (23.77) | 2.70 (23.19)
  Nausea and Vomiting C2D1: number analyzed (Participants) | 207 | 225
  Nausea and Vomiting C2D1 | 3.38 (25.90) | -3.70 (23.85)
  Nausea and Vomiting C2D22: number analyzed (Participants) | 150 | 181
  Nausea and Vomiting C2D22 | 4.33 (23.76) | 0.83 (26.25)
  Nausea and Vomiting C3D1: number analyzed (Participants) | 190 | 198
  Nausea and Vomiting C3D1 | 0.53 (27.43) | -5.13 (23.70)
  Nausea and Vomiting C3D22: number analyzed (Participants) | 152 | 149
  Nausea and Vomiting C3D22 | 4.61 (24.28) | -1.68 (28.19)
  Nausea and Vomiting C4D1: number analyzed (Participants) | 170 | 163
  Nausea and Vomiting C4D1 | 0.00 (26.46) | -4.19 (23.74)
  Nausea and Vomiting C4D22: number analyzed (Participants) | 123 | 128
  Nausea and Vomiting C4D22 | 2.30 (25.46) | -3.39 (25.48)
  Nausea and Vomiting C5D1: number analyzed (Participants) | 149 | 145
  Nausea and Vomiting C5D1 | -0.22 (23.00) | -6.78 (23.69)
  Nausea and Vomiting C5D22: number analyzed (Participants) | 111 | 116
  Nausea and Vomiting C5D22 | 2.40 (21.65) | -5.60 (22.08)
  Nausea and Vomiting C6D1: number analyzed (Participants) | 123 | 122
  Nausea and Vomiting C6D1 | -2.98 (19.33) | -3.42 (24.24)
  Nausea and Vomiting C6D22: number analyzed (Participants) | 103 | 94
  Nausea and Vomiting C6D22 | -1.13 (22.54) | -5.14 (24.32)
  Nausea and Vomiting C7D1: number analyzed (Participants) | 114 | 98
  Nausea and Vomiting C7D1 | -2.63 (19.40) | -4.25 (21.31)
  Nausea and Vomiting C7D22: number analyzed (Participants) | 81 | 74
  Nausea and Vomiting C7D22 | 2.06 (21.31) | -6.53 (22.21)
  Nausea and Vomiting C8D1: number analyzed (Participants) | 80 | 83
  Nausea and Vomiting C8D1 | -1.46 (18.41) | -3.61 (16.68)
  Nausea and Vomiting C8D22: number analyzed (Participants) | 72 | 65
  Nausea and Vomiting C8D22 | -1.85 (22.12) | -4.10 (21.86)
  Nausea and Vomiting C9D1: number analyzed (Participants) | 75 | 62
  Nausea and Vomiting C9D1 | -6.22 (20.46) | -4.57 (23.80)
  Nausea and Vomiting C9D22: number analyzed (Participants) | 60 | 55
  Nausea and Vomiting C9D22 | -0.56 (20.11) | -3.94 (21.98)
  Nausea and Vomiting C10D1: number analyzed (Participants) | 66 | 56
  Nausea and Vomiting C10D1 | -2.27 (21.26) | -3.87 (19.59)
  Nausea and Vomiting C10D22: number analyzed (Participants) | 57 | 43
  Nausea and Vomiting C10D22 | -1.17 (21.33) | -2.71 (25.18)
  Nausea and Vomiting C11D1: number analyzed (Participants) | 63 | 46
  Nausea and Vomiting C11D1 | -4.23 (20.95) | -1.81 (22.56)
  Nausea and Vomiting C11D22: number analyzed (Participants) | 44 | 31
  Nausea and Vomiting C11D22 | 0.38 (17.79) | -3.76 (24.23)
  Nausea and Vomiting C12D1: number analyzed (Participants) | 53 | 41
  Nausea and Vomiting C12D1 | -3.77 (19.51) | -1.63 (25.22)
  Nausea and Vomiting C12D22: number analyzed (Participants) | 38 | 25
  Nausea and Vomiting C12D22 | -1.75 (19.68) | -3.33 (24.06)
  Nausea and Vomiting C13D1: number analyzed (Participants) | 48 | 35
  Nausea and Vomiting C13D1 | -3.12 (19.34) | -3.33 (23.50)
  Nausea and Vomiting C13D22: number analyzed (Participants) | 41 | 21
  Nausea and Vomiting C13D22 | -1.63 (23.22) | -7.14 (24.48)
  Nausea and Vomiting C14D1: number analyzed (Participants) | 39 | 30
  Nausea and Vomiting C14D1 | -5.13 (22.99) | -2.78 (22.35)
  Nausea and Vomiting C14D22: number analyzed (Participants) | 32 | 19
  Nausea and Vomiting C14D22 | -2.08 (24.59) | -7.02 (24.42)
  Nausea and Vomiting C15D1: number analyzed (Participants) | 35 | 27
  Nausea and Vomiting C15D1 | -3.33 (23.50) | -3.09 (25.75)
  Nausea and Vomiting C15D22: number analyzed (Participants) | 30 | 17
  Nausea and Vomiting C15D22 | -3.89 (22.18) | -2.94 (31.31)
  Nausea and Vomiting C16D1: number analyzed (Participants) | 35 | 22
  Nausea and Vomiting C16D1 | -7.62 (22.63) | 1.52 (33.69)
  Nausea and Vomiting C16D22: number analyzed (Participants) | 29 | 14
  Nausea and Vomiting C16D22 | -1.72 (29.33) | -7.14 (30.46)
  Nausea and Vomiting C17D1: number analyzed (Participants) | 30 | 18
  Nausea and Vomiting C17D1 | -10.00 (21.71) | -4.63 (27.30)
  Nausea and Vomiting C17D22: number analyzed (Participants) | 23 | 0
  Nausea and Vomiting C17D22 | -1.45 (21.85) |
  Nausea and Vomiting C18D1: number analyzed (Participants) | 27 | 16
  Nausea and Vomiting C18D1 | -7.41 (20.84) | -4.17 (26.87)
  Nausea and Vomiting C18D22: number analyzed (Participants) | 21 | 10
  Nausea and Vomiting C18D22 | -3.17 (22.12) | -8.33 (29.66)
  Nausea and Vomiting C19D1: number analyzed (Participants) | 23 | 15
  Nausea and Vomiting C19D1 | -5.07 (21.58) | -1.11 (29.19)
  Nausea and Vomiting C19D22: number analyzed (Participants) | 20 | 11
  Nausea and Vomiting C19D22 | -5.00 (22.36) | -7.58 (31.94)
  Nausea and Vomiting C20D1: number analyzed (Participants) | 23 | 15
  Nausea and Vomiting C20D1 | -4.35 (22.60) | -3.33 (26.87)
  Nausea and Vomiting C20D22: number analyzed (Participants) | 18 | 10
  Nausea and Vomiting C20D22 | -4.63 (25.44) | -8.33 (32.63)
  Nausea and Vomiting C21D1: number analyzed (Participants) | 20 | 14
  Nausea and Vomiting C21D1 | -1.67 (16.13) | -3.57 (30.08)
  Nausea and Vomiting C21D22: number analyzed (Participants) | 14 | 0
  Nausea and Vomiting C21D22 | -4.76 (18.98) |
  Nausea and Vomiting C22D1: number analyzed (Participants) | 15 | 12
  Nausea and Vomiting C22D1 | -2.22 (20.77) | -9.72 (27.94)
  Nausea and Vomiting C22D22: number analyzed (Participants) | 11 | 0
  Nausea and Vomiting C22D22 | -6.06 (25.03) |
  Nausea and Vomiting C23D1: number analyzed (Participants) | 16 | 13
  Nausea and Vomiting C23D1 | -5.21 (19.92) | -3.85 (30.55)
  Nausea and Vomiting C23D22: number analyzed (Participants) | 11 | 0
  Nausea and Vomiting C23D22 | -6.06 (23.89) |
  Nausea and Vomiting C24D1: number analyzed (Participants) | 14 | 0
  Nausea and Vomiting C24D1 | -8.33 (21.43) |
  Nausea and Vomiting C24D22: number analyzed (Participants) | 0 | 0
  Nausea and Vomiting C25D1: number analyzed (Participants) | 12 | 0
  Nausea and Vomiting C25D1 | -8.33 (21.90) |
  Nausea and Vomiting C25D22: number analyzed (Participants) | 11 | 0
  Nausea and Vomiting C25D22 | -6.06 (25.03) |
  Nausea and Vomiting C26D1: number analyzed (Participants) | 13 | 0
  Nausea and Vomiting C26D1 | -10.26 (21.01) |
  Nausea and Vomiting C27D1: number analyzed (Participants) | 11 | 0
  Nausea and Vomiting C27D1 | -1.52 (8.99) |
  Nausea and Vomiting C28D1: number analyzed (Participants) | 12 | 0
  Nausea and Vomiting C28D1 | -4.17 (14.43) |
  Nausea and Vomiting 30 Day Follow up: number analyzed (Participants) | 72 | 91
  Nausea and Vomiting 30 Day Follow up | 3.24 (25.12) | -1.10 (27.19)
  Nausea and Vomiting 90 Day Follow up: number analyzed (Participants) | 86 | 83
  Nausea and Vomiting 90 Day Follow up | 0.39 (22.28) | -4.42 (29.34)
  Pain Baseline | 25.68 (25.51) | 26.61 (25.13)
  Pain C1D22: number analyzed (Participants) | 177 | 210
  Pain C1D22 | -2.54 (23.40) | -5.48 (19.23)
  Pain C2D1: number analyzed (Participants) | 207 | 225
  Pain C2D1 | -6.36 (24.77) | -9.19 (21.93)
  Pain C2D22: number analyzed (Participants) | 150 | 181
  Pain C2D22 | -7.67 (24.47) | -9.21 (23.27)
  Pain C3D1: number analyzed (Participants) | 190 | 198
  Pain C3D1 | -9.12 (25.92) | -9.18 (22.56)
  Pain C3D22: number analyzed (Participants) | 152 | 149
  Pain C3D22 | -8.44 (24.71) | -7.61 (22.13)
  Pain C4D1: number analyzed (Participants) | 170 | 163
  Pain C4D1 | -9.31 (24.46) | -9.41 (21.68)
  Pain C4D22: number analyzed (Participants) | 123 | 128
  Pain C4D22 | -5.69 (23.94) | -7.94 (22.91)
  Pain C5D1: number analyzed (Participants) | 149 | 145
  Pain C5D1 | -5.82 (26.91) | -6.55 (23.27)
  Pain C5D22: number analyzed (Participants) | 111 | 116
  Pain C5D22 | -5.41 (26.32) | -5.60 (24.27)
  Pain C6D1: number analyzed (Participants) | 123 | 122
  Pain C6D1 | -7.18 (27.25) | -4.64 (24.17)
  Pain C6D22: number analyzed (Participants) | 103 | 94
  Pain C6D22 | -5.34 (23.36) | -8.16 (18.89)
  Pain C7D1: number analyzed (Participants) | 114 | 98
  Pain C7D1 | -5.56 (24.15) | -6.80 (20.56)
  Pain C7D22: number analyzed (Participants) | 81 | 74
  Pain C7D22 | -1.65 (25.22) | -6.98 (20.65)
  Pain C8D1: number analyzed (Participants) | 80 | 83
  Pain C8D1 | -2.92 (25.13) | -7.83 (18.28)
  Pain C8D22: number analyzed (Participants) | 72 | 65
  Pain C8D22 | -8.10 (23.40) | -5.90 (17.04)
  Pain C9D1: number analyzed (Participants) | 75 | 62
  Pain C9D1 | -8.89 (22.48) | -6.99 (18.74)
  Pain C9D22: number analyzed (Participants) | 60 | 55
  Pain C9D22 | -6.11 (23.96) | -3.94 (21.75)
  Pain C10D1: number analyzed (Participants) | 66 | 56
  Pain C10D1 | -6.57 (24.09) | -2.38 (25.71)
  Pain C10D22: number analyzed (Participants) | 57 | 43
  Pain C10D22 | -2.92 (24.42) | -2.71 (24.65)
  Pain C11D1: number analyzed (Participants) | 63 | 46
  Pain C11D1 | -9.26 (23.91) | -3.62 (18.56)
  Pain C11D22: number analyzed (Participants) | 44 | 31
  Pain C11D22 | -7.20 (22.85) | -3.23 (15.17)
  Pain C12D1: number analyzed (Participants) | 53 | 41
  Pain C12D1 | -7.55 (22.54) | -1.22 (19.50)
  Pain C12D22: number analyzed (Participants) | 38 | 25
  Pain C12D22 | -0.88 (27.11) | -5.33 (20.25)
  Pain C13D1: number analyzed (Participants) | 48 | 35
  Pain C13D1 | -5.21 (25.76) | -2.86 (20.41)
  Pain C13D22: number analyzed (Participants) | 41 | 21
  Pain C13D22 | -2.03 (25.87) | -7.14 (21.46)
  Pain C14D1: number analyzed (Participants) | 39 | 30
  Pain C14D1 | -4.27 (24.10) | -1.11 (19.54)
  Pain C14D22: number analyzed (Participants) | 32 | 19
  Pain C14D22 | -5.73 (18.26) | -10.53 (26.18)
  Pain C15D1: number analyzed (Participants) | 35 | 27
  Pain C15D1 | -4.76 (23.07) | 1.85 (25.46)
  Pain C15D22: number analyzed (Participants) | 30 | 17
  Pain C15D22 | -5.00 (18.65) | -4.90 (28.73)
  Pain C16D1: number analyzed (Participants) | 35 | 22
  Pain C16D1 | -3.81 (24.95) | -4.55 (22.53)
  Pain C16D22: number analyzed (Participants) | 29 | 14
  Pain C16D22 | -6.32 (19.11) | -3.57 (11.65)
  Pain C17D1: number analyzed (Participants) | 30 | 18
  Pain C17D1 | 0.56 (29.84) | -4.63 (15.97)
  Pain C17D22: number analyzed (Participants) | 23 | 0
  Pain C17D22 | 2.17 (31.90) |
  Pain C18D1: number analyzed (Participants) | 27 | 16
  Pain C18D1 | -3.09 (28.13) | -6.25 (10.32)
  Pain C18D22: number analyzed (Participants) | 21 | 10
  Pain C18D22 | -1.59 (17.40) | -5.00 (15.81)
  Pain C19D1: number analyzed (Participants) | 23 | 15
  Pain C19D1 | 0.00 (20.72) | -1.11 (13.31)
  Pain C19D22: number analyzed (Participants) | 20 | 11
  Pain C19D22 | 0.00 (16.22) | -4.55 (10.78)
  Pain C20D1: number analyzed (Participants) | 23 | 15
  Pain C20D1 | -2.17 (26.26) | -3.33 (15.69)
  Pain C20D22: number analyzed (Participants) | 18 | 10
  Pain C20D22 | -3.70 (21.81) | 1.67 (16.57)
  Pain C21D1: number analyzed (Participants) | 20 | 14
  Pain C21D1 | -5.83 (18.95) | -4.76 (15.23)
  Pain C21D22: number analyzed (Participants) | 14 | 0
  Pain C21D22 | -2.38 (17.12) |
  Pain C22D1: number analyzed (Participants) | 15 | 12
  Pain C22D1 | -1.11 (14.73) | -4.17 (12.56)
  Pain C22D22: number analyzed (Participants) | 11 | 0
  Pain C22D22 | 0.00 (14.91) |
  Pain C23D1: number analyzed (Participants) | 16 | 13
  Pain C23D1 | 1.04 (21.49) | -6.41 (14.50)
  Pain C23D22: number analyzed (Participants) | 11 | 0
  Pain C23D22 | -1.52 (17.41) |
  Pain C24D1: number analyzed (Participants) | 14 | 0
  Pain C24D1 | 3.57 (26.29) |
  Pain C24D22: number analyzed (Participants) | 0 | 0
  Pain C25D1: number analyzed (Participants) | 12 | 0
  Pain C25D1 | 5.56 (14.79) |
  Pain C25D22: number analyzed (Participants) | 11 | 0
  Pain C25D22 | 6.06 (23.89) |
  Pain C26D1: number analyzed (Participants) | 13 | 0
  Pain C26D1 | 1.28 (14.37) |
  Pain C27D1: number analyzed (Participants) | 11 | 0
  Pain C27D1 | 0.00 (18.26) |
  Pain C28D1: number analyzed (Participants) | 12 | 0
  Pain C28D1 | 1.39 (19.41) |
  Pain 30 Follow up: number analyzed (Participants) | 72 | 91
  Pain 30 Follow up | 0.46 (29.33) | 7.33 (27.24)
  Pain 90 Day Follow up: number analyzed (Participants) | 86 | 83
  Pain 90 Day Follow up | 3.49 (28.37) | 6.02 (29.51)
  Dyspnoea Baseline | 13.23 (22.97) | 13.70 (23.20)
  Dyspnoea C1D22: number analyzed (Participants) | 177 | 210
  Dyspnoea C1D22 | 1.88 (22.67) | 1.43 (22.19)
  Dyspnoea C2D1: number analyzed (Participants) | 207 | 225
  Dyspnoea C2D1 | 0.48 (20.90) | 0.59 (20.88)
  Dyspnoea C2D22: number analyzed (Participants) | 150 | 181
  Dyspnoea C2D22 | -0.67 (20.96) | 0.18 (21.52)
  Dyspnoea C3D1: number analyzed (Participants) | 190 | 198
  Dyspnoea C3D1 | 0.35 (24.24) | 1.01 (20.13)
  Dyspnoea C3D22: number analyzed (Participants) | 152 | 149
  Dyspnoea C3D22 | 1.32 (21.32) | 2.24 (21.10)
  Dyspnoea C4D1: number analyzed (Participants) | 170 | 163
  Dyspnoea C4D1 | -0.20 (23.36) | 1.43 (21.07)
  Dyspnoea C4D22: number analyzed (Participants) | 123 | 128
  Dyspnoea C4D22 | 2.71 (20.29) | 0.26 (20.28)
  Dyspnoea C5D1: number analyzed (Participants) | 149 | 145
  Dyspnoea C5D1 | 2.24 (20.75) | -0.46 (24.21)
  Dyspnoea C5D22: number analyzed (Participants) | 111 | 116
  Dyspnoea C5D22 | 2.10 (22.15) | 1.44 (22.15)
  Dyspnoea C6D1: number analyzed (Participants) | 123 | 122
  Dyspnoea C6D1 | 0.81 (22.77) | 3.28 (22.02)
  Dyspnoea C6D22: number analyzed (Participants) | 103 | 94
  Dyspnoea C6D22 | 0.65 (20.86) | 1.42 (20.69)
  Dyspnoea C7D1: number analyzed (Participants) | 114 | 98
  Dyspnoea C7D1 | 4.09 (21.33) | -1.02 (19.42)
  Dyspnoea C7D22: number analyzed (Participants) | 81 | 74
  Dyspnoea C7D22 | 4.94 (19.80) | -2.25 (21.60)
  Dyspnoea C8D1: number analyzed (Participants) | 80 | 83
  Dyspnoea C8D1 | 3.75 (20.54) | -0.40 (21.77)
  Dyspnoea C8D22: number analyzed (Participants) | 72 | 65
  Dyspnoea C8D22 | 1.85 (18.46) | -3.59 (18.75)
  Dyspnoea C9D1: number analyzed (Participants) | 75 | 62
  Dyspnoea C9D1 | 1.78 (18.90) | -3.23 (19.75)
  Dyspnoea C9D22: number analyzed (Participants) | 60 | 55
  Dyspnoea C9D22 | 3.33 (27.92) | -3.64 (21.92)
  Dyspnoea C10D1: number analyzed (Participants) | 66 | 56
  Dyspnoea C10D1 | 1.52 (25.10) | 0.00 (22.92)
  Dyspnoea C10D22: number analyzed (Participants) | 57 | 43
  Dyspnoea C10D22 | 2.34 (18.75) | 1.55 (24.07)
  Dyspnoea C11D1: number analyzed (Participants) | 63 | 46
  Dyspnoea C11D1 | -0.53 (17.45) | 0.00 (17.21)
  Dyspnoea C11D22: number analyzed (Participants) | 44 | 31
  Dyspnoea C11D22 | 2.27 (18.18) | 2.15 (28.46)
  Dyspnoea C12D1: number analyzed (Participants) | 53 | 41
  Dyspnoea C12D1 | 4.40 (16.06) | 0.00 (21.08)
  Dyspnoea C12D22: number analyzed (Participants) | 38 | 25
  Dyspnoea C12D22 | 2.63 (16.22) | 5.33 (15.75)
  Dyspnoea C13D1: number analyzed (Participants) | 48 | 35
  Dyspnoea C13D1 | 2.78 (15.12) | 0.95 (22.12)
  Dyspnoea C13D22: number analyzed (Participants) | 41 | 21
  Dyspnoea C13D22 | 3.25 (16.34) | -1.59 (26.82)
  Dyspnoea C14D1: number analyzed (Participants) | 39 | 30
  Dyspnoea C14D1 | 0.85 (16.20) | 0.00 (24.76)
  Dyspnoea C14D22: number analyzed (Participants) | 32 | 19
  Dyspnoea C14D22 | 0.00 (16.93) | -3.51 (26.98)
  Dyspnoea C15D1: number analyzed (Participants) | 35 | 27
  Dyspnoea C15D1 | -0.95 (20.59) | -1.23 (26.92)
  Dyspnoea C15D22: number analyzed (Participants) | 30 | 17
  Dyspnoea C15D22 | -2.22 (14.99) | -3.92 (28.58)
  Dyspnoea C16D1: number analyzed (Participants) | 35 | 22
  Dyspnoea C16D1 | 1.90 (13.87) | -1.52 (26.18)
  Dyspnoea C16D22: number analyzed (Participants) | 29 | 14
  Dyspnoea C16D22 | 4.60 (19.36) | 4.76 (17.82)
  Dyspnoea C17D1: number analyzed (Participants) | 30 | 18
  Dyspnoea C17D1 | 2.22 (17.36) | 0.00 (16.17)
  Dyspnoea C17D22: number analyzed (Participants) | 23 | 0
  Dyspnoea C17D22 | 2.90 (19.88) |
  Dyspnoea C18D1: number analyzed (Participants) | 27 | 16
  Dyspnoea C18D1 | 0.00 (13.07) | 2.08 (19.12)
  Dyspnoea C18D22: number analyzed (Participants) | 21 | 10
  Dyspnoea C18D22 | 4.76 (19.11) | -3.33 (18.92)
  Dyspnoea C19D1: number analyzed (Participants) | 23 | 15
  Dyspnoea C19D1 | 2.90 (13.90) | -2.22 (15.26)
  Dyspnoea C19D22: number analyzed (Participants) | 20 | 11
  Dyspnoea C19D22 | 3.33 (14.91) | 0.00 (25.82)
  Dyspnoea C20D1: number analyzed (Participants) | 23 | 15
  Dyspnoea C20D1 | 1.45 (12.22) | 2.22 (23.46)
  Dyspnoea C20D22: number analyzed (Participants) | 18 | 10
  Dyspnoea C20D22 | 1.85 (7.86) | -6.67 (14.05)
  Dyspnoea C21D1: number analyzed (Participants) | 20 | 14
  Dyspnoea C21D1 | 0.00 (0.00) | 4.76 (25.68)
  Dyspnoea C21D22: number analyzed (Participants) | 14 | 0
  Dyspnoea C21D22 | 2.38 (8.91) |
  Dyspnoea C22D1: number analyzed (Participants) | 15 | 12
  Dyspnoea C22D1 | -2.22 (8.61) | 0.00 (20.10)
  Dyspnoea C22D22: number analyzed (Participants) | 11 | 0
  Dyspnoea C22D22 | 0.00 (14.91) |
  Dyspnoea C23D1: number analyzed (Participants) | 16 | 13
  Dyspnoea C23D1 | 6.25 (21.84) | 0.00 (19.25)
  Dyspnoea C23D22: number analyzed (Participants) | 11 | 0
  Dyspnoea C23D22 | 0.00 (14.91) |
  Dyspnoea C24D1: number analyzed (Participants) | 14 | 0
  Dyspnoea C24D1 | 0.00 (13.07) |
  Dyspnoea C24D22: number analyzed (Participants) | 0 | 0
  Dyspnoea C25D1: number analyzed (Participants) | 12 | 0
  Dyspnoea C25D1 | -5.56 (12.97) |
  Dyspnoea C25D22: number analyzed (Participants) | 11 | 0
  Dyspnoea C25D22 | -3.03 (10.05) |
  Dyspnoea C26D1: number analyzed (Participants) | 13 | 0
  Dyspnoea C26D1 | -2.56 (9.25) |
  Dyspnoea C27D1: number analyzed (Participants) | 11 | 0
  Dyspnoea C27D1 | 0.00 (14.91) |
  Dyspnoea C28D1: number analyzed (Participants) | 12 | 0
  Dyspnoea C28D1 | -2.78 (9.62) |
  Dyspnoea 30 Day Follow up: number analyzed (Participants) | 72 | 91
  Dyspnoea 30 Day Follow up | 4.63 (23.94) | 5.49 (21.81)
  Dyspnoea 90 Day Follow up: number analyzed (Participants) | 86 | 83
  Dyspnoea 90 Day Follow up | 13.57 (29.98) | 12.05 (27.83)
  Insomnia Baseline | 27.50 (28.50) | 29.59 (28.64)
  Insomnia C1D22: number analyzed (Participants) | 177 | 210
  Insomnia C1D22 | 0.00 (27.52) | -3.81 (29.28)
  Insomnia C2D1: number analyzed (Participants) | 207 | 225
  Insomnia C2D1 | -4.03 (29.92) | -6.22 (29.73)
  Insomnia C2D22: number analyzed (Participants) | 150 | 181
  Insomnia C2D22 | -5.33 (29.18) | -8.84 (28.68)
  Insomnia C3D1: number analyzed (Participants) | 190 | 198
  Insomnia C3D1 | -8.42 (30.85) | -10.27 (30.98)
  Insomnia C3D22: number analyzed (Participants) | 152 | 149
  Insomnia C3D22 | -5.26 (27.69) | -10.07 (31.17)
  Insomnia C4D1: number analyzed (Participants) | 170 | 163
  Insomnia C4D1 | -10.59 (29.55) | -11.86 (30.47)
  Insomnia C4D22: number analyzed (Participants) | 123 | 128
  Insomnia C4D22 | -5.42 (31.47) | -11.46 (29.11)
  Insomnia C5D1: number analyzed (Participants) | 149 | 145
  Insomnia C5D1 | -5.59 (32.28) | -8.97 (34.30)
  Insomnia C5D22: number analyzed (Participants) | 111 | 116
  Insomnia C5D22 | -6.01 (32.47) | -7.47 (30.16)
  Insomnia C6D1: number analyzed (Participants) | 123 | 122
  Insomnia C6D1 | -6.50 (32.13) | -8.47 (31.36)
  Insomnia C6D22: number analyzed (Participants) | 103 | 94
  Insomnia C6D22 | -4.21 (29.03) | -12.77 (30.57)
  Insomnia C7D1: number analyzed (Participants) | 114 | 98
  Insomnia C7D1 | -7.02 (27.86) | -11.90 (28.82)
  Insomnia C7D22: number analyzed (Participants) | 81 | 74
  Insomnia C7D22 | -4.94 (23.64) | -13.96 (25.29)
  Insomnia C8D1: number analyzed (Participants) | 80 | 83
  Insomnia C8D1 | -6.67 (26.73) | -8.84 (29.49)
  Insomnia C8D22: number analyzed (Participants) | 72 | 65
  Insomnia C8D22 | -6.94 (27.37) | -14.36 (24.98)
  Insomnia C9D1: number analyzed (Participants) | 75 | 62
  Insomnia C9D1 | -8.44 (29.05) | -13.98 (25.99)
  Insomnia C9D22: number analyzed (Participants) | 60 | 55
  Insomnia C9D22 | -8.89 (32.97) | -11.52 (30.24)
  Insomnia C10D1: number analyzed (Participants) | 66 | 56
  Insomnia C10D1 | -8.59 (27.62) | -8.33 (33.78)
  Insomnia C10D22: number analyzed (Participants) | 57 | 43
  Insomnia C10D22 | -9.94 (26.70) | -10.85 (29.74)
  Insomnia C11D1: number analyzed (Participants) | 63 | 46
  Insomnia C11D1 | -8.99 (27.57) | -10.14 (26.17)
  Insomnia C11D22: number analyzed (Participants) | 44 | 31
  Insomnia C11D22 | -11.36 (26.84) | -10.75 (29.04)
  Insomnia C12D1: number analyzed (Participants) | 53 | 41
  Insomnia C12D1 | -8.18 (29.17) | -12.20 (30.51)
  Insomnia C12D22: number analyzed (Participants) | 38 | 25
  Insomnia C12D22 | -3.51 (26.61) | -8.00 (25.96)
  Insomnia C13D1: number analyzed (Participants) | 48 | 35
  Insomnia C13D1 | -6.25 (32.73) | -10.48 (22.54)
  Insomnia C13D22: number analyzed (Participants) | 41 | 21
  Insomnia C13D22 | -9.76 (28.13) | -11.11 (19.25)
  Insomnia C14D1: number analyzed (Participants) | 39 | 30
  Insomnia C14D1 | -9.40 (25.30) | -5.56 (27.80)
  Insomnia C14D22: number analyzed (Participants) | 32 | 19
  Insomnia C14D22 | -7.29 (29.00) | -8.77 (26.86)
  Insomnia C15D1: number analyzed (Participants) | 35 | 27
  Insomnia C15D1 | -7.62 (30.34) | -6.17 (24.52)
  Insomnia C15D22: number analyzed (Participants) | 30 | 17
  Insomnia C15D22 | -8.89 (26.16) | -3.92 (26.04)
  Insomnia C16D1: number analyzed (Participants) | 35 | 22
  Insomnia C16D1 | -9.52 (28.66) | -1.52 (24.07)
  Insomnia C16D22: number analyzed (Participants) | 29 | 14
  Insomnia C16D22 | -9.20 (23.40) | -7.14 (29.75)
  Insomnia C17D1: number analyzed (Participants) | 30 | 18
  Insomnia C17D1 | -4.44 (33.60) | -7.41 (29.27)
  Insomnia C17D22: number analyzed (Participants) | 23 | 0
  Insomnia C17D22 | -4.35 (30.66) |
  Insomnia C18D1: number analyzed (Participants) | 27 | 16
  Insomnia C18D1 | -9.88 (28.96) | 0.00 (21.08)
  Insomnia C18D22: number analyzed (Participants) | 21 | 10
  Insomnia C18D22 | -1.59 (28.82) | 6.67 (21.08)
  Insomnia C19D1: number analyzed (Participants) | 23 | 15
  Insomnia C19D1 | -8.70 (28.81) | -2.22 (29.46)
  Insomnia C19D22: number analyzed (Participants) | 20 | 11
  Insomnia C19D22 | -8.33 (28.36) | 12.12 (22.47)
  Insomnia C20D1: number analyzed (Participants) | 23 | 15
  Insomnia C20D1 | -10.14 (29.19) | -4.44 (21.33)
  Insomnia C20D22: number analyzed (Participants) | 18 | 10
  Insomnia C20D22 | -9.26 (31.94) | 10.00 (27.44)
  Insomnia C21D1: number analyzed (Participants) | 20 | 14
  Insomnia C21D1 | -6.67 (25.59) | 2.38 (27.62)
  Insomnia C21D22: number analyzed (Participants) | 14 | 0
  Insomnia C21D22 | -9.52 (24.21) |
  Insomnia C22D1: number analyzed (Participants) | 15 | 12
  Insomnia C22D1 | -6.67 (25.82) | 2.78 (22.29)
  Insomnia C22D22: number analyzed (Participants) | 11 | 0
  Insomnia C22D22 | -3.03 (27.71) |
  Insomnia C23D1: number analyzed (Participants) | 16 | 13
  Insomnia C23D1 | -2.08 (28.46) | -2.56 (25.32)
  Insomnia C23D22: number analyzed (Participants) | 11 | 0
  Insomnia C23D22 | -6.06 (29.13) |
  Insomnia C24D1: number analyzed (Participants) | 14 | 0
  Insomnia C24D1 | -7.14 (26.73) |
  Insomnia C24D22: number analyzed (Participants) | 0 | 0
  Insomnia C25D1: number analyzed (Participants) | 12 | 0
  Insomnia C25D1 | 0.00 (24.62) |
  Insomnia C25D22: number analyzed (Participants) | 11 | 0
  Insomnia C25D22 | -3.03 (31.46) |
  Insomnia C26D1: number analyzed (Participants) | 13 | 0
  Insomnia C26D1 | -7.69 (27.74) |
  Insomnia C27D1: number analyzed (Participants) | 11 | 0
  Insomnia C27D1 | -9.09 (30.15) |
  Insomnia C28D1: number analyzed (Participants) | 12 | 0
  Insomnia C28D1 | -5.56 (27.83) |
  Insomnia 30 Day Follow up: number analyzed (Participants) | 72 | 91
  Insomnia 30 Day Follow up | -2.31 (28.71) | -2.93 (33.94)
  Insomnia 90 Day Follow up: number analyzed (Participants) | 86 | 83
  Insomnia 90 Day Follow up | 1.94 (29.53) | -3.21 (39.51)
  Appetite Loss Baseline | 32.81 (32.14) | 32.17 (31.44)
  Appetite Loss C1D22: number analyzed (Participants) | 177 | 210
  Appetite Loss C1D22 | 9.04 (33.05) | 4.13 (33.00)
  Appetite Loss C2D1: number analyzed (Participants) | 207 | 225
  Appetite Loss C2D1 | -4.99 (36.01) | -8.00 (31.74)
  Appetite Loss C2D22: number analyzed (Participants) | 150 | 181
  Appetite Loss C2D22 | -1.33 (34.08) | 0.18 (35.57)
  Appetite Loss C3D1: number analyzed (Participants) | 190 | 198
  Appetite Loss C3D1 | -8.07 (34.53) | -8.75 (31.18)
  Appetite Loss C3D22: number analyzed (Participants) | 152 | 149
  Appetite Loss C3D22 | 2.19 (35.71) | -2.68 (30.39)
  Appetite Loss C4D1: number analyzed (Participants) | 170 | 163
  Appetite Loss C4D1 | -6.08 (38.49) | -7.36 (34.35)
  Appetite Loss C4D22: number analyzed (Participants) | 123 | 128
  Appetite Loss C4D22 | 1.90 (38.01) | -4.95 (31.05)
  Appetite Loss C5D1: number analyzed (Participants) | 149 | 145
  Appetite Loss C5D1 | -4.03 (35.92) | -8.28 (30.31)
  Appetite Loss C5D22: number analyzed (Participants) | 111 | 116
  Appetite Loss C5D22 | -0.30 (37.20) | -6.03 (30.33)
  Appetite Loss C6D1: number analyzed (Participants) | 123 | 122
  Appetite Loss C6D1 | -6.50 (37.37) | -5.19 (31.50)
  Appetite Loss C6D22: number analyzed (Participants) | 103 | 94
  Appetite Loss C6D22 | -6.15 (39.81) | -8.51 (30.50)
  Appetite Loss C7D1: number analyzed (Participants) | 114 | 98
  Appetite Loss C7D1 | -9.65 (36.76) | -10.20 (28.48)
  Appetite Loss C7D22: number analyzed (Participants) | 81 | 74
  Appetite Loss C7D22 | -4.94 (39.48) | -11.26 (31.35)
  Appetite Loss C8D1: number analyzed (Participants) | 80 | 83
  Appetite Loss C8D1 | -8.75 (35.48) | -8.43 (28.91)
  Appetite Loss C8D22: number analyzed (Participants) | 72 | 65
  Appetite Loss C8D22 | -8.80 (38.76) | -4.10 (28.57)
  Appetite Loss C9D1: number analyzed (Participants) | 75 | 62
  Appetite Loss C9D1 | -15.56 (34.37) | -5.91 (32.24)
  Appetite Loss C9D22: number analyzed (Participants) | 60 | 55
  Appetite Loss C9D22 | -13.33 (41.26) | -1.82 (27.53)
  Appetite Loss C10D1: number analyzed (Participants) | 66 | 56
  Appetite Loss C10D1 | -10.10 (38.33) | -5.36 (27.54)
  Appetite Loss C10D22: number analyzed (Participants) | 57 | 43
  Appetite Loss C10D22 | -5.85 (37.86) | 0.78 (33.72)
  Appetite Loss C11D1: number analyzed (Participants) | 63 | 46
  Appetite Loss C11D1 | -15.34 (36.82) | -2.17 (28.46)
  Appetite Loss C11D22: number analyzed (Participants) | 44 | 31
  Appetite Loss C11D22 | -12.12 (33.79) | -6.45 (31.53)
  Appetite Loss C12D1: number analyzed (Participants) | 53 | 41
  Appetite Loss C12D1 | -10.69 (33.83) | -5.69 (28.77)
  Appetite Loss C12D22: number analyzed (Participants) | 38 | 25
  Appetite Loss C12D22 | 1.75 (31.90) | -5.33 (28.35)
  Appetite Loss C13D1: number analyzed (Participants) | 48 | 35
  Appetite Loss C13D1 | -9.72 (33.66) | -4.76 (30.40)
  Appetite Loss C13D22: number analyzed (Participants) | 41 | 21
  Appetite Loss C13D22 | -5.69 (39.37) | 7.94 (29.64)
  Appetite Loss C14D1: number analyzed (Participants) | 39 | 30
  Appetite Loss C14D1 | -10.26 (35.17) | 0.00 (27.68)
  Appetite Loss C14D22: number analyzed (Participants) | 32 | 19
  Appetite Loss C14D22 | -6.25 (39.20) | -7.02 (21.02)
  Appetite Loss C15D1: number analyzed (Participants) | 35 | 27
  Appetite Loss C15D1 | -6.67 (39.44) | -6.17 (27.79)
  Appetite Loss C15D22: number analyzed (Participants) | 30 | 17
  Appetite Loss C15D22 | -5.56 (42.96) | -7.84 (25.08)
  Appetite Loss C16D1: number analyzed (Participants) | 35 | 22
  Appetite Loss C16D1 | -14.29 (27.16) | -7.58 (22.84)
  Appetite Loss C16D22: number analyzed (Participants) | 29 | 14
  Appetite Loss C16D22 | -6.90 (39.22) | -7.14 (23.31)
  Appetite Loss C17D1: number analyzed (Participants) | 30 | 18
  Appetite Loss C17D1 | -12.22 (33.31) | -5.56 (23.57)
  Appetite Loss C17D22: number analyzed (Participants) | 23 | 0
  Appetite Loss C17D22 | -4.35 (32.26) |
  Appetite Loss C18D1: number analyzed (Participants) | 27 | 16
  Appetite Loss C18D1 | -14.81 (31.12) | -4.17 (29.50)
  Appetite Loss C18D22: number analyzed (Participants) | 21 | 10
  Appetite Loss C18D22 | -7.94 (27.70) | -10.00 (27.44)
  Appetite Loss C19D1: number analyzed (Participants) | 23 | 15
  Appetite Loss C19D1 | -11.59 (23.80) | -2.22 (29.46)
  Appetite Loss C19D22: number analyzed (Participants) | 20 | 11
  Appetite Loss C19D22 | -8.33 (23.88) | -6.06 (25.03)
  Appetite Loss C20D1: number analyzed (Participants) | 23 | 15
  Appetite Loss C20D1 | -10.14 (27.40) | -8.89 (23.46)
  Appetite Loss C20D22: number analyzed (Participants) | 18 | 10
  Appetite Loss C20D22 | 1.85 (33.28) | -10.00 (27.44)
  Appetite Loss C21D1: number analyzed (Participants) | 20 | 14
  Appetite Loss C21D1 | -6.67 (23.20) | -7.14 (19.30)
  Appetite Loss C21D22: number analyzed (Participants) | 14 | 0
  Appetite Loss C21D22 | -7.14 (23.31) |
  Appetite Loss C22D1: number analyzed (Participants) | 15 | 12
  Appetite Loss C22D1 | -13.33 (21.08) | -11.11 (25.95)
  Appetite Loss C22D22: number analyzed (Participants) | 11 | 0
  Appetite Loss C22D22 | -6.06 (32.72) |
  Appetite Loss C23D1: number analyzed (Participants) | 16 | 13
  Appetite Loss C23D1 | -6.25 (25.00) | -7.69 (27.74)
  Appetite Loss C2322: number analyzed (Participants) | 11 | 0
  Appetite Loss C2322 | -9.09 (26.21) |
  Appetite Loss C24D1: number analyzed (Participants) | 14 | 0
  Appetite Loss C24D1 | -11.90 (24.83) |
  Appetite Loss C24D22: number analyzed (Participants) | 0 | 0
  Appetite Loss C25D1: number analyzed (Participants) | 12 | 0
  Appetite Loss C25D1 | -2.78 (33.21) |
  Appetite Loss C25D22: number analyzed (Participants) | 11 | 0
  Appetite Loss C25D22 | -3.03 (27.71) |
  Appetite Loss C26D1: number analyzed (Participants) | 13 | 0
  Appetite Loss C26D1 | -10.26 (28.50) |
  Appetite Loss C27D1: number analyzed (Participants) | 11 | 0
  Appetite Loss C27D1 | -3.03 (17.98) |
  Appetite Loss C28D1: number analyzed (Participants) | 12 | 0
  Appetite Loss C28D1 | 0.00 (28.43) |
  Appetite Loss 30 Day Follow up: number analyzed (Participants) | 72 | 91
  Appetite Loss 30 Day Follow up | 2.31 (31.81) | 3.30 (32.60)
  Appetite Loss 90 Day Follow up: number analyzed (Participants) | 86 | 83
  Appetite Loss 90 Day Follow up | -5.04 (35.62) | 7.63 (39.07)
  Constipation Baseline | 19.33 (28.15) | 19.64 (28.39)
  Constipation C1D22: number analyzed (Participants) | 177 | 210
  Constipation C1D22 | 8.66 (32.96) | 4.44 (29.91)
  Constipation C2D1: number analyzed (Participants) | 207 | 225
  Constipation C2D1 | -0.48 (33.25) | -2.37 (32.80)
  Constipation C2D22: number analyzed (Participants) | 150 | 181
  Constipation C2D22 | -2.89 (31.12) | 0.37 (31.23)
  Constipation C3D1: number analyzed (Participants) | 190 | 198
  Constipation C3D1 | -5.09 (31.29) | -2.53 (30.40)
  Constipation C3D22: number analyzed (Participants) | 152 | 149
  Constipation C3D22 | -2.85 (28.18) | -0.89 (31.70)
  Constipation C4D1: number analyzed (Participants) | 170 | 163
  Constipation C4D1 | -2.75 (32.11) | -1.02 (28.79)
  Constipation C4D22: number analyzed (Participants) | 123 | 128
  Constipation C4D22 | 1.08 (31.92) | 2.08 (28.91)
  Constipation C5D1: number analyzed (Participants) | 149 | 145
  Constipation C5D1 | -2.24 (31.16) | -1.15 (30.79)
  Constipation C5D22: number analyzed (Participants) | 111 | 116
  Constipation C5D22 | 2.70 (31.83) | -1.44 (26.88)
  Constipation C6D1: number analyzed (Participants) | 123 | 122
  Constipation C6D1 | -2.44 (28.04) | 0.55 (28.42)
  Constipation C6D22: number analyzed (Participants) | 103 | 94
  Constipation C6D22 | -3.24 (27.82) | -1.77 (30.67)
  Constipation C7D1: number analyzed (Participants) | 114 | 98
  Constipation C7D1 | -2.63 (29.80) | -1.36 (29.08)
  Constipation C7D22: number analyzed (Participants) | 81 | 74
  Constipation C7D22 | -2.47 (25.70) | -4.05 (32.62)
  Constipation C8D1: number analyzed (Participants) | 80 | 83
  Constipation C8D1 | -4.17 (27.75) | -0.40 (29.67)
  Constipation C8D22: number analyzed (Participants) | 72 | 65
  Constipation C8D22 | -6.94 (29.04) | -2.56 (25.21)
  Constipation C9D1: number analyzed (Participants) | 75 | 62
  Constipation C9D1 | -8.44 (26.90) | 0.00 (28.95)
  Constipation C9D22: number analyzed (Participants) | 60 | 55
  Constipation C9D22 | -3.33 (32.88) | 2.42 (33.24)
  Constipation C10D1: number analyzed (Participants) | 66 | 56
  Constipation C10D1 | -2.02 (29.74) | 4.17 (30.53)
  Constipation C10D22: number analyzed (Participants) | 57 | 43
  Constipation C10D22 | -1.17 (22.68) | 7.75 (31.57)
  Constipation C11D1: number analyzed (Participants) | 63 | 46
  Constipation C11D1 | -4.23 (24.31) | 7.25 (31.36)
  Constipation C11D22: number analyzed (Participants) | 44 | 31
  Constipation C11D22 | -4.55 (26.50) | 6.45 (24.97)
  Constipation C12D1: number analyzed (Participants) | 53 | 41
  Constipation C12D1 | -6.29 (22.70) | 10.57 (32.86)
  Constipation C12D22: number analyzed (Participants) | 38 | 25
  Constipation C12D22 | 1.75 (29.96) | 18.67 (34.80)
  Constipation C13D1: number analyzed (Participants) | 48 | 35
  Constipation C13D1 | -3.47 (26.84) | 10.48 (35.95)
  Constipation C13D22: number analyzed (Participants) | 41 | 21
  Constipation C13D22 | -3.25 (28.68) | 11.11 (39.91)
  Constipation C14D1: number analyzed (Participants) | 39 | 30
  Constipation C14D1 | -8.55 (25.04) | 11.11 (36.44)
  Constipation C14D22: number analyzed (Participants) | 32 | 19
  Constipation C14D22 | -3.12 (30.95) | 3.51 (33.14)
  Constipation C15D1: number analyzed (Participants) | 35 | 27
  Constipation C15D1 | -8.57 (30.62) | 6.17 (32.08)
  Constipation C15D22: number analyzed (Participants) | 30 | 17
  Constipation C15D22 | -6.67 (25.37) | 3.92 (35.12)
  Constipation C16D1: number analyzed (Participants) | 35 | 22
  Constipation C16D1 | -5.71 (24.90) | 7.58 (36.99)
  Constipation C16D22: number analyzed (Participants) | 29 | 14
  Constipation C16D22 | -3.45 (27.23) | 14.29 (40.75)
  Constipation C17D1: number analyzed (Participants) | 30 | 18
  Constipation C17D1 | -5.56 (27.80) | 1.85 (29.09)
  Constipation C17D22: number analyzed (Participants) | 23 | 0
  Constipation C17D22 | -7.25 (26.51) |
  Constipation C18D1: number analyzed (Participants) | 27 | 16
  Constipation C18D1 | -8.64 (23.74) | 10.42 (33.82)
  Constipation C18D22: number analyzed (Participants) | 21 | 10
  Constipation C18D22 | -1.59 (24.67) | 6.67 (37.84)
  Constipation C19D1: number analyzed (Participants) | 23 | 15
  Constipation C19D1 | -2.90 (28.27) | 15.56 (37.52)
  Constipation C19D22: number analyzed (Participants) | 20 | 11
  Constipation C19D22 | -5.00 (22.36) | 18.18 (37.61)
  Constipation C20D1: number analyzed (Participants) | 23 | 15
  Constipation C20D1 | -2.90 (24.44) | 11.11 (34.88)
  Constipation C20D22: number analyzed (Participants) | 18 | 10
  Constipation C20D22 | -7.41 (26.95) | 3.33 (29.19)
  Constipation C21D1: number analyzed (Participants) | 20 | 14
  Constipation C21D1 | -3.33 (26.27) | 14.29 (33.88)
  Constipation C21D22: number analyzed (Participants) | 14 | 0
  Constipation C21D22 | 0.00 (29.24) |
  Constipation C22D1: number analyzed (Participants) | 15 | 12
  Constipation C22D1 | -6.67 (25.82) | 2.78 (30.01)
  Constipation C22D22: number analyzed (Participants) | 11 | 0
  Constipation C22D22 | -6.06 (29.13) |
  Constipation C23D1: number analyzed (Participants) | 16 | 13
  Constipation C23D1 | -4.17 (26.87) | 17.95 (35.00)
  Constipation C23D22: number analyzed (Participants) | 11 | 0
  Constipation C23D22 | -3.03 (17.98) |
  Constipation C24D1: number analyzed (Participants) | 14 | 0
  Constipation C24D1 | -9.52 (27.51) |
  Constipation C24D22: number analyzed (Participants) | 0 | 0
  Constipation C25D1: number analyzed (Participants) | 12 | 0
  Constipation C25D1 | 2.78 (30.01) |
  Constipation C25D22: number analyzed (Participants) | 11 | 0
  Constipation C25D22 | -3.03 (31.46) |
  Constipation C26D1: number analyzed (Participants) | 13 | 0
  Constipation C26D1 | -5.13 (32.90) |
  Constipation C27D1: number analyzed (Participants) | 11 | 0
  Constipation C27D1 | 0.00 (33.33) |
  Constipation C28D1: number analyzed (Participants) | 12 | 0
  Constipation C28D1 | -5.56 (31.25) |
  Constipation 30 Day Follow up: number analyzed (Participants) | 72 | 91
  Constipation 30 Day Follow up | 0.00 (32.14) | 2.56 (34.15)
  Constipation 90 Day Follow up: number analyzed (Participants) | 86 | 83
  Constipation 90 Day Follow up | -5.43 (33.86) | 1.20 (30.11)
  Diarrhoea Baseline | 7.91 (17.25) | 10.59 (19.94)
  Diarrhoea C1D22: number analyzed (Participants) | 177 | 210
  Diarrhoea C1D22 | 4.90 (23.05) | 2.86 (24.01)
  Diarrhoea C2D1: number analyzed (Participants) | 207 | 225
  Diarrhoea C2D1 | 6.28 (26.03) | 2.96 (22.52)
  Diarrhoea C2D22: number analyzed (Participants) | 150 | 181
  Diarrhoea C2D22 | 4.67 (24.74) | 0.92 (22.06)
  Diarrhoea C3D1: number analyzed (Participants) | 190 | 198
  Diarrhoea C3D1 | 2.11 (22.39) | 1.18 (24.99)
  Diarrhoea C3D22: number analyzed (Participants) | 152 | 149
  Diarrhoea C3D22 | 2.19 (24.16) | 1.57 (24.91)
  Diarrhoea C4D1: number analyzed (Participants) | 170 | 163
  Diarrhoea C4D1 | -0.20 (22.20) | 1.02 (24.12)
  Diarrhoea C4D22: number analyzed (Participants) | 123 | 128
  Diarrhoea C4D22 | 1.90 (23.49) | -0.78 (24.91)
  Diarrhoea C5D1: number analyzed (Participants) | 149 | 145
  Diarrhoea C5D1 | 3.58 (24.55) | -0.92 (25.44)
  Diarrhoea C5D22: number analyzed (Participants) | 111 | 116
  Diarrhoea C5D22 | 0.30 (20.84) | -4.31 (22.64)
  Diarrhoea C6D1: number analyzed (Participants) | 123 | 122
  Diarrhoea C6D1 | -2.17 (22.48) | -1.37 (24.01)
  Diarrhoea C6D22: number analyzed (Participants) | 103 | 94
  Diarrhoea C6D22 | -3.24 (17.16) | -1.77 (23.63)
  Diarrhoea C7D1: number analyzed (Participants) | 114 | 98
  Diarrhoea C7D1 | -3.51 (20.50) | -2.04 (24.32)
  Diarrhoea C7D22: number analyzed (Participants) | 81 | 74
  Diarrhoea C7D22 | 0.41 (22.04) | -7.66 (23.11)
  Diarrhoea C8D1: number analyzed (Participants) | 80 | 83
  Diarrhoea C8D1 | -2.08 (20.78) | -2.81 (22.81)
  Diarrhoea C8D22: number analyzed (Participants) | 72 | 65
  Diarrhoea C8D22 | -5.09 (22.14) | -2.05 (22.73)
  Diarrhoea C9D1: number analyzed (Participants) | 75 | 62
  Diarrhoea C9D1 | -2.22 (26.47) | -2.69 (18.40)
  Diarrhoea C9D22: number analyzed (Participants) | 60 | 55
  Diarrhoea C9D22 | -5.00 (20.19) | -3.03 (22.47)
  Diarrhoea C10D1: number analyzed (Participants) | 66 | 56
  Diarrhoea C10D1 | -5.05 (24.97) | -1.79 (19.51)
  Diarrhoea C10D22: number analyzed (Participants) | 57 | 43
  Diarrhoea C10D22 | -2.92 (24.62) | -1.55 (21.77)
  Diarrhoea C11D1: number analyzed (Participants) | 63 | 46
  Diarrhoea C11D1 | -4.76 (26.00) | 0.72 (22.76)
  Diarrhoea C11D22: number analyzed (Participants) | 44 | 31
  Diarrhoea C11D22 | -4.55 (18.46) | -2.15 (24.24)
  Diarrhoea C12D1: number analyzed (Participants) | 53 | 41
  Diarrhoea C12D1 | 0.00 (23.57) | -3.25 (19.44)
  Diarrhoea C12D22: number analyzed (Participants) | 38 | 25
  Diarrhoea C12D22 | -1.75 (20.43) | -4.00 (20.00)
  Diarrhoea C13D1: number analyzed (Participants) | 48 | 35
  Diarrhoea C13D1 | -3.47 (30.93) | 2.86 (27.26)
  Diarrhoea C13D22: number analyzed (Participants) | 41 | 21
  Diarrhoea C13D22 | -4.07 (23.80) | 4.76 (19.11)
  Diarrhoea C14D1: number analyzed (Participants) | 39 | 30
  Diarrhoea C14D1 | -1.71 (22.88) | 4.44 (29.99)
  Diarrhoea C14D22: number analyzed (Participants) | 32 | 19
  Diarrhoea C14D22 | -3.13 (21.35) | 1.75 (26.00)
  Diarrhoea C15D1: number analyzed (Participants) | 35 | 27
  Diarrhoea C15D1 | -4.76 (23.07) | -3.70 (21.35)
  Diarrhoea C15D22: number analyzed (Participants) | 30 | 17
  Diarrhoea C15D22 | -3.33 (20.25) | 0.00 (16.67)
  Diarrhoea C16D1: number analyzed (Participants) | 35 | 22
  Diarrhoea C16D1 | -6.67 (27.77) | 3.03 (32.38)
  Diarrhoea C16D22: number analyzed (Participants) | 29 | 14
  Diarrhoea C16D22 | 0.00 (25.20) | -4.76 (17.82)
  Diarrhoea C17D1: number analyzed (Participants) | 30 | 18
  Diarrhoea C17D1 | -6.67 (26.84) | -3.70 (19.43)
  Diarrhoea C17D22: number analyzed (Participants) | 23 | 0
  Diarrhoea C17D22 | -1.45 (23.52) |
  Diarrhoea C18D1: number analyzed (Participants) | 27 | 16
  Diarrhoea C18D1 | -4.94 (23.94) | -2.08 (25.73)
  Diarrhoea C18D22: number analyzed (Participants) | 21 | 10
  Diarrhoea C18D22 | 4.76 (33.81) | 0.00 (15.71)
  Diarrhoea C19D1: number analyzed (Participants) | 23 | 15
  Diarrhoea C19D1 | -1.45 (32.53) | 0.00 (25.20)
  Diarrhoea C19D22: number analyzed (Participants) | 20 | 11
  Diarrhoea C19D22 | -3.33 (21.36) | 0.00 (14.91)
  Diarrhoea C20D1: number analyzed (Participants) | 23 | 15
  Diarrhoea C20D1 | -4.35 (25.23) | -2.22 (23.46)
  Diarrhoea C20D22: number analyzed (Participants) | 18 | 10
  Diarrhoea C20D22 | -5.56 (20.61) | 3.33 (10.54)
  Diarrhoea C21D1: number analyzed (Participants) | 20 | 14
  Diarrhoea C21D1 | -5.00 (24.84) | 7.14 (19.30)
  Diarrhoea C21D22: number analyzed (Participants) | 14 | 0
  Diarrhoea C21D22 | -4.76 (22.10) |
  Diarrhoea C22D1: number analyzed (Participants) | 15 | 12
  Diarrhoea C22D1 | -8.89 (23.46) | -5.56 (23.92)
  Diarrhoea C22D22: number analyzed (Participants) | 11 | 0
  Diarrhoea C22D22 | -12.12 (22.47) |
  Diarrhoea C23D1: number analyzed (Participants) | 16 | 13
  Diarrhoea C23D1 | -8.33 (22.77) | -5.13 (22.96)
  Diarrhoea C23D22: number analyzed (Participants) | 11 | 0
  Diarrhoea C23D22 | -6.06 (25.03) |
  Diarrhoea C24D1: number analyzed (Participants) | 14 | 0
  Diarrhoea C24D1 | -11.90 (24.83) |
  Diarrhoea C24D22: number analyzed (Participants) | 0 | 0
  Diarrhoea C25D1: number analyzed (Participants) | 12 | 0
  Diarrhoea C25D1 | -16.67 (26.59) |
  Diarrhoea C25D22: number analyzed (Participants) | 11 | 0
  Diarrhoea C25D22 | -12.12 (22.47) |
  Diarrhoea C26D1: number analyzed (Participants) | 13 | 0
  Diarrhoea C26D1 | -15.38 (25.88) |
  Diarrhoea C27D1: number analyzed (Participants) | 11 | 0
  Diarrhoea C27D1 | -9.09 (21.56) |
  Diarrhoea C28D1: number analyzed (Participants) | 12 | 0
  Diarrhoea C28D1 | -11.11 (21.71) |
  Diarrhoea 30 Day Follow up: number analyzed (Participants) | 72 | 91
  Diarrhoea 30 Day Follow up | 3.24 (24.49) | 3.66 (20.76)
  Diarrhoea 90 Day Follow up: number analyzed (Participants) | 86 | 83
  Diarrhoea 90 Day Follow up | 3.88 (26.77) | 9.24 (30.49)
  Financial Difficulties Baseline | 19.58 (28.89) | 18.86 (27.38)
  Financial Difficulties C1D22: number analyzed (Participants) | 177 | 210
  Financial Difficulties C1D22 | 0.38 (24.62) | -0.48 (21.75)
  Financial Difficulties C2D1: number analyzed (Participants) | 207 | 225
  Financial Difficulties C2D1 | -1.45 (21.86) | -1.93 (24.01)
  Financial Difficulties C2D22: number analyzed (Participants) | 150 | 181
  Financial Difficulties C2D22 | -0.67 (20.96) | -1.84 (23.76)
  Financial Difficulties C3D1: number analyzed (Participants) | 190 | 198
  Financial Difficulties C3D1 | -0.88 (22.86) | -1.85 (24.26)
  Financial Difficulties C3D22: number analyzed (Participants) | 152 | 149
  Financial Difficulties C3D22 | 0.00 (21.36) | -1.12 (22.06)
  Financial Difficulties C4D1: number analyzed (Participants) | 170 | 163
  Financial Difficulties C4D1 | -2.55 (20.51) | -3.07 (22.77)
  Financial Difficulties C4D22: number analyzed (Participants) | 123 | 128
  Financial Difficulties C4D22 | -1.90 (26.41) | -0.78 (20.26)
  Financial Difficulties C5D1: number analyzed (Participants) | 149 | 145
  Financial Difficulties C5D1 | 0.67 (27.25) | -0.23 (26.79)
  Financial Difficulties C5D22: number analyzed (Participants) | 111 | 116
  Financial Difficulties C5D22 | 2.10 (23.04) | -1.72 (26.32)
  Financial Difficulties C6D1: number analyzed (Participants) | 123 | 122
  Financial Difficulties C6D1 | -1.63 (22.93) | 2.73 (25.92)
  Financial Difficulties C6D22: number analyzed (Participants) | 103 | 94
  Financial Difficulties C6D22 | -2.27 (21.52) | 0.00 (26.32)
  Financial Difficulties C7D1: number analyzed (Participants) | 114 | 98
  Financial Difficulties C7D1 | -1.46 (24.04) | 0.68 (23.92)
  Financial Difficulties C7D22: number analyzed (Participants) | 81 | 74
  Financial Difficulties C7D22 | -1.65 (22.91) | -2.70 (28.00)
  Financial Difficulties C8D1: number analyzed (Participants) | 80 | 83
  Financial Difficulties C8D1 | 0.42 (24.59) | 0.80 (26.02)
  Financial Difficulties C8D22: number analyzed (Participants) | 72 | 65
  Financial Difficulties C8D22 | -1.39 (24.67) | 1.54 (27.28)
  Financial Difficulties C9D1: number analyzed (Participants) | 75 | 62
  Financial Difficulties C9D1 | -1.33 (23.53) | -1.08 (27.64)
  Financial Difficulties C9D22: number analyzed (Participants) | 60 | 55
  Financial Difficulties C9D22 | -1.11 (28.10) | 1.82 (32.34)
  Financial Difficulties C10D1: number analyzed (Participants) | 66 | 56
  Financial Difficulties C10D1 | -1.01 (26.13) | 4.76 (31.42)
  Financial Difficulties C10D22: number analyzed (Participants) | 57 | 43
  Financial Difficulties C10D22 | -2.92 (26.19) | 3.88 (33.50)
  Financial Difficulties C11D1: number analyzed (Participants) | 63 | 46
  Financial Difficulties C11D1 | -3.17 (28.53) | 0.72 (31.02)
  Financial Difficulties C11D22: number analyzed (Participants) | 44 | 31
  Financial Difficulties C11D22 | -2.27 (31.66) | 6.45 (23.44)
  Financial Difficulties C12D1: number analyzed (Participants) | 53 | 41
  Financial Difficulties C12D1 | -1.26 (30.64) | 5.69 (23.45)
  Financial Difficulties C12D22: number analyzed (Participants) | 38 | 25
  Financial Difficulties C12D22 | -2.63 (30.39) | 2.67 (25.31)
  Financial Difficulties C13D1: number analyzed (Participants) | 48 | 35
  Financial Difficulties C13D1 | -2.78 (27.36) | 3.81 (22.54)
  Financial Difficulties C13D22: number analyzed (Participants) | 41 | 21
  Financial Difficulties C13D22 | 0.81 (30.27) | -4.76 (26.43)
  Financial Difficulties C14D1: number analyzed (Participants) | 39 | 30
  Financial Difficulties C14D1 | 0.85 (22.28) | 5.56 (26.38)
  Financial Difficulties C14D22: number analyzed (Participants) | 32 | 19
  Financial Difficulties C14D22 | 0.00 (23.95) | -5.26 (27.81)
  Financial Difficulties C15D1: number analyzed (Participants) | 35 | 27
  Financial Difficulties C15D1 | -5.71 (28.57) | 6.17 (30.71)
  Financial Difficulties C15D22: number analyzed (Participants) | 30 | 17
  Financial Difficulties C15D22 | -5.56 (26.38) | -1.96 (27.56)
  Financial Difficulties C16D1: number analyzed (Participants) | 35 | 22
  Financial Difficulties C16D1 | -1.90 (24.18) | 1.52 (26.18)
  Financial Difficulties C16D22: number analyzed (Participants) | 29 | 14
  Financial Difficulties C16D22 | -1.15 (28.84) | 2.38 (27.62)
  Financial Difficulties C17D1: number analyzed (Participants) | 30 | 18
  Financial Difficulties C17D1 | -1.11 (25.50) | 1.85 (24.18)
  Financial Difficulties C17D22: number analyzed (Participants) | 23 | 0
  Financial Difficulties C17D22 | 5.80 (16.37) |
  Financial Difficulties C18D1: number analyzed (Participants) | 27 | 16
  Financial Difficulties C18D1 | 1.23 (17.25) | 2.08 (25.73)
  Financial Difficulties C18D22: number analyzed (Participants) | 21 | 10
  Financial Difficulties C18D22 | 0.00 (14.91) | 3.33 (24.60)
  Financial Difficulties C19D1: number analyzed (Participants) | 23 | 15
  Financial Difficulties C19D1 | 0.00 (17.41) | 8.89 (26.63)
  Financial Difficulties C19D22: number analyzed (Participants) | 20 | 11
  Financial Difficulties C19D22 | 5.00 (16.31) | 6.06 (32.72)
  Financial Difficulties C20D1: number analyzed (Participants) | 23 | 15
  Financial Difficulties C20D1 | 0.00 (17.41) | 4.44 (24.77)
  Financial Difficulties C20D22: number analyzed (Participants) | 18 | 10
  Financial Difficulties C20D22 | 3.70 (19.43) | 6.67 (34.43)
  Financial Difficulties C21D1: number analyzed (Participants) | 20 | 14
  Financial Difficulties C21D1 | 1.67 (22.88) | 11.90 (28.06)
  Financial Difficulties C21D22: number analyzed (Participants) | 14 | 0
  Financial Difficulties C21D22 | -7.14 (19.30) |
  Financial Difficulties C22D1: number analyzed (Participants) | 15 | 12
  Financial Difficulties C22D1 | -2.22 (19.79) | 2.78 (26.43)
  Financial Difficulties C22D22: number analyzed (Participants) | 11 | 0
  Financial Difficulties C22D22 | 0.00 (25.82) |
  Financial Difficulties C23D1: number analyzed (Participants) | 16 | 13
  Financial Difficulties C23D1 | -2.08 (19.12) | 0.00 (23.57)
  Financial Difficulties C23D22: number analyzed (Participants) | 11 | 0
  Financial Difficulties C23D22 | -6.06 (20.10) |
  Financial Difficulties C24D1: number analyzed (Participants) | 14 | 0
  Financial Difficulties C24D1 | -4.76 (22.10) |
  Financial Difficulties C24D22: number analyzed (Participants) | 0 | 0
  Financial Difficulties C25D1: number analyzed (Participants) | 12 | 0
  Financial Difficulties C25D1 | -5.56 (19.25) |
  Financial Difficulties C25D22: number analyzed (Participants) | 11 | 0
  Financial Difficulties C25D22 | -6.06 (25.03) |
  Financial Difficulties C26D1: number analyzed (Participants) | 13 | 0
  Financial Difficulties C26D1 | -5.13 (22.96) |
  Financial Difficulties C27D1: number analyzed (Participants) | 11 | 0
  Financial Difficulties C27D1 | -3.03 (23.35) |
  Financial Difficulties C28D1: number analyzed (Participants) | 12 | 0
  Financial Difficulties C28D1 | -2.78 (22.29) |
  Financial Difficulties 30 Day Follow up: number analyzed (Participants) | 72 | 91
  Financial Difficulties 30 Day Follow up | 4.17 (26.79) | 5.13 (26.26)
  Financial Difficulties 90 Day Follow up: number analyzed (Participants) | 86 | 83
  Financial Difficulties 90 Day Follow up | 7.75 (24.35) | 4.02 (31.41)

11. Secondary Outcome: Change From Baseline in HRQoL Measured by the QLQ-OG25 Questionnaire
Description: The EORTC-QLQ-OG25 consists of a 25-item instrument that evaluates gastric and GEJ cancer-specific symptoms such as stomach discomfort, difficulties eating and swallowing and indigestion. This module consists of 6 scales: dysphagia (3 items), eating restrictions (4 items), reflux (2 items), odynophagia (2 items), pain and discomfort (2 items) and anxiety (2 items), as well as 10 single items: eating in front of others, dry mouth, trouble with taste, body image, trouble swallowing saliva, choked when swallowing, trouble with coughing, trouble talking, weight loss and hair loss. All questions have four response alternatives (1:not at all; 2:a little, 3:quite a bit, 4:very much). Questionnaire responses were transformed lineraly into scores ranging from 0 to 100 For symptom scales/items, higher scores indicate worse symptoms.
Time Frame: Baseline, C1D22, D1 and D22 of C2 through C25, C26D1, C27D1,C28D1 30 day follow up, 90 day follow up
Population: FAS with available data was analyzed.
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | mFOLFOX6 + Zolbetuximab | mFOLFOX6+ Placebo
Number analyzed (Participants) | 257 | 257
unit on a scale
  Dysphagia Baseline | 18.50 (24.39) | 20.02 (26.71)
  Dysphagia C1D22: number analyzed (Participants) | 176 | 208
  Dysphagia C1D22 | 2.90 (21.18) | -1.66 (22.31)
  Dysphagia C2D1: number analyzed (Participants) | 206 | 223
  Dysphagia C2D1 | -3.83 (23.11) | -7.92 (25.87)
  Dysphagia C2D22: number analyzed (Participants) | 150 | 180
  Dysphagia C2D22 | -4.00 (22.34) | -8.46 (23.70)
  Dysphagia C3D1: number analyzed (Participants) | 190 | 196
  Dysphagia C3D1 | -8.30 (23.64) | -8.45 (24.83)
  Dysphagia C3D22: number analyzed (Participants) | 152 | 148
  Dysphagia C3D22 | -4.02 (23.60) | -9.16 (26.55)
  Dysphagia C4D1: number analyzed (Participants) | 169 | 161
  Dysphagia C4D1 | -6.64 (23.49) | -8.70 (23.49)
  Dysphagia C4D22: number analyzed (Participants) | 122 | 127
  Dysphagia C4D22 | -2.82 (22.11) | -7.26 (24.74)
  Dysphagia C5D1: number analyzed (Participants) | 148 | 144
  Dysphagia C5D1 | -6.31 (22.64) | -8.02 (24.60)
  Dysphagia C5D22: number analyzed (Participants) | 110 | 115
  Dysphagia C5D22 | -4.85 (21.84) | -7.25 (22.94)
  Dysphagia C6D1: number analyzed (Participants) | 122 | 121
  Dysphagia C6D1 | -5.37 (20.46) | -5.42 (20.34)
  Dysphagia C6D22: number analyzed (Participants) | 103 | 92
  Dysphagia C6D22 | -5.07 (20.45) | -7.61 (21.28)
  Dysphagia C7D1: number analyzed (Participants) | 113 | 98
  Dysphagia C7D1 | -6.88 (19.66) | -6.35 (20.49)
  Dysphagia C7D22: number analyzed (Participants) | 81 | 73
  Dysphagia C7D22 | -6.04 (20.49) | -8.07 (20.73)
  Dysphagia C8D1: number analyzed (Participants) | 80 | 81
  Dysphagia C8D1 | -3.89 (18.38) | -5.62 (16.02)
  Dysphagia C8D22: number analyzed (Participants) | 71 | 65
  Dysphagia C8D22 | -5.63 (17.90) | -5.64 (20.42)
  Dysphagia C9D1: number analyzed (Participants) | 75 | 62
  Dysphagia C9D1 | -6.67 (17.62) | -6.81 (18.80)
  Dysphagia C9D22: number analyzed (Participants) | 60 | 55
  Dysphagia C9D22 | -5.93 (18.35) | -3.03 (19.65)
  Dysphagia C10D1: number analyzed (Participants) | 66 | 56
  Dysphagia C10D1 | -5.56 (18.92) | -4.76 (19.40)
  Dysphagia C10D22: number analyzed (Participants) | 57 | 43
  Dysphagia C10D22 | -8.38 (17.73) | -3.10 (20.19)
  Dysphagia C11D1: number analyzed (Participants) | 63 | 46
  Dysphagia C11D1 | -6.53 (20.32) | -0.24 (23.13)
  Dysphagia C11D22: number analyzed (Participants) | 44 | 31
  Dysphagia C11D22 | -8.59 (19.59) | -1.08 (10.48)
  Dysphagia C12D1: number analyzed (Participants) | 53 | 41
  Dysphagia C12D1 | -4.19 (16.19) | -4.34 (18.90)
  Dysphagia C12D22: number analyzed (Participants) | 37 | 25
  Dysphagia C12D22 | -6.61 (19.15) | -5.33 (14.74)
  Dysphagia C13D1: number analyzed (Participants) | 48 | 35
  Dysphagia C13D1 | -6.25 (18.47) | -4.76 (17.93)
  Dysphagia C13D22: number analyzed (Participants) | 40 | 21
  Dysphagia C13D22 | -4.72 (16.28) | -6.88 (24.21)
  Dysphagia C14D1: number analyzed (Participants) | 39 | 30
  Dysphagia C14D1 | -4.27 (12.39) | -5.56 (20.37)
  Dysphagia C14D22: number analyzed (Participants) | 32 | 19
  Dysphagia C14D22 | -4.17 (13.16) | -7.02 (25.45)
  Dysphagia C15D1: number analyzed (Participants) | 35 | 27
  Dysphagia C15D1 | -2.22 (12.58) | -5.76 (19.58)
  Dysphagia C15D22: number analyzed (Participants) | 29 | 17
  Dysphagia C15D22 | -4.98 (14.72) | -6.54 (27.23)
  Dysphagia C16D1: number analyzed (Participants) | 35 | 22
  Dysphagia C16D1 | -4.44 (15.29) | -4.55 (26.49)
  Dysphagia C16D22: number analyzed (Participants) | 29 | 14
  Dysphagia C16D22 | -2.30 (15.82) | -8.73 (28.97)
  Dysphagia C17D1: number analyzed (Participants) | 30 | 18
  Dysphagia C17D1 | -2.22 (15.82) | -6.79 (24.74)
  Dysphagia C17D22: number analyzed (Participants) | 23 | 0
  Dysphagia C17D22 | -4.35 (18.87) |
  Dysphagia C18D1: number analyzed (Participants) | 27 | 16
  Dysphagia C18D1 | -5.76 (15.83) | -7.64 (23.21)
  Dysphagia C18D22: number analyzed (Participants) | 20 | 10
  Dysphagia C18D22 | -6.11 (14.18) | -6.67 (16.73)
  Dysphagia C19D1: number analyzed (Participants) | 23 | 15
  Dysphagia C19D1 | -3.38 (14.38) | -2.22 (16.90)
  Dysphagia C19D22: number analyzed (Participants) | 20 | 11
  Dysphagia C19D22 | -3.89 (10.37) | -4.04 (16.68)
  Dysphagia C20D1: number analyzed (Participants) | 23 | 15
  Dysphagia C20D1 | -4.35 (11.96) | -3.70 (12.36)
  Dysphagia C20D22: number analyzed (Participants) | 18 | 10
  Dysphagia C20D22 | -6.17 (14.87) | -5.56 (15.04)
  Dysphagia C21D1: number analyzed (Participants) | 20 | 14
  Dysphagia C21D1 | -3.89 (10.37) | -4.76 (12.87)
  Dysphagia C21D22: number analyzed (Participants) | 14 | 0
  Dysphagia C21D22 | -4.76 (18.34) |
  Dysphagia C22D1: number analyzed (Participants) | 15 | 12
  Dysphagia C22D1 | -3.70 (12.36) | -5.56 (13.81)
  Dysphagia C22D22: number analyzed (Participants) | 10 | 0
  Dysphagia C22D22 | -2.22 (26.60) |
  Dysphagia C23D1: number analyzed (Participants) | 15 | 13
  Dysphagia C23D1 | -4.44 (18.69) | -4.27 (14.73)
  Dysphagia C23D22: number analyzed (Participants) | 11 | 0
  Dysphagia C23D22 | -7.07 (16.68) |
  Dysphagia C24D1: number analyzed (Participants) | 14 | 0
  Dysphagia C24D1 | -3.17 (19.21) |
  Dysphagia C25D1: number analyzed (Participants) | 12 | 0
  Dysphagia C25D1 | -4.63 (10.00) |
  Dysphagia C25D22: number analyzed (Participants) | 11 | 0
  Dysphagia C25D22 | 0.00 (12.17) |
  Dysphagia C26D1: number analyzed (Participants) | 13 | 0
  Dysphagia C26D1 | -1.71 (14.23) |
  Dysphagia C27D1: number analyzed (Participants) | 11 | 0
  Dysphagia C27D1 | 1.01 (12.62) |
  Dysphagia C28D1: number analyzed (Participants) | 12 | 0
  Dysphagia C28D1 | 0.00 (12.54) |
  Dysphagia 30 day follow-up: number analyzed (Participants) | 72 | 90
  Dysphagia 30 day follow-up | 0.93 (21.65) | -5.93 (28.47)
  Dysphagia 90 day follow-up: number analyzed (Participants) | 86 | 82
  Dysphagia 90 day follow-up | -2.20 (25.56) | -5.42 (34.62)
  Eating restrictions Baseline | 30.54 (29.05) | 33.01 (30.26)
  Eating restrictions C1D22: number analyzed (Participants) | 176 | 208
  Eating restrictions C1D22 | 4.40 (22.82) | -1.32 (23.11)
  Eating restrictions C2D1: number analyzed (Participants) | 206 | 223
  Eating restrictions C2D1 | -3.32 (27.60) | -9.94 (29.44)
  Eating restrictions C2D22: number analyzed (Participants) | 150 | 180
  Eating restrictions C2D22 | -5.00 (26.41) | -7.92 (30.90)
  Eating restrictions C3D1: number analyzed (Participants) | 190 | 196
  Eating restrictions C3D1 | -8.77 (27.65) | -13.52 (28.28)
  Eating restrictions C3D22: number analyzed (Participants) | 152 | 148
  Eating restrictions C3D22 | -0.38 (27.39) | -10.98 (29.80)
  Eating restrictions C4D1: number analyzed (Participants) | 169 | 161
  Eating restrictions C4D1 | -6.41 (29.50) | -13.15 (28.12)
  Eating restrictions C4D22: number analyzed (Participants) | 122 | 127
  Eating restrictions C4D22 | -1.09 (28.26) | -10.96 (28.79)
  Eating restrictions C5D1: number analyzed (Participants) | 148 | 144
  Eating restrictions C5D1 | -4.84 (27.80) | -13.43 (30.02)
  Eating restrictions C5D22: number analyzed (Participants) | 110 | 115
  Eating restrictions C5D22 | -3.86 (29.62) | -11.09 (28.33)
  Eating restrictions C6D1: number analyzed (Participants) | 122 | 121
  Eating restrictions C6D1 | -7.79 (26.48) | -9.92 (27.41)
  Eating restrictions C6D22: number analyzed (Participants) | 103 | 92
  Eating restrictions C6D22 | -8.25 (27.94) | -14.67 (26.99)
  Eating restrictions C7D1: number analyzed (Participants) | 113 | 98
  Eating restrictions C7D1 | -9.14 (26.63) | -12.16 (24.29)
  Eating restrictions C7D22: number analyzed (Participants) | 81 | 73
  Eating restrictions C7D22 | -8.13 (28.41) | -14.16 (25.26)
  Eating restrictions C8D1: number analyzed (Participants) | 80 | 81
  Eating restrictions C8D1 | -8.02 (21.72) | -10.60 (23.68)
  Eating restrictions C8D22: number analyzed (Participants) | 71 | 65
  Eating restrictions C8D22 | -8.92 (23.41) | -10.13 (26.62)
  Eating restrictions C9D1: number analyzed (Participants) | 75 | 62
  Eating restrictions C9D1 | -10.89 (24.12) | -12.63 (24.78)
  Eating restrictions C9D22: number analyzed (Participants) | 60 | 55
  Eating restrictions C9D22 | -5.97 (26.80) | -7.73 (25.60)
  Eating restrictions C10D1: number analyzed (Participants) | 66 | 56
  Eating restrictions C10D1 | -7.45 (25.20) | -9.97 (25.45)
  Eating restrictions C10D22: number analyzed (Participants) | 57 | 43
  Eating restrictions C10D22 | -7.60 (25.11) | -5.81 (29.07)
  Eating restrictions C11D1: number analyzed (Participants) | 63 | 46
  Eating restrictions C11D1 | -10.05 (24.05) | -6.16 (28.57)
  Eating restrictions C11D22: number analyzed (Participants) | 44 | 31
  Eating restrictions C11D22 | -8.33 (23.23) | -5.38 (20.25)
  Eating restrictions C12D1: number analyzed (Participants) | 53 | 41
  Eating restrictions C12D1 | -7.39 (21.10) | -7.32 (24.94)
  Eating restrictions C12D22: number analyzed (Participants) | 37 | 25
  Eating restrictions C12D22 | -4.95 (20.64) | -10.67 (20.91)
  Eating restrictions C13D1: number analyzed (Participants) | 48 | 35
  Eating restrictions C13D1 | -7.47 (20.72) | -9.52 (25.26)
  Eating restrictions C13D22: number analyzed (Participants) | 40 | 21
  Eating restrictions C13D22 | -4.17 (19.06) | -7.94 (30.79)
  Eating restrictions C14D1: number analyzed (Participants) | 39 | 30
  Eating restrictions C14D1 | -6.84 (22.45) | -8.61 (28.91)
  Eating restrictions C14D22: number analyzed (Participants) | 32 | 19
  Eating restrictions C14D22 | -7.29 (21.77) | -8.33 (28.87)
  Eating restrictions C15D1: number analyzed (Participants) | 35 | 27
  Eating restrictions C15D1 | -1.90 (20.32) | -6.17 (30.97)
  Eating restrictions C15D22: number analyzed (Participants) | 29 | 17
  Eating restrictions C15D22 | -5.17 (18.56) | -12.75 (35.49)
  Eating restrictions C16D1: number analyzed (Participants) | 35 | 22
  Eating restrictions C16D1 | -6.19 (18.89) | -5.68 (36.95)
  Eating restrictions C16D22: number analyzed (Participants) | 29 | 14
  Eating restrictions C16D22 | -2.30 (26.72) | -10.12 (37.15)
  Eating restrictions C17D1: number analyzed (Participants) | 30 | 18
  Eating restrictions C17D1 | -5.56 (16.86) | -13.89 (30.92)
  Eating restrictions C17D22: number analyzed (Participants) | 23 | 0
  Eating restrictions C17D22 | -2.17 (17.63) |
  Eating restrictions C18D1: number analyzed (Participants) | 27 | 16
  Eating restrictions C18D1 | -6.17 (17.54) | -12.50 (31.77)
  Eating restrictions C18D22: number analyzed (Participants) | 20 | 10
  Eating restrictions C18D22 | -5.00 (15.86) | -15.00 (23.17)
  Eating restrictions C19D1: number analyzed (Participants) | 23 | 15
  Eating restrictions C19D1 | -5.80 (13.63) | -8.89 (26.81)
  Eating restrictions C19D22: number analyzed (Participants) | 20 | 11
  Eating restrictions C19D22 | -3.33 (15.63) | -7.58 (20.23)
  Eating restrictions C20D1: number analyzed (Participants) | 23 | 15
  Eating restrictions C20D1 | -2.17 (21.35) | -10.00 (21.87)
  Eating restrictions C20D22: number analyzed (Participants) | 18 | 10
  Eating restrictions C20D22 | -4.63 (17.90) | -10.00 (19.16)
  Eating restrictions C21D1: number analyzed (Participants) | 20 | 14
  Eating restrictions C21D1 | -0.83 (15.74) | -11.31 (20.57)
  Eating restrictions C21D22: number analyzed (Participants) | 14 | 0
  Eating restrictions C21D22 | -3.57 (12.10) |
  Eating restrictions C22D1: number analyzed (Participants) | 15 | 12
  Eating restrictions C22D1 | -5.00 (12.52) | -9.72 (25.33)
  Eating restrictions C22D22: number analyzed (Participants) | 10 | 0
  Eating restrictions C22D22 | -2.50 (18.02) |
  Eating restrictions C23D1: number analyzed (Participants) | 15 | 13
  Eating restrictions C23D1 | -6.11 (11.12) | -8.97 (24.64)
  Eating restrictions C23D22: number analyzed (Participants) | 11 | 0
  Eating restrictions C23D22 | -4.55 (14.12) |
  Eating restrictions C24D1: number analyzed (Participants) | 14 | 0
  Eating restrictions C24D1 | 0.00 (19.88) |
  Eating restrictions C25D1: number analyzed (Participants) | 12 | 0
  Eating restrictions C25D1 | -4.86 (13.51) |
  Eating restrictions C25D22: number analyzed (Participants) | 11 | 0
  Eating restrictions C25D22 | -0.76 (13.15) |
  Eating restrictions C26D1: number analyzed (Participants) | 13 | 0
  Eating restrictions C26D1 | -4.49 (11.59) |
  Eating restrictions C27D1: number analyzed (Participants) | 11 | 0
  Eating restrictions C27D1 | -6.06 (10.60) |
  Eating restrictions C28D1: number analyzed (Participants) | 12 | 0
  Eating restrictions C28D1 | -4.17 (14.86) |
  Eating restrictions 30 day follow up: number analyzed (Participants) | 72 | 90
  Eating restrictions 30 day follow up | 2.31 (25.03) | -5.46 (33.57)
  Eating restrictions 90 day follow up: number analyzed (Participants) | 86 | 82
  Eating restrictions 90 day follow up | -5.62 (30.80) | -5.08 (38.53)
  Reflux Baseline | 17.64 (24.43) | 16.60 (24.00)
  Reflux C1D22: number analyzed (Participants) | 176 | 208
  Reflux C1D22 | -1.70 (21.61) | -1.28 (21.70)
  Reflux C2D1: number analyzed (Participants) | 206 | 223
  Reflux C2D1 | -2.99 (24.32) | -5.31 (26.20)
  Reflux C2D22: number analyzed (Participants) | 150 | 180
  Reflux C2D22 | -4.56 (23.00) | -5.00 (23.43)
  Reflux C3D1: number analyzed (Participants) | 190 | 196
  Reflux C3D1 | -5.61 (23.71) | -6.46 (23.10)
  Reflux C3D22: number analyzed (Participants) | 152 | 148
  Reflux C3D22 | -4.39 (21.16) | -5.86 (21.19)
  Reflux C4D1: number analyzed (Participants) | 169 | 161
  Reflux C4D1 | -5.52 (22.18) | -5.28 (20.95)
  Reflux C4D22: number analyzed (Participants) | 122 | 127
  Reflux C4D22 | -2.46 (21.18) | -5.64 (20.49)
  Reflux C5D1: number analyzed (Participants) | 148 | 144
  Reflux C5D1 | -4.95 (22.46) | -3.24 (22.92)
  Reflux C5D22: number analyzed (Participants) | 110 | 115
  Reflux C5D22 | -2.88 (21.76) | -2.75 (22.72)
  Reflux C6D1: number analyzed (Participants) | 122 | 121
  Reflux C6D1 | -5.87 (23.66) | -1.38 (20.82)
  Reflux C6D22: number analyzed (Participants) | 103 | 92
  Reflux C6D22 | -4.53 (20.50) | -1.81 (20.44)
  Reflux C7D1: number analyzed (Participants) | 113 | 98
  Reflux C7D1 | -4.13 (19.74) | 1.36 (18.64)
  Reflux C7D22: number analyzed (Participants) | 81 | 73
  Reflux C7D22 | -5.14 (21.99) | -1.14 (16.97)
  Reflux C8D1: number analyzed (Participants) | 80 | 81
  Reflux C8D1 | -5.63 (21.37) | 0.41 (14.19)
  Reflux C8D22: number analyzed (Participants) | 71 | 65
  Reflux C8D22 | -6.34 (22.95) | 1.03 (18.13)
  Reflux C9D1: number analyzed (Participants) | 75 | 62
  Reflux C9D1 | -6.00 (23.19) | -0.81 (16.65)
  Reflux C9D22: number analyzed (Participants) | 60 | 55
  Reflux C9D22 | -2.22 (18.27) | 1.82 (14.58)
  Reflux C10D1: number analyzed (Participants) | 66 | 56
  Reflux C10D1 | -4.80 (23.16) | 0.30 (17.26)
  Reflux C10D22: number analyzed (Participants) | 57 | 43
  Reflux C10D22 | -6.43 (20.11) | 5.04 (19.43)
  Reflux C11D1: number analyzed (Participants) | 63 | 46
  Reflux C11D1 | -7.41 (21.54) | 7.97 (24.02)
  Reflux C11D22: number analyzed (Participants) | 44 | 31
  Reflux C11D22 | -6.82 (17.36) | 7.53 (21.45)
  Reflux C12D1: number analyzed (Participants) | 53 | 41
  Reflux C12D1 | -4.40 (19.38) | 8.13 (24.75)
  Reflux C12D22: number analyzed (Participants) | 37 | 25
  Reflux C12D22 | -5.86 (21.95) | 2.67 (19.65)
  Reflux C13D1: number analyzed (Participants) | 48 | 35
  Reflux C13D1 | -4.17 (20.48) | 4.76 (21.23)
  Reflux C13D22: number analyzed (Participants) | 40 | 21
  Reflux C13D22 | -2.08 (18.94) | 5.56 (13.26)
  Reflux C14D1: number analyzed (Participants) | 39 | 30
  Reflux C14D1 | -1.71 (21.90) | -0.56 (15.46)
  Reflux C14D22: number analyzed (Participants) | 32 | 19
  Reflux C14D22 | -5.73 (21.00) | 7.02 (13.96)
  Reflux C15D1: number analyzed (Participants) | 35 | 27
  Reflux C15D1 | -0.95 (14.54) | 2.47 (21.03)
  Reflux C15D22: number analyzed (Participants) | 29 | 17
  Reflux C15D22 | -4.60 (19.36) | 2.94 (15.85)
  Reflux C16D1: number analyzed (Participants) | 35 | 22
  Reflux C16D1 | -3.33 (17.99) | 6.06 (22.74)
  Reflux C16D22: number analyzed (Participants) | 29 | 14
  Reflux C16D22 | -8.62 (21.65) | 7.14 (28.28)
  Reflux C17D1: number analyzed (Participants) | 30 | 18
  Reflux C17D1 | -1.11 (21.86) | 1.85 (20.52)
  Reflux C17D22: number analyzed (Participants) | 23 | 0
  Reflux C17D22 | -1.45 (21.27) |
  Reflux C18D1: number analyzed (Participants) | 27 | 16
  Reflux C18D1 | -4.32 (20.46) | -3.13 (17.45)
  Reflux C18D22: number analyzed (Participants) | 20 | 10
  Reflux C18D22 | 0.83 (22.60) | 0.00 (23.57)
  Reflux C19D1: number analyzed (Participants) | 23 | 15
  Reflux C19D1 | -0.72 (15.47) | -1.11 (20.38)
  Reflux C19D22: number analyzed (Participants) | 20 | 11
  Reflux C19D22 | -1.67 (14.20) | 3.03 (14.56)
  Reflux C20D1: number analyzed (Participants) | 23 | 15
  Reflux C20D1 | 0.00 (15.08) | -3.33 (14.36)
  Reflux C20D22: number analyzed (Participants) | 18 | 10
  Reflux C20D22 | -2.78 (15.39) | 1.67 (14.59)
  Reflux C21D1: number analyzed (Participants) | 20 | 14
  Reflux C21D1 | 0.00 (9.37) | -1.19 (12.17)
  Reflux C21D22: number analyzed (Participants) | 14 | 0
  Reflux C21D22 | 0.00 (11.32) |
  Reflux C22D1: number analyzed (Participants) | 15 | 12
  Reflux C22D1 | 0.00 (19.92) | -6.94 (16.60)
  Reflux C22D22: number analyzed (Participants) | 10 | 0
  Reflux C22D22 | -6.67 (19.56) |
  Reflux C23D1: number analyzed (Participants) | 15 | 13
  Reflux C23D1 | -5.56 (15.00) | 0.00 (19.25)
  Reflux C23D22: number analyzed (Participants) | 11 | 0
  Reflux C23D22 | -6.06 (18.67) |
  Reflux C24D1: number analyzed (Participants) | 14 | 0
  Reflux C24D1 | -4.76 (16.57) |
  Reflux C25D1: number analyzed (Participants) | 12 | 0
  Reflux C25D1 | -5.56 (19.25) |
  Reflux C25D22: number analyzed (Participants) | 11 | 0
  Reflux C25D22 | -4.55 (15.08) |
  Reflux C26D1: number analyzed (Participants) | 13 | 0
  Reflux C26D1 | -1.28 (17.30) |
  Reflux C27D1: number analyzed (Participants) | 11 | 0
  Reflux C27D1 | 0.00 (14.91) |
  Reflux C28D1: number analyzed (Participants) | 12 | 0
  Reflux C28D1 | 0.00 (12.31) |
  Reflux 30 day follow up: number analyzed (Participants) | 72 | 90
  Reflux 30 day follow up | -1.85 (26.32) | -2.96 (26.63)
  Reflux 90 day follow up: number analyzed (Participants) | 86 | 82
  Reflux 90 day follow up | -0.78 (24.91) | 1.02 (26.49)
  Odynophagia Baseline | 22.18 (25.96) | 22.44 (26.60)
  Odynophagia C1D22: number analyzed (Participants) | 176 | 208
  Odynophagia C1D22 | -2.37 (24.22) | -5.69 (22.72)
  Odynophagia C2D1: number analyzed (Participants) | 206 | 223
  Odynophagia C2D1 | -4.77 (24.64) | -9.19 (24.94)
  Odynophagia C2D22: number analyzed (Participants) | 150 | 180
  Odynophagia C2D22 | -6.22 (24.62) | -9.35 (25.05)
  Odynophagia C3D1: number analyzed (Participants) | 190 | 196
  Odynophagia C3D1 | -9.39 (24.63) | -11.39 (24.00)
  Odynophagia C3D22: number analyzed (Participants) | 152 | 148
  Odynophagia C3D22 | -6.36 (22.77) | -12.50 (23.56)
  Odynophagia C4D1: number analyzed (Participants) | 169 | 161
  Odynophagia C4D1 | -9.66 (24.84) | -11.18 (23.26)
  Odynophagia C4D22: number analyzed (Participants) | 122 | 127
  Odynophagia C4D22 | -3.69 (25.67) | -9.19 (22.29)
  Odynophagia C5D1: number analyzed (Participants) | 148 | 144
  Odynophagia C5D1 | -4.73 (23.49) | -11.23 (23.14)
  Odynophagia C5D22: number analyzed (Participants) | 110 | 115
  Odynophagia C5D22 | -4.85 (26.17) | -11.01 (23.87)
  Odynophagia C6D1: number analyzed (Participants) | 122 | 121
  Odynophagia C6D1 | -7.92 (20.24) | -8.13 (20.98)
  Odynophagia C6D22: number analyzed (Participants) | 103 | 92
  Odynophagia C6D22 | -8.41 (22.49) | -12.32 (21.52)
  Odynophagia C7D1: number analyzed (Participants) | 113 | 98
  Odynophagia C7D1 | -9.44 (21.92) | -7.99 (19.77)
  Odynophagia C7D22: number analyzed (Participants) | 81 | 73
  Odynophagia C7D22 | -8.23 (22.99) | -7.31 (18.84)
  Odynophagia C8D1: number analyzed (Participants) | 80 | 81
  Odynophagia C8D1 | -5.21 (20.81) | -6.58 (16.39)
  Odynophagia C8D22: number analyzed (Participants) | 71 | 65
  Odynophagia C8D22 | -8.69 (22.16) | -7.44 (19.99)
  Odynophagia C9D1: number analyzed (Participants) | 75 | 62
  Odynophagia C9D1 | -8.67 (20.20) | -8.06 (20.63)
  Odynophagia C9D22: number analyzed (Participants) | 60 | 55
  Odynophagia C9D22 | -5.56 (20.74) | -2.42 (19.36)
  Odynophagia C10D1: number analyzed (Participants) | 66 | 56
  Odynophagia C10D1 | -6.31 (18.89) | -4.17 (17.48)
  Odynophagia C10D22: number analyzed (Participants) | 57 | 43
  Odynophagia C10D22 | -4.09 (18.44) | -3.49 (18.74)
  Odynophagia C11D1: number analyzed (Participants) | 63 | 46
  Odynophagia C11D1 | -5.56 (17.96) | -2.54 (16.84)
  Odynophagia C11D22: number analyzed (Participants) | 44 | 31
  Odynophagia C11D22 | -3.41 (14.19) | 0.54 (11.77)
  Odynophagia C12D1: number analyzed (Participants) | 53 | 41
  Odynophagia C12D1 | -4.40 (20.45) | -1.22 (15.09)
  Odynophagia C12D22: number analyzed (Participants) | 37 | 25
  Odynophagia C12D22 | -2.25 (17.64) | -2.00 (17.56)
  Odynophagia C13D1: number analyzed (Participants) | 48 | 35
  Odynophagia C13D1 | -3.82 (16.93) | -3.33 (13.89)
  Odynophagia C13D22: number analyzed (Participants) | 40 | 21
  Odynophagia C13D22 | -4.17 (18.78) | 0.79 (15.34)
  Odynophagia C14D1: number analyzed (Participants) | 39 | 30
  Odynophagia C14D1 | -2.56 (23.43) | -0.00 (13.13)
  Odynophagia C14D22: number analyzed (Participants) | 32 | 19
  Odynophagia C14D22 | -5.73 (15.03) | -1.75 (15.61)
  Odynophagia C15D1: number analyzed (Participants) | 35 | 27
  Odynophagia C15D1 | -1.43 (15.85) | 2.47 (18.89)
  Odynophagia C15D22: number analyzed (Participants) | 29 | 17
  Odynophagia C15D22 | -1.72 (16.87) | -1.96 (18.52)
  Odynophagia C16D1: number analyzed (Participants) | 35 | 22
  Odynophagia C16D1 | -3.81 (13.46) | 1.52 (18.48)
  Odynophagia C16D22: number analyzed (Participants) | 29 | 14
  Odynophagia C16D22 | -4.02 (15.21) | 1.19 (21.15)
  Odynophagia C17D1: number analyzed (Participants) | 30 | 18
  Odynophagia C17D1 | -4.44 (16.34) | -0.93 (12.09)
  Odynophagia C17D22: number analyzed (Participants) | 23 | 0
  Odynophagia C17D22 | 1.45 (25.08) |
  Odynophagia C18D1: number analyzed (Participants) | 27 | 16
  Odynophagia C18D1 | -5.56 (16.67) | -1.04 (14.23)
  Odynophagia C18D22: number analyzed (Participants) | 20 | 10
  Odynophagia C18D22 | -2.50 (13.55) | -5.00 (13.72)
  Odynophagia C19D1: number analyzed (Participants) | 23 | 15
  Odynophagia C19D1 | -5.80 (13.86) | -2.22 (12.39)
  Odynophagia C19D22: number analyzed (Participants) | 20 | 11
  Odynophagia C19D22 | -5.00 (13.36) | -3.03 (17.98)
  Odynophagia C20D1: number analyzed (Participants) | 23 | 15
  Odynophagia C20D1 | -0.72 (25.37) | -5.56 (16.27)
  Odynophagia C20D22: number analyzed (Participants) | 18 | 10
  Odynophagia C20D22 | -6.48 (14.16) | 0.00 (15.71)
  Odynophagia C21D1: number analyzed (Participants) | 20 | 14
  Odynophagia C21D1 | -3.33 (8.72) | -3.57 (13.36)
  Odynophagia C21D22: number analyzed (Participants) | 14 | 0
  Odynophagia C21D22 | -1.19 (10.26) |
  Odynophagia C22D1: number analyzed (Participants) | 15 | 12
  Odynophagia C22D1 | -2.22 (10.67) | -2.78 (9.62)
  Odynophagia C22D22: number analyzed (Participants) | 10 | 0
  Odynophagia C22D22 | 0.00 (13.61) |
  Odynophagia C23D1: number analyzed (Participants) | 15 | 13
  Odynophagia C23D1 | -4.44 (9.89) | -5.13 (8.01)
  Odynophagia C23D22: number analyzed (Participants) | 11 | 0
  Odynophagia C23D22 | 0.00 (14.91) |
  Odynophagia C24D1: number analyzed (Participants) | 14 | 0
  Odynophagia C24D1 | 1.19 (21.15) |
  Odynophagia C25D1: number analyzed (Participants) | 12 | 0
  Odynophagia C25D1 | -1.39 (4.81) |
  Odynophagia C25D22: number analyzed (Participants) | 11 | 0
  Odynophagia C25D22 | 4.55 (7.78) |
  Odynophagia C26D1: number analyzed (Participants) | 13 | 0
  Odynophagia C26D1 | -1.28 (10.68) |
  Odynophagia C27D1: number analyzed (Participants) | 11 | 0
  Odynophagia C27D1 | -4.55 (10.78) |
  Odynophagia C28D1: number analyzed (Participants) | 12 | 0
  Odynophagia C28D1 | 1.39 (4.81) |
  Odynophagia 30 day follow up: number analyzed (Participants) | 72 | 90
  Odynophagia 30 day follow up | -3.01 (25.53) | -4.44 (24.20)
  Odynophagia 90 day follow up: number analyzed (Participants) | 86 | 82
  Odynophagia 90 day follow up | -5.62 (27.49) | -3.46 (29.01)
  Pain and Discomfort Baseline | 27.04 (26.61) | 26.39 (27.45)
  Pain and Discomfort C1D22: number analyzed (Participants) | 176 | 208
  Pain and Discomfort C1D22 | -4.55 (21.78) | -3.45 (23.17)
  Pain and Discomfort C2D1: number analyzed (Participants) | 206 | 223
  Pain and Discomfort C2D1 | -4.94 (26.72) | -8.37 (28.25)
  Pain and Discomfort C2D22: number analyzed (Participants) | 150 | 180
  Pain and Discomfort C2D22 | -8.00 (25.01) | -8.89 (26.04)
  Pain and Discomfort C3D1: number analyzed (Participants) | 190 | 196
  Pain and Discomfort C3D1 | -9.56 (24.26) | -8.50 (23.48)
  Pain and Discomfort C3D22: number analyzed (Participants) | 152 | 148
  Pain and Discomfort C3D22 | -6.14 (23.93) | -8.67 (24.86)
  Pain and Discomfort C4D1: number analyzed (Participants) | 169 | 161
  Pain and Discomfort C4D1 | -9.76 (24.30) | -8.70 (23.13)
  Pain and Discomfort C4D22: number analyzed (Participants) | 122 | 127
  Pain and Discomfort C4D22 | -6.56 (21.70) | -8.79 (23.93)
  Pain and Discomfort C5D1: number analyzed (Participants) | 148 | 144
  Pain and Discomfort C5D1 | -5.29 (22.84) | -8.68 (24.14)
  Pain and Discomfort C5D22: number analyzed (Participants) | 110 | 115
  Pain and Discomfort C5D22 | -7.42 (26.58) | -8.99 (22.44)
  Pain and Discomfort C6D1: number analyzed (Participants) | 122 | 121
  Pain and Discomfort C6D1 | -7.51 (23.77) | -5.79 (23.64)
  Pain and Discomfort C6D22: number analyzed (Participants) | 103 | 92
  Pain and Discomfort C6D22 | -9.87 (26.24) | -12.68 (24.51)
  Pain and Discomfort C7D1: number analyzed (Participants) | 113 | 98
  Pain and Discomfort C7D1 | -8.41 (23.05) | -8.50 (21.30)
  Pain and Discomfort C7D22: number analyzed (Participants) | 81 | 73
  Pain and Discomfort C7D22 | -9.67 (21.55) | -8.68 (20.43)
  Pain and Discomfort C8D1: number analyzed (Participants) | 80 | 81
  Pain and Discomfort C8D1 | -5.42 (24.42) | -7.82 (23.29)
  Pain and Discomfort C8D22: number analyzed (Participants) | 71 | 65
  Pain and Discomfort C8D22 | -10.09 (23.48) | -9.23 (23.39)
  Pain and Discomfort C9D1: number analyzed (Participants) | 75 | 62
  Pain and Discomfort C9D1 | -10.00 (22.26) | -7.53 (22.11)
  Pain and Discomfort C9D22: number analyzed (Participants) | 60 | 55
  Pain and Discomfort C9D22 | -6.94 (22.82) | -7.27 (21.93)
  Pain and Discomfort C10D1: number analyzed (Participants) | 66 | 56
  Pain and Discomfort C10D1 | -10.35 (22.22) | -7.14 (19.81)
  Pain and Discomfort C10D22: number analyzed (Participants) | 57 | 43
  Pain and Discomfort C10D22 | -6.14 (22.85) | -3.49 (21.07)
  Pain and Discomfort C11D1: number analyzed (Participants) | 63 | 46
  Pain and Discomfort C11D1 | -8.47 (19.37) | -0.72 (20.47)
  Pain and Discomfort C11D22: number analyzed (Participants) | 44 | 31
  Pain and Discomfort C11D22 | -7.95 (19.52) | -2.15 (17.07)
  Pain and Discomfort C12D1: number analyzed (Participants) | 53 | 41
  Pain and Discomfort C12D1 | -4.40 (20.71) | -1.63 (21.67)
  Pain and Discomfort C12D22: number analyzed (Participants) | 37 | 25
  Pain and Discomfort C12D22 | -4.95 (19.98) | -1.33 (19.20)
  Pain and Discomfort C13D1: number analyzed (Participants) | 48 | 35
  Pain and Discomfort C13D1 | -4.86 (21.18) | -2.38 (21.44)
  Pain and Discomfort C13D22: number analyzed (Participants) | 40 | 21
  Pain and Discomfort C13D22 | -4.58 (22.32) | 0.79 (23.26)
  Pain and Discomfort C14D1: number analyzed (Participants) | 39 | 30
  Pain and Discomfort C14D1 | -2.99 (22.58) | -1.67 (21.15)
  Pain and Discomfort C14D22: number analyzed (Participants) | 32 | 19
  Pain and Discomfort C14D22 | -9.38 (17.42) | -5.26 (20.07)
  Pain and Discomfort C15D1: number analyzed (Participants) | 35 | 27
  Pain and Discomfort C15D1 | -1.90 (24.51) | -1.23 (24.43)
  Pain and Discomfort C15D22: number analyzed (Participants) | 29 | 17
  Pain and Discomfort C15D22 | -6.32 (24.16) | -2.94 (25.16)
  Pain and Discomfort C16D1: number analyzed (Participants) | 35 | 22
  Pain and Discomfort C16D1 | -7.14 (25.34) | -3.03 (20.98)
  Pain and Discomfort C16D22: number analyzed (Participants) | 29 | 14
  Pain and Discomfort C16D22 | -8.62 (22.55) | -3.57 (23.73)
  Pain and Discomfort C17D1: number analyzed (Participants) | 30 | 18
  Pain and Discomfort C17D1 | -3.89 (22.61) | 1.85 (18.86)
  Pain and Discomfort C17D22: number analyzed (Participants) | 23 | 0
  Pain and Discomfort C17D22 | -4.35 (21.45) |
  Pain and Discomfort C18D1: number analyzed (Participants) | 27 | 16
  Pain and Discomfort C18D1 | -8.02 (22.35) | -4.17 (20.64)
  Pain and Discomfort C18D22: number analyzed (Participants) | 20 | 10
  Pain and Discomfort C18D22 | -8.33 (22.62) | -6.67 (11.65)
  Pain and Discomfort C19D1: number analyzed (Participants) | 23 | 15
  Pain and Discomfort C19D1 | -13.77 (18.57) | -6.67 (23.40)
  Pain and Discomfort C19D22: number analyzed (Participants) | 20 | 11
  Pain and Discomfort C19D22 | -7.50 (21.95) | -4.55 (21.20)
  Pain and Discomfort C20D1: number analyzed (Participants) | 23 | 15
  Pain and Discomfort C20D1 | -11.59 (17.72) | -7.78 (20.77)
  Pain and Discomfort C20D22: number analyzed (Participants) | 18 | 10
  Pain and Discomfort C20D22 | -11.11 (18.96) | -5.00 (15.81)
  Pain and Discomfort C21D1: number analyzed (Participants) | 20 | 14
  Pain and Discomfort C21D1 | -8.33 (19.12) | -10.71 (19.18)
  Pain and Discomfort C21D22: number analyzed (Participants) | 14 | 0
  Pain and Discomfort C21D22 | -9.52 (21.40) |
  Pain and Discomfort C22D1: number analyzed (Participants) | 15 | 12
  Pain and Discomfort C22D1 | -13.33 (19.11) | -4.17 (16.09)
  Pain and Discomfort C22D22: number analyzed (Participants) | 10 | 0
  Pain and Discomfort C22D22 | -13.33 (21.94) |
  Pain and Discomfort C23D1: number analyzed (Participants) | 15 | 13
  Pain and Discomfort C23D1 | -14.44 (18.76) | -7.69 (21.10)
  Pain and Discomfort C23D22: number analyzed (Participants) | 11 | 0
  Pain and Discomfort C23D22 | -10.61 (18.67) |
  Pain and Discomfort C24D1: number analyzed (Participants) | 14 | 0
  Pain and Discomfort C24D1 | -13.10 (19.81) |
  Pain and Discomfort C25D1: number analyzed (Participants) | 12 | 0
  Pain and Discomfort C25D1 | -11.11 (19.25) |
  Pain and Discomfort C25D22: number analyzed (Participants) | 11 | 0
  Pain and Discomfort C25D22 | -10.61 (20.10) |
  Pain and Discomfort C26D1: number analyzed (Participants) | 13 | 0
  Pain and Discomfort C26D1 | -14.10 (20.24) |
  Pain and Discomfort C27D1: number analyzed (Participants) | 11 | 0
  Pain and Discomfort C27D1 | -10.61 (15.41) |
  Pain and Discomfort C28D1: number analyzed (Participants) | 12 | 0
  Pain and Discomfort C28D1 | -6.94 (16.60) |
  Pain and Discomfort 30 day follow up: number analyzed (Participants) | 72 | 90
  Pain and Discomfort 30 day follow up | -6.02 (29.11) | -1.85 (27.08)
  Pain and Discomfort 90 day follow up: number analyzed (Participants) | 86 | 82
  Pain and Discomfort 90 day follow up | -6.59 (30.17) | -1.83 (32.50)
  Anxiety Baseline | 51.30 (28.99) | 52.92 (30.74)
  Anxiety C1D22: number analyzed (Participants) | 176 | 208
  Anxiety C1D22 | -8.33 (24.69) | -6.09 (25.60)
  Anxiety C2D1: number analyzed (Participants) | 206 | 223
  Anxiety C2D1 | -10.19 (26.31) | -11.29 (29.40)
  Anxiety C2D22: number analyzed (Participants) | 150 | 180
  Anxiety C2D22 | -11.67 (24.33) | -11.85 (30.33)
  Anxiety C3D1: number analyzed (Participants) | 190 | 196
  Anxiety C3D1 | -12.63 (26.19) | -13.44 (28.71)
  Anxiety C3D22: number analyzed (Participants) | 152 | 148
  Anxiety C3D22 | -9.65 (26.48) | -14.30 (27.90)
  Anxiety C4D1: number analyzed (Participants) | 169 | 161
  Anxiety C4D1 | -14.60 (24.61) | -12.63 (26.21)
  Anxiety C4D22: number analyzed (Participants) | 122 | 127
  Anxiety C4D22 | -11.34 (26.87) | -12.99 (26.97)
  Anxiety C5D1: number analyzed (Participants) | 148 | 144
  Anxiety C5D1 | -12.16 (28.61) | -7.75 (28.42)
  Anxiety C5D22: number analyzed (Participants) | 110 | 115
  Anxiety C5D22 | -10.30 (29.61) | -8.12 (25.59)
  Anxiety C6D1: number analyzed (Participants) | 122 | 121
  Anxiety C6D1 | -13.39 (31.68) | -9.09 (28.22)
  Anxiety C6D22: number analyzed (Participants) | 103 | 92
  Anxiety C6D22 | -11.65 (26.59) | -14.67 (25.30)
  Anxiety C7D1: number analyzed (Participants) | 113 | 98
  Anxiety C7D1 | -12.68 (28.46) | -17.18 (25.49)
  Anxiety C7D22: number analyzed (Participants) | 81 | 73
  Anxiety C7D22 | -13.79 (27.99) | -15.98 (27.84)
  Anxiety C8D1: number analyzed (Participants) | 80 | 81
  Anxiety C8D1 | -11.46 (28.51) | -14.20 (25.97)
  Anxiety C8D22: number analyzed (Participants) | 71 | 65
  Anxiety C8D22 | -13.62 (26.92) | -16.92 (28.79)
  Anxiety C9D1: number analyzed (Participants) | 75 | 62
  Anxiety C9D1 | -18.22 (25.14) | -15.86 (27.06)
  Anxiety C9D22: number analyzed (Participants) | 60 | 55
  Anxiety C9D22 | -16.94 (25.76) | -20.30 (26.97)
  Anxiety C10D1: number analyzed (Participants) | 66 | 56
  Anxiety C10D1 | -16.67 (25.15) | -18.15 (31.51)
  Anxiety C10D22: number analyzed (Participants) | 57 | 43
  Anxiety C10D22 | -18.71 (27.65) | -13.95 (29.08)
  Anxiety C11D1: number analyzed (Participants) | 63 | 46
  Anxiety C11D1 | -18.25 (30.78) | -9.06 (24.77)
  Anxiety C11D22: number analyzed (Participants) | 44 | 31
  Anxiety C11D22 | -20.83 (27.40) | -14.52 (29.73)
  Anxiety C12D1: number analyzed (Participants) | 53 | 41
  Anxiety C12D1 | -17.30 (30.13) | -10.57 (22.59)
  Anxiety C12D22: number analyzed (Participants) | 37 | 25
  Anxiety C12D22 | -13.06 (28.64) | -19.33 (29.53)
  Anxiety C13D1: number analyzed (Participants) | 48 | 35
  Anxiety C13D1 | -15.63 (29.26) | -15.24 (25.36)
  Anxiety C13D22: number analyzed (Participants) | 40 | 21
  Anxiety C13D22 | -9.58 (25.84) | -10.32 (26.07)
  Anxiety C14D1: number analyzed (Participants) | 39 | 30
  Anxiety C14D1 | -13.68 (25.33) | -15.00 (24.11)
  Anxiety C14D22: number analyzed (Participants) | 32 | 19
  Anxiety C14D22 | -18.75 (28.95) | -10.53 (23.71)
  Anxiety C15D1: number analyzed (Participants) | 35 | 27
  Anxiety C15D1 | -13.33 (27.65) | -16.67 (30.66)
  Anxiety C15D22: number analyzed (Participants) | 29 | 17
  Anxiety C15D22 | -14.37 (27.72) | -17.65 (33.06)
  Anxiety C16D1: number analyzed (Participants) | 35 | 22
  Anxiety C16D1 | -17.14 (31.95) | -15.91 (29.76)
  Anxiety C16D22: number analyzed (Participants) | 29 | 14
  Anxiety C16D22 | -14.94 (26.48) | -20.24 (31.47)
  Anxiety C17D1: number analyzed (Participants) | 30 | 18
  Anxiety C17D1 | -12.78 (33.53) | -20.37 (29.46)
  Anxiety C17D22: number analyzed (Participants) | 23 | 0
  Anxiety C17D22 | -11.59 (22.15) |
  Anxiety C18D1: number analyzed (Participants) | 27 | 16
  Anxiety C18D1 | -14.81 (27.48) | -15.63 (25.44)
  Anxiety C18D22: number analyzed (Participants) | 20 | 10
  Anxiety C18D22 | -15.83 (24.47) | -16.67 (30.43)
  Anxiety C19D1: number analyzed (Participants) | 23 | 15
  Anxiety C19D1 | -19.57 (30.42) | -21.11 (32.41)
  Anxiety C19D22: number analyzed (Participants) | 20 | 11
  Anxiety C19D22 | -10.00 (30.78) | -16.67 (29.81)
  Anxiety C20D1: number analyzed (Participants) | 23 | 15
  Anxiety C20D1 | -21.01 (28.52) | -21.11 (26.33)
  Anxiety C20D22: number analyzed (Participants) | 18 | 10
  Anxiety C20D22 | -16.67 (25.57) | -18.33 (22.84)
  Anxiety C21D1: number analyzed (Participants) | 20 | 14
  Anxiety C21D1 | -19.17 (29.75) | -15.48 (33.63)
  Anxiety C21D22: number analyzed (Participants) | 14 | 0
  Anxiety C21D22 | -14.29 (21.54) |
  Anxiety C22D1: number analyzed (Participants) | 15 | 12
  Anxiety C22D1 | -18.89 (33.25) | -16.67 (26.59)
  Anxiety C22D22: number analyzed (Participants) | 10 | 0
  Anxiety C22D22 | -3.33 (42.16) |
  Anxiety C23D1: number analyzed (Participants) | 15 | 13
  Anxiety C23D1 | -22.22 (38.14) | -23.08 (29.30)
  Anxiety C23D22: number analyzed (Participants) | 11 | 0
  Anxiety C23D22 | -16.67 (29.81) |
  Anxiety C24D1: number analyzed (Participants) | 14 | 0
  Anxiety C24D1 | -20.24 (35.91) |
  Anxiety C25D1: number analyzed (Participants) | 12 | 0
  Anxiety C25D1 | -19.44 (38.82) |
  Anxiety C25D22: number analyzed (Participants) | 11 | 0
  Anxiety C25D22 | -12.12 (38.07) |
  Anxiety C26D1: number analyzed (Participants) | 13 | 0
  Anxiety C26D1 | -21.79 (36.25) |
  Anxiety C27D1: number analyzed (Participants) | 11 | 0
  Anxiety C27D1 | -30.30 (30.57) |
  Anxiety C28D1: number analyzed (Participants) | 12 | 0
  Anxiety C28D1 | -20.83 (33.43) |
  Anxiety 30 day follow up: number analyzed (Participants) | 72 | 90
  Anxiety 30 day follow up | -3.47 (30.25) | -6.30 (33.39)
  Anxiety 90 day follow up: number analyzed (Participants) | 86 | 82
  Anxiety 90 day follow up | -2.52 (31.88) | -2.44 (33.86)
  Eating in front of others Baseline | 14.66 (25.11) | 15.95 (26.85)
  Eating in front of others C1D22: number analyzed (Participants) | 176 | 208
  Eating in front of others C1D22 | -1.14 (25.42) | -0.64 (23.16)
  Eating in front of others C2D1: number analyzed (Participants) | 206 | 223
  Eating in front of others C2D1 | -1.46 (25.57) | -4.04 (23.86)
  Eating in front of others C2D22: number analyzed (Participants) | 150 | 180
  Eating in front of others C2D22 | -2.00 (28.96) | -3.52 (25.28)
  Eating in front of others C3D1: number analyzed (Participants) | 190 | 196
  Eating in front of others C3D1 | -5.79 (25.11) | -5.27 (27.23)
  Eating in front of others C3D22: number analyzed (Participants) | 152 | 148
  Eating in front of others C3D22 | -2.19 (26.21) | -6.08 (26.38)
  Eating in front of others C4D1: number analyzed (Participants) | 169 | 161
  Eating in front of others C4D1 | -4.93 (27.13) | -7.45 (23.86)
  Eating in front of others C4D22: number analyzed (Participants) | 122 | 127
  Eating in front of others C4D22 | -0.82 (25.16) | -4.99 (26.25)
  Eating in front of others C5D1: number analyzed (Participants) | 148 | 144
  Eating in front of others C5D1 | -3.83 (25.94) | -4.63 (25.43)
  Eating in front of others C5D22: number analyzed (Participants) | 110 | 115
  Eating in front of others C5D22 | -2.42 (26.22) | -4.06 (22.14)
  Eating in front of others C6D1: number analyzed (Participants) | 122 | 121
  Eating in front of others C6D1 | -5.74 (22.14) | -1.93 (24.83)
  Eating in front of others C6D22: number analyzed (Participants) | 103 | 92
  Eating in front of others C6D22 | -2.27 (21.52) | -4.71 (23.48)
  Eating in front of others C7D1: number analyzed (Participants) | 113 | 98
  Eating in front of others C7D1 | -2.36 (26.99) | -4.76 (23.93)
  Eating in front of others C7D22: number analyzed (Participants) | 81 | 73
  Eating in front of others C7D22 | -2.88 (20.55) | -3.65 (22.61)
  Eating in front of others C8D1: number analyzed (Participants) | 80 | 81
  Eating in front of others C8D1 | -1.25 (23.98) | -4.94 (18.34)
  Eating in front of others C8D22: number analyzed (Participants) | 71 | 65
  Eating in front of others C8D22 | -3.29 (21.93) | -3.59 (20.52)
  Eating in front of others C9D1: number analyzed (Participants) | 75 | 62
  Eating in front of others C9D1 | -6.67 (19.76) | -4.84 (23.26)
  Eating in front of others C9D22: number analyzed (Participants) | 60 | 55
  Eating in front of others C9D22 | -2.22 (22.85) | -0.61 (27.59)
  Eating in front of others C10D1: number analyzed (Participants) | 66 | 56
  Eating in front of others C10D1 | -6.06 (26.09) | -2.98 (22.27)
  Eating in front of others C10D22: number analyzed (Participants) | 57 | 43
  Eating in front of others C10D22 | -3.51 (21.53) | -2.33 (21.08)
  Eating in front of others C11D1: number analyzed (Participants) | 63 | 46
  Eating in front of others C11D1 | -6.35 (23.84) | -1.45 (22.17)
  Eating in front of others C11D22: number analyzed (Participants) | 44 | 31
  Eating in front of others C11D22 | -8.33 (22.87) | -2.15 (17.07)
  Eating in front of others C12D1: number analyzed (Participants) | 53 | 41
  Eating in front of others C12D1 | -5.03 (20.04) | -2.44 (18.84)
  Eating in front of others C12D22: number analyzed (Participants) | 37 | 25
  Eating in front of others C12D22 | -9.91 (27.06) | -5.33 (18.46)
  Eating in front of others C13D1: number analyzed (Participants) | 48 | 35
  Eating in front of others C13D1 | -4.17 (27.18) | -3.81 (17.66)
  Eating in front of others C13D22: number analyzed (Participants) | 40 | 21
  Eating in front of others C13D22 | -3.33 (21.08) | -0.00 (25.82)
  Eating in front of others C14D1: number analyzed (Participants) | 39 | 30
  Eating in front of others C14D1 | -4.27 (20.49) | -2.22 (21.32)
  Eating in front of others C14D22: number analyzed (Participants) | 32 | 19
  Eating in front of others C14D22 | -2.08 (22.30) | -3.51 (18.90)
  Eating in front of others C15D1: number analyzed (Participants) | 35 | 27
  Eating in front of others C15D1 | -0.95 (18.94) | -2.47 (15.81)
  Eating in front of others C15D22: number analyzed (Participants) | 29 | 17
  Eating in front of others C15D22 | 1.15 (25.95) | -1.96 (21.96)
  Eating in front of others C16D1: number analyzed (Participants) | 35 | 22
  Eating in front of others C16D1 | -2.86 (18.74) | -1.52 (21.77)
  Eating in front of others C16D22: number analyzed (Participants) | 29 | 14
  Eating in front of others C16D22 | -2.30 (17.66) | -4.76 (17.82)
  Eating in front of others C17D1: number analyzed (Participants) | 30 | 18
  Eating in front of others C17D1 | -2.22 (21.32) | -3.70 (15.71)
  Eating in front of others C17D22: number analyzed (Participants) | 23 | 0
  Eating in front of others C17D22 | -1.45 (23.52) |
  Eating in front of others C18D1: number analyzed (Participants) | 27 | 16
  Eating in front of others C18D1 | -3.70 (16.88) | -4.17 (16.67)
  Eating in front of others C18D22: number analyzed (Participants) | 20 | 10
  Eating in front of others C18D22 | -3.33 (18.42) | -10.00 (16.10)
  Eating in front of others C19D1: number analyzed (Participants) | 23 | 15
  Eating in front of others C19D1 | -5.80 (16.37) | -4.44 (17.21)
  Eating in front of others C19D22: number analyzed (Participants) | 20 | 11
  Eating in front of others C19D22 | -6.67 (17.44) | -6.06 (13.48)
  Eating in front of others C20D1: number analyzed (Participants) | 23 | 15
  Eating in front of others C20D1 | -4.35 (15.26) | -4.44 (17.21)
  Eating in front of others C20D22: number analyzed (Participants) | 18 | 10
  Eating in front of others C20D22 | -3.70 (19.43) | -6.67 (21.08)
  Eating in Front of Other C21D1: number analyzed (Participants) | 20 | 14
  Eating in Front of Other C21D1 | -3.33 (14.91) | -7.14 (19.30)
  Eating in front of others C21D22: number analyzed (Participants) | 14 | 0
  Eating in front of others C21D22 | -4.76 (17.82) |
  Eating in front of others C22D1: number analyzed (Participants) | 15 | 12
  Eating in front of others C22D1 | -2.22 (15.26) | -5.56 (19.25)
  Eating in front of others C22D22: number analyzed (Participants) | 10 | 0
  Eating in front of others C22D22 | 0.00 (15.71) |
  Eating in front of others C23D1: number analyzed (Participants) | 15 | 13
  Eating in front of others C23D1 | -4.44 (17.21) | -2.56 (21.35)
  Eating in front of others C23D22: number analyzed (Participants) | 11 | 0
  Eating in front of others C23D22 | -3.03 (10.05) |
  Eating in front of others C24D1: number analyzed (Participants) | 14 | 0
  Eating in front of others C24D1 | -4.76 (17.82) |
  Eating in front of others C25D1: number analyzed (Participants) | 12 | 0
  Eating in front of others C25D1 | -8.33 (15.08) |
  Eating in front of others C25D22: number analyzed (Participants) | 11 | 0
  Eating in front of others C25D22 | -3.03 (17.98) |
  Eating in front of others C26D1: number analyzed (Participants) | 13 | 0
  Eating in front of others C26D1 | -7.69 (19.97) |
  Eating in front of others C27D1: number analyzed (Participants) | 11 | 0
  Eating in front of others C27D1 | -6.06 (20.10) |
  Eating in front of others C28D1: number analyzed (Participants) | 12 | 0
  Eating in front of others C28D1 | -5.56 (19.25) |
  Eating in front of others 30 day follow up: number analyzed (Participants) | 72 | 90
  Eating in front of others 30 day follow up | 3.24 (24.49) | 0.37 (33.70)
  Eating in front of others 90 day follow up: number analyzed (Participants) | 86 | 82
  Eating in front of others 90 day follow up | 1.94 (25.23) | 0.81 (34.34)
  Dry Mouth Baseline | 21.92 (26.99) | 22.70 (26.83)
  Dry Mouth C1D22: number analyzed (Participants) | 176 | 208
  Dry Mouth C1D22 | 5.68 (27.01) | 4.33 (27.17)
  Dry Mouth C2D1: number analyzed (Participants) | 206 | 223
  Dry Mouth C2D1 | 1.78 (31.10) | 0.45 (28.03)
  Dry Mouth C2D22: number analyzed (Participants) | 150 | 180
  Dry Mouth C2D22 | 3.56 (26.80) | 1.11 (29.67)
  Dry Mouth C3D1: number analyzed (Participants) | 190 | 196
  Dry Mouth C3D1 | 1.05 (31.03) | -1.53 (29.68)
  Dry Mouth C3D22: number analyzed (Participants) | 152 | 148
  Dry Mouth C3D22 | 4.39 (30.85) | 1.13 (29.46)
  Dry Mouth C4D1: number analyzed (Participants) | 169 | 161
  Dry Mouth C4D1 | -0.39 (30.43) | -0.62 (29.22)
  Dry Mouth C4D22: number analyzed (Participants) | 122 | 127
  Dry Mouth C4D22 | 1.09 (29.36) | 1.57 (29.05)
  Dry Mouth C5D1: number analyzed (Participants) | 148 | 144
  Dry Mouth C5D1 | 3.15 (32.14) | 1.16 (27.43)
  Dry Mouth C5D22: number analyzed (Participants) | 110 | 115
  Dry Mouth C5D22 | -1.91 (26.87) | -0.58 (25.74)
  Dry Mouth C6D1: number analyzed (Participants) | 122 | 121
  Dry Mouth C6D1 | -0.87 (25.92) | 0.28 (29.66)
  Dry Mouth C6D22: number analyzed (Participants) | 103 | 92
  Dry Mouth C6D22 | -3.56 (27.97) | -3.99 (25.60)
  Dry Mouth C7D1: number analyzed (Participants) | 113 | 98
  Dry Mouth C7D1 | -2.06 (25.31) | -2.38 (29.21)
  Dry Mouth C7D22: number analyzed (Participants) | 81 | 73
  Dry Mouth C7D22 | -0.82 (29.33) | -3.65 (31.21)
  Dry Mouth C8D1: number analyzed (Participants) | 80 | 81
  Dry Mouth C8D1 | -0.83 (28.05) | -3.29 (29.16)
  Dry Mouth C8D22: number analyzed (Participants) | 71 | 65
  Dry Mouth C8D22 | -0.94 (28.16) | 0.51 (30.33)
  Dry Mouth C9D1: number analyzed (Participants) | 75 | 62
  Dry Mouth C9D1 | -0.44 (27.67) | -0.54 (30.47)
  Dry Mouth C9D22: number analyzed (Participants) | 60 | 55
  Dry Mouth C9D22 | 2.22 (29.98) | -1.21 (31.40)
  Dry Mouth C10D1: number analyzed (Participants) | 66 | 56
  Dry Mouth C10D1 | -0.51 (30.66) | -2.38 (28.33)
  Dry Mouth C10D22: number analyzed (Participants) | 57 | 43
  Dry Mouth C10D22 | -0.58 (25.58) | -0.78 (31.28)
  Dry Mouth C11D1: number analyzed (Participants) | 63 | 46
  Dry Mouth C11D1 | 1.59 (27.06) | -2.17 (27.58)
  Dry Mouth C11D22: number analyzed (Participants) | 44 | 31
  Dry Mouth C11D22 | 2.27 (24.27) | -1.08 (21.92)
  Dry Mouth C12D1: number analyzed (Participants) | 53 | 41
  Dry Mouth C12D1 | 2.52 (29.12) | -0.81 (29.33)
  Dry Mouth C12D22: number analyzed (Participants) | 37 | 25
  Dry Mouth C12D22 | 0.90 (25.44) | 2.67 (27.08)
  Dry Mouth C13D1: number analyzed (Participants) | 48 | 35
  Dry Mouth C13D1 | 2.08 (26.10) | -1.90 (29.09)
  Dry Mouth C13D22: number analyzed (Participants) | 40 | 21
  Dry Mouth C13D22 | 4.17 (25.25) | -1.59 (34.12)
  Dry Mouth C14D1: number analyzed (Participants) | 39 | 30
  Dry Mouth C14D1 | 0.00 (26.49) | -4.44 (29.99)
  Dry Mouth C14D22: number analyzed (Participants) | 32 | 19
  Dry Mouth C14D22 | 0.00 (26.77) | -5.26 (31.94)
  Dry Mouth C15D1: number analyzed (Participants) | 35 | 27
  Dry Mouth C15D1 | 0.00 (29.15) | -9.88 (28.96)
  Dry Mouth C15D22: number analyzed (Participants) | 29 | 17
  Dry Mouth C15D22 | 0.00 (26.73) | -13.73 (33.46)
  Dry Mouth C16D1: number analyzed (Participants) | 35 | 22
  Dry Mouth C16D1 | -1.90 (27.94) | -12.12 (30.07)
  Dry Mouth C16D22: number analyzed (Participants) | 29 | 14
  Dry Mouth C16D22 | 2.30 (26.62) | -7.14 (41.71)
  Dry Mouth C17D1: number analyzed (Participants) | 30 | 18
  Dry Mouth C17D1 | 5.56 (30.43) | -9.26 (31.94)
  Dry Mouth C17D22: number analyzed (Participants) | 23 | 0
  Dry Mouth C17D22 | 1.45 (27.48) |
  Dry Mouth C18D1: number analyzed (Participants) | 27 | 16
  Dry Mouth C18D1 | -3.70 (23.27) | -8.33 (35.49)
  Dry Mouth C18D22: number analyzed (Participants) | 20 | 10
  Dry Mouth C18D22 | -1.67 (22.88) | -6.67 (30.63)
  Dry Mouth C19D1: number analyzed (Participants) | 23 | 15
  Dry Mouth C19D1 | -2.90 (26.43) | -2.22 (23.46)
  Dry Mouth C19D22: number analyzed (Participants) | 20 | 11
  Dry Mouth C19D22 | -3.33 (18.42) | 0.00 (29.81)
  Dry Mouth C20D1: number analyzed (Participants) | 23 | 15
  Dry Mouth C20D1 | -5.80 (25.92) | -4.44 (24.77)
  Dry Mouth C20D22: number analyzed (Participants) | 18 | 10
  Dry Mouth C20D22 | -5.56 (23.57) | -6.67 (30.63)
  Dry Mouth C21D1: number analyzed (Participants) | 20 | 14
  Dry Mouth C21D1 | -10.00 (24.42) | -2.38 (27.62)
  Dry Mouth C21D22: number analyzed (Participants) | 14 | 12
  Dry Mouth C21D22 | -4.76 (22.10) | -11.11 (21.71)
  Dry Mouth C22D1: number analyzed (Participants) | 15 | 13
  Dry Mouth C22D1 | -11.11 (24.12) | -2.56 (28.74)
  Dry Mouth C22D22: number analyzed (Participants) | 10 | 0
  Dry Mouth C22D22 | -10.00 (22.50) |
  Dry Mouth C23D1: number analyzed (Participants) | 15 | 13
  Dry Mouth C23D1 | -13.33 (27.60) | -2.56 (28.74)
  Dry Mouth C23D22: number analyzed (Participants) | 11 | 0
  Dry Mouth C23D22 | -12.12 (22.47) |
  Dry Mouth C24D1: number analyzed (Participants) | 14 | 0
  Dry Mouth C24D1 | -14.29 (25.20) |
  Dry Mouth C25D1: number analyzed (Participants) | 12 | 0
  Dry Mouth C25D1 | -11.11 (21.71) |
  Dry Mouth C25D22: number analyzed (Participants) | 11 | 0
  Dry Mouth C25D22 | -12.12 (22.47) |
  Dry Mouth C26D1: number analyzed (Participants) | 13 | 0
  Dry Mouth C26D1 | -17.95 (25.88) |
  Dry Mouth C27D1: number analyzed (Participants) | 11 | 0
  Dry Mouth C27D1 | -21.21 (26.97) |
  Dry Mouth C28D1: number analyzed (Participants) | 12 | 0
  Dry Mouth C28D1 | -19.44 (26.43) |
  Dry Mouth 30 day follow up: number analyzed (Participants) | 72 | 90
  Dry Mouth 30 day follow up | 5.09 (28.89) | 5.19 (36.69)
  Dry Mouth 90 Day follow up: number analyzed (Participants) | 86 | 82
  Dry Mouth 90 Day follow up | 1.94 (30.83) | 4.47 (33.85)
  Trouble with taste Baseline | 12.06 (23.32) | 11.54 (22.07)
  Trouble with taste C1D22: number analyzed (Participants) | 176 | 208
  Trouble with taste C1D22 | 10.80 (29.66) | 8.17 (27.46)
  Trouble with taste C2D1: number analyzed (Participants) | 206 | 223
  Trouble with taste C2D1 | 12.62 (29.49) | 4.19 (28.69)
  Trouble with taste C2D22: number analyzed (Participants) | 150 | 180
  Trouble with taste C2D22 | 15.78 (33.60) | 10.56 (31.01)
  Trouble with taste C3D1: number analyzed (Participants) | 190 | 196
  Trouble with taste C3D1 | 14.56 (34.52) | 9.35 (30.53)
  Trouble with taste C3D22: number analyzed (Participants) | 152 | 148
  Trouble with taste C3D22 | 21.93 (31.66) | 13.51 (31.31)
  Trouble with taste C4D1: number analyzed (Participants) | 169 | 161
  Trouble with taste C4D1 | 17.75 (35.46) | 15.94 (34.78)
  Trouble with taste C4D22: number analyzed (Participants) | 122 | 127
  Trouble with taste C4D22 | 20.49 (32.48) | 16.01 (35.10)
  Trouble with taste C5D1: number analyzed (Participants) | 148 | 144
  Trouble with taste C5D1 | 19.59 (31.81) | 15.05 (29.98)
  Trouble with taste C5D22: number analyzed (Participants) | 110 | 115
  Trouble with taste C5D22 | 20.00 (28.98) | 16.52 (30.71)
  Trouble with taste C6D1: number analyzed (Participants) | 122 | 121
  Trouble with taste C6D1 | 12.02 (27.46) | 15.70 (26.90)
  Trouble with taste C6D22: number analyzed (Participants) | 103 | 92
  Trouble with taste C6D22 | 9.71 (29.38) | 10.87 (28.86)
  Trouble with taste C7D1: number analyzed (Participants) | 113 | 98
  Trouble with taste C7D1 | 8.55 (24.71) | 9.18 (23.83)
  Trouble with taste C7D22: number analyzed (Participants) | 81 | 73
  Trouble with taste C7D22 | 10.70 (26.78) | 10.50 (24.77)
  Trouble with taste C8D1: number analyzed (Participants) | 80 | 81
  Trouble with taste C8D1 | 6.25 (22.56) | 10.70 (22.25)
  Trouble with taste C8D22: number analyzed (Participants) | 71 | 65
  Trouble with taste C8D22 | 3.76 (22.22) | 11.28 (22.26)
  Trouble with taste C9D1: number analyzed (Participants) | 75 | 62
  Trouble with taste C9D1 | 3.56 (20.92) | 12.37 (28.46)
  Trouble with taste C9D22: number analyzed (Participants) | 60 | 55
  Trouble with taste C9D22 | 12.78 (28.85) | 11.52 (27.38)
  Trouble with taste C10D1: number analyzed (Participants) | 66 | 56
  Trouble with taste C10D1 | 7.07 (23.76) | 8.33 (21.32)
  Trouble with taste C10D22: number analyzed (Participants) | 57 | 43
  Trouble with taste C10D22 | 7.02 (22.48) | 9.30 (23.37)
  Trouble with taste C11D1: number analyzed (Participants) | 63 | 46
  Trouble with taste C11D1 | 6.35 (26.00) | 7.25 (20.98)
  Trouble with taste C11D22: number analyzed (Participants) | 44 | 31
  Trouble with taste C11D22 | 4.55 (18.46) | 8.60 (24.29)
  Trouble with taste C12D1: number analyzed (Participants) | 53 | 41
  Trouble with taste C12D1 | 6.29 (26.20) | 8.13 (17.92)
  Trouble with taste C12D22: number analyzed (Participants) | 37 | 25
  Trouble with taste C12D22 | 11.71 (25.11) | 16.00 (27.42)
  Trouble with taste C13D1: number analyzed (Participants) | 48 | 35
  Trouble with taste C13D1 | 7.64 (20.90) | 10.48 (25.27)
  Trouble with taste C13D22: number analyzed (Participants) | 40 | 21
  Trouble with taste C13D22 | 10.00 (27.43) | 22.22 (30.43)
  Trouble with taste C14D1: number analyzed (Participants) | 39 | 30
  Trouble with taste C14D1 | 4.27 (24.40) | 14.44 (27.24)
  Trouble with taste C14D22: number analyzed (Participants) | 32 | 19
  Trouble with taste C14D22 | 9.37 (22.77) | 12.28 (22.80)
  Trouble with taste C15D1: number analyzed (Participants) | 35 | 27
  Trouble with taste C15D1 | 3.81 (26.53) | 6.17 (18.58)
  Trouble with taste C15D22: number analyzed (Participants) | 29 | 17
  Trouble with taste C15D22 | 11.49 (28.56) | 3.92 (20.01)
  Trouble with taste C16D1: number analyzed (Participants) | 35 | 22
  Trouble with taste C16D1 | 7.62 (21.52) | 4.55 (18.67)
  Trouble with taste C16D22: number analyzed (Participants) | 29 | 14
  Trouble with taste C16D22 | 6.90 (24.20) | 4.76 (22.10)
  Trouble with taste C17D1: number analyzed (Participants) | 30 | 18
  Trouble with taste C17D1 | 4.44 (24.34) | 5.56 (20.61)
  Trouble with taste C17D22: number analyzed (Participants) | 23 | 0
  Trouble with taste C17D22 | 11.59 (29.49) |
  Trouble with taste C18D1: number analyzed (Participants) | 27 | 16
  Trouble with taste C18D1 | 1.23 (19.57) | 4.17 (20.64)
  Trouble with taste C18D22: number analyzed (Participants) | 20 | 10
  Trouble with taste C18D22 | 3.33 (18.42) | 6.67 (26.29)
  Trouble with taste C19D1: number analyzed (Participants) | 23 | 15
  Trouble with taste C19D1 | 2.90 (17.15) | 4.44 (17.21)
  Trouble with taste C19D22: number analyzed (Participants) | 20 | 11
  Trouble with taste C19D22 | 5.00 (22.36) | 6.06 (25.03)
  Trouble with taste C20D1: number analyzed (Participants) | 23 | 15
  Trouble with taste C20D1 | 1.45 (15.82) | 6.67 (22.54)
  Trouble with taste C20D22: number analyzed (Participants) | 18 | 10
  Trouble with taste C20D22 | 3.70 (15.71) | 0.00 (15.71)
  Trouble with taste C21D1: number analyzed (Participants) | 20 | 14
  Trouble with taste C21D1 | 6.67 (17.44) | 0.00 (13.07)
  Trouble with Taste C21D22: number analyzed (Participants) | 14 | 0
  Trouble with Taste C21D22 | -2.38 (20.52) |
  Trouble with taste C22D1: number analyzed (Participants) | 15 | 12
  Trouble with taste C22D1 | 2.22 (15.26) | 5.56 (23.92)
  Trouble with taste C22D22: number analyzed (Participants) | 10 | 0
  Trouble with taste C22D22 | 0.00 (15.71) |
  Trouble with taste C23D1: number analyzed (Participants) | 15 | 13
  Trouble with taste C23D1 | 2.22 (15.26) | 5.13 (22.96)
  Trouble with taste C23D22: number analyzed (Participants) | 11 | 0
  Trouble with taste C23D22 | 6.06 (13.48) |
  Trouble with taste C24D1: number analyzed (Participants) | 14 | 0
  Trouble with taste C24D1 | 2.38 (15.82) |
  Trouble with taste C25D1: number analyzed (Participants) | 12 | 0
  Trouble with taste C25D1 | 0.00 (20.10) |
  Trouble with taste C25D22: number analyzed (Participants) | 11 | 0
  Trouble with taste C25D22 | 3.03 (17.98) |
  Trouble with taste C26D1: number analyzed (Participants) | 13 | 0
  Trouble with taste C26D1 | 2.56 (16.45) |
  Trouble with taste C27D1: number analyzed (Participants) | 11 | 0
  Trouble with taste C27D1 | 0.00 (14.91) |
  Trouble with taste C28D1: number analyzed (Participants) | 12 | 0
  Trouble with taste C28D1 | 2.78 (22.29) |
  Trouble with taste 30 day follow up: number analyzed (Participants) | 72 | 90
  Trouble with taste 30 day follow up | 12.96 (27.15) | 15.93 (32.08)
  Trouble with taste 90 day follow up: number analyzed (Participants) | 86 | 82
  Trouble with taste 90 day follow up | 14.73 (28.29) | 13.82 (32.69)
  Body Image Baseline | 22.57 (29.62) | 24.90 (30.80)
  Body Image C1D22: number analyzed (Participants) | 176 | 208
  Body Image C1D22 | 3.60 (25.06) | -0.96 (26.60)
  Body Image C2D1: number analyzed (Participants) | 206 | 223
  Body Image C2D1 | 3.56 (26.91) | 0.00 (31.00)
  Body Image C2D22: number analyzed (Participants) | 150 | 180
  Body Image C2D22 | 5.11 (26.96) | 2.78 (30.08)
  Body Image C3D1: number analyzed (Participants) | 190 | 196
  Body Image C3D1 | 4.21 (25.54) | -0.51 (29.33)
  Body Image C3D22: number analyzed (Participants) | 152 | 148
  Body Image C3D22 | 7.46 (25.21) | -0.90 (28.02)
  Body Image C4D1: number analyzed (Participants) | 169 | 161
  Body Image C4D1 | 1.58 (24.07) | -4.35 (28.90)
  Body Image C4D22: number analyzed (Participants) | 122 | 127
  Body Image C4D22 | 9.29 (27.53) | -3.41 (26.84)
  Body Image C5D1: number analyzed (Participants) | 148 | 144
  Body Image C5D1 | 5.63 (28.67) | -3.01 (26.42)
  Body Image C5D22: number analyzed (Participants) | 110 | 115
  Body Image C5D22 | 5.76 (30.91) | -2.32 (34.69)
  Body Image C6D1: number analyzed (Participants) | 122 | 121
  Body Image C6D1 | 4.64 (31.00) | -1.93 (28.32)
  Body Image C6D22: number analyzed (Participants) | 103 | 92
  Body Image C6D22 | 1.62 (27.76) | -4.71 (29.06)
  Body Image C7D1: number analyzed (Participants) | 113 | 98
  Body Image C7D1 | -0.29 (29.04) | -2.72 (31.27)
  Body Image C7D22: number analyzed (Participants) | 81 | 73
  Body Image C7D22 | 3.70 (30.28) | -5.48 (34.25)
  Body Image C8D1: number analyzed (Participants) | 80 | 81
  Body Image C8D1 | -1.25 (28.29) | -2.88 (30.82)
  Body Image C8D22: number analyzed (Participants) | 71 | 65
  Body Image C8D22 | -0.47 (31.11) | -6.15 (29.98)
  Body Image C9D1: number analyzed (Participants) | 75 | 62
  Body Image C9D1 | -4.44 (30.67) | -8.06 (32.33)
  Body Image C9D22: number analyzed (Participants) | 60 | 55
  Body Image C9D22 | -1.11 (32.46) | -8.48 (32.21)
  Body Image C10D1: number analyzed (Participants) | 66 | 56
  Body Image C10D1 | -1.01 (32.54) | -4.17 (33.67)
  Body Image C10D22: number analyzed (Participants) | 57 | 43
  Body Image C10D22 | -0.58 (31.80) | -10.08 (31.32)
  Body Image C11D1: number analyzed (Participants) | 63 | 46
  Body Image C11D1 | -2.65 (31.28) | -5.07 (31.40)
  Body Image C11D22: number analyzed (Participants) | 44 | 31
  Body Image C11D22 | -7.58 (27.72) | -7.53 (33.01)
  Body Image C12D1: number analyzed (Participants) | 53 | 41
  Body Image C12D1 | -0.63 (28.86) | -7.32 (30.29)
  Body Image C12D22: number analyzed (Participants) | 37 | 25
  Body Image C12D22 | 0.00 (33.33) | -4.00 (26.03)
  Body Image C13D1: number analyzed (Participants) | 48 | 35
  Body Image C13D1 | -2.08 (31.81) | -5.71 (27.40)
  Body Image C13D22: number analyzed (Participants) | 40 | 21
  Body Image C13D22 | -5.00 (28.79) | -12.70 (32.45)
  Body Image C14D1: number analyzed (Participants) | 39 | 30
  Body Image C14D1 | -4.27 (30.76) | -11.11 (33.14)
  Body Image C14D22: number analyzed (Participants) | 32 | 19
  Body Image C14D22 | -1.04 (31.09) | -12.28 (33.72)
  Body Image C15D1: number analyzed (Participants) | 35 | 27
  Body Image C15D1 | -3.81 (27.74) | -12.35 (33.52)
  Body Image C15D22: number analyzed (Participants) | 29 | 17
  Body Image C15D22 | 29.08 (8.05) | -17.65 (33.58)
  Body Image C16D1: number analyzed (Participants) | 35 | 22
  Body Image C16D1 | -5.71 (28.57) | -10.61 (37.64)
  Body Image C16D22: number analyzed (Participants) | 29 | 14
  Body Image C16D22 | -8.05 (26.21) | -14.29 (33.88)
  Body Image C17D1: number analyzed (Participants) | 30 | 18
  Body Image C17D1 | 0.00 (36.09) | -7.41 (26.95)
  Body Image C17D22: number analyzed (Participants) | 23 | 0
  Body Image C17D22 | -2.90 (30.01) |
  Body Image C18D1: number analyzed (Participants) | 27 | 16
  Body Image C18D1 | -7.41 (21.35) | -4.17 (31.91)
  Body Image C18D22: number analyzed (Participants) | 20 | 10
  Body Image C18D22 | -5.00 (27.09) | -20.00 (28.11)
  Body Image C19D1: number analyzed (Participants) | 23 | 15
  Body Image C19D1 | -1.45 (25.58) | -4.44 (30.52)
  Body Image C19D22: number analyzed (Participants) | 20 | 11
  Body Image C19D22 | -5.00 (24.84) | -12.12 (34.23)
  Body Image C20D1: number analyzed (Participants) | 23 | 15
  Body Image C20D1 | -2.90 (28.27) | -8.89 (29.46)
  Body Image C20D22: number analyzed (Participants) | 18 | 10
  Body Image C20D22 | -3.70 (27.75) | -16.67 (32.39)
  Body Image C21D1: number analyzed (Participants) | 20 | 14
  Body Image C21D1 | -6.67 (17.44) | 2.38 (40.22)
  Body Image C21D22: number analyzed (Participants) | 14 | 0
  Body Image C21D22 | -4.76 (22.10) |
  Body Image C22D1: number analyzed (Participants) | 15 | 12
  Body Image C22D1 | 0.00 (28.17) | -13.89 (36.12)
  Body Image C22D22: number analyzed (Participants) | 10 | 0
  Body Image C22D22 | -6.67 (30.63) |
  Body Image C23D1: number analyzed (Participants) | 15 | 13
  Body Image C23D1 | -6.67 (22.54) | -5.13 (35.61)
  Body Image C23D22: number analyzed (Participants) | 11 | 0
  Body Image C23D22 | -6.06 (20.10) |
  Body Image C24D1: number analyzed (Participants) | 14 | 0
  Body Image C24D1 | -4.76 (22.10) |
  Body Image C25D1: number analyzed (Participants) | 12 | 0
  Body Image C25D1 | -8.33 (28.87) |
  Body Image C25D22: number analyzed (Participants) | 11 | 0
  Body Image C25D22 | -9.09 (30.15) |
  Body Image C26D1: number analyzed (Participants) | 13 | 0
  Body Image C26D1 | -5.13 (26.69) |
  Body Image C27D1: number analyzed (Participants) | 11 | 0
  Body Image C27D1 | -12.12 (16.82) |
  Body Image C28D1: number analyzed (Participants) | 12 | 0
  Body Image C28D1 | -11.11 (16.41) |
  Body Image 30 day follow up: number analyzed (Participants) | 72 | 90
  Body Image 30 day follow up | 9.72 (28.77) | 5.56 (31.70)
  Body Image 90 Day follow up: number analyzed (Participants) | 86 | 82
  Body Image 90 Day follow up | 6.98 (32.39) | 8.94 (29.65)
  Trouble swallowing saliva Baseline | 7.65 (17.36) | 9.08 (20.93)
  Trouble swallowing saliva C1D22: number analyzed (Participants) | 176 | 208
  Trouble swallowing saliva C1D22 | 0.95 (21.51) | -2.40 (19.65)
  Trouble swallowing saliva C2D1: number analyzed (Participants) | 206 | 223
  Trouble swallowing saliva C2D1 | 1.46 (21.91) | -3.44 (24.57)
  Trouble swallowing saliva C2D22: number analyzed (Participants) | 150 | 180
  Trouble swallowing saliva C2D22 | 1.56 (19.44) | -2.41 (24.16)
  Trouble swallowing saliva C3D1: number analyzed (Participants) | 190 | 196
  Trouble swallowing saliva C3D1 | -0.18 (20.72) | -2.89 (22.59)
  Trouble swallowing saliva C3D22: number analyzed (Participants) | 152 | 148
  Trouble swallowing saliva C3D22 | 3.73 (25.02) | -2.25 (21.88)
  Trouble swallowing saliva C4D1: number analyzed (Participants) | 169 | 161
  Trouble swallowing saliva C4D1 | -0.59 (21.66) | -3.11 (21.34)
  Trouble swallowing saliva C4D22: number analyzed (Participants) | 122 | 127
  Trouble swallowing saliva C4D22 | 1.64 (23.41) | 0.26 (21.62)
  Trouble swallowing saliva C5D1: number analyzed (Participants) | 148 | 144
  Trouble swallowing saliva C5D1 | 3.60 (24.01) | -2.78 (19.51)
  Trouble swallowing saliva C5D22: number analyzed (Participants) | 110 | 115
  Trouble swallowing saliva C5D22 | 2.12 (21.31) | -1.45 (21.81)
  Trouble swallowing saliva C6D1: number analyzed (Participants) | 122 | 121
  Trouble swallowing saliva C6D1 | -0.82 (18.41) | -0.55 (20.63)
  Trouble swallowing saliva C6D22: number analyzed (Participants) | 103 | 92
  Trouble swallowing saliva C6D22 | -1.29 (18.03) | -1.45 (20.32)
  Trouble swallowing saliva C7D1: number analyzed (Participants) | 113 | 98
  Trouble swallowing saliva C7D1 | -1.77 (19.33) | -1.70 (18.77)
  Trouble swallowing saliva C7D22: number analyzed (Participants) | 81 | 73
  Trouble swallowing saliva C7D22 | -0.41 (20.75) | -0.91 (20.77)
  Trouble swallowing saliva C8D1: number analyzed (Participants) | 80 | 81
  Trouble swallowing saliva C8D1 | 0.00 (19.12) | -2.47 (18.09)
  Trouble swallowing saliva C8D22: number analyzed (Participants) | 71 | 65
  Trouble swallowing saliva C8D22 | -0.47 (17.36) | -3.59 (22.14)
  Trouble swallowing saliva C9D1: number analyzed (Participants) | 75 | 62
  Trouble swallowing saliva C9D1 | -0.44 (17.75) | -2.15 (19.90)
  Trouble swallowing saliva C9D22: number analyzed (Participants) | 60 | 55
  Trouble swallowing saliva C9D22 | 0.56 (19.88) | -2.42 (20.14)
  Trouble swallowing saliva C10D1: number analyzed (Participants) | 66 | 56
  Trouble swallowing saliva C10D1 | -1.52 (21.43) | -2.38 (19.96)
  Trouble swallowing saliva C10D22: number analyzed (Participants) | 57 | 43
  Trouble swallowing saliva C10D22 | -1.17 (20.86) | -0.78 (21.19)
  Trouble swallowing saliva C11D1: number analyzed (Participants) | 63 | 46
  Trouble swallowing saliva C11D1 | 0.00 (19.86) | 1.45 (23.26)
  Trouble swallowing saliva C11D22: number analyzed (Participants) | 44 | 31
  Trouble swallowing saliva C11D22 | -4.55 (21.07) | 4.30 (11.36)
  Trouble swallowing saliva C12D1: number analyzed (Participants) | 53 | 41
  Trouble swallowing saliva C12D1 | 0.00 (14.62) | 0.00 (21.08)
  Trouble swallowing saliva C12D22: number analyzed (Participants) | 37 | 25
  Trouble swallowing saliva C12D22 | -3.60 (21.92) | 2.67 (16.44)
  Trouble swallowing saliva C13D1: number analyzed (Participants) | 48 | 35
  Trouble swallowing saliva C13D1 | -1.39 (22.76) | 0.00 (22.87)
  Trouble swallowing saliva C13D22: number analyzed (Participants) | 40 | 21
  Trouble swallowing saliva C13D22 | 0.00 (23.87) | 0.00 (25.82)
  Trouble swallowing saliva C14D1: number analyzed (Participants) | 39 | 30
  Trouble swallowing saliva C14D1 | 1.71 (17.01) | -3.33 (20.25)
  Trouble swallowing saliva C14D22: number analyzed (Participants) | 32 | 19
  Trouble swallowing saliva C14D22 | -2.08 (14.51) | -3.51 (24.58)
  Trouble swallowing saliva C15D1: number analyzed (Participants) | 35 | 27
  Trouble swallowing saliva C15D1 | -0.95 (15.09) | -6.17 (20.75)
  Trouble swallowing saliva C15D22: number analyzed (Participants) | 29 | 17
  Trouble swallowing saliva C15D22 | -2.30 (12.38) | -5.88 (24.25)
  Trouble swallowing saliva C16D1: number analyzed (Participants) | 35 | 22
  Trouble swallowing saliva C16D1 | 0.95 (15.09) | -3.03 (22.79)
  Trouble swallowing saliva C16D22: number analyzed (Participants) | 29 | 14
  Trouble swallowing saliva C16D22 | -1.15 (14.04) | -7.14 (26.73)
  Trouble swallowing saliva C17D1: number analyzed (Participants) | 30 | 18
  Trouble swallowing saliva C17D1 | 1.11 (16.34) | -5.56 (23.57)
  Trouble swallowing saliva C17D22: number analyzed (Participants) | 23 | 0
  Trouble swallowing saliva C17D22 | 0.00 (17.41) |
  Trouble swallowing saliva C18D1: number analyzed (Participants) | 27 | 16
  Trouble swallowing saliva C18D1 | -1.23 (17.25) | -6.25 (25.00)
  Trouble swallowing saliva C18D22: number analyzed (Participants) | 20 | 10
  Trouble swallowing saliva C18D22 | -1.67 (13.13) | 3.33 (10.54)
  Trouble swallowing saliva C19D1: number analyzed (Participants) | 23 | 15
  Trouble swallowing saliva C19D1 | -1.45 (12.22) | 0.00 (0.00)
  Trouble swallowing saliva C19D22: number analyzed (Participants) | 20 | 11
  Trouble swallowing saliva C19D22 | 0.00 (10.81) | 0.00 (0.00)
  Trouble swallowing saliva C20D1: number analyzed (Participants) | 23 | 15
  Trouble swallowing saliva C20D1 | 0.00 (10.05) | 0.00 (0.00)
  Trouble swallowing saliva C20D22: number analyzed (Participants) | 18 | 10
  Trouble swallowing saliva C20D22 | 0.00 (11.43) | 3.33 (10.54)
  Trouble swallowing saliva C21D1: number analyzed (Participants) | 20 | 14
  Trouble swallowing saliva C21D1 | 1.67 (13.13) | 0.00 (0.00)
  Trouble swallowing saliva C21D22: number analyzed (Participants) | 14 | 0
  Trouble swallowing saliva C21D22 | 0.00 (13.07) |
  Trouble swallowing saliva C22D1: number analyzed (Participants) | 15 | 12
  Trouble swallowing saliva C22D1 | -4.44 (17.21) | 0.00 (0.00)
  Trouble swallowing saliva C22D22: number analyzed (Participants) | 10 | 0
  Trouble swallowing saliva C22D22 | -6.67 (21.08) |
  Trouble swallowing saliva C23D1: number analyzed (Participants) | 15 | 13
  Trouble swallowing saliva C23D1 | -4.44 (17.21) | 0.00 (0.00)
  Trouble swallowing saliva C23D22: number analyzed (Participants) | 11 | 0
  Trouble swallowing saliva C23D22 | -9.09 (15.57) |
  Trouble swallowing saliva C24D1: number analyzed (Participants) | 14 | 0
  Trouble swallowing saliva C24D1 | -2.38 (15.82) |
  Trouble swallowing saliva C25D1: number analyzed (Participants) | 12 | 0
  Trouble swallowing saliva C25D1 | -8.33 (15.08) |
  Trouble swallowing saliva C25D22: number analyzed (Participants) | 11 | 0
  Trouble swallowing saliva C25D22 | -3.03 (17.98) |
  Trouble swallowing saliva C26D1: number analyzed (Participants) | 13 | 0
  Trouble swallowing saliva C26D1 | -2.56 (21.35) |
  Trouble swallowing saliva C27D1: number analyzed (Participants) | 11 | 0
  Trouble swallowing saliva C27D1 | -3.03 (17.98) |
  Trouble swallowing saliva C28D1: number analyzed (Participants) | 12 | 0
  Trouble swallowing saliva C28D1 | -2.78 (17.16) |
  Trouble swallowing saliva 30 Day follow up: number analyzed (Participants) | 72 | 90
  Trouble swallowing saliva 30 Day follow up | 6.94 (24.35) | -0.37 (24.73)
  Trouble swallowing saliva 90 Day follow up: number analyzed (Participants) | 86 | 82
  Trouble swallowing saliva 90 Day follow up | 2.33 (24.94) | -1.63 (24.51)
  Choked when swallowing Baseline | 7.00 (18.24) | 6.10 (15.65)
  Choked when swallowing C1D22: number analyzed (Participants) | 176 | 208
  Choked when swallowing C1D22 | 1.52 (17.75) | -1.28 (16.98)
  Choked when swallowing C2D1: number analyzed (Participants) | 206 | 223
  Choked when swallowing C2D1 | -0.49 (17.26) | -1.05 (13.93)
  Choked when swallowing C2D22: number analyzed (Participants) | 150 | 180
  Choked when swallowing C2D22 | -2.67 (19.12) | -1.30 (16.29)
  Choked when swallowing C3D1: number analyzed (Participants) | 190 | 196
  Choked when swallowing C3D1 | -1.23 (18.90) | -0.34 (15.47)
  Choked when swallowing C3D22: number analyzed (Participants) | 152 | 148
  Choked when swallowing C3D22 | 2.19 (19.81) | -2.93 (16.46)
  Choked when swallowing C4D1: number analyzed (Participants) | 169 | 161
  Choked when swallowing C4D1 | -0.99 (17.22) | -1.86 (16.77)
  Choked when swallowing C4D22: number analyzed (Participants) | 122 | 127
  Choked when swallowing C4D22 | 1.09 (18.15) | -0.26 (17.57)
  Choked when swallowing C5D1: number analyzed (Participants) | 148 | 144
  Choked when swallowing C5D1 | 0.45 (18.64) | -2.08 (15.88)
  Choked when swallowing C5D22: number analyzed (Participants) | 110 | 115
  Choked when swallowing C5D22 | 0.91 (18.87) | 0.29 (18.47)
  Choked when swallowing C6D1: number analyzed (Participants) | 122 | 121
  Choked when swallowing C6D1 | -1.37 (17.87) | 0.83 (17.98)
  Choked when swallowing C6D22: number analyzed (Participants) | 103 | 92
  Choked when swallowing C6D22 | -1.62 (16.42) | -2.90 (14.54)
  Choked when swallowing C7D1: number analyzed (Participants) | 113 | 98
  Choked when swallowing C7D1 | -2.95 (17.00) | -2.04 (15.00)
  Choked when swallowing C7D22: number analyzed (Participants) | 81 | 73
  Choked when swallowing C7D22 | 0.41 (17.07) | -1.37 (16.14)
  Choked when swallowing C8D1: number analyzed (Participants) | 80 | 81
  Choked when swallowing C8D1 | -0.83 (18.35) | 0.00 (14.91)
  Choked when swallowing C8D22: number analyzed (Participants) | 71 | 65
  Choked when swallowing C8D22 | -1.88 (16.80) | -0.51 (15.01)
  Choked when swallowing C9D1: number analyzed (Participants) | 75 | 62
  Choked when swallowing C9D1 | -2.22 (14.84) | -1.61 (16.45)
  Choked when swallowing C9D22: number analyzed (Participants) | 60 | 55
  Choked when swallowing C9D22 | -0.56 (17.88) | -0.61 (17.56)
  Choked when swallowing C10D1: number analyzed (Participants) | 66 | 56
  Choked when swallowing C10D1 | -0.51 (17.04) | -2.38 (17.82)
  Choked when swallowing C10D22: number analyzed (Participants) | 57 | 43
  Choked when swallowing C10D22 | -1.17 (16.62) | -2.33 (18.40)
  Choked when swallowing C11D1: number analyzed (Participants) | 63 | 46
  Choked when swallowing C11D1 | 0.53 (15.25) | -1.45 (19.82)
  Choked when swallowing C11D22: number analyzed (Participants) | 44 | 31
  Choked when swallowing C11D22 | -1.52 (18.96) | 2.15 (14.75)
  Choked when swallowing C12D1: number analyzed (Participants) | 53 | 41
  Choked when swallowing C12D1 | 0.00 (16.01) | -0.81 (13.92)
  Choked when swallowing C12D22: number analyzed (Participants) | 37 | 25
  Choked when swallowing C12D22 | -1.80 (17.47) | -1.33 (15.15)
  Choked when swallowing C13D1: number analyzed (Participants) | 48 | 35
  Choked when swallowing C13D1 | -0.69 (16.11) | 0.95 (22.12)
  Choked when swallowing C13D22: number analyzed (Participants) | 40 | 21
  Choked when swallowing C13D22 | 0.83 (19.23) | 1.59 (16.59)
  Choked when swallowing C14D1: number analyzed (Participants) | 39 | 30
  Choked when swallowing C14D1 | -2.56 (16.01) | 0.00 (15.16)
  Choked when swallowing C14D22: number analyzed (Participants) | 32 | 19
  Choked when swallowing C14D22 | -6.25 (15.70) | -1.75 (13.49)
  Choked when swallowing C15D1: number analyzed (Participants) | 35 | 27
  Choked when swallowing C15D1 | -0.95 (12.75) | -2.47 (12.83)
  Choked when swallowing C15D22: number analyzed (Participants) | 29 | 17
  Choked when swallowing C15D22 | -4.60 (11.70) | -3.92 (11.07)
  Choked when swallowing C16D1: number analyzed (Participants) | 35 | 22
  Choked when swallowing C16D1 | -1.90 (13.87) | 0.00 (10.29)
  Choked when swallowing C16D22: number analyzed (Participants) | 29 | 14
  Choked when swallowing C16D22 | -2.30 (12.38) | -2.38 (8.91)
  Choked when swallowing C17D1: number analyzed (Participants) | 30 | 18
  Choked when swallowing C17D1 | -2.22 (17.36) | -3.70 (10.78)
  Choked when swallowing C17D22: number analyzed (Participants) | 23 | 0
  Choked when swallowing C17D22 | -1.45 (21.27) |
  Choked when swallowing C18D1: number analyzed (Participants) | 27 | 16
  Choked when swallowing C18D1 | -2.47 (18.32) | 0.00 (12.17)
  Choked when swallowing C18D22: number analyzed (Participants) | 20 | 10
  Choked when swallowing C18D22 | 1.67 (13.13) | 0.00 (22.22)
  Choked when swallowing C19D1: number analyzed (Participants) | 23 | 15
  Choked when swallowing C19D1 | 0.00 (17.41) | -2.22 (15.26)
  Choked when swallowing C19D22: number analyzed (Participants) | 20 | 11
  Choked when swallowing C19D22 | 0.00 (10.81) | -3.03 (17.98)
  Choked when swallowing C20D1: number analyzed (Participants) | 23 | 15
  Choked when swallowing C20D1 | 0.00 (10.05) | -4.44 (11.73)
  Choked when swallowing C20D22: number analyzed (Participants) | 18 | 10
  Choked when swallowing C20D22 | 0.00 (11.43) | -3.33 (18.92)
  Choked when swallowing C21D1: number analyzed (Participants) | 20 | 14
  Choked when swallowing C21D1 | -1.67 (17.01) | -4.76 (12.10)
  Choked when swallowing C21D22: number analyzed (Participants) | 14 | 0
  Choked when swallowing C21D22 | -4.76 (17.82) |
  Choked when swallowing C22D1: number analyzed (Participants) | 15 | 12
  Choked when swallowing C22D1 | -2.22 (15.26) | -2.78 (17.16)
  Choked when swallowing C22D22: number analyzed (Participants) | 10 | 0
  Choked when swallowing C22D22 | -10.00 (22.50) |
  Choked when swallowing C23D1: number analyzed (Participants) | 15 | 13
  Choked when swallowing C23D1 | -4.44 (21.33) | 2.56 (16.45)
  Choked when swallowing C23D22: number analyzed (Participants) | 11 | 0
  Choked when swallowing C23D22 | -9.09 (21.56) |
  Choked when swallowing C24D1: number analyzed (Participants) | 14 | 0
  Choked when swallowing C24D1 | -4.76 (22.10) |
  Choked when swallowing C25D1: number analyzed (Participants) | 12 | 0
  Choked when swallowing C25D1 | -8.33 (20.72) |
  Choked when swallowing C25D22: number analyzed (Participants) | 11 | 0
  Choked when swallowing C25D22 | -6.06 (25.03) |
  Choked when swallowing C26D1: number analyzed (Participants) | 13 | 0
  Choked when swallowing C26D1 | -5.13 (22.96) |
  Choked when swallowing C27D1: number analyzed (Participants) | 11 | 0
  Choked when swallowing C27D1 | 0.00 (14.91) |
  Choked when swallowing C28D1: number analyzed (Participants) | 12 | 0
  Choked when swallowing C28D1 | 0.00 (14.21) |
  Choked when swallowing 30 Day follow up: number analyzed (Participants) | 72 | 90
  Choked when swallowing 30 Day follow up | 1.39 (20.51) | 0.00 (17.31)
  Choked when swallowing 90 Day follow up: number analyzed (Participants) | 86 | 82
  Choked when swallowing 90 Day follow up | 2.71 (19.28) | 1.63 (22.77)
  Trouble with coughing Baseline | 12.06 (19.69) | 16.73 (22.85)
  Trouble with coughing C1D22: number analyzed (Participants) | 176 | 208
  Trouble with coughing C1D22 | 4.17 (23.27) | -3.04 (21.14)
  Trouble with coughing C2D1: number analyzed (Participants) | 206 | 223
  Trouble with coughing C2D1 | 2.75 (23.47) | -4.19 (24.56)
  Trouble with coughing C2D22: number analyzed (Participants) | 150 | 180
  Trouble with coughing C2D22 | 2.22 (20.31) | -3.70 (27.04)
  Trouble with coughing C3D1: number analyzed (Participants) | 190 | 196
  Trouble with coughing C3D1 | 4.74 (26.24) | -5.78 (24.12)
  Trouble with coughing C3D22: number analyzed (Participants) | 152 | 148
  Trouble with coughing C3D22 | 3.29 (24.19) | -4.28 (23.74)
  Trouble with coughing C4D1: number analyzed (Participants) | 169 | 161
  Trouble with coughing C4D1 | 1.97 (23.77) | -7.04 (23.40)
  Trouble with coughing C4D22: number analyzed (Participants) | 122 | 127
  Trouble with coughing C4D22 | 1.37 (18.87) | -4.20 (23.75)
  Trouble with coughing C5D1: number analyzed (Participants) | 148 | 144
  Trouble with coughing C5D1 | 1.80 (20.86) | -5.32 (22.18)
  Trouble with coughing C5D22: number analyzed (Participants) | 110 | 115
  Trouble with coughing C5D22 | 1.21 (20.66) | -3.48 (23.93)
  Trouble with coughing C6D1: number analyzed (Participants) | 122 | 121
  Trouble with coughing C6D1 | -0.82 (22.05) | -3.03 (22.77)
  Trouble with coughing C6D22: number analyzed (Participants) | 103 | 92
  Trouble with coughing C6D22 | -0.65 (19.79) | -5.80 (22.97)
  Trouble with coughing C7D1: number analyzed (Participants) | 113 | 98
  Trouble with coughing C7D1 | 0.29 (20.65) | -4.42 (19.52)
  Trouble with coughing C7D22: number analyzed (Participants) | 81 | 73
  Trouble with coughing C7D22 | -1.65 (18.18) | -7.31 (20.22)
  Trouble with coughing C8D1: number analyzed (Participants) | 80 | 81
  Trouble with coughing C8D1 | 0.83 (21.85) | -3.29 (20.14)
  Trouble with coughing C8D22: number analyzed (Participants) | 71 | 65
  Trouble with coughing C8D22 | 2.35 (18.96) | -5.64 (21.71)
  Trouble with coughing C9D1: number analyzed (Participants) | 75 | 62
  Trouble with coughing C9D1 | -2.22 (17.62) | -1.61 (22.93)
  Trouble with coughing C9D22: number analyzed (Participants) | 60 | 55
  Trouble with coughing C9D22 | 2.22 (22.01) | -1.82 (22.61)
  Trouble with coughing C10D1: number analyzed (Participants) | 66 | 56
  Trouble with coughing C10D1 | -1.01 (18.46) | -4.17 (22.97)
  Trouble with coughing C10D22: number analyzed (Participants) | 57 | 43
  Trouble with coughing C10D22 | 0.58 (17.24) | -3.88 (25.42)
  Trouble with coughing C11D1: number analyzed (Participants) | 63 | 46
  Trouble with coughing C11D1 | 0.00 (17.96) | -1.45 (26.25)
  Trouble with coughing C11D22: number analyzed (Participants) | 44 | 31
  Trouble with coughing C11D22 | -1.52 (16.00) | 0.00 (22.77)
  Trouble with coughing C12D1: number analyzed (Participants) | 53 | 41
  Trouble with coughing C12D1 | -0.63 (16.65) | -4.88 (24.22)
  Trouble with coughing C12D22: number analyzed (Participants) | 37 | 25
  Trouble with coughing C12D22 | 0.90 (12.39) | -6.67 (23.57)
  Trouble with coughing C13D1: number analyzed (Participants) | 48 | 35
  Trouble with coughing C13D1 | 2.08 (17.40) | -8.57 (21.91)
  Trouble with coughing C13D22: number analyzed (Participants) | 40 | 21
  Trouble with coughing C13D22 | 4.17 (15.45) | -4.76 (28.45)
  Trouble with coughing C14D1: number analyzed (Participants) | 39 | 30
  Trouble with coughing C14D1 | 2.56 (16.01) | -2.22 (26.16)
  Trouble with coughing C14D22: number analyzed (Participants) | 32 | 19
  Trouble with coughing C14D22 | -3.12 (13.01) | -7.02 (26.24)
  Trouble with coughing C15D1: number analyzed (Participants) | 35 | 27
  Trouble with coughing C15D1 | 2.86 (23.39) | -1.23 (25.29)
  Trouble with coughing C15D22: number analyzed (Participants) | 29 | 17
  Trouble with coughing C15D22 | 0.00 (15.43) | -7.84 (25.08)
  Trouble with coughing C16D1: number analyzed (Participants) | 35 | 22
  Trouble with coughing C16D1 | 1.90 (16.05) | -9.09 (21.04)
  Trouble with coughing C16D22: number analyzed (Participants) | 29 | 14
  Trouble with coughing C16D22 | 4.60 (19.36) | -9.52 (27.51)
  Trouble with coughing C17D1: number analyzed (Participants) | 30 | 18
  Trouble with coughing C17D1 | 3.33 (16.02) | -3.70 (25.28)
  Trouble with coughing C17D22: number analyzed (Participants) | 23 | 0
  Trouble with coughing C17D22 | -1.45 (15.82) |
  Trouble with coughing C18D1: number analyzed (Participants) | 27 | 16
  Trouble with coughing C18D1 | 0.00 (16.01) | -6.25 (27.81)
  Trouble with coughing C18D22: number analyzed (Participants) | 20 | 10
  Trouble with coughing C18D22 | 1.67 (13.13) | -10.00 (22.50)
  Trouble with coughing C19D1: number analyzed (Participants) | 23 | 15
  Trouble with coughing C19D1 | -1.45 (12.22) | -4.44 (21.33)
  Trouble with coughing C19D22: number analyzed (Participants) | 20 | 11
  Trouble with coughing C19D22 | 3.33 (14.91) | -6.06 (25.03)
  Trouble with coughing C20D1: number analyzed (Participants) | 23 | 15
  Trouble with coughing C20D1 | 0.00 (14.21) | -4.44 (17.21)
  Trouble with coughing C20D22: number analyzed (Participants) | 18 | 10
  Trouble with coughing C20D22 | 1.85 (13.87) | -6.67 (21.08)
  Trouble with coughing C21D1: number analyzed (Participants) | 20 | 14
  Trouble with coughing C21D1 | -3.33 (10.26) | 0.00 (26.15)
  Trouble with coughing C21D22: number analyzed (Participants) | 14 | 0
  Trouble with coughing C21D22 | 2.38 (8.91) |
  Trouble with coughing C22D1: number analyzed (Participants) | 15 | 12
  Trouble with coughing C22D1 | -4.44 (11.73) | -2.78 (26.43)
  Trouble with coughing C22D22: number analyzed (Participants) | 10 | 0
  Trouble with coughing C22D22 | 0.00 (15.71) |
  Trouble with coughing C23D1: number analyzed (Participants) | 15 | 13
  Trouble with coughing C23D1 | -2.22 (15.26) | 0.00 (23.57)
  Trouble with coughing C23D22: number analyzed (Participants) | 11 | 0
  Trouble with coughing C23D22 | -6.06 (13.48) |
  Trouble with coughing C24D1: number analyzed (Participants) | 14 | 0
  Trouble with coughing C24D1 | -4.76 (12.10) |
  Trouble with coughing C25D1: number analyzed (Participants) | 12 | 0
  Trouble with coughing C25D1 | -8.33 (15.08) |
  Trouble with coughing C25D22: number analyzed (Participants) | 11 | 0
  Trouble with coughing C25D22 | -3.03 (10.05) |
  Trouble with coughing C26D1: number analyzed (Participants) | 13 | 0
  Trouble with coughing C26D1 | -7.69 (14.62) |
  Trouble with coughing C27D1: number analyzed (Participants) | 11 | 0
  Trouble with coughing C27D1 | -6.06 (13.48) |
  Trouble with coughing C28D1: number analyzed (Participants) | 12 | 0
  Trouble with coughing C28D1 | -8.33 (15.08) |
  Trouble with coughing 30 day follow up: number analyzed (Participants) | 72 | 90
  Trouble with coughing 30 day follow up | -0.93 (27.96) | -5.93 (26.24)
  Trouble with coughing 90 Day follow up: number analyzed (Participants) | 86 | 82
  Trouble with coughing 90 Day follow up | 2.33 (22.75) | -2.85 (21.72)
  Trouble talking Baseline | 5.45 (14.00) | 5.97 (15.28)
  Trouble talking C1D22: number analyzed (Participants) | 176 | 208
  Trouble talking C1D22 | 3.03 (19.93) | 1.60 (14.56)
  Trouble talking C2D1: number analyzed (Participants) | 206 | 223
  Trouble talking C2D1 | 0.81 (16.28) | -0.75 (15.96)
  Trouble talking C2D22: number analyzed (Participants) | 150 | 180
  Trouble talking C2D22 | 0.89 (16.81) | 0.93 (15.93)
  Trouble talking C3D1: number analyzed (Participants) | 190 | 196
  Trouble talking C3D1 | -0.18 (15.52) | -0.34 (15.09)
  Trouble talking C3D22: number analyzed (Participants) | 152 | 148
  Trouble talking C3D22 | 0.66 (16.93) | 0.23 (15.31)
  Trouble talking C4D1: number analyzed (Participants) | 169 | 161
  Trouble talking C4D1 | 0.59 (16.05) | -0.21 (14.67)
  Trouble talking C4D22: number analyzed (Participants) | 122 | 127
  Trouble talking C4D22 | 2.19 (19.04) | -0.52 (17.81)
  Trouble talking C5D1: number analyzed (Participants) | 148 | 144
  Trouble talking C5D1 | -0.68 (15.29) | 1.16 (17.81)
  Trouble talking C5D22: number analyzed (Participants) | 110 | 115
  Trouble talking C5D22 | 1.21 (16.23) | 1.45 (19.94)
  Trouble talking C6D1: number analyzed (Participants) | 122 | 121
  Trouble talking C6D1 | -0.27 (15.74) | 1.10 (16.63)
  Trouble talking C6D22: number analyzed (Participants) | 103 | 92
  Trouble talking C6D22 | -1.62 (16.42) | 1.09 (16.72)
  Trouble talking C7D1: number analyzed (Participants) | 113 | 98
  Trouble talking C7D1 | -1.47 (17.47) | 0.34 (14.75)
  Trouble talking C7D22: number analyzed (Participants) | 81 | 73
  Trouble talking C7D22 | -1.65 (15.72) | 0.46 (15.21)
  Trouble talking C8D1: number analyzed (Participants) | 80 | 81
  Trouble talking C8D1 | 1.25 (20.16) | 5.35 (17.84)
  Trouble talking C8D22: number analyzed (Participants) | 71 | 65
  Trouble talking C8D22 | -1.41 (15.36) | 3.59 (18.75)
  Trouble talking C9D1: number analyzed (Participants) | 75 | 62
  Trouble talking C9D1 | -2.67 (11.96) | 3.23 (17.81)
  Trouble talking C9D22: number analyzed (Participants) | 60 | 55
  Trouble talking C9D22 | -0.56 (15.64) | 1.82 (13.48)
  Trouble talking C10D1: number analyzed (Participants) | 66 | 56
  Trouble talking C10D1 | -1.01 (13.03) | 2.38 (12.48)
  Trouble talking C10D22: number analyzed (Participants) | 57 | 43
  Trouble talking C10D22 | 0.58 (13.35) | 4.65 (18.66)
  Trouble talking C11D1: number analyzed (Participants) | 63 | 46
  Trouble talking C11D1 | 0.53 (14.03) | 4.35 (19.38)
  Trouble talking C11D22: number analyzed (Participants) | 44 | 31
  Trouble talking C11D22 | -3.03 (14.05) | 4.30 (22.35)
  Trouble talking C12D1: number analyzed (Participants) | 53 | 41
  Trouble talking C12D1 | -0.63 (13.85) | 2.44 (17.30)
  Trouble talking C12D22: number analyzed (Participants) | 37 | 25
  Trouble talking C12D22 | -2.70 (12.12) | 8.00 (24.11)
  Trouble talking C13D1: number analyzed (Participants) | 48 | 35
  Trouble talking C13D1 | -0.69 (14.57) | 4.76 (21.61)
  Trouble talking C13D22: number analyzed (Participants) | 40 | 21
  Trouble talking C13D22 | -0.83 (14.10) | 6.35 (22.65)
  Trouble talking C14D1: number analyzed (Participants) | 39 | 30
  Trouble talking C14D1 | -0.85 (14.28) | 3.33 (13.42)
  Trouble talking C14D22: number analyzed (Participants) | 32 | 19
  Trouble talking C14D22 | -2.08 (11.79) | 1.75 (7.65)
  Trouble talking C15D1: number analyzed (Participants) | 35 | 27
  Trouble talking C15D1 | 0.00 (14.00) | 1.23 (11.25)
  Trouble talking C15D22: number analyzed (Participants) | 29 | 17
  Trouble talking C15D22 | 0.00 (12.60) | -1.96 (8.08)
  Trouble talking C16D1: number analyzed (Participants) | 35 | 22
  Trouble talking C16D1 | -1.90 (13.87) | 1.52 (12.50)
  Trouble talking C16D22: number analyzed (Participants) | 29 | 14
  Trouble talking C16D22 | -3.45 (13.64) | 0.00 (13.07)
  Trouble talking C17D1: number analyzed (Participants) | 30 | 18
  Trouble talking C17D1 | 1.11 (13.79) | 0.00 (11.43)
  Trouble talking C17D22: number analyzed (Participants) | 23 | 0
  Trouble talking C17D22 | -4.35 (15.26) |
  Trouble talking C18D1: number analyzed (Participants) | 27 | 16
  Trouble talking C18D1 | -2.47 (8.90) | 0.00 (12.17)
  Trouble talking C18D22: number analyzed (Participants) | 20 | 10
  Trouble talking C18D22 | 0.00 (10.81) | -3.33 (10.54)
  Trouble talking C19D1: number analyzed (Participants) | 23 | 15
  Trouble talking C19D1 | -1.45 (6.95) | 2.22 (15.26)
  Trouble talking C19D22: number analyzed (Participants) | 20 | 11
  Trouble talking C19D22 | 0.00 (0.00) | -3.03 (10.05)
  Trouble talking C20D1: number analyzed (Participants) | 23 | 15
  Trouble talking C20D1 | 4.35 (23.15) | 0.00 (12.60)
  Trouble Talking C20D22: number analyzed (Participants) | 18 | 10
  Trouble Talking C20D22 | -1.85 (7.86) | 0.00 (0.00)
  Trouble talking C21D1: number analyzed (Participants) | 20 | 14
  Trouble talking C21D1 | -1.67 (7.45) | -2.38 (8.91)
  Trouble talking C21D22: number analyzed (Participants) | 14 | 0
  Trouble talking C21D22 | 0.00 (0.00) |
  Trouble talking C22D1: number analyzed (Participants) | 15 | 12
  Trouble talking C22D1 | -2.22 (15.26) | 0.00 (14.21)
  Trouble talking C22D22: number analyzed (Participants) | 10 | 13
  Trouble talking C22D22 | -3.33 (10.54) | 0.00 (13.61)
  Trouble talking C23D1: number analyzed (Participants) | 15 | 0
  Trouble talking C23D1 | 0.00 (12.60) |
  Trouble talking C23D22: number analyzed (Participants) | 11 | 0
  Trouble talking C23D22 | -3.03 (10.05) |
  Trouble talking C24D1: number analyzed (Participants) | 14 | 0
  Trouble talking C24D1 | -4.76 (12.10) |
  Trouble talking C25D1: number analyzed (Participants) | 12 | 0
  Trouble talking C25D1 | -5.56 (12.97) |
  Trouble talking C25D22: number analyzed (Participants) | 11 | 0
  Trouble talking C25D22 | 3.03 (23.35) |
  Trouble talking C26D1: number analyzed (Participants) | 13 | 0
  Trouble talking C26D1 | -2.56 (9.25) |
  Trouble talking C27D1: number analyzed (Participants) | 11 | 0
  Trouble talking C27D1 | -3.03 (10.05) |
  Trouble talking C28D1: number analyzed (Participants) | 12 | 0
  Trouble talking C28D1 | -2.78 (9.62) |
  Trouble talking 30 day follow up: number analyzed (Participants) | 72 | 90
  Trouble talking 30 day follow up | 1.85 (21.59) | 2.59 (15.98)
  Trouble talking 90 Day follow up: number analyzed (Participants) | 86 | 82
  Trouble talking 90 Day follow up | 1.16 (18.75) | 4.88 (14.93)
  Weight loss Baseline | 29.70 (32.47) | 34.24 (31.38)
  Weight loss C1D22: number analyzed (Participants) | 176 | 208
  Weight loss C1D22 | 0.95 (28.60) | -2.72 (28.34)
  Weight loss C2D1: number analyzed (Participants) | 206 | 223
  Weight loss C2D1 | -0.65 (31.23) | -7.92 (28.33)
  Weight loss C2D22: number analyzed (Participants) | 150 | 180
  Weight loss C2D22 | 0.00 (30.41) | -6.11 (30.41)
  Weight loss C3D1: number analyzed (Participants) | 190 | 196
  Weight loss C3D1 | -2.46 (31.14) | -9.35 (30.34)
  Weight loss C3D22: number analyzed (Participants) | 152 | 148
  Weight loss C3D22 | -1.75 (31.59) | -9.46 (29.62)
  Weight loss C4D1: number analyzed (Participants) | 169 | 161
  Weight loss C4D1 | -5.72 (29.32) | -13.87 (29.71)
  Weight loss C4D22: number analyzed (Participants) | 122 | 127
  Weight loss C4D22 | -2.19 (32.84) | -12.34 (29.04)
  Weight loss C5D1: number analyzed (Participants) | 148 | 144
  Weight loss C5D1 | -3.15 (35.49) | -12.04 (28.32)
  Weight loss C5D22: number analyzed (Participants) | 110 | 115
  Weight loss C5D22 | -5.76 (33.44) | -13.33 (32.08)
  Weight loss C6D1: number analyzed (Participants) | 122 | 121
  Weight loss C6D1 | -6.01 (31.79) | -11.02 (30.24)
  Weight loss C6D22: number analyzed (Participants) | 103 | 92
  Weight loss C6D22 | -9.39 (34.11) | -15.58 (30.64)
  Weight loss C7D1: number analyzed (Participants) | 113 | 98
  Weight loss C7D1 | -11.80 (31.79) | -15.31 (28.38)
  Weight loss C7D22: number analyzed (Participants) | 81 | 73
  Weight loss C7D22 | -8.64 (34.47) | -21.00 (31.18)
  Weight loss C8D1: number analyzed (Participants) | 80 | 81
  Weight loss C8D1 | -10.83 (31.28) | -13.58 (27.27)
  Weight loss C8D22: number analyzed (Participants) | 71 | 65
  Weight loss C8D22 | -11.27 (33.78) | -14.87 (27.66)
  Weight loss C9D1: number analyzed (Participants) | 75 | 62
  Weight loss C9D1 | -15.56 (32.11) | -13.98 (25.28)
  Weight loss C9D22: number analyzed (Participants) | 60 | 55
  Weight loss C9D22 | -9.44 (34.77) | -19.39 (28.47)
  Weight loss C10D1: number analyzed (Participants) | 66 | 56
  Weight loss C10D1 | -10.61 (33.67) | -16.07 (31.78)
  Weight loss C10D22: number analyzed (Participants) | 57 | 43
  Weight loss C10D22 | -11.11 (30.43) | -20.93 (30.88)
  Weight loss C11D1: number analyzed (Participants) | 63 | 46
  Weight loss C11D1 | -12.17 (34.03) | -15.94 (32.00)
  Weight loss C11D22: number analyzed (Participants) | 44 | 31
  Weight loss C11D22 | -17.42 (29.19) | -17.20 (29.65)
  Weight loss C12D1: number analyzed (Participants) | 53 | 41
  Weight loss C12D1 | -10.06 (33.71) | -18.70 (28.91)
  Weight loss C12D22: number analyzed (Participants) | 37 | 25
  Weight loss C12D22 | -11.71 (27.46) | -20.00 (30.43)
  Weight loss C13D1: number analyzed (Participants) | 48 | 35
  Weight loss C13D1 | -10.42 (29.30) | -21.90 (33.28)
  Weight loss C13D22: number analyzed (Participants) | 40 | 21
  Weight loss C13D22 | -10.00 (26.37) | -25.40 (23.34)
  Weight loss C14D1: number analyzed (Participants) | 39 | 30
  Weight loss C14D1 | -11.97 (25.92) | -21.11 (29.66)
  Weight loss C14D22: number analyzed (Participants) | 32 | 19
  Weight loss C14D22 | -8.33 (28.08) | -26.32 (30.59)
  Weight loss C15D1: number analyzed (Participants) | 35 | 27
  Weight loss C15D1 | -6.67 (26.57) | -23.46 (34.36)
  Weight loss C15D22: number analyzed (Participants) | 29 | 17
  Weight loss C15D22 | -8.05 (26.21) | -23.53 (38.67)
  Weight loss C16D1: number analyzed (Participants) | 35 | 22
  Weight loss C16D1 | -13.33 (23.15) | -18.18 (38.11)
  Weight loss C16D22: number analyzed (Participants) | 29 | 14
  Weight loss C16D22 | -8.05 (30.41) | -23.81 (27.51)
  Weight loss C17D1: number analyzed (Participants) | 30 | 18
  Weight loss C17D1 | -10.00 (26.48) | -20.37 (30.55)
  Weight loss C17D22: number analyzed (Participants) | 23 | 0
  Weight loss C17D22 | -8.70 (25.06) |
  Weight loss C18D1: number analyzed (Participants) | 27 | 16
  Weight loss C18D1 | -14.81 (23.27) | -16.67 (32.20)
  Weight loss C18D22: number analyzed (Participants) | 20 | 10
  Weight loss C18D22 | -15.00 (25.31) | -30.00 (29.19)
  Weight loss C19D1: number analyzed (Participants) | 23 | 15
  Weight loss C19D1 | -17.39 (22.18) | -17.78 (33.01)
  Weight loss C19D22: number analyzed (Participants) | 20 | 11
  Weight loss C19D22 | -11.67 (29.17) | -27.27 (32.72)
  Weight loss C20D1: number analyzed (Participants) | 23 | 15
  Weight loss C20D1 | -15.94 (24.35) | -17.78 (27.79)
  Weight loss C20D22: number analyzed (Participants) | 18 | 10
  Weight loss C20D22 | -14.81 (26.13) | -30.00 (33.15)
  Weight loss C21D1: number analyzed (Participants) | 20 | 14
  Weight loss C21D1 | -16.67 (25.36) | -23.81 (30.46)
  Weight loss C21D22: number analyzed (Participants) | 14 | 0
  Weight loss C21D22 | -16.67 (28.50) |
  Weight loss C22D1: number analyzed (Participants) | 15 | 12
  Weight loss C22D1 | -15.56 (27.79) | -16.67 (36.24)
  Weight loss C22D22: number analyzed (Participants) | 10 | 0
  Weight loss C22D22 | -20.00 (28.11) |
  Weight loss C23D1: number analyzed (Participants) | 15 | 13
  Weight loss C23D1 | -15.56 (24.77) | -15.38 (37.55)
  Weight loss C23D22: number analyzed (Participants) | 11 | 0
  Weight loss C23D22 | -9.09 (30.15) |
  Weight loss C24D1: number analyzed (Participants) | 14 | 0
  Weight loss C24D1 | -16.67 (28.50) |
  Weight loss C25D1: number analyzed (Participants) | 12 | 0
  Weight loss C25D1 | -11.11 (25.95) |
  Weight loss C25D22: number analyzed (Participants) | 11 | 0
  Weight loss C25D22 | -12.12 (22.47) |
  Weight loss C26D1: number analyzed (Participants) | 13 | 0
  Weight loss C26D1 | -17.95 (22.01) |
  Weight loss C27D1: number analyzed (Participants) | 11 | 0
  Weight loss C27D1 | -24.24 (15.57) |
  Weight loss C28D1: number analyzed (Participants) | 12 | 0
  Weight loss C28D1 | -16.67 (22.47) |
  Weight loss 30 day follow up: number analyzed (Participants) | 72 | 90
  Weight loss 30 day follow up | 3.24 (34.10) | -9.63 (33.98)
  Weight Loss 90 Day follow up: number analyzed (Participants) | 86 | 82
  Weight Loss 90 Day follow up | -2.71 (37.99) | -6.91 (37.31)
  Hair loss Baseline: number analyzed (Participants) | 64 | 66
  Hair loss Baseline | 15.62 (26.54) | 14.14 (29.27)
  Hair loss C1D22: number analyzed (Participants) | 24 | 41
  Hair loss C1D22 | 11.11 (25.38) | 4.07 (29.05)
  Hair loss C2D1: number analyzed (Participants) | 38 | 43
  Hair loss C2D1 | 0.88 (27.39) | 3.10 (28.00)
  Hair loss C2D22: number analyzed (Participants) | 33 | 29
  Hair loss C2D22 | 4.04 (32.01) | 3.45 (24.14)
  Hair loss C3D1: number analyzed (Participants) | 34 | 37
  Hair loss C3D1 | 8.82 (26.35) | 2.70 (30.81)
  Hair loss C3D22: number analyzed (Participants) | 29 | 28
  Hair loss C3D22 | 10.34 (25.36) | 0.00 (27.22)
  Hair loss C4D1: number analyzed (Participants) | 31 | 30
  Hair loss C4D1 | 9.68 (23.08) | 7.78 (34.67)
  Hair loss C4D22: number analyzed (Participants) | 26 | 23
  Hair loss C4D22 | 11.54 (22.98) | 11.59 (21.58)
  Hair loss C5D1: number analyzed (Participants) | 27 | 25
  Hair loss C5D1 | 6.17 (24.52) | 10.67 (26.74)
  Hair loss C5D22: number analyzed (Participants) | 19 | 17
  Hair loss C5D22 | 10.53 (27.34) | 0.00 (37.27)
  Hair loss C6D1: number analyzed (Participants) | 23 | 21
  Hair loss C6D1 | 8.70 (25.06) | 9.52 (28.17)
  Hair loss C6D22: number analyzed (Participants) | 16 | 14
  Hair loss C6D22 | 4.17 (23.96) | 4.76 (38.91)
  Hair loss C7D1: number analyzed (Participants) | 15 | 17
  Hair loss C7D1 | 2.22 (23.46) | 7.84 (30.11)
  Hair loss C7D22: number analyzed (Participants) | 17 | 12
  Hair loss C7D22 | 1.96 (18.52) | 5.56 (37.15)
  Hair loss C8D1: number analyzed (Participants) | 18 | 15
  Hair loss C8D1 | 5.56 (17.15) | 0.00 (30.86)
  Hair loss C8D22: number analyzed (Participants) | 11 | 12
  Hair loss C8D22 | 9.09 (15.57) | 2.78 (26.43)
  Hair loss C9D1: number analyzed (Participants) | 11 | 11
  Hair loss C9D1 | 0.00 (14.91) | 0.00 (36.51)
  Hair loss C9D22: number analyzed (Participants) | 10 | 9
  Hair loss C9D22 | 13.33 (17.21) | 0.00 (40.82)
  Hair loss C10D1: number analyzed (Participants) | 9 | 10
  Hair loss C10D1 | 11.11 (28.87) | 6.67 (40.98)
  Hair loss C10D22: number analyzed (Participants) | 8 | 7
  Hair loss C10D22 | 12.50 (17.25) | -9.52 (53.45)
  Hair loss C11D1: number analyzed (Participants) | 11 | 8
  Hair loss C11D1 | 15.15 (17.41) | 0.00 (43.64)
  Hair loss C11D22: number analyzed (Participants) | 8 | 7
  Hair loss C11D22 | 12.50 (17.25) | 4.76 (23.00)
  Hair loss C12D1: number analyzed (Participants) | 10 | 6
  Hair loss C12D1 | 13.33 (23.31) | -5.56 (49.07)
  Hair loss C12D22: number analyzed (Participants) | 8 | 6
  Hair loss C12D22 | 12.50 (35.36) | -16.67 (40.82)
  Hair loss C13D1: number analyzed (Participants) | 9 | 0
  Hair loss C13D1 | 7.41 (14.70) |
  Hair loss C13D22: number analyzed (Participants) | 5 | 7
  Hair loss C13D22 | 13.33 (18.26) | 4.76 (29.99)
  Hair loss C14D1: number analyzed (Participants) | 7 | 5
  Hair loss C14D1 | 9.52 (16.27) | 6.67 (27.89)
  Hair loss C14D22: number analyzed (Participants) | 5 | 0
  Hair loss C14D22 | 33.33 (40.82) |
  Hair loss C15D1: number analyzed (Participants) | 7 | 0
  Hair loss C15D1 | 23.81 (37.09) |
  Hair loss C15D22: number analyzed (Participants) | 4 | 0
  Hair loss C15D22 | 16.67 (19.25) |
  Hair loss C16D1: number analyzed (Participants) | 5 | 0
  Hair loss C16D1 | 13.33 (18.26) |
  Hair loss C16D22: number analyzed (Participants) | 4 | 0
  Hair loss C16D22 | 16.67 (19.25) |
  Hair loss C17D1: number analyzed (Participants) | 4 | 0
  Hair loss C17D1 | 8.33 (31.91) |
  Hair loss C17D22: number analyzed (Participants) | 4 | 0
  Hair loss C17D22 | 0.00 (27.22) |
  Hair loss C18D1: number analyzed (Participants) | 4 | 0
  Hair loss C18D1 | 0.00 (27.22) |
  Hair loss C18D22: number analyzed (Participants) | 0 | 0
  Hair loss C19D1: number analyzed (Participants) | 0 | 0
  Hair loss C19D22: number analyzed (Participants) | 4 | 0
  Hair loss C19D22 | 41.67 (31.91) |
  Hair loss 30 day follow up: number analyzed (Participants) | 6 | 11
  Hair loss 30 day follow up | -11.11 (45.54) | 18.18 (22.92)
  Hair loss 90 day follow up: number analyzed (Participants) | 14 | 14
  Hair loss 90 day follow up | 21.43 (33.61) | 16.67 (25.32)

12. Secondary Outcome: Change From Baseline in HRQoL Measured by Global Pain (GP)
Description: The GP instrument is a single assessment of overall pain. Participants were assessed in global pain according to the following response categories: 1= no pain (anymore), 2 = less pain, 3 = no change and 4 = more pain.
Time Frame: Baseline, C1D22, D1 and D22 of C2 through C25, C26D1, C27D1,C28D1 30 day follow up, 90 day follow up
Population: FAS with available data was analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | mFOLFOX6 + Zolbetuximab | mFOLFOX6+ Placebo
Number analyzed (Participants) | 257 | 257
units on a scale
  Baseline | 2.87 (2.67) | 2.96 (2.74)
  C1D22: number analyzed (Participants) | 175 | 208
  C1D22 | -0.55 (2.85) | -0.74 (2.32)
  C2D1: number analyzed (Participants) | 205 | 223
  C2D1 | -0.75 (2.94) | -0.75 (2.98)
  C2D22: number analyzed (Participants) | 150 | 178
  C2D22 | -0.67 (3.11) | -1.01 (2.70)
  C3D1: number analyzed (Participants) | 189 | 195
  C3D1 | -0.87 (2.88) | -0.90 (2.70)
  C3D22: number analyzed (Participants) | 151 | 148
  C3D22 | -0.62 (3.16) | -0.83 (2.60)
  C4D1: number analyzed (Participants) | 169 | 161
  C4D1 | -0.86 (2.61) | -0.66 (2.81)
  C4D22: number analyzed (Participants) | 122 | 126
  C4D22 | -0.51 (3.02) | -0.78 (2.55)
  C5D1: number analyzed (Participants) | 148 | 144
  C5D1 | -0.53 (2.91) | -0.81 (2.91)
  C5D22: number analyzed (Participants) | 110 | 115
  C5D22 | -0.54 (2.89) | -0.84 (3.00)
  C6D1: number analyzed (Participants) | 122 | 120
  C6D1 | -0.63 (3.13) | -0.32 (3.33)
  C6D22: number analyzed (Participants) | 103 | 92
  C6D22 | -0.68 (2.91) | -0.98 (2.52)
  C7D1: number analyzed (Participants) | 113 | 96
  C7D1 | -0.46 (2.87) | -0.86 (2.88)
  C7D22: number analyzed (Participants) | 81 | 73
  C7D22 | -0.31 (3.00) | -1.01 (2.60)
  C8D1: number analyzed (Participants) | 80 | 81
  C8D1 | -0.69 (2.54) | -0.67 (3.17)
  C8D22: number analyzed (Participants) | 71 | 65
  C8D22 | -0.79 (3.28) | -1.09 (2.30)
  C9D1: number analyzed (Participants) | 75 | 62
  C9D1 | -0.71 (3.05) | -1.18 (2.04)
  C9D22: number analyzed (Participants) | 60 | 55
  C9D22 | -1.02 (2.76) | -1.13 (2.71)
  C10D1: number analyzed (Participants) | 65 | 56
  C10D1 | -0.54 (2.84) | -0.75 (2.91)
  C10D22: number analyzed (Participants) | 56 | 43
  C10D22 | -0.50 (3.12) | -0.74 (3.09)
  C11D1: number analyzed (Participants) | 63 | 46
  C11D1 | -0.38 (3.58) | -0.96 (2.16)
  C11D22: number analyzed (Participants) | 44 | 31
  C11D22 | -0.59 (3.27) | -0.77 (1.89)
  C12D1: number analyzed (Participants) | 53 | 41
  C12D1 | -0.30 (3.42) | -0.54 (2.81)
  C12D22: number analyzed (Participants) | 36 | 24
  C12D22 | -0.14 (2.82) | -0.88 (2.17)
  C13D1: number analyzed (Participants) | 47 | 35
  C13D1 | -0.79 (3.51) | -0.66 (2.52)
  C13D22: number analyzed (Participants) | 40 | 21
  C13D22 | -0.63 (3.01) | -1.19 (3.23)
  C14D1: number analyzed (Participants) | 39 | 30
  C14D1 | -0.21 (2.91) | -0.37 (2.46)
  C14D22: number analyzed (Participants) | 32 | 19
  C14D22 | -0.44 (3.70) | -0.84 (3.34)
  C15D1: number analyzed (Participants) | 35 | 27
  C15D1 | 0.09 (3.49) | 0.22 (3.63)
  C15D22: number analyzed (Participants) | 29 | 17
  C15D22 | -0.38 (3.81) | -0.71 (3.62)
  C16D1: number analyzed (Participants) | 35 | 22
  C16D1 | -0.60 (3.91) | -0.45 (3.66)
  C16D22: number analyzed (Participants) | 29 | 14
  C16D22 | -0.97 (3.23) | -0.71 (2.46)
  C17D1: number analyzed (Participants) | 30 | 17
  C17D1 | -0.03 (2.94) | -0.53 (2.62)
  C17D22: number analyzed (Participants) | 23 | 0
  C17D22 | 0.22 (3.00) |
  C18D1: number analyzed (Participants) | 26 | 16
  C18D1 | -0.62 (3.11) | -0.31 (2.91)
  C18D22: number analyzed (Participants) | 21 | 10
  C18D22 | -1.14 (2.87) | -0.40 (2.32)
  C19D1: number analyzed (Participants) | 23 | 15
  C19D1 | -1.04 (3.24) | -0.73 (2.22)
  C19D22: number analyzed (Participants) | 20 | 11
  C19D22 | -0.50 (2.33) | -0.45 (2.34)
  C20D1: number analyzed (Participants) | 23 | 15
  C20D1 | -0.43 (3.26) | 0.60 (3.07)
  C20D22: number analyzed (Participants) | 18 | 10
  C20D22 | -0.17 (3.70) | -0.20 (2.74)
  C21D1: number analyzed (Participants) | 20 | 14
  C21D1 | -0.50 (3.66) | -0.79 (2.36)
  C21D22: number analyzed (Participants) | 14 | 0
  C21D22 | 0.57 (2.90) |
  C22D1: number analyzed (Participants) | 15 | 12
  C22D1 | 0.07 (3.47) | -0.42 (2.78)
  C22D22: number analyzed (Participants) | 10 | 0
  C22D22 | 0.60 (3.24) |
  C23D1: number analyzed (Participants) | 15 | 13
  C23D1 | 1.07 (4.13) | -0.54 (2.63)
  C23D22: number analyzed (Participants) | 11 | 0
  C23D22 | 1.27 (4.13) |
  C24D1: number analyzed (Participants) | 14 | 0
  C24D1 | 1.43 (4.54) |
  C24D22: number analyzed (Participants) | 0 | 0
  C25D1: number analyzed (Participants) | 12 | 0
  C25D1 | 2.33 (3.03) |
  C25D22: number analyzed (Participants) | 11 | 0
  C25D22 | 1.45 (3.30) |
  C26D1: number analyzed (Participants) | 13 | 0
  C26D1 | 1.08 (3.77) |
  C27D1: number analyzed (Participants) | 11 | 0
  C27D1 | 1.55 (3.75) |
  C28D1: number analyzed (Participants) | 12 | 0
  C28D1 | 1.42 (3.55) |
  30 day follow up: number analyzed (Participants) | 72 | 90
  30 day follow up | -0.19 (2.99) | 0.39 (3.16)
  90 Day follow up: number analyzed (Participants) | 84 | 81
  90 Day follow up | -0.27 (2.94) | 0.31 (3.12)

13. Secondary Outcome: Change From Baseline in HRQoL Measured by the EuroQOL Five Dimensions Questionnaire 5L (EQ-5D-5L) Questionnaire
Description: EQ-5D-5L is a standardized instrument for use as a measure of health outcomes consisting of 6 items that cover 5 main domains (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and a general visual analog scale for health status.It was developed by the EuroQol Group for use as a generic, preference-based measure of health outcomes. Each dimension comprises 5 levels (no problems, slight problems, moderate problems, severe problems, extreme problems). A unique EQ-5D-5L health state is defined by combining 1 level from each of the 5 dimensions. This questionnaire also records the respondent's self-rated health status on a vertical graduated (0 = the worst health a participant can imagine to 100 = the best health a participant can imagine) visual analogue scale. Responses to the 5 items will also be converted to a weighted health state index (utility score) based on values derived from general population samples.
Time Frame: Baseline, C1D22, D1 and D22 of C2 through C25, C26D1, C27D1,C28D1 30 day follow up, 90 day follow up
Population: FAS with available data was analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | mFOLFOX6 + Zolbetuximab | mFOLFOX6+ Placebo
Number analyzed (Participants) | 258 | 258
units on a scale
  Mobility Baseline | 1.40 (0.73) | 1.40 (0.74)
  Mobility C1D22: number analyzed (Participants) | 178 | 212
  Mobility C1D22 | 0.15 (0.67) | -0.01 (0.68)
  Mobility C2D1: number analyzed (Participants) | 207 | 226
  Mobility C2D1 | 0.09 (0.76) | -0.05 (0.77)
  Mobility C2D22: number analyzed (Participants) | 152 | 181
  Mobility C2D22 | 0.03 (0.76) | -0.05 (0.64)
  Mobility C3D1: number analyzed (Participants) | 190 | 198
  Mobility C3D1 | 0.09 (0.85) | -0.02 (0.82)
  Mobility C3D22: number analyzed (Participants) | 154 | 149
  Mobility C3D22 | 0.21 (0.88) | -0.04 (0.70)
  Mobility C4D1: number analyzed (Participants) | 172 | 164
  Mobility C4D1 | 0.16 (0.94) | 0.01 (0.76)
  Mobility C4D22: number analyzed (Participants) | 125 | 128
  Mobility C4D22 | 0.16 (0.90) | 0.13 (0.82)
  Mobility C5D1: number analyzed (Participants) | 150 | 146
  Mobility C5D1 | 0.15 (0.89) | 0.18 (0.80)
  Mobility C5D22: number analyzed (Participants) | 114 | 116
  Mobility C5D22 | 0.27 (0.96) | 0.16 (0.81)
  Mobility C6D1: number analyzed (Participants) | 123 | 122
  Mobility C6D1 | 0.20 (0.82) | 0.20 (0.72)
  Mobility C6D22: number analyzed (Participants) | 103 | 95
  Mobility C6D22 | 0.17 (0.90) | 0.23 (0.69)
  Mobility C7D1: number analyzed (Participants) | 114 | 98
  Mobility C7D1 | 0.17 (0.90) | 0.10 (0.63)
  Mobility C7D22: number analyzed (Participants) | 81 | 74
  Mobility C7D22 | 0.26 (0.91) | 0.24 (0.72)
  Mobility C8D1: number analyzed (Participants) | 82 | 83
  Mobility C8D1 | 0.17 (0.78) | 0.20 (0.68)
  Mobility C8D22: number analyzed (Participants) | 72 | 65
  Mobility C8D22 | 0.10 (0.61) | 0.12 (0.67)
  Mobility C9D1: number analyzed (Participants) | 75 | 62
  Mobility C9D1 | 0.13 (0.78) | 0.10 (0.65)
  Mobility C9D22: number analyzed (Participants) | 61 | 55
  Mobility C9D22 | 0.11 (0.82) | 0.09 (0.62)
  Mobility C10D1: number analyzed (Participants) | 66 | 56
  Mobility C10D1 | 0.12 (0.85) | 0.11 (0.87)
  Mobility C10D22: number analyzed (Participants) | 57 | 43
  Mobility C10D22 | 0.00 (0.73) | 0.09 (0.75)
  Mobility C11D1: number analyzed (Participants) | 63 | 46
  Mobility C11D1 | 0.16 (0.88) | 0.17 (0.74)
  Mobility C11D22: number analyzed (Participants) | 45 | 31
  Mobility C11D22 | 0.11 (0.83) | 0.23 (0.56)
  Mobility C12D1: number analyzed (Participants) | 53 | 41
  Mobility C12D1 | 0.08 (0.76) | 0.32 (0.72)
  Mobility C12D22: number analyzed (Participants) | 38 | 26
  Mobility C12D22 | 0.21 (0.81) | 0.31 (0.74)
  Mobility C13D1: number analyzed (Participants) | 48 | 35
  Mobility C13D1 | 0.02 (0.73) | 0.20 (0.68)
  Mobility C13D22: number analyzed (Participants) | 41 | 21
  Mobility C13D22 | 0.20 (0.68) | 0.24 (0.77)
  Mobility C14D1: number analyzed (Participants) | 39 | 30
  Mobility C14D1 | 0.05 (0.72) | 0.23 (0.73)
  Mobility C14D22: number analyzed (Participants) | 32 | 19
  Mobility C14D22 | 0.16 (0.81) | 0.16 (0.69)
  Mobility C15D1: number analyzed (Participants) | 35 | 27
  Mobility C15D1 | 0.23 (0.84) | 0.15 (0.66)
  Mobility C15D22: number analyzed (Participants) | 30 | 17
  Mobility C15D22 | 0.30 (0.75) | 0.06 (0.56)
  Mobility C16D1: number analyzed (Participants) | 35 | 22
  Mobility C16D1 | 0.20 (0.83) | 0.14 (0.64)
  Mobility C16D22: number analyzed (Participants) | 29 | 14
  Mobility C16D22 | 0.03 (0.68) | 0.29 (0.73)
  Mobility C17D1: number analyzed (Participants) | 30 | 18
  Mobility C17D1 | 0.23 (0.86) | 0.17 (0.51)
  Mobility C17D22: number analyzed (Participants) | 23 | 0
  Mobility C17D22 | 0.17 (0.83) |
  Mobility C18D1: number analyzed (Participants) | 27 | 16
  Mobility C18D1 | 0.15 (1.10) | 0.19 (0.40)
  Mobility C18D22: number analyzed (Participants) | 21 | 10
  Mobility C18D22 | 0.05 (0.67) | 0.20 (0.42)
  Mobility C19D1: number analyzed (Participants) | 23 | 15
  Mobility C19D1 | 0.09 (0.51) | 0.27 (0.46)
  Mobility C19D22: number analyzed (Participants) | 20 | 11
  Mobility C19D22 | 0.20 (0.52) | 0.27 (0.47)
  Mobility C20D1: number analyzed (Participants) | 23 | 15
  Mobility C20D1 | 0.13 (0.63) | 0.13 (0.52)
  Mobility C20D22: number analyzed (Participants) | 18 | 10
  Mobility C20D22 | 0.17 (0.71) | 0.10 (0.32)
  Mobility C21D1: number analyzed (Participants) | 20 | 14
  Mobility C21D1 | 0.15 (0.49) | 0.07 (0.27)
  Mobility C21D22: number analyzed (Participants) | 14 | 0
  Mobility C21D22 | 0.14 (0.53) |
  Mobility C22D1: number analyzed (Participants) | 15 | 12
  Mobility C22D1 | 0.20 (0.77) | 0.00 (0.43)
  Mobility C22D22: number analyzed (Participants) | 11 | 0
  Mobility C22D22 | 0.55 (0.82) |
  Mobility C23D1: number analyzed (Participants) | 16 | 13
  Mobility C23D1 | 0.31 (0.70) | 0.00 (0.41)
  Mobility C23D22: number analyzed (Participants) | 11 | 0
  Mobility C23D22 | 0.09 (0.54) |
  Mobility C24D1: number analyzed (Participants) | 14 | 0
  Mobility C24D1 | 0.14 (0.36) |
  Mobility C25D1: number analyzed (Participants) | 12 | 0
  Mobility C25D1 | 0.25 (0.62) |
  Mobility C25D22: number analyzed (Participants) | 11 | 0
  Mobility C25D22 | 0.27 (0.47) |
  Mobility C26D1: number analyzed (Participants) | 13 | 0
  Mobility C26D1 | 0.23 (0.44) |
  Mobility C27D1: number analyzed (Participants) | 11 | 0
  Mobility C27D1 | 0.00 (0.00) |
  Mobility C28D1: number analyzed (Participants) | 12 | 0
  Mobility C28D1 | 0.17 (0.39) |
  Mobility 30 Day follow up: number analyzed (Participants) | 72 | 92
  Mobility 30 Day follow up | 0.38 (1.11) | 0.47 (0.99)
  Mobility 90 Day follow up: number analyzed (Participants) | 86 | 83
  Mobility 90 Day follow up | 0.51 (1.09) | 0.53 (0.99)
  Self-care Baseline | 1.23 (0.57) | 1.21 (0.56)
  Self-care C1DD22: number analyzed (Participants) | 178 | 212
  Self-care C1DD22 | 0.11 (0.66) | 0.07 (0.49)
  Self-care C2D1: number analyzed (Participants) | 207 | 226
  Self-care C2D1 | 0.08 (0.65) | -0.04 (0.52)
  Self-care C2D22: number analyzed (Participants) | 152 | 181
  Self-care C2D22 | 0.09 (0.77) | -0.01 (0.56)
  Self-care C3D1: number analyzed (Participants) | 190 | 198
  Self-care C3D1 | 0.06 (0.69) | 0.06 (0.61)
  Self-care C3D22: number analyzed (Participants) | 154 | 149
  Self-care C3D22 | 0.06 (0.72) | -0.01 (0.43)
  Self-care C4D1: number analyzed (Participants) | 172 | 164
  Self-care C4D1 | 0.08 (0.81) | 0.03 (0.54)
  Self-care C4D22: number analyzed (Participants) | 125 | 128
  Self-care C4D22 | 0.05 (0.72) | 0.03 (0.49)
  Self-care C5D1: number analyzed (Participants) | 150 | 146
  Self-care C5D1 | 0.10 (0.86) | 0.05 (0.50)
  Self-care C5D22: number analyzed (Participants) | 114 | 116
  Self-care C5D22 | 0.16 (0.82) | 0.09 (0.57)
  Self-care C6D1: number analyzed (Participants) | 123 | 122
  Self-care C6D1 | 0.07 (0.66) | 0.10 (0.54)
  Self-care C6D22: number analyzed (Participants) | 103 | 95
  Self-care C6D22 | 0.07 (0.74) | 0.05 (0.55)
  Self-care C7D1: number analyzed (Participants) | 114 | 98
  Self-care C7D1 | 0.11 (0.75) | 0.11 (0.49)
  Self-care C7D22: number analyzed (Participants) | 81 | 74
  Self-care C7D22 | 0.01 (0.78) | 0.04 (0.48)
  Self-care C8D1: number analyzed (Participants) | 82 | 83
  Self-care C8D1 | 0.09 (0.95) | 0.10 (0.55)
  Self-care C8D22: number analyzed (Participants) | 72 | 65
  Self-care C8D22 | -0.01 (0.64) | 0.08 (0.62)
  Self-care C9D1: number analyzed (Participants) | 75 | 62
  Self-care C9D1 | 0.08 (0.87) | 0.02 (0.46)
  Self-care C9D22: number analyzed (Participants) | 61 | 55
  Self-care C9D22 | -0.02 (0.81) | 0.04 (0.61)
  Self-care C10D1: number analyzed (Participants) | 66 | 56
  Self-care C10D1 | -0.03 (0.80) | 0.11 (0.65)
  Self-care C10D22: number analyzed (Participants) | 57 | 43
  Self-care C10D22 | -0.04 (0.80) | 0.09 (0.48)
  Self-care C11D1: number analyzed (Participants) | 63 | 46
  Self-care C11D1 | 0.00 (0.93) | 0.11 (0.43)
  Self-care C11D22: number analyzed (Participants) | 45 | 31
  Self-care C11D22 | -0.04 (0.64) | 0.10 (0.30)
  Self-care C12D1: number analyzed (Participants) | 53 | 41
  Self-care C12D1 | -0.04 (0.76) | 0.20 (0.40)
  Self-care C12D22: number analyzed (Participants) | 38 | 26
  Self-care C12D22 | -0.05 (0.73) | 0.15 (0.37)
  Self-care C13DD1: number analyzed (Participants) | 48 | 35
  Self-care C13DD1 | -0.06 (0.76) | 0.14 (0.43)
  Self-care C13D22: number analyzed (Participants) | 41 | 21
  Self-care C13D22 | -0.02 (0.85) | 0.14 (0.36)
  Self-care C14D1: number analyzed (Participants) | 39 | 30
  Self-care C14D1 | -0.08 (0.74) | 0.10 (0.31)
  Self-care C14D22: number analyzed (Participants) | 32 | 19
  Self-care C14D22 | 0.03 (0.86) | 0.16 (0.37)
  Self-care C15D1: number analyzed (Participants) | 35 | 27
  Self-care C15D1 | -0.03 (0.79) | 0.19 (0.40)
  Self-care C15D22: number analyzed (Participants) | 30 | 17
  Self-care C15D22 | -0.03 (0.85) | 0.12 (0.33)
  Self-care C16D1: number analyzed (Participants) | 35 | 22
  Self-care C16D1 | 0.00 (0.84) | 0.09 (0.29)
  Self-care C16D22: number analyzed (Participants) | 29 | 14
  Self-care C16D22 | -0.10 (0.82) | 0.07 (0.27)
  Self-care C17D1: number analyzed (Participants) | 30 | 18
  Self-care C17D1 | 0.03 (1.00) | 0.00 (0.00)
  Self-care C17D22: number analyzed (Participants) | 23 | 0
  Self-care C17D22 | 0.13 (0.92) |
  Self-care C18D1: number analyzed (Participants) | 27 | 16
  Self-care C18D1 | 0.00 (0.92) | 0.06 (0.25)
  Self-care C18D22: number analyzed (Participants) | 21 | 10
  Self-care C18D22 | -0.10 (0.94) | 0.10 (0.32)
  Self-care C19D1: number analyzed (Participants) | 23 | 15
  Self-care C19D1 | 0.04 (0.77) | 0.20 (0.41)
  Self-care C19D22: number analyzed (Participants) | 20 | 11
  Self-care C19D22 | 0.20 (1.06) | 0.09 (0.30)
  Self-care C20D1: number analyzed (Participants) | 23 | 15
  Self-care C20D1 | 0.09 (0.85) | 0.13 (0.35)
  Self-care C20D22: number analyzed (Participants) | 18 | 10
  Self-care C20D22 | 0.06 (0.80) | 0.00 (0.00)
  Self-care C21D1: number analyzed (Participants) | 20 | 14
  Self-care C21D1 | 0.10 (0.64) | 0.14 (0.36)
  Self-care C21D22: number analyzed (Participants) | 14 | 0
  Self-care C21D22 | 0.29 (0.73) |
  Self-care C22D1: number analyzed (Participants) | 15 | 12
  Self-care C22D1 | 0.20 (0.77) | 0.00 (0.00)
  Self-care C22D22: number analyzed (Participants) | 11 | 0
  Self-care C22D22 | 0.18 (0.60) |
  Self-care C23D1: number analyzed (Participants) | 16 | 13
  Self-care C23D1 | 0.31 (0.87) | 0.08 (0.28)
  Self-care C23D22: number analyzed (Participants) | 11 | 0
  Self-care C23D22 | 0.27 (0.79) |
  Self-care C24D1: number analyzed (Participants) | 14 | 0
  Self-care C24D1 | 0.21 (0.89) |
  Self-care C25D1: number analyzed (Participants) | 12 | 0
  Self-care C25D1 | 0.00 (0.43) |
  Self-care C25D22: number analyzed (Participants) | 11 | 0
  Self-care C25D22 | 0.09 (0.54) |
  Self-care C26D1: number analyzed (Participants) | 13 | 0
  Self-care C26D1 | -0.08 (0.49) |
  Self-care C27D1: number analyzed (Participants) | 11 | 0
  Self-care C27D1 | -0.18 (0.40) |
  Self-care C28D1: number analyzed (Participants) | 12 | 0
  Self-care C28D1 | -0.08 (0.51) |
  Self-Care 30 Day follow up: number analyzed (Participants) | 72 | 92
  Self-Care 30 Day follow up | 0.21 (0.90) | 0.30 (0.72)
  Self-care 90 Day follow up: number analyzed (Participants) | 86 | 83
  Self-care 90 Day follow up | 0.35 (0.90) | 0.39 (0.78)
  Usual Activities Baseline | 1.68 (0.97) | 1.56 (0.88)
  Usual Activities C1D22: number analyzed (Participants) | 178 | 212
  Usual Activities C1D22 | 0.24 (0.80) | 0.14 (0.89)
  Usual Activities C2D1: number analyzed (Participants) | 207 | 226
  Usual Activities C2D1 | 0.08 (0.87) | -0.01 (0.82)
  Usual Activities C2D22: number analyzed (Participants) | 152 | 181
  Usual Activities C2D22 | 0.05 (0.86) | -0.01 (0.77)
  Usual Activities C3D1: number analyzed (Participants) | 190 | 198
  Usual Activities C3D1 | 0.05 (0.91) | 0.01 (0.82)
  Usual Activities C3D22: number analyzed (Participants) | 154 | 149
  Usual Activities C3D22 | 0.23 (0.90) | 0.05 (0.89)
  Usual Activities C4D1: number analyzed (Participants) | 172 | 164
  Usual Activities C4D1 | 0.06 (0.92) | 0.04 (0.83)
  Usual Activities C4D22: number analyzed (Participants) | 125 | 128
  Usual Activities C4D22 | 0.11 (0.85) | 0.16 (0.80)
  Usual Activities C5D1: number analyzed (Participants) | 150 | 146
  Usual Activities C5D1 | 0.13 (0.93) | 0.15 (0.80)
  Usual Activities C5D22: number analyzed (Participants) | 114 | 116
  Usual Activities C5D22 | 0.17 (0.94) | 0.18 (0.84)
  Usual Activities C6D1: number analyzed (Participants) | 123 | 122
  Usual Activities C6D1 | 0.14 (0.94) | 0.25 (0.84)
  Usual Activities C6D22: number analyzed (Participants) | 103 | 95
  Usual Activities C6D22 | 0.15 (1.02) | 0.15 (0.81)
  Usual Activities C7D1: number analyzed (Participants) | 114 | 98
  Usual Activities C7D1 | 0.15 (1.05) | 0.12 (0.80)
  Usual Activities C7D22: number analyzed (Participants) | 81 | 74
  Usual Activities C7D22 | 0.15 (1.10) | 0.05 (0.76)
  Usual Activities C8D1: number analyzed (Participants) | 82 | 83
  Usual Activities C8D1 | 0.18 (0.97) | 0.18 (0.87)
  Usual Activities C8D22: number analyzed (Participants) | 72 | 65
  Usual Activities C8D22 | 0.03 (1.05) | 0.09 (0.86)
  Usual Activities C9D1: number analyzed (Participants) | 75 | 62
  Usual Activities C9D1 | 0.07 (0.96) | 0.03 (0.75)
  Usual Activities C9D22: number analyzed (Participants) | 61 | 55
  Usual Activities C9D22 | 0.13 (0.99) | 0.07 (0.72)
  Usual Activities C10D1: number analyzed (Participants) | 66 | 56
  Usual Activities C10D1 | -0.02 (1.00) | 0.07 (0.95)
  Usual Activities C10D22: number analyzed (Participants) | 57 | 43
  Usual Activities C10D22 | -0.02 (0.88) | 0.09 (0.87)
  Usual Activities C11D1: number analyzed (Participants) | 63 | 46
  Usual Activities C11D1 | -0.05 (0.87) | 0.04 (0.82)
  Usual Activities C11D22: number analyzed (Participants) | 45 | 31
  Usual Activities C11D22 | 0.09 (0.95) | 0.23 (0.67)
  Usual Activities C12D1: number analyzed (Participants) | 53 | 41
  Usual Activities C12D1 | -0.08 (1.00) | 0.12 (0.60)
  Usual Activities C12D22: number analyzed (Participants) | 38 | 26
  Usual Activities C12D22 | 0.00 (0.93) | 0.23 (0.71)
  Usual Activities C13D1: number analyzed (Participants) | 48 | 35
  Usual Activities C13D1 | 0.04 (0.82) | 0.14 (0.81)
  Usual Activities C13D22: number analyzed (Participants) | 41 | 21
  Usual Activities C13D22 | 0.15 (0.88) | 0.10 (0.89)
  Usual Activities C14D1: number analyzed (Participants) | 39 | 30
  Usual Activities C14D1 | 0.03 (0.84) | 0.27 (0.91)
  Usual Activities C14D22: number analyzed (Participants) | 32 | 19
  Usual Activities C14D22 | 0.06 (0.76) | 0.00 (0.88)
  Usual Activities C15D1: number analyzed (Participants) | 35 | 27
  Usual Activities C15D1 | 0.09 (0.74) | 0.07 (0.68)
  Usual Activities C15D22: number analyzed (Participants) | 30 | 17
  Usual Activities C15D22 | 0.13 (1.04) | -0.12 (0.86)
  Usual Activities C16D1: number analyzed (Participants) | 35 | 22
  Usual Activities C16D1 | 0.20 (1.08) | 0.05 (0.84)
  Usual Activities C16D22: number analyzed (Participants) | 29 | 14
  Usual Activities C16D22 | -0.10 (0.72) | 0.14 (0.86)
  Usual Activities C17D1: number analyzed (Participants) | 30 | 18
  Usual Activities C17D1 | 0.23 (0.97) | 0.00 (0.69)
  Usual Activities C17D22: number analyzed (Participants) | 23 | 0
  Usual Activities C17D22 | 0.26 (0.86) |
  Usual Activities C18D1: number analyzed (Participants) | 27 | 16
  Usual Activities C18D1 | -0.07 (0.68) | 0.00 (0.37)
  Usual Activities C18D22: number analyzed (Participants) | 21 | 10
  Usual Activities C18D22 | 0.00 (0.84) | 0.10 (0.57)
  Usual Activities C19D1: number analyzed (Participants) | 23 | 15
  Usual Activities C19D1 | 0.13 (0.76) | 0.13 (0.52)
  Usual Activities C19D22: number analyzed (Participants) | 20 | 11
  Usual Activities C19D22 | 0.20 (0.77) | 0.00 (0.45)
  Usual Activities C20D1: number analyzed (Participants) | 23 | 15
  Usual Activities C20D1 | 0.04 (0.64) | 0.07 (0.46)
  Usual Activities C20D22: number analyzed (Participants) | 18 | 10
  Usual Activities C20D22 | 0.11 (0.83) | -0.10 (0.32)
  Usual Activities C21D1: number analyzed (Participants) | 20 | 14
  Usual Activities C21D1 | 0.10 (0.31) | 0.07 (0.47)
  Usual Activities C21D22: number analyzed (Participants) | 14 | 0
  Usual Activities C21D22 | 0.14 (0.36) |
  Usual Activities C22D1: number analyzed (Participants) | 15 | 12
  Usual Activities C22D1 | 0.13 (0.52) | 0.08 (0.51)
  Usual Activities C22D22: number analyzed (Participants) | 11 | 0
  Usual Activities C22D22 | 0.36 (0.67) |
  Usual Activities C23D1: number analyzed (Participants) | 16 | 13
  Usual Activities C23D1 | 0.50 (0.63) | 0.00 (0.41)
  Usual Activities C23D22: number analyzed (Participants) | 11 | 0
  Usual Activities C23D22 | 0.18 (0.40) |
  Usual Activities C24D1: number analyzed (Participants) | 14 | 0
  Usual Activities C24D1 | 0.36 (0.63) |
  Usual Activities C24D22: number analyzed (Participants) | 0 | 0
  Usual Activities C25D1: number analyzed (Participants) | 12 | 0
  Usual Activities C25D1 | 0.17 (0.58) |
  Usual Activities C25D22: number analyzed (Participants) | 11 | 0
  Usual Activities C25D22 | 0.18 (0.40) |
  Usual Activities C26D1: number analyzed (Participants) | 13 | 0
  Usual Activities C26D1 | 0.15 (0.38) |
  Usual Activities C27D1: number analyzed (Participants) | 11 | 0
  Usual Activities C27D1 | 0.27 (0.47) |
  Usual Activities C28D1: number analyzed (Participants) | 12 | 0
  Usual Activities C28D1 | 0.17 (0.39) |
  Usual Activities 30 Day follow up: number analyzed (Participants) | 72 | 92
  Usual Activities 30 Day follow up | 0.29 (1.13) | 0.40 (1.02)
  Usual Activities 90 Day follow up: number analyzed (Participants) | 86 | 83
  Usual Activities 90 Day follow up | 0.41 (1.12) | 0.59 (1.06)
  Pain/Discomfort Baseline | 1.93 (0.87) | 1.98 (0.91)
  Pain/Discomfort C1D22: number analyzed (Participants) | 178 | 212
  Pain/Discomfort C1D22 | 0.08 (0.93) | -0.15 (0.84)
  Pain/Discomfort C2D1: number analyzed (Participants) | 207 | 226
  Pain/Discomfort C2D1 | -0.14 (0.91) | -0.36 (0.87)
  Pain/Discomfort C2D22: number analyzed (Participants) | 152 | 181
  Pain/Discomfort C2D22 | -0.14 (0.88) | -0.24 (0.90)
  Pain/Discomfort C3D1: number analyzed (Participants) | 190 | 198
  Pain/Discomfort C3D1 | -0.23 (0.94) | -0.31 (0.96)
  Pain/Discomfort C3D22: number analyzed (Participants) | 154 | 149
  Pain/Discomfort C3D22 | -0.11 (0.88) | -0.31 (0.85)
  Pain/Discomfort C4D1: number analyzed (Participants) | 172 | 164
  Pain/Discomfort C4D1 | -0.16 (0.93) | -0.28 (0.90)
  Pain/Discomfort C4D22: number analyzed (Participants) | 125 | 128
  Pain/Discomfort C4D22 | -0.14 (0.89) | -0.28 (0.85)
  Pain/Discomfort C5D1: number analyzed (Participants) | 150 | 146
  Pain/Discomfort C5D1 | -0.19 (0.88) | -0.22 (0.97)
  Pain/Discomfort C5D22: number analyzed (Participants) | 114 | 116
  Pain/Discomfort C5D22 | -0.02 (1.04) | -0.19 (0.95)
  Pain/Discomfort C6D1: number analyzed (Participants) | 123 | 122
  Pain/Discomfort C6D1 | -0.18 (0.87) | -0.19 (0.92)
  Pain/Discomfort C6D22: number analyzed (Participants) | 103 | 95
  Pain/Discomfort C6D22 | -0.08 (0.96) | -0.26 (0.80)
  Pain/Discomfort C7D1: number analyzed (Participants) | 114 | 98
  Pain/Discomfort C7D1 | -0.15 (0.91) | -0.21 (0.92)
  Pain/Discomfort C7D22: number analyzed (Participants) | 81 | 74
  Pain/Discomfort C7D22 | -0.12 (0.97) | -0.30 (0.90)
  Pain/Discomfort C8D1: number analyzed (Participants) | 82 | 83
  Pain/Discomfort C8D1 | -0.12 (0.91) | -0.18 (0.98)
  Pain/Discomfort C8D22: number analyzed (Participants) | 72 | 65
  Pain/Discomfort C8D22 | -0.14 (0.88) | -0.34 (0.73)
  Pain/Discomfort C9D1: number analyzed (Participants) | 75 | 62
  Pain/Discomfort C9D1 | -0.21 (1.02) | -0.29 (0.78)
  Pain/Discomfort C9D22: number analyzed (Participants) | 61 | 55
  Pain/Discomfort C9D22 | -0.05 (0.80) | -0.31 (0.88)
  Pain/Discomfort C10D1: number analyzed (Participants) | 66 | 56
  Pain/Discomfort C10D1 | -0.20 (0.95) | -0.30 (1.03)
  Pain/Discomfort C10D22: number analyzed (Participants) | 57 | 43
  Pain/Discomfort C10D22 | -0.14 (0.88) | -0.35 (0.87)
  Pain/Discomfort C11D1: number analyzed (Participants) | 63 | 46
  Pain/Discomfort C11D1 | -0.22 (0.89) | -0.17 (0.71)
  Pain/Discomfort C11D22: number analyzed (Participants) | 45 | 31
  Pain/Discomfort C11D22 | -0.11 (0.83) | -0.32 (0.79)
  Pain/Discomfort C12D1: number analyzed (Participants) | 53 | 41
  Pain/Discomfort C12D1 | -0.19 (0.81) | -0.15 (0.79)
  Pain/Discomfort C12D22: number analyzed (Participants) | 38 | 26
  Pain/Discomfort C12D22 | -0.18 (0.95) | -0.27 (0.72)
  Pain/Discomfort C13D1: number analyzed (Participants) | 48 | 35
  Pain/Discomfort C13D1 | -0.13 (0.89) | -0.20 (0.93)
  Pain/Discomfort C13D22: number analyzed (Participants) | 41 | 21
  Pain/Discomfort C13D22 | 0.07 (0.93) | -0.19 (1.12)
  Pain/Discomfort C14D1: number analyzed (Participants) | 39 | 30
  Pain/Discomfort C14D1 | -0.05 (0.83) | -0.33 (0.66)
  Pain/Discomfort C14D22: number analyzed (Participants) | 32 | 19
  Pain/Discomfort C14D22 | -0.09 (0.89) | -0.47 (1.02)
  Pain/Discomfort C15D1: number analyzed (Participants) | 35 | 27
  Pain/Discomfort C15D1 | -0.14 (0.73) | -0.07 (0.92)
  Pain/Discomfort C15D22: number analyzed (Participants) | 30 | 17
  Pain/Discomfort C15D22 | -0.17 (0.83) | -0.35 (1.27)
  Pain/Discomfort C16D1: number analyzed (Participants) | 35 | 22
  Pain/Discomfort C16D1 | -0.17 (0.71) | -0.14 (1.04)
  Pain/Discomfort C16D22: number analyzed (Participants) | 29 | 14
  Pain/Discomfort C16D22 | -0.28 (0.80) | -0.29 (0.61)
  Pain/Discomfort C17D1: number analyzed (Participants) | 30 | 18
  Pain/Discomfort C17D1 | -0.23 (0.73) | -0.33 (0.69)
  Pain/Discomfort C17D22: number analyzed (Participants) | 23 | 0
  Pain/Discomfort C17D22 | -0.13 (0.92) |
  Pain/Discomfort C18D1: number analyzed (Participants) | 27 | 16
  Pain/Discomfort C18D1 | -0.26 (0.90) | 0.00 (0.73)
  Pain/Discomfort C18D22: number analyzed (Participants) | 21 | 10
  Pain/Discomfort C18D22 | -0.43 (0.81) | -0.20 (0.79)
  Pain/Discomfort C19D1: number analyzed (Participants) | 23 | 15
  Pain/Discomfort C19D1 | -0.30 (0.70) | -0.07 (0.70)
  Pain/Discomfort C19D22: number analyzed (Participants) | 20 | 11
  Pain/Discomfort C19D22 | -0.10 (0.72) | -0.18 (0.75)
  Pain/Discomfort C20D1: number analyzed (Participants) | 23 | 15
  Pain/Discomfort C20D1 | -0.22 (0.80) | 0.00 (0.76)
  Pain/Discomfort C20D22: number analyzed (Participants) | 18 | 10
  Pain/Discomfort C20D22 | -0.28 (0.75) | 0.10 (0.74)
  Pain/Discomfort C21D1: number analyzed (Participants) | 20 | 14
  Pain/Discomfort C21D1 | -0.25 (0.64) | -0.14 (0.66)
  Pain/Discomfort C21D22: number analyzed (Participants) | 14 | 0
  Pain/Discomfort C21D22 | 0.21 (0.58) |
  Pain/Discomfort C22D1: number analyzed (Participants) | 15 | 12
  Pain/Discomfort C22D1 | -0.20 (0.68) | -0.17 (0.72)
  Pain/Discomfort C22D22: number analyzed (Participants) | 11 | 0
  Pain/Discomfort C22D22 | 0.00 (0.77) |
  Pain/Discomfort C23D1: number analyzed (Participants) | 16 | 13
  Pain/Discomfort C23D1 | -0.13 (0.89) | -0.23 (0.73)
  Pain/Discomfort C23D22: number analyzed (Participants) | 11 | 0
  Pain/Discomfort C23D22 | -0.09 (0.83) |
  Pain/Discomfort C24D1: number analyzed (Participants) | 14 | 0
  Pain/Discomfort C24D1 | -0.07 (1.14) |
  Pain/Discomfort C24D22: number analyzed (Participants) | 0 | 0
  Pain/Discomfort C25D1: number analyzed (Participants) | 12 | 0
  Pain/Discomfort C25D1 | -0.17 (0.72) |
  Pain/Discomfort C25D22: number analyzed (Participants) | 11 | 0
  Pain/Discomfort C25D22 | -0.09 (0.70) |
  Pain/Discomfort C26D1: number analyzed (Participants) | 13 | 0
  Pain/Discomfort C26D1 | -0.08 (0.76) |
  Pain/Discomfort C27D1: number analyzed (Participants) | 11 | 0
  Pain/Discomfort C27D1 | -0.27 (0.79) |
  Pain/Discomfort C28D1: number analyzed (Participants) | 12 | 0
  Pain/Discomfort C28D1 | -0.25 (0.97) |
  Pain/Discomfort 30 Day follow up: number analyzed (Participants) | 72 | 92
  Pain/Discomfort 30 Day follow up | -0.06 (0.96) | 0.17 (0.99)
  Pain/Discomfort 90 day follow up: number analyzed (Participants) | 86 | 83
  Pain/Discomfort 90 day follow up | 0.02 (1.04) | 0.07 (1.06)
  Anxiety/Depression Baseline | 1.76 (0.84) | 1.80 (0.83)
  Anxiety/Depression C1D22: number analyzed (Participants) | 178 | 212
  Anxiety/Depression C1D22 | -0.03 (0.81) | -0.09 (0.70)
  Anxiety/Depression C2D1: number analyzed (Participants) | 207 | 226
  Anxiety/Depression C2D1 | -0.09 (0.82) | -0.22 (0.73)
  Anxiety/Depression C2D22: number analyzed (Participants) | 152 | 181
  Anxiety/Depression C2D22 | -0.09 (0.78) | -0.12 (0.78)
  Anxiety/Depression C3D1: number analyzed (Participants) | 190 | 198
  Anxiety/Depression C3D1 | -0.14 (0.80) | -0.24 (0.76)
  Anxiety/Depression C3D22: number analyzed (Participants) | 154 | 149
  Anxiety/Depression C3D22 | -0.10 (0.85) | -0.24 (0.80)
  Anxiety/Depression C4D1: number analyzed (Participants) | 172 | 164
  Anxiety/Depression C4D1 | -0.22 (0.78) | -0.23 (0.84)
  Anxiety/Depression C4D22: number analyzed (Participants) | 125 | 128
  Anxiety/Depression C4D22 | -0.10 (0.87) | -0.17 (0.88)
  Anxiety/Depression C5D1: number analyzed (Participants) | 150 | 146
  Anxiety/Depression C5D1 | -0.15 (0.80) | -0.16 (0.81)
  Anxiety/Depression C5D22: number analyzed (Participants) | 114 | 116
  Anxiety/Depression C5D22 | -0.11 (0.97) | -0.05 (0.79)
  Anxiety/Depression C6D1: number analyzed (Participants) | 123 | 122
  Anxiety/Depression C6D1 | -0.20 (0.82) | -0.18 (0.86)
  Anxiety/Depression C6D22: number analyzed (Participants) | 103 | 95
  Anxiety/Depression C6D22 | -0.08 (0.82) | -0.14 (0.94)
  Anxiety/Depression C7D1: number analyzed (Participants) | 114 | 98
  Anxiety/Depression C7D1 | -0.12 (0.94) | -0.28 (0.77)
  Anxiety/Depression C7D22: number analyzed (Participants) | 81 | 74
  Anxiety/Depression C7D22 | -0.06 (0.83) | -0.19 (0.77)
  Anxiety/Depression C8D1: number analyzed (Participants) | 82 | 83
  Anxiety/Depression C8D1 | -0.18 (0.83) | -0.11 (0.86)
  Anxiety/Depression C8D22: number analyzed (Participants) | 72 | 65
  Anxiety/Depression C8D22 | -0.10 (0.87) | -0.22 (0.80)
  Anxiety/Depression C9D1: number analyzed (Participants) | 75 | 62
  Anxiety/Depression C9D1 | -0.17 (1.07) | -0.19 (0.83)
  Anxiety/Depression C9D22: number analyzed (Participants) | 61 | 55
  Anxiety/Depression C9D22 | -0.08 (0.97) | -0.15 (0.87)
  Anxiety/Depression C10D1: number analyzed (Participants) | 66 | 56
  Anxiety/Depression C10D1 | -0.17 (0.94) | -0.27 (0.88)
  Anxiety/Depression C10D22: number analyzed (Participants) | 57 | 43
  Anxiety/Depression C10D22 | -0.16 (0.86) | -0.19 (0.96)
  Anxiety/Depression C11D1: number analyzed (Participants) | 63 | 46
  Anxiety/Depression C11D1 | -0.21 (0.97) | -0.15 (0.89)
  Anxiety/Depression C11D22: number analyzed (Participants) | 45 | 31
  Anxiety/Depression C11D22 | -0.20 (0.94) | -0.03 (1.17)
  Anxiety/Depression C12D1: number analyzed (Participants) | 53 | 41
  Anxiety/Depression C12D1 | -0.09 (0.97) | -0.07 (0.93)
  Anxiety/Depression C12D22: number analyzed (Participants) | 38 | 26
  Anxiety/Depression C12D22 | -0.11 (0.86) | 0.08 (0.98)
  Anxiety/Depression C13D1: number analyzed (Participants) | 48 | 35
  Anxiety/Depression C13D1 | -0.10 (1.02) | 0.00 (1.08)
  Anxiety/Depression C13D22: number analyzed (Participants) | 41 | 21
  Anxiety/Depression C13D22 | -0.10 (1.07) | 0.19 (0.98)
  Anxiety/Depression C14D1: number analyzed (Participants) | 39 | 30
  Anxiety/Depression C14D1 | -0.03 (1.04) | 0.00 (1.11)
  Anxiety/Depression C14D22: number analyzed (Participants) | 32 | 19
  Anxiety/Depression C14D22 | -0.19 (1.03) | -0.05 (1.13)
  Anxiety/Depression C15D1: number analyzed (Participants) | 35 | 27
  Anxiety/Depression C15D1 | -0.26 (0.92) | -0.15 (0.86)
  Anxiety/Depression C15D22: number analyzed (Participants) | 30 | 17
  Anxiety/Depression C15D22 | -0.17 (1.05) | -0.12 (0.99)
  Anxiety/Depression C16D1: number analyzed (Participants) | 35 | 22
  Anxiety/Depression C16D1 | -0.29 (1.05) | -0.14 (0.99)
  Anxiety/Depression C16D22: number analyzed (Participants) | 29 | 14
  Anxiety/Depression C16D22 | -0.41 (0.91) | -0.14 (0.66)
  Anxiety/Depression C17D1: number analyzed (Participants) | 30 | 18
  Anxiety/Depression C17D1 | -0.10 (0.96) | -0.33 (0.69)
  Anxiety/Depression C17D22: number analyzed (Participants) | 23 | 0
  Anxiety/Depression C17D22 | -0.26 (1.01) |
  Anxiety/Depression C18D1: number analyzed (Participants) | 27 | 16
  Anxiety/Depression C18D1 | -0.48 (0.85) | -0.06 (0.93)
  Anxiety/Depression C18D22: number analyzed (Participants) | 21 | 10
  Anxiety/Depression C18D22 | -0.33 (0.73) | -0.40 (0.97)
  Anxiety/Depression C19D1: number analyzed (Participants) | 23 | 15
  Anxiety/Depression C19D1 | -0.30 (0.56) | -0.13 (0.74)
  Anxiety/Depression C19D22: number analyzed (Participants) | 20 | 11
  Anxiety/Depression C19D22 | -0.25 (0.72) | -0.18 (1.08)
  Anxiety/Depression C20D1: number analyzed (Participants) | 23 | 15
  Anxiety/Depression C20D1 | -0.26 (0.62) | -0.20 (0.77)
  Anxiety/Depression C20D22: number analyzed (Participants) | 18 | 10
  Anxiety/Depression C20D22 | -0.39 (0.78) | -0.20 (0.79)
  Anxiety/Depression C21D1: number analyzed (Participants) | 20 | 14
  Anxiety/Depression C21D1 | -0.35 (0.75) | -0.21 (0.89)
  Anxiety/Depression C21D22: number analyzed (Participants) | 14 | 0
  Anxiety/Depression C21D22 | -0.36 (0.63) |
  Anxiety/Depression C22D1: number analyzed (Participants) | 15 | 12
  Anxiety/Depression C22D1 | -0.27 (0.80) | -0.33 (0.78)
  Anxiety/Depression C22D22: number analyzed (Participants) | 11 | 0
  Anxiety/Depression C22D22 | 0.00 (1.00) |
  Anxiety/Depression C23D1: number analyzed (Participants) | 16 | 13
  Anxiety/Depression C23D1 | -0.06 (1.06) | -0.15 (0.69)
  Anxiety/Depression C23D22: number analyzed (Participants) | 11 | 0
  Anxiety/Depression C23D22 | -0.18 (1.08) |
  Anxiety/Depression C24D1: number analyzed (Participants) | 14 | 0
  Anxiety/Depression C24D1 | 0.00 (1.04) |
  Anxiety/Depression C24D22: number analyzed (Participants) | 0 | 0
  Anxiety/Depression C25D1: number analyzed (Participants) | 12 | 0
  Anxiety/Depression C25D1 | -0.17 (0.72) |
  Anxiety/Depression C25D22: number analyzed (Participants) | 11 | 0
  Anxiety/Depression C25D22 | -0.27 (0.65) |
  Anxiety/Depression C26D1: number analyzed (Participants) | 13 | 0
  Anxiety/Depression C26D1 | -0.23 (0.73) |
  Anxiety/Depression C27D1: number analyzed (Participants) | 11 | 0
  Anxiety/Depression C27D1 | -0.27 (0.79) |
  Anxiety/Depression C28D1: number analyzed (Participants) | 12 | 0
  Anxiety/Depression C28D1 | -0.33 (0.78) |
  Anxiety/Depression 30 Day follow up: number analyzed (Participants) | 72 | 92
  Anxiety/Depression 30 Day follow up | 0.04 (1.01) | 0.12 (0.98)
  Anxiety/Depression 90 Day follow up: number analyzed (Participants) | 86 | 83
  Anxiety/Depression 90 Day follow up | 0.01 (1.02) | 0.00 (0.96)
  Visual Analog Scale Baseline | 68.91 (19.15) | 67.95 (19.78)
  Visual Analog Scale C1D22: number analyzed (Participants) | 178 | 212
  Visual Analog Scale C1D22 | -3.44 (18.53) | -0.21 (15.63)
  Visual Analog Scale C2D1: number analyzed (Participants) | 207 | 226
  Visual Analog Scale C2D1 | 0.05 (18.05) | 4.10 (17.43)
  Visual Analog Scale C2D22: number analyzed (Participants) | 152 | 181
  Visual Analog Scale C2D22 | 0.63 (18.37) | 2.25 (19.26)
  Visual Analog Scale C3D1: number analyzed (Participants) | 190 | 198
  Visual Analog Scale C3D1 | 1.16 (18.61) | 5.57 (18.23)
  Visual Analog Scale C3D22: number analyzed (Participants) | 154 | 149
  Visual Analog Scale C3D22 | -1.69 (18.39) | 2.73 (19.27)
  Visual Analog Scale C4D1: number analyzed (Participants) | 172 | 164
  Visual Analog Scale C4D1 | 0.35 (17.10) | 5.89 (17.65)
  Visual Analog Scale C4D22: number analyzed (Participants) | 125 | 128
  Visual Analog Scale C4D22 | -1.11 (19.16) | 3.39 (17.41)
  Visual Analog Scale C5D1: number analyzed (Participants) | 150 | 146
  Visual Analog Scale C5D1 | -0.54 (19.36) | 5.14 (17.26)
  Visual Analog Scale C5D22: number analyzed (Participants) | 114 | 116
  Visual Analog Scale C5D22 | 0.37 (22.01) | 2.29 (18.00)
  Visual Analog Scale C6D1: number analyzed (Participants) | 123 | 122
  Visual Analog Scale C6D1 | 1.28 (19.67) | 2.48 (20.43)
  Visual Analog Scale C6D22: number analyzed (Participants) | 103 | 95
  Visual Analog Scale C6D22 | 4.33 (18.56) | 5.21 (16.71)
  Visual Analog Scale C7D1: number analyzed (Participants) | 114 | 98
  Visual Analog Scale C7D1 | 1.32 (20.58) | 6.15 (15.20)
  Visual Analog Scale C7D22: number analyzed (Participants) | 81 | 74
  Visual Analog Scale C7D22 | 3.51 (17.92) | 5.14 (14.60)
  Visual Analog Scale C8D1: number analyzed (Participants) | 82 | 83
  Visual Analog Scale C8D1 | 3.77 (21.13) | 6.60 (14.65)
  Visual Analog Scale C8D22: number analyzed (Participants) | 72 | 65
  Visual Analog Scale C8D22 | 2.71 (19.07) | 7.65 (14.13)
  Visual Analog Scale C9D1: number analyzed (Participants) | 75 | 62
  Visual Analog Scale C9D1 | 5.05 (19.16) | 5.24 (13.63)
  Visual Analog Scale C9D22: number analyzed (Participants) | 61 | 55
  Visual Analog Scale C9D22 | 2.44 (21.10) | 6.42 (15.96)
  Visual Analog Scale C10D1: number analyzed (Participants) | 66 | 56
  Visual Analog Scale C10D1 | 2.52 (18.65) | 5.86 (18.29)
  C10D22: number analyzed (Participants) | 57 | 43
  C10D22 | 3.23 (17.27) | 6.72 (15.81)
  Visual Analog Scale C11D1: number analyzed (Participants) | 63 | 46
  Visual Analog Scale C11D1 | 5.10 (17.23) | 7.33 (14.98)
  Visual Analog Scale C11D22: number analyzed (Participants) | 45 | 31
  Visual Analog Scale C11D22 | 3.96 (15.63) | 5.58 (15.74)
  Visual Analog Scale C12D1: number analyzed (Participants) | 53 | 41
  Visual Analog Scale C12D1 | 1.06 (18.03) | 3.95 (17.66)
  Visual Analog Scale C12D22: number analyzed (Participants) | 38 | 26
  Visual Analog Scale C12D22 | -1.55 (17.56) | 3.69 (16.11)
  Visual Analog Scale C13D1: number analyzed (Participants) | 48 | 35
  Visual Analog Scale C13D1 | 3.27 (17.64) | 3.34 (17.40)
  Visual Analog Scale C13D22: number analyzed (Participants) | 41 | 21
  Visual Analog Scale C13D22 | -0.29 (18.30) | 1.67 (17.02)
  Visual Analog Scale C14D1: number analyzed (Participants) | 39 | 30
  Visual Analog Scale C14D1 | -0.15 (16.81) | 5.83 (13.93)
  Visual Analog Scale C14D22: number analyzed (Participants) | 32 | 19
  Visual Analog Scale C14D22 | -0.25 (18.75) | 3.53 (14.98)
  Visual Analog Scale C15D1: number analyzed (Participants) | 35 | 27
  Visual Analog Scale C15D1 | -0.09 (16.90) | 7.11 (14.91)
  Visual Analog Scale C15D22: number analyzed (Participants) | 30 | 17
  Visual Analog Scale C15D22 | -2.63 (23.87) | 2.29 (17.85)
  Visual Analog Scale C16D1: number analyzed (Participants) | 35 | 22
  Visual Analog Scale C16D1 | 2.43 (16.37) | 3.86 (15.94)
  Visual Analog Scale C16D22: number analyzed (Participants) | 29 | 14
  Visual Analog Scale C16D22 | 2.00 (15.26) | 0.36 (12.34)
  Visual Analog Scale C17D1: number analyzed (Participants) | 30 | 18
  Visual Analog Scale C17D1 | 2.50 (16.74) | 1.72 (14.90)
  Visual Analog Scale C17D22: number analyzed (Participants) | 23 | 0
  Visual Analog Scale C17D22 | -2.61 (17.26) |
  Visual Analog Scale C18D1: number analyzed (Participants) | 27 | 16
  Visual Analog Scale C18D1 | 2.85 (18.61) | 2.69 (12.72)
  Visual Analog Scale C18D22: number analyzed (Participants) | 21 | 10
  Visual Analog Scale C18D22 | 0.86 (18.74) | 2.90 (12.08)
  Visual Analog Scale C19D1: number analyzed (Participants) | 23 | 15
  Visual Analog Scale C19D1 | 5.39 (16.57) | 3.33 (14.11)
  Visual Analog Scale C19D22: number analyzed (Participants) | 20 | 11
  Visual Analog Scale C19D22 | -0.25 (19.05) | 3.73 (10.36)
  Visual Analog Scale C20D1: number analyzed (Participants) | 23 | 15
  Visual Analog Scale C20D1 | 1.57 (21.46) | 3.67 (13.97)
  Visual Analog Scale C20D22: number analyzed (Participants) | 18 | 10
  Visual Analog Scale C20D22 | 0.78 (16.00) | 7.00 (14.24)
  Visual Analog Scale C21D1: number analyzed (Participants) | 20 | 14
  Visual Analog Scale C21D1 | 2.80 (15.83) | 4.00 (15.06)
  Visual Analog Scale C21D22: number analyzed (Participants) | 14 | 0
  Visual Analog Scale C21D22 | -4.64 (12.29) |
  Visual Analog Scale C22D1: number analyzed (Participants) | 15 | 12
  Visual Analog Scale C22D1 | 1.33 (17.37) | 4.25 (16.19)
  Visual Analog Scale C22D22: number analyzed (Participants) | 11 | 0
  Visual Analog Scale C22D22 | -6.00 (19.20) |
  Visual Analog Scale C23D1: number analyzed (Participants) | 16 | 13
  Visual Analog Scale C23D1 | -2.25 (18.36) | 5.31 (17.77)
  Visual Analog Scale C23D22: number analyzed (Participants) | 11 | 0
  Visual Analog Scale C23D22 | -3.09 (16.57) |
  Visual Analog Scale C24D1: number analyzed (Participants) | 14 | 0
  Visual Analog Scale C24D1 | -3.43 (18.81) |
  Visual Analog Scale C24D22: number analyzed (Participants) | 0 | 0
  Visual Analog Scale C25D1: number analyzed (Participants) | 12 | 0
  Visual Analog Scale C25D1 | -4.08 (15.32) |
  Visual Analog Scale C25D22: number analyzed (Participants) | 11 | 0
  Visual Analog Scale C25D22 | -4.64 (14.43) |
  Visual Analog Scale C26D1: number analyzed (Participants) | 13 | 0
  Visual Analog Scale C26D1 | 1.69 (16.79) |
  Visual Analog Scale C27D1: number analyzed (Participants) | 11 | 0
  Visual Analog Scale C27D1 | 1.45 (17.15) |
  Visual Analog Scale C28D1: number analyzed (Participants) | 12 | 0
  Visual Analog Scale C28D1 | -0.42 (17.61) |
  Visual Analog Scale 30 Day follow up: number analyzed (Participants) | 72 | 92
  Visual Analog Scale 30 Day follow up | -1.33 (18.53) | -2.07 (17.67)
  Visual Analog Scale 90 Day follow up: number analyzed (Participants) | 86 | 83
  Visual Analog Scale 90 Day follow up | -3.79 (20.59) | -4.84 (19.73)

14. Secondary Outcome: Pharmacokinetics (PK) of Zolbetuximab in Serum: Trough Concentration (Ctrough)
Description: Ctrough was defined as the predose concentration at the end of dosing interval.
Time Frame: Predose on C1D22, C3D1, C5D1, C7D1, C9D1
Population: PKAS consisted of the subset of the SAF for which at least 1 zolbetuximab concentration measurement was available. Participants with available data at each timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: micrograms/mililiter (ug/mL)
Arm/Group | mFOLFOX6 + Zolbetuximab
Number analyzed (Participants) | 184
micrograms/mililiter (ug/mL)
  C1D22: number analyzed (Participants) | 181
  C1D22 | 40.9 (37.2)
  C3D1 | 70.1 (49.8)
  C5D1: number analyzed (Participants) | 139
  C5D1 | 97.4 (50.8)
  C7D1: number analyzed (Participants) | 97
  C7D1 | 118.0 (64.9)
  C9D1: number analyzed (Participants) | 58
  C9D1 | 135.0 (56.2)

15. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADA)
Description: Immunogenicity will be measured by the number of participants that are ADA positive.
Time Frame: Predose on C1D1, C1D22, C3D1, C5D1, C7D1, C9D1, 30-day follow up, 90-day follow up
Population: Participants who were randomized to zolbetuximab + mFOLFOX6 Arm with at least One Valid Result for ADA.
Measure: Number; unit: Participants
Arm/Group | mFOLFOX6 + Zolbetuximab
Number analyzed (Participants) | 283
Participants
  C1D1: number analyzed (Participants) | 265
  C1D1 | 2
  C1D22: number analyzed (Participants) | 182
  C1D22 | 2
  C3D1: number analyzed (Participants) | 189
  C3D1 | 3
  C5D1: number analyzed (Participants) | 139
  C5D1 | 2
  C7D1: number analyzed (Participants) | 101
  C7D1 | 2
  C9D1: number analyzed (Participants) | 59
  C9D1 | 1
  30 day follow up: number analyzed (Participants) | 85
  30 day follow up | 4
  90 day follow up: number analyzed (Participants) | 76
  90 day follow up | 1

ADVERSE EVENTS:
Time Frame: All- cause mortality (ACM): From randomization up to 62 months and 18 days Adverse events: From first dose until 62 months and 18 days
Description: Serious adverse events: SAF defined as all participants who received at least one dose of the study drug. Participants may have been repeated in the arm groups.
  ACM was analyzed for all randomized population.
Groups:
- Zolbetuximab: Participants received an IV infusion (as a minimum of 2-hourinfusion) ofzolbetuximab at a loading dose of 800mg/m^2 on C1D1followed by subsequent doses of 600 mg/m^2every 3 weeks starting from C1D22 until participant meets study treatment discontinuation criteria .Each cycle wasapproximately 42 days.
- 5-fluorouracil: Participants received up to 12 treatments of5-fluorouracil over 4 or more cycles administered by IV bolus 400 mg/m^2 over5 to 15 minutes followed by 2400mg/m^2 over46-48 hours continuous IV infusion every 2weeks for 4 cycles. Participants could continue to receive 5-fluorouracil on Days 1,15 and 29 of each cycle at the investigator's discretion or until the participant met the study treatment discontinuation criteria. Each cycle was approximately 42 days.
- Folinic Acid / Leucovorin: Participants received up to 12 treatments of folinic acid administered 400mg/m^2 IV infusion over 2 hours 4 or more cycles on Days 1, 15 and29 of each cycle. Participants could continue to receive folinic acid on Days 1,15 and 29 of each cycle at the investigator's discretion or until the participant met the study treatment discontinuation criteria. Each cycle was approximately 42 days.
- Oxaliplatin: Participants received up to 12 treatments of oxaliplatin administered 85 mg/m^2 IV infusion over 2 hours) on Days 1,15 and 29 of each cycle.. A maximum of 12 doses of oxaliplatin was permitted. Each cycle was approximately 42days.
- Placebo: Participants received anIV infusion (as a minimum of 2-hourinfusion) of placebo matched to zolbetuximab on C1D1followed by subsequent doses every 3 weeks starting from C1D22until participant met study treatment discontinuation criteria. Each cycle was approximately 42 days.
Arm/Group | Zolbetuximab | 5-fluorouracil | Folinic Acid / Leucovorin | Oxaliplatin | Placebo
All-Cause Mortality (participants affected / at risk) | 197/283 | 414/565 | 414/565 | 414/565 | 217/282
Serious Adverse Events (participants affected / at risk) | 133/279 | 262/557 | 262/557 | 262/557 | 129/278
Other Adverse Events (participants affected / at risk) | 276/279 | 550/557 | 550/557 | 550/557 | 274/278
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zolbetuximab (N=279) | 5-fluorouracil (N=557) | Folinic Acid / Leucovorin (N=557) | Oxaliplatin (N=557) | Placebo (N=278)
Anaemia (Blood and lymphatic system disorders) | 5 (6) | 9 (10) | 9 (10) | 9 (10) | 4 (4)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 8 (8) | 9 (9) | 9 (9) | 9 (9) | 1 (1)
Microangiopathic haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 6 (6) | 9 (9) | 9 (9) | 9 (9) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 3 (3) | 3 (3) | 3 (3) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (3) | 2 (3) | 2 (3) | 2 (3) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 3 (3) | 3 (3) | 3 (3) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Dihydropyrimidine dehydrogenase deficiency (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 14 (17) | 14 (17) | 14 (17) | 9 (12)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (3) | 3 (3) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 13 (14) | 13 (14) | 13 (14) | 5 (6)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 6 (9) | 6 (9) | 6 (9) | 4 (7)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Gastric stenosis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (3) | 2 (3) | 2 (3) | 2 (3)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (2) | 1 (2) | 1 (2)
Haematemesis (Gastrointestinal disorders) | 1 (2) | 3 (4) | 3 (4) | 3 (4) | 2 (2)
Haemorrhagic ascites (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 4 (4) | 4 (4) | 4 (4) | 4 (4)
Intestinal obstruction (Gastrointestinal disorders) | 7 (13) | 12 (21) | 12 (21) | 12 (21) | 5 (8)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 2 (3) | 2 (3) | 2 (3) | 1 (2)
Lip swelling (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 19 (25) | 31 (39) | 31 (39) | 31 (39) | 12 (14)
Obstruction gastric (Gastrointestinal disorders) | 2 (2) | 3 (3) | 3 (3) | 3 (3) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 2 (2)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (2) | 1 (2) | 1 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Retching (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (3) | 5 (7) | 5 (7) | 5 (7) | 3 (4)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (4) | 3 (4) | 3 (4) | 3 (4) | 0 (0)
Volvulus (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 24 (36) | 38 (59) | 38 (59) | 38 (59) | 14 (23)
Asthenia (General disorders) | 6 (6) | 9 (9) | 9 (9) | 9 (9) | 3 (3)
Chest pain (General disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Chills (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Complication associated with device (General disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Death (General disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Device related thrombosis (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Discomfort (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Fatigue (General disorders) | 4 (4) | 7 (7) | 7 (7) | 7 (7) | 3 (3)
General physical health deterioration (General disorders) | 2 (2) | 8 (9) | 8 (9) | 8 (9) | 6 (7)
Inflammation (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Pneumatosis (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 7 (7) | 13 (14) | 13 (14) | 13 (14) | 6 (7)
Acute hepatic failure (Hepatobiliary disorders) | 1 (2) | 1 (2) | 1 (2) | 1 (2) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Biliary dilatation (Hepatobiliary disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Biliary obstruction (Hepatobiliary disorders) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 4 (5) | 4 (5) | 4 (5) | 3 (4)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 4 (4) | 4 (4) | 4 (4) | 3 (3)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 3 (3) | 3 (3) | 3 (3) | 3 (3)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Abscess soft tissue (Infections and infestations) | 0 (0) | 1 (2) | 1 (2) | 1 (2) | 1 (2)
Appendicitis (Infections and infestations) | 1 (2) | 3 (4) | 3 (4) | 3 (4) | 2 (2)
Atypical pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 3 (4) | 3 (4) | 3 (4) | 2 (3)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 1 (2) | 2 (3) | 2 (3) | 2 (3) | 1 (1)
Campylobacter infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 2 (2) | 4 (4) | 4 (4) | 4 (4) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Large intestine infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (2) | 1 (2) | 1 (2) | 1 (2) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 7 (7) | 15 (16) | 15 (16) | 15 (16) | 8 (9)
Pneumonia aspiration (Infections and infestations) | 3 (3) | 4 (4) | 4 (4) | 4 (4) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 5 (6) | 6 (7) | 6 (7) | 6 (7) | 1 (1)
Septic shock (Infections and infestations) | 2 (3) | 2 (3) | 2 (3) | 2 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 2 (2) | 3 (3) | 3 (3) | 3 (3) | 1 (1)
Urinary tract infection fungal (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal anastomotic stenosis (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (2) | 1 (2) | 1 (2) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 4 (4) | 4 (4) | 4 (4) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 4 (4) | 4 (4) | 4 (4) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 2 (5) | 2 (5) | 2 (5) | 1 (4)
Blood potassium decreased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Electrocardiogram T wave inversion (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
General physical condition abnormal (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 5 (5) | 5 (5) | 5 (5) | 4 (4)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Adult failure to thrive (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 3 (3) | 3 (3) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 4 (4) | 4 (4) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 3 (3) | 3 (3) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (8) | 7 (10) | 7 (10) | 7 (10) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10) | 22 (23) | 22 (23) | 22 (23) | 12 (13)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 2 (2)
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4) | 4 (4) | 4 (4) | 1 (1)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 2 (2)
Ataxia (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 2 (2)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Embolic stroke (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (2) | 1 (2) | 1 (2) | 1 (2) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Slow speech (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 3 (3) | 4 (4) | 4 (4) | 4 (4) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Wernicke's encephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 2 (2)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 3 (3) | 3 (3) | 3 (3) | 3 (3) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Renal artery occlusion (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (2) | 1 (2) | 1 (2) | 1 (2) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (4) | 3 (4) | 3 (4) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 6 (7) | 6 (7) | 6 (7) | 5 (5)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5) | 5 (5) | 5 (5) | 3 (3)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 10 (10) | 10 (10) | 10 (10) | 4 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (4) | 3 (4) | 3 (4) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 4 (4) | 5 (5) | 5 (5) | 5 (5) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Embolism venous (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (3) | 3 (4) | 3 (4) | 3 (4) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Abdominal sepsis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Clostridial sepsis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Varicella (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Fat embolism (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Post procedural bile leak (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Euthanasia (Surgical and medical procedures) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zolbetuximab (N=279) | 5-fluorouracil (N=557) | Folinic Acid / Leucovorin (N=557) | Oxaliplatin (N=557) | Placebo (N=278)
Anaemia (Blood and lymphatic system disorders) | 105 (309) | 211 (616) | 211 (616) | 211 (616) | 106 (307)
Leukopenia (Blood and lymphatic system disorders) | 17 (34) | 30 (57) | 30 (57) | 30 (57) | 13 (23)
Neutropenia (Blood and lymphatic system disorders) | 101 (340) | 195 (674) | 195 (674) | 195 (674) | 94 (334)
Thrombocytopenia (Blood and lymphatic system disorders) | 29 (67) | 74 (180) | 74 (180) | 74 (180) | 45 (113)
Abdominal distension (Gastrointestinal disorders) | 16 (23) | 39 (50) | 39 (50) | 39 (50) | 23 (27)
Abdominal pain (Gastrointestinal disorders) | 68 (137) | 154 (274) | 154 (274) | 154 (274) | 86 (137)
Abdominal pain upper (Gastrointestinal disorders) | 47 (76) | 80 (124) | 80 (124) | 80 (124) | 33 (48)
Constipation (Gastrointestinal disorders) | 101 (154) | 212 (334) | 212 (334) | 212 (334) | 111 (180)
Diarrhoea (Gastrointestinal disorders) | 112 (202) | 237 (477) | 237 (477) | 237 (477) | 125 (275)
Dyspepsia (Gastrointestinal disorders) | 28 (35) | 48 (60) | 48 (60) | 48 (60) | 20 (25)
Dysphagia (Gastrointestinal disorders) | 22 (28) | 43 (62) | 43 (62) | 43 (62) | 21 (34)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 14 (16) | 30 (32) | 30 (32) | 30 (32) | 16 (16)
Nausea (Gastrointestinal disorders) | 226 (816) | 396 (1221) | 396 (1221) | 396 (1221) | 170 (405)
Stomatitis (Gastrointestinal disorders) | 60 (133) | 119 (226) | 119 (226) | 119 (226) | 59 (93)
Vomiting (Gastrointestinal disorders) | 180 (557) | 278 (732) | 278 (732) | 278 (732) | 98 (175)
Asthenia (General disorders) | 69 (198) | 131 (339) | 131 (339) | 131 (339) | 62 (141)
Chills (General disorders) | 16 (18) | 26 (29) | 26 (29) | 26 (29) | 10 (11)
Fatigue (General disorders) | 83 (190) | 175 (414) | 175 (414) | 175 (414) | 92 (224)
Malaise (General disorders) | 21 (55) | 30 (76) | 30 (76) | 30 (76) | 9 (21)
Oedema peripheral (General disorders) | 51 (70) | 78 (104) | 78 (104) | 78 (104) | 27 (34)
Pyrexia (General disorders) | 55 (102) | 102 (175) | 102 (175) | 102 (175) | 47 (73)
COVID-19 (Infections and infestations) | 24 (26) | 48 (53) | 48 (53) | 48 (53) | 24 (27)
Oral candidiasis (Infections and infestations) | 5 (5) | 19 (30) | 19 (30) | 19 (30) | 14 (25)
Urinary tract infection (Infections and infestations) | 15 (20) | 24 (33) | 24 (33) | 24 (33) | 9 (13)
Alanine aminotransferase increased (Investigations) | 35 (74) | 83 (204) | 83 (204) | 83 (204) | 48 (130)
Aspartate aminotransferase increased (Investigations) | 50 (99) | 95 (225) | 95 (225) | 95 (225) | 45 (126)
Blood alkaline phosphatase increased (Investigations) | 21 (32) | 46 (95) | 46 (95) | 46 (95) | 25 (63)
Neutrophil count decreased (Investigations) | 96 (359) | 185 (772) | 185 (772) | 185 (772) | 89 (413)
Platelet count decreased (Investigations) | 41 (107) | 90 (257) | 90 (257) | 90 (257) | 49 (150)
Weight decreased (Investigations) | 57 (81) | 113 (170) | 113 (170) | 113 (170) | 56 (89)
White blood cell count decreased (Investigations) | 51 (236) | 97 (492) | 97 (492) | 97 (492) | 46 (256)
Decreased appetite (Metabolism and nutrition disorders) | 136 (259) | 233 (458) | 233 (458) | 233 (458) | 97 (199)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 46 (117) | 64 (153) | 64 (153) | 64 (153) | 18 (36)
Hypocalcaemia (Metabolism and nutrition disorders) | 30 (72) | 39 (82) | 39 (82) | 39 (82) | 9 (10)
Hypokalaemia (Metabolism and nutrition disorders) | 49 (101) | 89 (167) | 89 (167) | 89 (167) | 40 (66)
Hyponatraemia (Metabolism and nutrition disorders) | 15 (26) | 27 (41) | 27 (41) | 27 (41) | 12 (15)
Hypophosphataemia (Metabolism and nutrition disorders) | 18 (27) | 32 (60) | 32 (60) | 32 (60) | 14 (33)
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 (28) | 47 (63) | 47 (63) | 47 (63) | 25 (35)
Back pain (Musculoskeletal and connective tissue disorders) | 36 (47) | 70 (89) | 70 (89) | 70 (89) | 34 (42)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (12) | 25 (30) | 25 (30) | 25 (30) | 15 (18)
Dizziness (Nervous system disorders) | 37 (61) | 64 (96) | 64 (96) | 64 (96) | 27 (35)
Dysgeusia (Nervous system disorders) | 44 (60) | 84 (112) | 84 (112) | 84 (112) | 40 (52)
Headache (Nervous system disorders) | 34 (60) | 69 (113) | 69 (113) | 69 (113) | 35 (53)
Neuropathy peripheral (Nervous system disorders) | 23 (57) | 45 (94) | 45 (94) | 45 (94) | 22 (37)
Paraesthesia (Nervous system disorders) | 44 (88) | 91 (175) | 91 (175) | 91 (175) | 47 (87)
Peripheral sensory neuropathy (Nervous system disorders) | 107 (261) | 226 (549) | 226 (549) | 226 (549) | 119 (288)
Insomnia (Psychiatric disorders) | 31 (44) | 56 (73) | 56 (73) | 56 (73) | 25 (29)
Cough (Respiratory, thoracic and mediastinal disorders) | 30 (42) | 60 (80) | 60 (80) | 60 (80) | 30 (38)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 (35) | 53 (79) | 53 (79) | 53 (79) | 32 (44)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14 (15) | 40 (45) | 40 (45) | 40 (45) | 26 (30)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 17 (21) | 29 (35) | 29 (35) | 29 (35) | 12 (14)
Alopecia (Skin and subcutaneous tissue disorders) | 21 (21) | 42 (43) | 42 (43) | 42 (43) | 21 (22)
Dry skin (Skin and subcutaneous tissue disorders) | 22 (26) | 35 (39) | 35 (39) | 35 (39) | 13 (13)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 25 (43) | 47 (74) | 47 (74) | 47 (74) | 22 (31)
Pruritus (Skin and subcutaneous tissue disorders) | 24 (32) | 50 (65) | 50 (65) | 50 (65) | 26 (33)
Rash (Skin and subcutaneous tissue disorders) | 17 (20) | 40 (48) | 40 (48) | 40 (48) | 23 (28)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 (13) | 23 (31) | 23 (31) | 23 (31) | 15 (18)
Hypertension (Vascular disorders) | 33 (82) | 54 (115) | 54 (115) | 54 (115) | 21 (33)
Dry mouth (Gastrointestinal disorders) | 14 (16) | 24 (30) | 24 (30) | 24 (30) | 10 (14)
Mucosal inflammation (General disorders) | 6 (7) | 20 (23) | 20 (23) | 20 (23) | 14 (16)
Blood bilirubin increased (Investigations) | 7 (7) | 22 (34) | 22 (34) | 22 (34) | 15 (27)
Hyperglycaemia (Metabolism and nutrition disorders) | 15 (29) | 26 (52) | 26 (52) | 26 (52) | 11 (23)
Anxiety (Psychiatric disorders) | 14 (16) | 22 (25) | 22 (25) | 22 (25) | 8 (9)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 17 (19) | 17 (19) | 17 (19) | 14 (15)
Hypotension (Vascular disorders) | 13 (20) | 27 (36) | 27 (36) | 27 (36) | 14 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2024-11-14): https://cdn.clinicaltrials.gov/large-docs/97/NCT03504397/Prot_002.pdf
  • Statistical Analysis Plan (2023-05-02): https://cdn.clinicaltrials.gov/large-docs/97/NCT03504397/SAP_003.pdf